CLINICAL TRIAL: NCT03688620
Title: Enhanced Safety Surveillance of GSK's Quadrivalent Seasonal Influenza Vaccines
Brief Title: Enhanced Safety Surveillance of GlaxoSmithKline's (GSK's) Quadrivalent Seasonal Influenza Vaccines During the 2018/19 Influenza Season
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 207737
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Influenza, Human
Keywords: Pilot study; Safety surveillance; Quadrivalent seasonal influenza vaccine; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccinated_AlphaRix Tetra Group (Other): Volunteered male and female subjects, 18 years of age and above, who received in Belgium one dose of GlaxoSmithKline's (GSK's) quadrivalent seasonal influenza vaccine (AlphaRix Tetra) between 01 October and 31 December 2018.
  Interventions: Other: Passive enhanced safety surveillance
- Vaccinated_Influsplit Tetra Group (Other): Volunteered subjects male and female subjects, 18 years of age and above, who received in Germany one dose of GSK's quadrivalent seasonal influenza vaccine (Influsplit Tetra) between 01 October and 31 December 2018.
  Interventions: Other: Passive enhanced safety surveillance
- Vaccinated_Fluarix Tetra Group (Other): Volunteered male and female subjects, between 6 months and 65 years of age, who received in Spain one or two dose(s) of GSK's quadrivalent seasonal influenza vaccine (Fluarix Tetra) between 01 October and 31 December 2018.
  Interventions: Other: Passive enhanced safety surveillance

INTERVENTIONS:
Other: Passive enhanced safety surveillance — Prospective data collection starting at Visit 1 (Day 1) and ending at Visit 2 (Day 8 or when the ADR card was returned by mail) for all subjects who have previously been vaccinated against influenza in preceding seasons or aged ≥9 years at the time of vaccination, or ending at Visit 4 (Day 36 or when the last ADR card was returned by mail) for children aged <9 years who have not previously been vaccinated against influenza in preceding seasons). Subjects had up to 14 days post vaccination to return their ADR card (at the next study visit or by mail).

SUMMARY:
The purpose of this study is to comply with the European Medicines Agency (EMA) guidance on enhanced safety surveillance for seasonal influenza vaccines in the European Union (EU) and aims to assess adverse events of interest (AEIs) experienced within 7 days post vaccination with GSK's quadrivalent seasonal influenza vaccine (AlphaRix Tetra in Belgium; Influsplit Tetra in Germany, Fluarix Tetra in Spain).

This study may help to inform decisions regarding future influenza vaccine safety surveillance for influenza vaccines in Europe.

DETAILED DESCRIPTION:
The key objective of the EMA enhanced safety surveillance is to rapidly detect a significant increase in the frequency and/or severity of expected reactions (local, systemic or allergic reactions) that may indicate a potential risk.

The study is a passive enhanced safety surveillance aiming to collect prospectively AEIs and/or other AEs experienced within 7 days post vaccination with GSK's quadrivalent seasonal influenza vaccine, using customized Adverse Drug Reaction cards. Data will be collected via the healthcare provide (HCP) or study medical staff who administer the seasonal influenza vaccination or who provide the inform consent form and the ADR cards.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., complete the ADR card, return for the next scheduled visit or return the ADR card by mail within a timely manner).
* A male or female subject vaccinated with GSK's quadrivalent seasonal influenza vaccine (one or two dose schedule) according to the routine medical practices between 01 October 2018 and 31 December 2018.
* Subjects aged 6 months or above at the time of the vaccination according to the countries' specificities.
* Written informed consent/informed assent obtained from the subjects/subjects' parent(s)/Legally Acceptable Representative(s) (LARs).

Exclusion Criteria:

• Child in care.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Belgium (3):
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Steenokkerzeel
  - GSK Investigational Site, Tessenderlo
- Germany (3):
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
- Spain (3):
  - GSK Investigational Site, Marbella - Málaga, Andalusia
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dos Santos G, Nguyen BY, Damaso S, Godderis L, Martinez-Gomez X, Eckermann T, Loos H, Salamanca de la Cueva I, Shende V, Schmidt AC, Yeakey A. Brand-Specific Enhanced Safety Surveillance of GSK's Quadrivalent Seasonal Influenza Vaccine in Belgium, Germany and Spain for the 2018/2019 Season. Drug Saf. 2020 Mar;43(3):265-279. doi: 10.1007/s40264-019-00893-4. PMID 31884676
- [Background] Dos Santos G, Shende V, Damaso S, Yeakey A. Enhanced Safety Surveillance of GSK's Quadrivalent Seasonal Influenza Vaccine in Belgium, Germany, and Spain for the 2018/19 Season: Interim Analysis. Adv Ther. 2019 Dec;36(12):3340-3355. doi: 10.1007/s12325-019-01105-2. Epub 2019 Oct 8. PMID 31595482
- [Background] Dos Santos G, Yeakey A, Shende V, Smith K, Lin F, Zandman-van-Dijk E, Damaso S, Schmidt A. Passive enhanced safety surveillance of GSK's quadrivalent seasonal influenza vaccine in Belgium, Germany and Spain, an observational study: protocol for the 2018/2019 influenza season. BMJ Open. 2019 Aug 18;9(8):e028043. doi: 10.1136/bmjopen-2018-028043. PMID 31427321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GSK's quadrivalent seasonal influenza vaccine (AlphaRix Tetra in Belgium; Influsplit Tetra in Germany, Fluarix Tetra in Spain) was administered to subjects in this study
Pre-assignment Details: Subjects aged <9 years in Vaccinated_Fluarix Tetra Group (Spain) who were not vaccinated against influenza in preceding seasons received 2 doses of quadrivalent seasonal influenza vaccine in this study. Subjects from other groups received only 1 dose of the vaccine. Dose 2 results correspond to only some subjects in Vaccinated_Fluarix Tetra Group.
Period: Overall Study
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group
Started | 329 | 278 | 453
Completed | 313 | 277 | 445
Not Completed | 16 | 1 | 8
Not completed — Other | 0 | 0 | 1
Not completed — Unwilling to attend the scheduled visit | 0 | 1 | 0
Not completed — Lost to Follow-up | 16 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (18.2) | 65.0 (15.1) | 15.7 (18.7) | 42.8 (29.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 166 | 231 | 544
  Male | 182 | 112 | 222 | 516
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or african american | 0 | 2 | 1 | 3
  Asian - central / south asian heritage | 1 | 1 | 1 | 3
  Asian - east asian heritage | 4 | 1 | 0 | 5
  Asian - south east asian heritage | 2 | 0 | 0 | 2
  White - arabic / north african heritage | 1 | 0 | 3 | 4
  White - caucasian / european heritage | 321 | 274 | 444 | 1039
  Other, Not specified | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Weekly Percentage of Subjects Reporting Any AEIs and/or Other Aes, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: Analysis was performed on the enrolled subjects who were vaccinated with the first dose of GSK's quadrivalent seasonal influenza vaccine and who returned the ADR card.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Total Group: Volunteered male and female subjects from Vaccinated_AlphaRix Tetra Group, Vaccinated_Influsplit Tetra Group and Vaccinated_Fluarix Tetra Group were pooled into the Total Group. Therefore, subjects included in the Total Group received GSK's quadrivalent seasonal influenza vaccine, as follows: one dose of AlphaRix Tetra vaccine (first group) or one dose of Influsplit Tetra (second group) or one or two dose(s) of Fluarix Tetra vaccine (third group), between 1 October and 31 December 2018.
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Week 40 |  | 32.86 [12.23 to 59.90] |  | 32.86 [12.23 to 59.90]
  Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Week 41 |  | 36.26 [0.95 to 92.78] |  | 36.26 [0.95 to 92.78]
  Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Week 42 | 45.39 [36.99 to 53.98] | 32.56 [19.08 to 48.54] | 44.23 [0.11 to 99.54] | 42.80 [35.52 to 50.31]
  Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Week 43 | 45.16 [27.32 to 63.97] | 38.46 [13.86 to 68.42] | 47.44 [36.01 to 59.07] | 45.90 [36.85 to 55.16]
  Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Week 44 | 55.56 [0.01 to 100] | 20.00 [4.33 to 48.09] | 35.38 [7.27 to 74.31] | 39.66 [19.21 to 63.16]
  Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Week 45 | 35.14 [0.51 to 94.16] | 66.67 [40.99 to 86.66] | 50.97 [22.51 to 78.97] | 47.37 [32.15 to 62.96]
  Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Week 46 | 26.92 [11.57 to 47.79] | 42.31 [23.35 to 63.08] | 38.81 [27.14 to 51.50] | 36.97 [28.01 to 46.66]
  Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Week 47 | 38.10 [18.11 to 61.56] | 50.00 [1.26 to 98.74] | 70.00 [0.00 to 100] | 53.49 [16.09 to 88.07]
  Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Week 48 |  |  | 81.25 [0.01 to 100] | 81.25 [0.01 to 100]

2. Secondary Outcome: Weekly Percentage of Subjects Reporting Any AEIs and/or AEs Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: Analysis was performed on the enrolled subjects who were vaccinated with a second dose of GSK's quadrivalent seasonal influenza vaccine and who returned the ADR card. This analysis was performed only for the Fluarix Tetra Group, and not on the other groups who did not received this second dose.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Week 46: number analyzed (Participants) | 3
  Week 46 | 33.33 [0.84 to 90.57]
  Week 47: number analyzed (Participants) | 19
  Week 47 | 47.37 [24.45 to 71.14]
  Week 48: number analyzed (Participants) | 25
  Week 48 | 44.00 [24.40 to 65.07]
  Week 49: number analyzed (Participants) | 34
  Week 49 | 11.76 [0.58 to 44.96]
  Week 50: number analyzed (Participants) | 42
  Week 50 | 9.52 [2.66 to 22.62]
  Week 51: number analyzed (Participants) | 12
  Week 51 | 25.00 [0.00 to 100]
  Week 52: number analyzed (Participants) | 4
  Week 52 | 25.00 [0.63 to 80.59]

3. Secondary Outcome: Weekly Percentage of Subjects Reporting Gastrointestinal Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were diarrhoea, nausea, and vomiting.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 2.20 [0.01 to 16.50] |  | 2.20 [0.01 to 16.50]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 2.13 [0.00 to 57.89] | 11.63 [0.00 to 97.87] | 7.69 [0.19 to 36.17] | 5.08 [0.60 to 17.38]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 9.68 [2.04 to 25.75] | 7.69 [0.19 to 36.03] | 8.97 [0.05 to 50.25] | 9.02 [4.59 to 15.56]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 13.89 [0.00 to 87.39] | 6.67 [0.17 to 31.95] | 4.62 [0.40 to 17.47] | 7.76 [2.02 to 19.22]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 9.46 [3.89 to 18.52] | 11.11 [1.38 to 34.71] | 3.87 [0.04 to 23.24] | 6.07 [1.97 to 13.71]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 7.69 [0.95 to 25.13] | 3.85 [0.10 to 19.64] | 10.45 [1.35 to 32.48] | 8.40 [2.93 to 18.07]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 84.19] | 10.00 [1.23 to 31.70] | 9.30 [2.59 to 22.14]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  Diarrhoea,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Diarrhoea,Week 40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Diarrhoea,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Diarrhoea,Week 41 |  | 2.20 [0.01 to 16.50] |  | 2.20 [0.01 to 16.50]
  Diarrhoea,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Diarrhoea,Week 42 | 0.00 [0.00 to 2.58] | 6.98 [0.00 to 87.92] | 3.85 [0.11 to 19.24] | 2.12 [0.03 to 12.28]
  Diarrhoea,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Diarrhoea,Week 43 | 6.45 [0.79 to 21.42] | 0.00 [0.00 to 24.71] | 5.13 [0.00 to 75.69] | 4.92 [1.81 to 10.44]
  Diarrhoea,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Diarrhoea,Week 44 | 2.78 [0.00 to 84.65] | 6.67 [0.17 to 31.95] | 3.08 [0.00 to 24.91] | 3.45 [0.95 to 8.59]
  Diarrhoea,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Diarrhoea,Week 45 | 2.70 [0.00 to 85.98] | 5.56 [0.14 to 27.29] | 3.23 [0.00 to 33.25] | 3.24 [0.60 to 9.60]
  Diarrhoea,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Diarrhoea,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 13.23] | 5.97 [0.15 to 29.14] | 4.20 [0.40 to 15.52]
  Diarrhoea,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Diarrhoea,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Diarrhoea,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Diarrhoea,Week 48 |  |  | 6.25 [0.00 to 89.64] | 6.25 [0.00 to 89.64]
  Nausea,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Nausea,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Nausea,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Nausea,Week 41 |  | 1.10 [0.00 to 21.06] |  | 1.10 [0.00 to 21.06]
  Nausea,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Nausea,Week 42 | 2.13 [0.00 to 57.89] | 4.65 [0.00 to 74.17] | 3.85 [0.11 to 19.24] | 2.97 [0.90 to 7.05]
  Nausea,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Nausea,Week 43 | 3.23 [0.08 to 16.70] | 7.69 [0.19 to 36.03] | 2.56 [0.31 to 8.96] | 3.28 [0.90 to 8.18]
  Nausea,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Nausea,Week 44 | 8.33 [1.75 to 22.47] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 24.91] | 4.31 [0.90 to 12.07]
  Nausea,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Nausea,Week 45 | 5.41 [0.00 to 64.32] | 0.00 [0.00 to 18.53] | 1.29 [0.00 to 12.14] | 2.43 [0.24 to 9.10]
  Nausea,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Nausea,Week 46 | 3.85 [0.10 to 19.64] | 3.85 [0.10 to 19.64] | 5.97 [0.15 to 29.14] | 5.04 [1.43 to 12.26]
  Nausea,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Nausea,Week 47 | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.98] | 6.98 [1.18 to 20.68]
  Nausea,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Nausea,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Vomiting,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Vomiting,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Vomiting,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Vomiting,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Vomiting,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Vomiting,Week 42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 8.22] | 5.77 [0.15 to 27.99] | 1.69 [0.07 to 8.20]
  Vomiting,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Vomiting,Week 43 | 3.23 [0.08 to 16.70] | 0.00 [0.00 to 24.71] | 3.85 [0.57 to 12.37] | 3.28 [0.90 to 8.18]
  Vomiting,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Vomiting,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 24.91] | 2.59 [0.54 to 7.37]
  Vomiting,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Vomiting,Week 45 | 2.70 [0.00 to 39.00] | 0.00 [0.00 to 18.53] | 1.94 [0.00 to 28.41] | 2.02 [0.25 to 7.13]
  Vomiting,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Vomiting,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 1.49 [0.00 to 42.07] | 0.84 [0.00 to 9.95]
  Vomiting,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Vomiting,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 2.33 [0.00 to 25.06]
  Vomiting,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Vomiting,Week 48 |  |  | 6.25 [0.00 to 89.64] | 6.25 [0.00 to 89.64]
  Abdominal discomfort,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Abdominal discomfort,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Abdominal discomfort,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Abdominal discomfort,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Abdominal discomfort,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Abdominal discomfort,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Abdominal discomfort,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Abdominal discomfort,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Abdominal discomfort,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Abdominal discomfort,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Abdominal discomfort,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Abdominal discomfort,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Abdominal discomfort,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Abdominal discomfort,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 1.49 [0.04 to 8.04] | 0.84 [0.01 to 5.12]
  Abdominal discomfort,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Abdominal discomfort,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Abdominal discomfort,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Abdominal discomfort,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Abdominal pain,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Abdominal pain,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Abdominal pain,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Abdominal pain,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Abdominal pain,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Abdominal pain,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Abdominal pain,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Abdominal pain,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 3.85 [0.57 to 12.37] | 2.46 [0.11 to 11.37]
  Abdominal pain,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Abdominal pain,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Abdominal pain,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Abdominal pain,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Abdominal pain,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Abdominal pain,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Abdominal pain,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Abdominal pain,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Abdominal pain,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Abdominal pain,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Gingival bleeding,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Gingival bleeding,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Gingival bleeding,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Gingival bleeding,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Gingival bleeding,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Gingival bleeding,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Gingival bleeding,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Gingival bleeding,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Gingival bleeding,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Gingival bleeding,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Gingival bleeding,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Gingival bleeding,Week 45 | 0.00 [0.00 to 4.86] | 5.56 [0.14 to 27.29] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 4.05]
  Gingival bleeding,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Gingival bleeding,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Gingival bleeding,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Gingival bleeding,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Gingival bleeding,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Gingival bleeding,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Lip swelling,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Lip swelling,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Lip swelling,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Lip swelling,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Lip swelling,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Lip swelling,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Lip swelling,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Lip swelling,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Lip swelling,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Lip swelling,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Lip swelling,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Lip swelling,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Lip swelling,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Lip swelling,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Lip swelling,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Lip swelling,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Lip swelling,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Lip swelling,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Stomatitis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Stomatitis,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Stomatitis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Stomatitis,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Stomatitis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Stomatitis,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Stomatitis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Stomatitis,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Stomatitis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Stomatitis,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Stomatitis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Stomatitis,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Stomatitis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Stomatitis,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Stomatitis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Stomatitis,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Stomatitis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Stomatitis,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Tongue discomfort,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tongue discomfort,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Tongue discomfort,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Tongue discomfort,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Tongue discomfort,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Tongue discomfort,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Tongue discomfort,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Tongue discomfort,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Tongue discomfort,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Tongue discomfort,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Tongue discomfort,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Tongue discomfort,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Tongue discomfort,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Tongue discomfort,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Tongue discomfort,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Tongue discomfort,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Tongue discomfort,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Tongue discomfort,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

4. Secondary Outcome: Weekly Percentage of Subjects Reporting Gastrointestinal Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were diarrhoea, nausea, and vomiting.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 33.33 [0.84 to 90.57]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 10.53 [0.00 to 91.11]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 0.00 [0.00 to 13.72]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 0.00 [0.00 to 10.28]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 2.38 [0.00 to 58.03]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 0.00 [0.00 to 26.46]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Diarrhoea,Week 46: number analyzed (Participants) | 3
  Diarrhoea,Week 46 | 33.33 [0.84 to 90.57]
  Diarrhoea,Week 47: number analyzed (Participants) | 19
  Diarrhoea,Week 47 | 0.00 [0.00 to 17.65]
  Diarrhoea,Week 48: number analyzed (Participants) | 25
  Diarrhoea,Week 48 | 0.00 [0.00 to 13.72]
  Diarrhoea,Week 49: number analyzed (Participants) | 34
  Diarrhoea,Week 49 | 0.00 [0.00 to 10.28]
  Diarrhoea,Week 50: number analyzed (Participants) | 42
  Diarrhoea,Week 50 | 2.38 [0.00 to 58.03]
  Diarrhoea,Week 51: number analyzed (Participants) | 12
  Diarrhoea,Week 51 | 0.00 [0.00 to 26.46]
  Diarrhoea,Week 52: number analyzed (Participants) | 4
  Diarrhoea,Week 52 | 0.00 [0.00 to 60.24]
  Nausea,Week 46: number analyzed (Participants) | 3
  Nausea,Week 46 | 0.00 [0.00 to 70.76]
  Nausea,Week 47: number analyzed (Participants) | 19
  Nausea,Week 47 | 0.00 [0.00 to 17.65]
  Nausea,Week 48: number analyzed (Participants) | 25
  Nausea,Week 48 | 0.00 [0.00 to 13.72]
  Nausea,Week 49: number analyzed (Participants) | 34
  Nausea,Week 49 | 0.00 [0.00 to 10.28]
  Nausea,Week 50: number analyzed (Participants) | 42
  Nausea,Week 50 | 0.00 [0.00 to 8.41]
  Nausea,Week 51: number analyzed (Participants) | 12
  Nausea,Week 51 | 0.00 [0.00 to 26.46]
  Nausea,Week 52: number analyzed (Participants) | 4
  Nausea,Week 52 | 0.00 [0.00 to 60.24]
  Vomiting,Week 46: number analyzed (Participants) | 3
  Vomiting,Week 46 | 0.00 [0.00 to 70.76]
  Vomiting,Week 47: number analyzed (Participants) | 19
  Vomiting,Week 47 | 5.26 [0.00 to 100]
  Vomiting,Week 48: number analyzed (Participants) | 25
  Vomiting,Week 48 | 0.00 [0.00 to 13.72]
  Vomiting,Week 49: number analyzed (Participants) | 34
  Vomiting,Week 49 | 0.00 [0.00 to 10.28]
  Vomiting,Week 50: number analyzed (Participants) | 42
  Vomiting,Week 50 | 0.00 [0.00 to 8.41]
  Vomiting,Week 51: number analyzed (Participants) | 12
  Vomiting,Week 51 | 0.00 [0.00 to 26.46]
  Vomiting,Week 52: number analyzed (Participants) | 4
  Vomiting,Week 52 | 0.00 [0.00 to 60.24]
  Abdominal pain,Week 46: number analyzed (Participants) | 3
  Abdominal pain,Week 46 | 0.00 [0.00 to 70.76]
  Abdominal pain,Week 47: number analyzed (Participants) | 19
  Abdominal pain,Week 47 | 5.26 [0.00 to 95.26]
  Abdominal pain,Week 48: number analyzed (Participants) | 25
  Abdominal pain,Week 48 | 0.00 [0.00 to 13.72]
  Abdominal pain,Week 49: number analyzed (Participants) | 34
  Abdominal pain,Week 49 | 0.00 [0.00 to 10.28]
  Abdominal pain,Week 50: number analyzed (Participants) | 42
  Abdominal pain,Week 50 | 0.00 [0.00 to 8.41]
  Abdominal pain,Week 51: number analyzed (Participants) | 12
  Abdominal pain,Week 51 | 0.00 [0.00 to 26.46]
  Abdominal pain,Week 52: number analyzed (Participants) | 4
  Abdominal pain,Week 52 | 0.00 [0.00 to 60.24]

5. Secondary Outcome: Weekly Percentage of Subjects Reporting General Disorders and Administration Site Conditions by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were chills, face oedema, fatigue, injection site erythema, injection site pain, injection site swelling, and pyrexia.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 25.71 [16.01 to 37.56] |  | 25.71 [16.01 to 37.56]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 29.67 [0.86 to 86.02] |  | 29.67 [0.86 to 86.02]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 31.21 [18.49 to 46.39] | 25.58 [1.10 to 77.48] | 26.92 [0.28 to 88.26] | 29.24 [23.52 to 35.49]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 19.35 [7.45 to 37.47] | 15.38 [1.92 to 45.45] | 26.92 [17.50 to 38.16] | 23.77 [15.38 to 33.97]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 41.67 [0.00 to 100] | 20.00 [4.33 to 48.09] | 18.46 [2.70 to 50.43] | 25.86 [8.25 to 52.11]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 17.57 [0.00 to 96.81] | 50.00 [26.02 to 73.98] | 32.90 [6.71 to 70.97] | 29.55 [14.19 to 49.27]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 15.38 [4.36 to 34.87] | 26.92 [11.57 to 47.79] | 28.36 [13.66 to 47.42] | 25.21 [15.92 to 36.52]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 28.57 [11.28 to 52.18] | 0.00 [0.00 to 84.19] | 50.00 [3.46 to 96.54] | 37.21 [16.09 to 62.67]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 62.50 [2.31 to 99.81] | 62.50 [2.31 to 99.81]
  Chills,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Chills,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Chills,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Chills,Week 41 |  | 3.30 [0.00 to 51.97] |  | 3.30 [0.00 to 51.97]
  Chills,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Chills,Week 42 | 0.71 [0.01 to 4.40] | 4.65 [0.00 to 74.17] | 1.92 [0.05 to 10.26] | 1.69 [0.24 to 5.71]
  Chills,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Chills,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 3.85 [0.57 to 12.37] | 2.46 [0.11 to 11.37]
  Chills,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Chills,Week 44 | 5.56 [0.00 to 98.06] | 0.00 [0.00 to 21.80] | 1.54 [0.00 to 49.55] | 2.59 [0.04 to 14.92]
  Chills,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Chills,Week 45 | 1.35 [0.00 to 21.52] | 5.56 [0.14 to 27.29] | 1.94 [0.40 to 5.55] | 2.02 [0.66 to 4.66]
  Chills,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Chills,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 5.97 [0.15 to 29.14] | 4.20 [0.40 to 15.52]
  Chills,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Chills,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.98] | 4.65 [0.54 to 16.09]
  Chills,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Chills,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Face oedema,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Face oedema,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Face oedema,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Face oedema,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Face oedema,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Face oedema,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Face oedema,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Face oedema,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 1.28 [0.03 to 6.94] | 0.82 [0.02 to 4.48]
  Face oedema,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Face oedema,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.86 [0.00 to 7.14]
  Face oedema,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Face oedema,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Face oedema,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Face oedema,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Face oedema,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Face oedema,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Face oedema,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Face oedema,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Fatigue,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Fatigue,Week 40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Fatigue,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Fatigue,Week 41 |  | 6.59 [0.04 to 39.62] |  | 6.59 [0.04 to 39.62]
  Fatigue,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Fatigue,Week 42 | 2.84 [0.04 to 16.88] | 9.30 [0.00 to 94.72] | 3.85 [0.11 to 19.24] | 4.24 [1.42 to 9.50]
  Fatigue,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Fatigue,Week 43 | 3.23 [0.08 to 16.70] | 15.38 [1.92 to 45.45] | 8.97 [0.05 to 50.25] | 8.20 [3.43 to 15.98]
  Fatigue,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Fatigue,Week 44 | 11.11 [0.00 to 99.99] | 13.33 [1.66 to 40.46] | 7.69 [0.14 to 37.96] | 9.48 [3.06 to 21.05]
  Fatigue,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Fatigue,Week 45 | 4.05 [0.00 to 53.08] | 16.67 [3.58 to 41.42] | 6.45 [0.01 to 45.16] | 6.48 [1.76 to 15.92]
  Fatigue,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Fatigue,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 10.45 [4.30 to 20.35] | 6.72 [1.58 to 17.54]
  Fatigue,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Fatigue,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 15.00 [0.01 to 81.57] | 9.30 [1.44 to 27.75]
  Fatigue,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Fatigue,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Injection site erythema,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site erythema,Week 40 |  | 8.57 [0.03 to 50.40] |  | 8.57 [0.03 to 50.40]
  Injection site erythema,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Injection site erythema,Week 41 |  | 7.69 [3.15 to 15.21] |  | 7.69 [3.15 to 15.21]
  Injection site erythema,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Injection site erythema,Week 42 | 0.71 [0.01 to 4.40] | 11.63 [0.00 to 100] | 5.77 [0.15 to 27.99] | 3.81 [0.30 to 14.98]
  Injection site erythema,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Injection site erythema,Week 43 | 3.23 [0.08 to 16.70] | 0.00 [0.00 to 24.71] | 6.41 [0.92 to 20.26] | 4.92 [1.32 to 12.25]
  Injection site erythema,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Injection site erythema,Week 44 | 2.78 [0.00 to 99.94] | 6.67 [0.17 to 31.95] | 6.15 [1.70 to 15.01] | 5.17 [1.92 to 10.92]
  Injection site erythema,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Injection site erythema,Week 45 | 2.70 [0.00 to 85.98] | 0.00 [0.00 to 18.53] | 5.16 [0.14 to 25.09] | 4.05 [1.00 to 10.57]
  Injection site erythema,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Injection site erythema,Week 46 | 7.69 [0.95 to 25.13] | 7.69 [0.95 to 25.13] | 5.97 [1.65 to 14.59] | 6.72 [2.95 to 12.82]
  Injection site erythema,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Injection site erythema,Week 47 | 14.29 [3.05 to 36.34] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 6.98 [0.07 to 38.51]
  Injection site erythema,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Injection site erythema,Week 48 |  |  | 6.25 [0.00 to 89.64] | 6.25 [0.00 to 89.64]
  Injection site pain,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site pain,Week 40 |  | 17.14 [9.18 to 28.03] |  | 17.14 [9.18 to 28.03]
  Injection site pain,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Injection site pain,Week 41 |  | 18.68 [0.45 to 69.26] |  | 18.68 [0.45 to 69.26]
  Injection site pain,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Injection site pain,Week 42 | 28.37 [7.46 to 59.80] | 11.63 [3.89 to 25.08] | 15.38 [0.28 to 63.30] | 22.46 [11.43 to 37.26]
  Injection site pain,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Injection site pain,Week 43 | 16.13 [5.45 to 33.73] | 7.69 [0.19 to 36.03] | 6.41 [0.92 to 20.26] | 9.02 [2.58 to 21.26]
  Injection site pain,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Injection site pain,Week 44 | 22.22 [0.17 to 83.21] | 13.33 [1.66 to 40.46] | 6.15 [1.57 to 15.56] | 12.07 [3.94 to 26.25]
  Injection site pain,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Injection site pain,Week 45 | 10.81 [0.08 to 55.52] | 33.33 [13.34 to 59.01] | 20.00 [1.69 to 60.38] | 18.22 [7.78 to 33.71]
  Injection site pain,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Injection site pain,Week 46 | 3.85 [0.10 to 19.64] | 11.54 [2.45 to 30.15] | 17.91 [9.61 to 29.20] | 13.45 [6.23 to 24.24]
  Injection site pain,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Injection site pain,Week 47 | 14.29 [3.05 to 36.34] | 0.00 [0.00 to 84.19] | 30.00 [0.00 to 100] | 20.93 [4.47 to 50.12]
  Injection site pain,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Injection site pain,Week 48 |  |  | 62.50 [2.31 to 99.81] | 62.50 [2.31 to 99.81]
  Injection site swelling,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site swelling,Week 40 |  | 11.43 [1.34 to 36.13] |  | 11.43 [1.34 to 36.13]
  Injection site swelling,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Injection site swelling,Week 41 |  | 9.89 [2.71 to 23.60] |  | 9.89 [2.71 to 23.60]
  Injection site swelling,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Injection site swelling,Week 42 | 4.96 [0.48 to 18.09] | 9.30 [0.00 to 100] | 5.77 [0.15 to 27.99] | 5.93 [2.76 to 10.94]
  Injection site swelling,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Injection site swelling,Week 43 | 12.90 [3.63 to 29.83] | 0.00 [0.00 to 24.71] | 6.41 [0.92 to 20.26] | 7.38 [2.54 to 16.06]
  Injection site swelling,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Injection site swelling,Week 44 | 0.00 [0.00 to 9.74] | 13.33 [1.66 to 40.46] | 3.08 [0.37 to 10.68] | 3.45 [0.57 to 10.72]
  Injection site swelling,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Injection site swelling,Week 45 | 2.70 [0.00 to 100] | 16.67 [3.58 to 41.42] | 6.45 [2.78 to 12.43] | 6.07 [1.95 to 13.77]
  Injection site swelling,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Injection site swelling,Week 46 | 3.85 [0.10 to 19.64] | 15.38 [4.36 to 34.87] | 8.96 [1.32 to 27.23] | 9.24 [3.77 to 18.19]
  Injection site swelling,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Injection site swelling,Week 47 | 14.29 [3.05 to 36.34] | 0.00 [0.00 to 84.19] | 20.00 [0.00 to 99.87] | 16.28 [6.50 to 31.42]
  Injection site swelling,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Injection site swelling,Week 48 |  |  | 18.75 [0.00 to 100] | 18.75 [0.00 to 100]
  Pyrexia,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pyrexia,Week 40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Pyrexia,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Pyrexia,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Pyrexia,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Pyrexia,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 5.77 [0.15 to 27.99] | 1.27 [0.00 to 11.17]
  Pyrexia,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Pyrexia,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 12.82 [1.67 to 38.65] | 8.20 [0.32 to 35.08]
  Pyrexia,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Pyrexia,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 28.63] | 2.59 [0.54 to 7.37]
  Pyrexia,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Pyrexia,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 4.52 [0.41 to 16.82] | 2.83 [0.61 to 7.92]
  Pyrexia,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Pyrexia,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 13.23] | 7.46 [1.19 to 22.48] | 5.04 [0.91 to 14.89]
  Pyrexia,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Pyrexia,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 2.33 [0.00 to 25.06]
  Pyrexia,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Pyrexia,Week 48 |  |  | 6.25 [0.00 to 89.64] | 6.25 [0.00 to 89.64]
  Discomfort,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Discomfort,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Discomfort,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Discomfort,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Discomfort,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Discomfort,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Discomfort,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Discomfort,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Discomfort,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Discomfort,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Discomfort,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Discomfort,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 7.91] | 0.40 [0.00 to 2.58]
  Discomfort,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Discomfort,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Discomfort,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Discomfort,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Discomfort,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Discomfort,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Feeling cold,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Feeling cold,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Feeling cold,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Feeling cold,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Feeling cold,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Feeling cold,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Feeling cold,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Feeling cold,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Feeling cold,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Feeling cold,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Feeling cold,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Feeling cold,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Feeling cold,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Feeling cold,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Feeling cold,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Feeling cold,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Feeling cold,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Feeling cold,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Feeling hot,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Feeling hot,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Feeling hot,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Feeling hot,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Feeling hot,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Feeling hot,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Feeling hot,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Feeling hot,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Feeling hot,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Feeling hot,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Feeling hot,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Feeling hot,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Feeling hot,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Feeling hot,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Feeling hot,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Feeling hot,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Feeling hot,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Feeling hot,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Influenza like illness,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Influenza like illness,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Influenza like illness,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Influenza like illness,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Influenza like illness,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Influenza like illness,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Influenza like illness,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Influenza like illness,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Influenza like illness,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Influenza like illness,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Influenza like illness,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Influenza like illness,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Influenza like illness,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Influenza like illness,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 13.23] | 1.49 [0.04 to 8.04] | 1.68 [0.20 to 5.94]
  Influenza like illness,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Influenza like illness,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Influenza like illness,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Influenza like illness,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Injection site haematoma,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site haematoma,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Injection site haematoma,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Injection site haematoma,Week 41 |  | 1.10 [0.00 to 20.56] |  | 1.10 [0.00 to 20.56]
  Injection site haematoma,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Injection site haematoma,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Injection site haematoma,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Injection site haematoma,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Injection site haematoma,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Injection site haematoma,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Injection site haematoma,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Injection site haematoma,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Injection site haematoma,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Injection site haematoma,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Injection site haematoma,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Injection site haematoma,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Injection site haematoma,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Injection site haematoma,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Injection site pruritus,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site pruritus,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Injection site pruritus,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Injection site pruritus,Week 41 |  | 1.10 [0.00 to 21.06] |  | 1.10 [0.00 to 21.06]
  Injection site pruritus,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Injection site pruritus,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Injection site pruritus,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Injection site pruritus,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Injection site pruritus,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Injection site pruritus,Week 44 | 2.78 [0.00 to 99.94] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.86 [0.00 to 8.39]
  Injection site pruritus,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Injection site pruritus,Week 45 | 0.00 [0.00 to 4.86] | 11.11 [1.38 to 34.71] | 0.65 [0.00 to 7.91] | 1.21 [0.03 to 6.55]
  Injection site pruritus,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Injection site pruritus,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Injection site pruritus,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Injection site pruritus,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Injection site pruritus,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Injection site pruritus,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Injection site warmth,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site warmth,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Injection site warmth,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Injection site warmth,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Injection site warmth,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Injection site warmth,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Injection site warmth,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Injection site warmth,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Injection site warmth,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Injection site warmth,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Injection site warmth,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Injection site warmth,Week 45 | 1.35 [0.00 to 99.69] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 4.19]
  Injection site warmth,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Injection site warmth,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Injection site warmth,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Injection site warmth,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Injection site warmth,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Injection site warmth,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Malaise,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Malaise,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Malaise,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Malaise,Week 41 |  | 1.10 [0.00 to 20.56] |  | 1.10 [0.00 to 20.56]
  Malaise,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Malaise,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Malaise,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Malaise,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Malaise,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Malaise,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Malaise,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Malaise,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Malaise,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Malaise,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Malaise,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Malaise,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Malaise,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Malaise,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Mucous membrane disorder,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Mucous membrane disorder,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Mucous membrane disorder,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Mucous membrane disorder,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Mucous membrane disorder,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Mucous membrane disorder,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Mucous membrane disorder,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Mucous membrane disorder,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Mucous membrane disorder,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Mucous membrane disorder,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 1.54 [0.00 to 47.01] | 0.86 [0.00 to 8.91]
  Mucous membrane disorder,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Mucous membrane disorder,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 11.49] | 0.40 [0.00 to 3.03]
  Mucous membrane disorder,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Mucous membrane disorder,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Mucous membrane disorder,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Mucous membrane disorder,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Mucous membrane disorder,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Mucous membrane disorder,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Peripheral swelling,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Peripheral swelling,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Peripheral swelling,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Peripheral swelling,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Peripheral swelling,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Peripheral swelling,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Peripheral swelling,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Peripheral swelling,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Peripheral swelling,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Peripheral swelling,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.86 [0.00 to 7.14]
  Peripheral swelling,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Peripheral swelling,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Peripheral swelling,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Peripheral swelling,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 1.49 [0.00 to 42.07] | 0.84 [0.00 to 9.95]
  Peripheral swelling,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Peripheral swelling,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Peripheral swelling,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Peripheral swelling,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

6. Secondary Outcome: Weekly Percentage of Subjects Reporting General Disorders and Administration Site Conditions by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were chills, face oedema, fatigue, injection site erythema, injection site pain, injection site swelling, and pyrexia.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 36.84 [0.00 to 100]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 4.00 [0.10 to 20.35]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 2.94 [0.07 to 15.33]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 4.76 [0.58 to 16.16]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 8.33 [0.21 to 38.48]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 25.00 [0.63 to 80.59]
  Chills,Week 46: number analyzed (Participants) | 3
  Chills,Week 46 | 0.00 [0.00 to 70.76]
  Chills,Week 47: number analyzed (Participants) | 19
  Chills,Week 47 | 0.00 [0.00 to 17.65]
  Chills,Week 48: number analyzed (Participants) | 25
  Chills,Week 48 | 0.00 [0.00 to 13.72]
  Chills,Week 49: number analyzed (Participants) | 34
  Chills,Week 49 | 0.00 [0.00 to 10.28]
  Chills,Week 50: number analyzed (Participants) | 42
  Chills,Week 50 | 0.00 [0.00 to 8.41]
  Chills,Week 51: number analyzed (Participants) | 12
  Chills,Week 51 | 0.00 [0.00 to 26.46]
  Chills,Week 52: number analyzed (Participants) | 4
  Chills,Week 52 | 0.00 [0.00 to 60.24]
  Face oedema,Week 46: number analyzed (Participants) | 3
  Face oedema,Week 46 | 0.00 [0.00 to 70.76]
  Face oedema,Week 47: number analyzed (Participants) | 19
  Face oedema,Week 47 | 0.00 [0.00 to 17.65]
  Face oedema,Week 48: number analyzed (Participants) | 25
  Face oedema,Week 48 | 0.00 [0.00 to 13.72]
  Face oedema,Week 49: number analyzed (Participants) | 34
  Face oedema,Week 49 | 0.00 [0.00 to 10.28]
  Face oedema,Week 50: number analyzed (Participants) | 42
  Face oedema,Week 50 | 0.00 [0.00 to 8.41]
  Face oedema,Week 51: number analyzed (Participants) | 12
  Face oedema,Week 51 | 0.00 [0.00 to 26.46]
  Face oedema,Week 52: number analyzed (Participants) | 4
  Face oedema,Week 52 | 0.00 [0.00 to 60.24]
  Fatigue,Week 46: number analyzed (Participants) | 3
  Fatigue,Week 46 | 0.00 [0.00 to 70.76]
  Fatigue,Week 47: number analyzed (Participants) | 19
  Fatigue,Week 47 | 0.00 [0.00 to 17.65]
  Fatigue,Week 48: number analyzed (Participants) | 25
  Fatigue,Week 48 | 0.00 [0.00 to 13.72]
  Fatigue,Week 49: number analyzed (Participants) | 34
  Fatigue,Week 49 | 0.00 [0.00 to 10.28]
  Fatigue,Week 50: number analyzed (Participants) | 42
  Fatigue,Week 50 | 0.00 [0.00 to 8.41]
  Fatigue,Week 51: number analyzed (Participants) | 12
  Fatigue,Week 51 | 8.33 [0.21 to 38.48]
  Fatigue,Week 52: number analyzed (Participants) | 4
  Fatigue,Week 52 | 0.00 [0.00 to 60.24]
  Injection site erythema,Week 46: number analyzed (Participants) | 3
  Injection site erythema,Week 46 | 0.00 [0.00 to 70.76]
  Injection site erythema,Week 47: number analyzed (Participants) | 19
  Injection site erythema,Week 47 | 0.00 [0.00 to 17.65]
  Injection site erythema,Week 48: number analyzed (Participants) | 25
  Injection site erythema,Week 48 | 0.00 [0.00 to 13.72]
  Injection site erythema,Week 49: number analyzed (Participants) | 34
  Injection site erythema,Week 49 | 0.00 [0.00 to 10.28]
  Injection site erythema,Week 50: number analyzed (Participants) | 42
  Injection site erythema,Week 50 | 0.00 [0.00 to 8.41]
  Injection site erythema,Week 51: number analyzed (Participants) | 12
  Injection site erythema,Week 51 | 0.00 [0.00 to 26.46]
  Injection site erythema,Week 52: number analyzed (Participants) | 4
  Injection site erythema,Week 52 | 0.00 [0.00 to 60.24]
  Injection site pain,Week 46: number analyzed (Participants) | 3
  Injection site pain,Week 46 | 0.00 [0.00 to 70.76]
  Injection site pain,Week 47: number analyzed (Participants) | 19
  Injection site pain,Week 47 | 31.58 [0.00 to 99.96]
  Injection site pain,Week 48: number analyzed (Participants) | 25
  Injection site pain,Week 48 | 4.00 [0.10 to 20.35]
  Injection site pain,Week 49: number analyzed (Participants) | 34
  Injection site pain,Week 49 | 0.00 [0.00 to 10.28]
  Injection site pain,Week 50: number analyzed (Participants) | 42
  Injection site pain,Week 50 | 0.00 [0.00 to 8.41]
  Injection site pain,Week 51: number analyzed (Participants) | 12
  Injection site pain,Week 51 | 0.00 [0.00 to 26.46]
  Injection site pain,Week 52: number analyzed (Participants) | 4
  Injection site pain,Week 52 | 0.00 [0.00 to 60.24]
  Injection site swelling,Week 46: number analyzed (Participants) | 3
  Injection site swelling,Week 46 | 0.00 [0.00 to 70.76]
  Injection site swelling,Week 47: number analyzed (Participants) | 19
  Injection site swelling,Week 47 | 0.00 [0.00 to 17.65]
  Injection site swelling,Week 48: number analyzed (Participants) | 25
  Injection site swelling,Week 48 | 0.00 [0.00 to 13.72]
  Injection site swelling,Week 49: number analyzed (Participants) | 34
  Injection site swelling,Week 49 | 0.00 [0.00 to 10.28]
  Injection site swelling,Week 50: number analyzed (Participants) | 42
  Injection site swelling,Week 50 | 0.00 [0.00 to 8.41]
  Injection site swelling,Week 51: number analyzed (Participants) | 12
  Injection site swelling,Week 51 | 0.00 [0.00 to 26.46]
  Injection site swelling,Week 52: number analyzed (Participants) | 4
  Injection site swelling,Week 52 | 0.00 [0.00 to 60.24]
  Pyrexia,Week 46: number analyzed (Participants) | 3
  Pyrexia,Week 46 | 0.00 [0.00 to 70.76]
  Pyrexia,Week 47: number analyzed (Participants) | 19
  Pyrexia,Week 47 | 10.53 [0.00 to 99.89]
  Pyrexia,Week 48: number analyzed (Participants) | 25
  Pyrexia,Week 48 | 4.00 [0.10 to 20.35]
  Pyrexia,Week 49: number analyzed (Participants) | 34
  Pyrexia,Week 49 | 2.94 [0.07 to 15.33]
  Pyrexia,Week 50: number analyzed (Participants) | 42
  Pyrexia,Week 50 | 4.76 [0.58 to 16.16]
  Pyrexia,Week 51: number analyzed (Participants) | 12
  Pyrexia,Week 51 | 0.00 [0.00 to 26.46]
  Pyrexia,Week 52: number analyzed (Participants) | 4
  Pyrexia,Week 52 | 25.00 [0.63 to 80.59]

7. Secondary Outcome: Weekly Percentage of Subjects Reporting Immune System Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were anaphylactic reaction and hypersensitivity.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Anaphylactic reaction,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Anaphylactic reaction,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Anaphylactic reaction,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Anaphylactic reaction,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Anaphylactic reaction,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Anaphylactic reaction,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Anaphylactic reaction,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Anaphylactic reaction,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Anaphylactic reaction,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Anaphylactic reaction,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Anaphylactic reaction,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Anaphylactic reaction,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Anaphylactic reaction,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Anaphylactic reaction,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Anaphylactic reaction,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Anaphylactic reaction,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Anaphylactic reaction,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Anaphylactic reaction,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Hypersensitivity,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hypersensitivity,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Hypersensitivity,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Hypersensitivity,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Hypersensitivity,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Hypersensitivity,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Hypersensitivity,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Hypersensitivity,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Hypersensitivity,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Hypersensitivity,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Hypersensitivity,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Hypersensitivity,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Hypersensitivity,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Hypersensitivity,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Hypersensitivity,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Hypersensitivity,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Hypersensitivity,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Hypersensitivity,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

8. Secondary Outcome: Weekly Percentage of Subjects Reporting Immune System Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: as for outcome 2
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

9. Secondary Outcome: Weekly Percentage of Subjects Reporting Infections and Infestations by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were conjunctivitis and rhinitis.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 8.57 [0.31 to 37.07] |  | 8.57 [0.31 to 37.07]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 8.79 [0.32 to 37.74] |  | 8.79 [0.32 to 37.74]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.71 [0.01 to 4.40] | 4.65 [0.00 to 74.17] | 1.92 [0.05 to 10.26] | 1.69 [0.24 to 5.71]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 6.45 [0.79 to 21.42] | 7.69 [0.19 to 36.03] | 5.13 [0.75 to 16.35] | 5.74 [2.34 to 11.46]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 8.33 [1.75 to 22.47] | 6.67 [0.17 to 31.95] | 6.15 [0.05 to 35.17] | 6.90 [2.81 to 13.71]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 9.46 [0.00 to 69.82] | 11.11 [1.38 to 34.71] | 5.81 [0.09 to 30.59] | 7.29 [3.51 to 13.08]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 3.85 [0.10 to 19.64] | 7.69 [0.95 to 25.13] | 8.96 [1.32 to 27.23] | 7.56 [3.17 to 14.77]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 15.00 [0.01 to 81.57] | 9.30 [1.44 to 27.75]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  Conjunctivitis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Conjunctivitis,Week 40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Conjunctivitis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Conjunctivitis,Week 41 |  | 3.30 [0.00 to 27.97] |  | 3.30 [0.00 to 27.97]
  Conjunctivitis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Conjunctivitis,Week 42 | 0.71 [0.01 to 4.40] | 4.65 [0.00 to 74.17] | 0.00 [0.00 to 6.85] | 1.27 [0.07 to 5.72]
  Conjunctivitis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Conjunctivitis,Week 43 | 3.23 [0.08 to 16.70] | 7.69 [0.19 to 36.03] | 1.28 [0.03 to 6.94] | 2.46 [0.33 to 8.30]
  Conjunctivitis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Conjunctivitis,Week 44 | 5.56 [0.00 to 65.52] | 0.00 [0.00 to 21.80] | 1.54 [0.00 to 49.55] | 2.59 [0.11 to 12.18]
  Conjunctivitis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Conjunctivitis,Week 45 | 8.11 [0.00 to 83.19] | 0.00 [0.00 to 18.53] | 3.23 [0.09 to 16.57] | 4.45 [1.83 to 8.91]
  Conjunctivitis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Conjunctivitis,Week 46 | 3.85 [0.10 to 19.64] | 7.69 [0.95 to 25.13] | 5.97 [0.87 to 18.86] | 5.88 [2.40 to 11.74]
  Conjunctivitis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Conjunctivitis,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 4.65 [0.57 to 15.81]
  Conjunctivitis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Conjunctivitis,Week 48 |  |  | 6.25 [0.00 to 89.64] | 6.25 [0.00 to 89.64]
  Rhinitis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rhinitis,Week 40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Rhinitis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Rhinitis,Week 41 |  | 6.59 [0.04 to 39.62] |  | 6.59 [0.04 to 39.62]
  Rhinitis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Rhinitis,Week 42 | 0.71 [0.01 to 4.40] | 2.33 [0.00 to 47.90] | 1.92 [0.05 to 10.26] | 1.27 [0.26 to 3.67]
  Rhinitis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Rhinitis,Week 43 | 3.23 [0.08 to 16.70] | 0.00 [0.00 to 24.71] | 2.56 [0.31 to 8.96] | 2.46 [0.51 to 7.02]
  Rhinitis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Rhinitis,Week 44 | 5.56 [0.00 to 98.06] | 6.67 [0.17 to 31.95] | 3.08 [0.00 to 24.91] | 4.31 [0.97 to 11.71]
  Rhinitis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Rhinitis,Week 45 | 2.70 [0.00 to 39.00] | 11.11 [1.38 to 34.71] | 2.58 [0.00 to 28.73] | 3.24 [0.81 to 8.44]
  Rhinitis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Rhinitis,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 4.48 [0.34 to 17.63] | 2.52 [0.20 to 10.12]
  Rhinitis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Rhinitis,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.98] | 2.33 [0.00 to 27.06]
  Rhinitis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Rhinitis,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Bronchitis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Bronchitis,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Bronchitis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Bronchitis,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Bronchitis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Bronchitis,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Bronchitis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Bronchitis,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Bronchitis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Bronchitis,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 1.54 [0.04 to 8.28] | 0.86 [0.02 to 4.71]
  Bronchitis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Bronchitis,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Bronchitis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Bronchitis,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Bronchitis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Bronchitis,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Bronchitis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Bronchitis,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Ear infection,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear infection,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear infection,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Ear infection,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Ear infection,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Ear infection,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Ear infection,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Ear infection,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Ear infection,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Ear infection,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 1.54 [0.04 to 8.28] | 0.86 [0.02 to 4.71]
  Ear infection,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Ear infection,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Ear infection,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Ear infection,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Ear infection,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Ear infection,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Ear infection,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Ear infection,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Herpes simplex,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Herpes simplex,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Herpes simplex,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Herpes simplex,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Herpes simplex,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Herpes simplex,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Herpes simplex,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Herpes simplex,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Herpes simplex,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Herpes simplex,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Herpes simplex,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Herpes simplex,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Herpes simplex,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Herpes simplex,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Herpes simplex,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Herpes simplex,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Herpes simplex,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Herpes simplex,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Hordeolum,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hordeolum,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Hordeolum,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Hordeolum,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Hordeolum,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Hordeolum,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Hordeolum,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Hordeolum,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Hordeolum,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Hordeolum,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Hordeolum,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Hordeolum,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Hordeolum,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Hordeolum,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Hordeolum,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Hordeolum,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 2.33 [0.00 to 25.06]
  Hordeolum,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Hordeolum,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Laryngitis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Laryngitis,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Laryngitis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Laryngitis,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Laryngitis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Laryngitis,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Laryngitis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Laryngitis,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Laryngitis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Laryngitis,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Laryngitis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Laryngitis,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 19.47] | 0.40 [0.00 to 4.07]
  Laryngitis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Laryngitis,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Laryngitis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Laryngitis,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Laryngitis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Laryngitis,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Nasopharyngitis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Nasopharyngitis,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Nasopharyngitis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Nasopharyngitis,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Nasopharyngitis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Nasopharyngitis,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Nasopharyngitis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Nasopharyngitis,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Nasopharyngitis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Nasopharyngitis,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Nasopharyngitis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Nasopharyngitis,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Nasopharyngitis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Nasopharyngitis,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Nasopharyngitis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Nasopharyngitis,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Nasopharyngitis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Nasopharyngitis,Week 48 |  |  | 6.25 [0.00 to 100] | 6.25 [0.00 to 100]
  Oral herpes,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Oral herpes,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Oral herpes,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Oral herpes,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Oral herpes,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Oral herpes,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Oral herpes,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Oral herpes,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Oral herpes,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Oral herpes,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Oral herpes,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Oral herpes,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Oral herpes,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Oral herpes,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Oral herpes,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Oral herpes,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Oral herpes,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Oral herpes,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Upper respiratory tract infection,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Upper respiratory tract infection,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Upper respiratory tract infection,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Upper respiratory tract infection,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Upper respiratory tract infection,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Upper respiratory tract infection,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Upper respiratory tract infection,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Upper respiratory tract infection,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 1.28 [0.03 to 6.94] | 0.82 [0.02 to 4.48]
  Upper respiratory tract infection,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Upper respiratory tract infection,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Upper respiratory tract infection,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Upper respiratory tract infection,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Upper respiratory tract infection,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Upper respiratory tract infection,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Upper respiratory tract infection,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Upper respiratory tract infection,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Upper respiratory tract infection,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Upper respiratory tract infection,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

10. Secondary Outcome: Weekly Percentage of Subjects Reporting Infections and Infestations by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were conjunctivitis and rhinitis.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 0.00 [0.00 to 17.65]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 12.00 [2.55 to 31.22]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 0.00 [0.00 to 10.28]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 2.38 [0.06 to 12.57]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 0.00 [0.00 to 26.46]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Conjunctivitis,Week 46: number analyzed (Participants) | 3
  Conjunctivitis,Week 46 | 0.00 [0.00 to 70.76]
  Conjunctivitis,Week 47: number analyzed (Participants) | 19
  Conjunctivitis,Week 47 | 0.00 [0.00 to 17.65]
  Conjunctivitis,Week 48: number analyzed (Participants) | 25
  Conjunctivitis,Week 48 | 8.00 [0.98 to 26.03]
  Conjunctivitis,Week 49: number analyzed (Participants) | 34
  Conjunctivitis,Week 49 | 0.00 [0.00 to 10.28]
  Conjunctivitis,Week 50: number analyzed (Participants) | 42
  Conjunctivitis,Week 50 | 2.38 [0.06 to 12.57]
  Conjunctivitis,Week 51: number analyzed (Participants) | 12
  Conjunctivitis,Week 51 | 0.00 [0.00 to 26.46]
  Conjunctivitis,Week 52: number analyzed (Participants) | 4
  Conjunctivitis,Week 52 | 0.00 [0.00 to 60.24]
  Rhinitis,Week 46: number analyzed (Participants) | 3
  Rhinitis,Week 46 | 0.00 [0.00 to 70.76]
  Rhinitis,Week 47: number analyzed (Participants) | 19
  Rhinitis,Week 47 | 0.00 [0.00 to 17.65]
  Rhinitis,Week 48: number analyzed (Participants) | 25
  Rhinitis,Week 48 | 4.00 [0.10 to 20.35]
  Rhinitis,Week 49: number analyzed (Participants) | 34
  Rhinitis,Week 49 | 0.00 [0.00 to 10.28]
  Rhinitis,Week 50: number analyzed (Participants) | 42
  Rhinitis,Week 50 | 0.00 [0.00 to 8.41]
  Rhinitis,Week 51: number analyzed (Participants) | 12
  Rhinitis,Week 51 | 0.00 [0.00 to 26.46]
  Rhinitis,Week 52: number analyzed (Participants) | 4
  Rhinitis,Week 52 | 0.00 [0.00 to 60.24]

11. Secondary Outcome: Weekly Percentage of Subjects Reporting Metabolism and Nutrition Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card was decreased appetite.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 1.10 [0.00 to 20.56] |  | 1.10 [0.00 to 20.56]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 8.22] | 3.85 [0.11 to 19.24] | 1.27 [0.12 to 4.95]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 11.54 [1.53 to 35.14] | 7.38 [0.30 to 31.94]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 7.69 [2.54 to 17.05] | 5.17 [1.92 to 10.92]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 4.05 [0.00 to 53.08] | 0.00 [0.00 to 18.53] | 3.87 [0.00 to 38.62] | 3.64 [0.66 to 10.89]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 2.33 [0.03 to 14.14]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  Decreased appetite,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Decreased appetite,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Decreased appetite,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Decreased appetite,Week 41 |  | 1.10 [0.00 to 20.56] |  | 1.10 [0.00 to 20.56]
  Decreased appetite,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Decreased appetite,Week 42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 8.22] | 3.85 [0.11 to 19.24] | 1.27 [0.12 to 4.95]
  Decreased appetite,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Decreased appetite,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 11.54 [1.53 to 35.14] | 7.38 [0.30 to 31.94]
  Decreased appetite,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Decreased appetite,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 7.69 [2.54 to 17.05] | 5.17 [1.92 to 10.92]
  Decreased appetite,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Decreased appetite,Week 45 | 4.05 [0.00 to 53.08] | 0.00 [0.00 to 18.53] | 3.87 [0.00 to 38.62] | 3.64 [0.66 to 10.89]
  Decreased appetite,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Decreased appetite,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Decreased appetite,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Decreased appetite,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 2.33 [0.03 to 14.14]
  Decreased appetite,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Decreased appetite,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]

12. Secondary Outcome: Weekly Percentage of Subjects Reporting Metabolism and Nutrition Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card was decreased appetite.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 5.26 [0.00 to 95.26]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 4.00 [0.10 to 20.35]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 0.00 [0.00 to 10.28]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 2.38 [0.06 to 12.57]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 0.00 [0.00 to 26.46]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Decreased appetite,Week 46: number analyzed (Participants) | 3
  Decreased appetite,Week 46 | 0.00 [0.00 to 70.76]
  Decreased appetite,Week 47: number analyzed (Participants) | 19
  Decreased appetite,Week 47 | 5.26 [0.00 to 95.26]
  Decreased appetite,Week 48: number analyzed (Participants) | 25
  Decreased appetite,Week 48 | 4.00 [0.10 to 20.35]
  Decreased appetite,Week 49: number analyzed (Participants) | 34
  Decreased appetite,Week 49 | 0.00 [0.00 to 10.28]
  Decreased appetite,Week 50: number analyzed (Participants) | 42
  Decreased appetite,Week 50 | 2.38 [0.06 to 12.57]
  Decreased appetite,Week 51: number analyzed (Participants) | 12
  Decreased appetite,Week 51 | 0.00 [0.00 to 26.46]
  Decreased appetite,Week 52: number analyzed (Participants) | 4
  Decreased appetite,Week 52 | 0.00 [0.00 to 60.24]

13. Secondary Outcome: Weekly Percentage of Subjects Reporting Musculoskeletal and Connective Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were arthropathy and myalgia.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 7.69 [0.00 to 71.12] |  | 7.69 [0.00 to 71.12]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 11.35 [0.10 to 56.46] | 2.33 [0.00 to 47.90] | 7.69 [0.19 to 36.17] | 8.90 [3.78 to 17.15]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 23.08 [5.04 to 53.81] | 7.69 [1.08 to 24.10] | 7.38 [1.08 to 22.89]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 19.44 [0.05 to 83.92] | 6.67 [0.17 to 31.95] | 3.08 [0.00 to 72.80] | 8.62 [0.56 to 32.97]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 10.81 [0.08 to 55.52] | 16.67 [3.58 to 41.42] | 8.39 [0.37 to 34.98] | 9.72 [5.35 to 15.89]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 11.54 [2.45 to 30.15] | 15.38 [4.36 to 34.87] | 8.96 [1.32 to 27.23] | 10.92 [5.95 to 17.96]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 4.65 [0.57 to 15.81]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 37.50 [0.00 to 100] | 37.50 [0.00 to 100]
  Arthropathy,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Arthropathy,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Arthropathy,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Arthropathy,Week 41 |  | 2.20 [0.00 to 37.37] |  | 2.20 [0.00 to 37.37]
  Arthropathy,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Arthropathy,Week 42 | 1.42 [0.02 to 8.68] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 1.27 [0.26 to 3.67]
  Arthropathy,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Arthropathy,Week 43 | 0.00 [0.00 to 11.22] | 15.38 [1.92 to 45.45] | 0.00 [0.00 to 4.62] | 1.64 [0.00 to 25.52]
  Arthropathy,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Arthropathy,Week 44 | 13.89 [0.70 to 50.99] | 0.00 [0.00 to 21.80] | 1.54 [0.00 to 47.01] | 5.17 [0.23 to 22.97]
  Arthropathy,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Arthropathy,Week 45 | 2.70 [0.00 to 85.98] | 11.11 [1.38 to 34.71] | 3.23 [0.09 to 16.57] | 3.64 [1.29 to 7.95]
  Arthropathy,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Arthropathy,Week 46 | 3.85 [0.10 to 19.64] | 7.69 [0.95 to 25.13] | 1.49 [0.04 to 8.04] | 3.36 [0.80 to 8.99]
  Arthropathy,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Arthropathy,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 4.65 [0.57 to 15.81]
  Arthropathy,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Arthropathy,Week 48 |  |  | 18.75 [0.00 to 99.99] | 18.75 [0.00 to 99.99]
  Myalgia,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Myalgia,Week 40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Myalgia,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Myalgia,Week 41 |  | 5.49 [0.00 to 52.38] |  | 5.49 [0.00 to 52.38]
  Myalgia,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Myalgia,Week 42 | 9.93 [0.09 to 50.96] | 0.00 [0.00 to 8.22] | 7.69 [0.19 to 36.17] | 7.63 [2.78 to 16.09]
  Myalgia,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Myalgia,Week 43 | 0.00 [0.00 to 11.22] | 7.69 [0.19 to 36.03] | 6.41 [0.92 to 20.26] | 4.92 [0.74 to 15.51]
  Myalgia,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Myalgia,Week 44 | 8.33 [1.75 to 22.47] | 6.67 [0.17 to 31.95] | 1.54 [0.00 to 47.01] | 4.31 [0.36 to 16.52]
  Myalgia,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Myalgia,Week 45 | 9.46 [0.00 to 69.82] | 11.11 [1.38 to 34.71] | 6.45 [0.15 to 31.44] | 7.69 [3.98 to 13.17]
  Myalgia,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Myalgia,Week 46 | 11.54 [2.45 to 30.15] | 7.69 [0.95 to 25.13] | 7.46 [1.19 to 22.48] | 8.40 [4.10 to 14.91]
  Myalgia,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Myalgia,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 2.33 [0.00 to 25.06]
  Myalgia,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Myalgia,Week 48 |  |  | 31.25 [0.00 to 100] | 31.25 [0.00 to 100]
  Limb discomfort,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Limb discomfort,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Limb discomfort,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Limb discomfort,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Limb discomfort,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Limb discomfort,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Limb discomfort,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Limb discomfort,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Limb discomfort,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Limb discomfort,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Limb discomfort,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Limb discomfort,Week 45 | 0.00 [0.00 to 4.86] | 5.56 [0.14 to 27.29] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 4.05]
  Limb discomfort,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Limb discomfort,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Limb discomfort,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Limb discomfort,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Limb discomfort,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Limb discomfort,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Musculoskeletal pain,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Musculoskeletal pain,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Musculoskeletal pain,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Musculoskeletal pain,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Musculoskeletal pain,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Musculoskeletal pain,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Musculoskeletal pain,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Musculoskeletal pain,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Musculoskeletal pain,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Musculoskeletal pain,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Musculoskeletal pain,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Musculoskeletal pain,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Musculoskeletal pain,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Musculoskeletal pain,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Musculoskeletal pain,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Musculoskeletal pain,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Musculoskeletal pain,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Musculoskeletal pain,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Pain in extremity,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pain in extremity,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Pain in extremity,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Pain in extremity,Week 41 |  | 1.10 [0.00 to 20.56] |  | 1.10 [0.00 to 20.56]
  Pain in extremity,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Pain in extremity,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Pain in extremity,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Pain in extremity,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 1.28 [0.03 to 6.94] | 0.82 [0.02 to 4.48]
  Pain in extremity,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Pain in extremity,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Pain in extremity,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Pain in extremity,Week 45 | 0.00 [0.00 to 4.86] | 5.56 [0.14 to 27.29] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 4.05]
  Pain in extremity,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Pain in extremity,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Pain in extremity,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Pain in extremity,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Pain in extremity,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Pain in extremity,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Rheumatic disorder,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rheumatic disorder,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Rheumatic disorder,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Rheumatic disorder,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Rheumatic disorder,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Rheumatic disorder,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Rheumatic disorder,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Rheumatic disorder,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Rheumatic disorder,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Rheumatic disorder,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Rheumatic disorder,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Rheumatic disorder,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Rheumatic disorder,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Rheumatic disorder,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Rheumatic disorder,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Rheumatic disorder,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Rheumatic disorder,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Rheumatic disorder,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Synovial cyst,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Synovial cyst,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Synovial cyst,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Synovial cyst,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Synovial cyst,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Synovial cyst,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Synovial cyst,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Synovial cyst,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Synovial cyst,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Synovial cyst,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 1.54 [0.00 to 47.01] | 0.86 [0.00 to 8.91]
  Synovial cyst,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Synovial cyst,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Synovial cyst,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Synovial cyst,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Synovial cyst,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Synovial cyst,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Synovial cyst,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Synovial cyst,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

14. Secondary Outcome: Weekly Percentage of Subjects Reporting Musculoskeletal and Connective Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were arthropathy and myalgia.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 5.26 [0.00 to 95.26]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 0.00 [0.00 to 13.72]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 0.00 [0.00 to 10.28]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 0.00 [0.00 to 8.41]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 0.00 [0.00 to 26.46]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Arthropathy,Week 46: number analyzed (Participants) | 3
  Arthropathy,Week 46 | 0.00 [0.00 to 70.76]
  Arthropathy,Week 47: number analyzed (Participants) | 19
  Arthropathy,Week 47 | 0.00 [0.00 to 17.65]
  Arthropathy,Week 48: number analyzed (Participants) | 25
  Arthropathy,Week 48 | 0.00 [0.00 to 13.72]
  Arthropathy,Week 49: number analyzed (Participants) | 34
  Arthropathy,Week 49 | 0.00 [0.00 to 10.28]
  Arthropathy,Week 50: number analyzed (Participants) | 42
  Arthropathy,Week 50 | 0.00 [0.00 to 8.41]
  Arthropathy,Week 51: number analyzed (Participants) | 12
  Arthropathy,Week 51 | 0.00 [0.00 to 26.46]
  Arthropathy,Week 52: number analyzed (Participants) | 4
  Arthropathy,Week 52 | 0.00 [0.00 to 60.24]
  Myalgia,Week 46: number analyzed (Participants) | 3
  Myalgia,Week 46 | 0.00 [0.00 to 70.76]
  Myalgia,Week 47: number analyzed (Participants) | 19
  Myalgia,Week 47 | 5.26 [0.00 to 95.26]
  Myalgia,Week 48: number analyzed (Participants) | 25
  Myalgia,Week 48 | 0.00 [0.00 to 13.72]
  Myalgia,Week 49: number analyzed (Participants) | 34
  Myalgia,Week 49 | 0.00 [0.00 to 10.28]
  Myalgia,Week 50: number analyzed (Participants) | 42
  Myalgia,Week 50 | 0.00 [0.00 to 8.41]
  Myalgia,Week 51: number analyzed (Participants) | 12
  Myalgia,Week 51 | 0.00 [0.00 to 26.46]
  Myalgia,Week 52: number analyzed (Participants) | 4
  Myalgia,Week 52 | 0.00 [0.00 to 60.24]

15. Secondary Outcome: Weekly Percentage of Subjects Reporting Nervous System Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were febrile convulsion and headache.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 7.69 [0.47 to 30.27] |  | 7.69 [0.47 to 30.27]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 5.67 [0.00 to 68.10] | 4.65 [0.00 to 74.17] | 1.92 [0.05 to 10.26] | 4.66 [2.35 to 8.19]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 9.68 [2.04 to 25.75] | 7.69 [0.19 to 36.03] | 7.69 [1.08 to 24.10] | 8.20 [4.00 to 14.56]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 16.67 [0.00 to 98.03] | 6.67 [0.17 to 31.95] | 1.54 [0.04 to 8.28] | 6.90 [0.53 to 25.99]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 13.51 [0.84 to 47.92] | 11.11 [1.38 to 34.71] | 9.68 [2.09 to 25.51] | 10.93 [7.16 to 15.78]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 15.38 [4.36 to 34.87] | 8.96 [1.32 to 27.23] | 8.40 [2.11 to 21.07]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 50.00 [1.26 to 98.74] | 5.00 [0.00 to 99.71] | 4.65 [0.01 to 34.34]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 37.50 [0.19 to 97.69] | 37.50 [0.19 to 97.69]
  Febrile convulsion,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Febrile convulsion,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Febrile convulsion,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Febrile convulsion,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Febrile convulsion,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Febrile convulsion,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Febrile convulsion,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Febrile convulsion,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Febrile convulsion,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Febrile convulsion,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Febrile convulsion,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Febrile convulsion,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Febrile convulsion,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Febrile convulsion,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Febrile convulsion,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Febrile convulsion,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Febrile convulsion,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Febrile convulsion,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Headache,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Headache,Week 40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Headache,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Headache,Week 41 |  | 7.69 [0.47 to 30.27] |  | 7.69 [0.47 to 30.27]
  Headache,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Headache,Week 42 | 4.96 [0.48 to 18.09] | 4.65 [0.00 to 74.17] | 1.92 [0.05 to 10.26] | 4.24 [2.05 to 7.65]
  Headache,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Headache,Week 43 | 9.68 [2.04 to 25.75] | 7.69 [0.19 to 36.03] | 7.69 [1.08 to 24.10] | 8.20 [4.00 to 14.56]
  Headache,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Headache,Week 44 | 16.67 [0.00 to 98.03] | 6.67 [0.17 to 31.95] | 1.54 [0.04 to 8.28] | 6.90 [0.53 to 25.99]
  Headache,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Headache,Week 45 | 10.81 [3.04 to 25.35] | 11.11 [1.38 to 34.71] | 7.74 [3.11 to 15.48] | 8.91 [5.67 to 13.17]
  Headache,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Headache,Week 46 | 0.00 [0.00 to 13.23] | 15.38 [4.36 to 34.87] | 8.96 [1.32 to 27.23] | 8.40 [2.11 to 21.07]
  Headache,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Headache,Week 47 | 0.00 [0.00 to 16.11] | 50.00 [1.26 to 98.74] | 5.00 [0.00 to 99.71] | 4.65 [0.01 to 34.34]
  Headache,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Headache,Week 48 |  |  | 37.50 [0.19 to 97.69] | 37.50 [0.19 to 97.69]
  Aphonia,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Aphonia,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Aphonia,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Aphonia,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Aphonia,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Aphonia,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Aphonia,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Aphonia,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Aphonia,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Aphonia,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Aphonia,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Aphonia,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 7.91] | 0.40 [0.00 to 2.58]
  Aphonia,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Aphonia,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Aphonia,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Aphonia,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Aphonia,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Aphonia,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Dizziness,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dizziness,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Dizziness,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Dizziness,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Dizziness,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Dizziness,Week 42 | 0.71 [0.00 to 97.40] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.77]
  Dizziness,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Dizziness,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Dizziness,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Dizziness,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Dizziness,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Dizziness,Week 45 | 2.70 [0.00 to 39.00] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 7.91] | 1.21 [0.15 to 4.34]
  Dizziness,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Dizziness,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Dizziness,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Dizziness,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Dizziness,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Dizziness,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Poor quality sleep,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Poor quality sleep,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Poor quality sleep,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Poor quality sleep,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Poor quality sleep,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Poor quality sleep,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Poor quality sleep,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Poor quality sleep,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Poor quality sleep,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Poor quality sleep,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Poor quality sleep,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Poor quality sleep,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Poor quality sleep,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Poor quality sleep,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Poor quality sleep,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Poor quality sleep,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Poor quality sleep,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Poor quality sleep,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Somnolence,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Somnolence,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Somnolence,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Somnolence,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Somnolence,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Somnolence,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Somnolence,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Somnolence,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Somnolence,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Somnolence,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Somnolence,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Somnolence,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 7.91] | 0.40 [0.00 to 2.58]
  Somnolence,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Somnolence,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Somnolence,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Somnolence,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Somnolence,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Somnolence,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Tremor,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tremor,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Tremor,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Tremor,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Tremor,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Tremor,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Tremor,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Tremor,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Tremor,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Tremor,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Tremor,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Tremor,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Tremor,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Tremor,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Tremor,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Tremor,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Tremor,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Tremor,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

16. Secondary Outcome: Weekly Percentage of Subjects Reporting Nervous System Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were febrile convulsion and headache.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

17. Secondary Outcome: Weekly Percentage of Subjects Reporting Psychiatric Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEI listed on the ADR card was irritability.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 9.30 [0.00 to 94.72] | 1.92 [0.05 to 10.26] | 2.12 [0.01 to 14.95]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 7.69 [0.19 to 36.03] | 5.13 [0.75 to 16.35] | 4.10 [0.69 to 12.52]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 24.91] | 2.59 [0.54 to 7.37]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 11.49] | 0.81 [0.10 to 2.89]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 13.23] | 2.99 [0.00 to 47.77] | 2.52 [0.10 to 12.03]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.98] | 2.33 [0.00 to 27.06]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Irritability,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Irritability,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Irritability,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Irritability,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Irritability,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Irritability,Week 42 | 0.00 [0.00 to 2.58] | 6.98 [0.00 to 87.92] | 1.92 [0.05 to 10.26] | 1.69 [0.01 to 11.37]
  Irritability,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Irritability,Week 43 | 0.00 [0.00 to 11.22] | 7.69 [0.19 to 36.03] | 5.13 [0.75 to 16.35] | 4.10 [0.69 to 12.52]
  Irritability,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Irritability,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 24.91] | 2.59 [0.54 to 7.37]
  Irritability,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Irritability,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 11.49] | 0.81 [0.10 to 2.89]
  Irritability,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Irritability,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 13.23] | 2.99 [0.00 to 47.77] | 2.52 [0.10 to 12.03]
  Irritability,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Irritability,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.98] | 2.33 [0.00 to 27.06]
  Irritability,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Irritability,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Insomnia,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Insomnia,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Insomnia,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Insomnia,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Insomnia,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Insomnia,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Insomnia,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Insomnia,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Insomnia,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Insomnia,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Insomnia,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Insomnia,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Insomnia,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Insomnia,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Insomnia,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Insomnia,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Insomnia,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Insomnia,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Mood swings,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Mood swings,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Mood swings,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Mood swings,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Mood swings,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Mood swings,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Mood swings,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Mood swings,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Mood swings,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Mood swings,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 1.54 [0.00 to 47.01] | 0.86 [0.00 to 8.91]
  Mood swings,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Mood swings,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Mood swings,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Mood swings,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Mood swings,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Mood swings,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Mood swings,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Mood swings,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Sleep disorder,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Sleep disorder,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Sleep disorder,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Sleep disorder,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Sleep disorder,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Sleep disorder,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Sleep disorder,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Sleep disorder,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Sleep disorder,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Sleep disorder,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Sleep disorder,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Sleep disorder,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Sleep disorder,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Sleep disorder,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Sleep disorder,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Sleep disorder,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Sleep disorder,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Sleep disorder,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

18. Secondary Outcome: Weekly Percentage of Subjects Reporting Psychiatric Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEI listed on the ADR card was irritability.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 0.00 [0.00 to 17.65]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 8.00 [0.98 to 26.03]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 5.88 [0.01 to 40.78]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 0.00 [0.00 to 8.41]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 0.00 [0.00 to 26.46]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Irritability,Week 46: number analyzed (Participants) | 3
  Irritability,Week 46 | 0.00 [0.00 to 70.76]
  Irritability,Week 47: number analyzed (Participants) | 19
  Irritability,Week 47 | 0.00 [0.00 to 17.65]
  Irritability,Week 48: number analyzed (Participants) | 25
  Irritability,Week 48 | 8.00 [0.98 to 26.03]
  Irritability,Week 49: number analyzed (Participants) | 34
  Irritability,Week 49 | 5.88 [0.01 to 40.78]
  Irritability,Week 50: number analyzed (Participants) | 42
  Irritability,Week 50 | 0.00 [0.00 to 8.41]
  Irritability,Week 51: number analyzed (Participants) | 12
  Irritability,Week 51 | 0.00 [0.00 to 26.46]
  Irritability,Week 52: number analyzed (Participants) | 4
  Irritability,Week 52 | 0.00 [0.00 to 60.24]

19. Secondary Outcome: Weekly Percentage of Subjects Reporting Respiratory, Thoracic and Mediastinal Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were cough, dysphonia, epistaxis, nasal congestion, oropharyngeal pain, rhinorrhoea, and wheezing.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 8.57 [0.31 to 37.07] |  | 8.57 [0.31 to 37.07]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 13.19 [0.09 to 63.62] |  | 13.19 [0.09 to 63.62]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 9.93 [0.87 to 34.53] | 9.30 [0.00 to 94.72] | 26.92 [0.28 to 88.26] | 13.56 [4.50 to 29.03]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 19.35 [7.45 to 37.47] | 23.08 [5.04 to 53.81] | 25.64 [16.42 to 36.79] | 23.77 [16.53 to 32.32]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 25.00 [12.12 to 42.20] | 6.67 [0.17 to 31.95] | 18.46 [8.54 to 32.71] | 18.97 [12.28 to 27.29]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 20.27 [7.81 to 39.06] | 22.22 [6.41 to 47.64] | 21.29 [6.33 to 45.42] | 21.05 [15.27 to 27.84]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 7.69 [0.95 to 25.13] | 7.69 [0.95 to 25.13] | 20.90 [11.92 to 32.57] | 15.13 [6.18 to 29.01]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 84.19] | 30.00 [0.00 to 100] | 18.60 [0.88 to 63.28]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 31.25 [0.00 to 99.95] | 31.25 [0.00 to 99.95]
  Cough,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Cough,Week 40 |  | 7.14 [0.27 to 31.53] |  | 7.14 [0.27 to 31.53]
  Cough,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Cough,Week 41 |  | 2.20 [0.01 to 16.50] |  | 2.20 [0.01 to 16.50]
  Cough,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Cough,Week 42 | 2.84 [0.04 to 16.88] | 4.65 [0.00 to 74.17] | 15.38 [0.28 to 63.30] | 5.93 [0.85 to 18.82]
  Cough,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Cough,Week 43 | 6.45 [0.79 to 21.42] | 0.00 [0.00 to 24.71] | 15.38 [5.28 to 32.08] | 11.48 [3.55 to 25.67]
  Cough,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Cough,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 12.31 [5.47 to 22.82] | 7.76 [2.75 to 16.60]
  Cough,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Cough,Week 45 | 5.41 [0.00 to 64.32] | 11.11 [1.38 to 34.71] | 6.45 [1.05 to 19.50] | 6.48 [3.75 to 10.31]
  Cough,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Cough,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 8.96 [3.36 to 18.48] | 5.04 [0.67 to 16.58]
  Cough,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Cough,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 10.00 [0.00 to 100] | 6.98 [0.30 to 29.98]
  Cough,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Cough,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  Dysphonia,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dysphonia,Week 40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Dysphonia,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Dysphonia,Week 41 |  | 1.10 [0.00 to 21.06] |  | 1.10 [0.00 to 21.06]
  Dysphonia,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Dysphonia,Week 42 | 1.42 [0.02 to 8.68] | 6.98 [0.00 to 87.92] | 3.85 [0.11 to 19.24] | 2.97 [0.61 to 8.45]
  Dysphonia,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Dysphonia,Week 43 | 3.23 [0.08 to 16.70] | 0.00 [0.00 to 24.71] | 2.56 [0.31 to 8.96] | 2.46 [0.51 to 7.02]
  Dysphonia,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Dysphonia,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 1.54 [0.00 to 47.01] | 0.86 [0.00 to 8.91]
  Dysphonia,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Dysphonia,Week 45 | 0.00 [0.00 to 4.86] | 11.11 [1.38 to 34.71] | 2.58 [0.71 to 6.48] | 2.43 [0.55 to 6.66]
  Dysphonia,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Dysphonia,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 1.49 [0.00 to 42.07] | 0.84 [0.00 to 9.95]
  Dysphonia,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Dysphonia,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 2.33 [0.03 to 14.14]
  Dysphonia,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Dysphonia,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Epistaxis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Epistaxis,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Epistaxis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Epistaxis,Week 41 |  | 2.20 [0.01 to 16.50] |  | 2.20 [0.01 to 16.50]
  Epistaxis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Epistaxis,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Epistaxis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Epistaxis,Week 43 | 3.23 [0.08 to 16.70] | 7.69 [0.19 to 36.03] | 0.00 [0.00 to 4.62] | 1.64 [0.00 to 14.48]
  Epistaxis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Epistaxis,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Epistaxis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Epistaxis,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 2.58 [0.01 to 19.41] | 1.62 [0.17 to 5.98]
  Epistaxis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Epistaxis,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Epistaxis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Epistaxis,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Epistaxis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Epistaxis,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Nasal congestion,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Nasal congestion,Week 40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Nasal congestion,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Nasal congestion,Week 41 |  | 2.20 [0.00 to 37.37] |  | 2.20 [0.00 to 37.37]
  Nasal congestion,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Nasal congestion,Week 42 | 2.84 [0.04 to 16.88] | 4.65 [0.00 to 74.17] | 15.38 [0.28 to 63.30] | 5.93 [0.85 to 18.82]
  Nasal congestion,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Nasal congestion,Week 43 | 3.23 [0.08 to 16.70] | 7.69 [0.19 to 36.03] | 7.69 [1.08 to 24.10] | 6.56 [2.69 to 13.00]
  Nasal congestion,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Nasal congestion,Week 44 | 8.33 [0.00 to 99.81] | 6.67 [0.17 to 31.95] | 9.23 [1.68 to 26.07] | 8.62 [4.21 to 15.28]
  Nasal congestion,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Nasal congestion,Week 45 | 2.70 [0.00 to 39.00] | 0.00 [0.00 to 18.53] | 5.16 [1.41 to 12.74] | 4.05 [1.96 to 7.32]
  Nasal congestion,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Nasal congestion,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 8.96 [2.78 to 20.33] | 5.04 [0.28 to 21.29]
  Nasal congestion,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Nasal congestion,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 2.33 [0.00 to 25.06]
  Nasal congestion,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Nasal congestion,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  Oropharyngeal pain,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Oropharyngeal pain,Week 40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Oropharyngeal pain,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Oropharyngeal pain,Week 41 |  | 5.49 [0.00 to 49.36] |  | 5.49 [0.00 to 49.36]
  Oropharyngeal pain,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Oropharyngeal pain,Week 42 | 3.55 [0.04 to 20.80] | 6.98 [0.00 to 87.92] | 1.92 [0.05 to 10.26] | 3.81 [1.76 to 7.12]
  Oropharyngeal pain,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Oropharyngeal pain,Week 43 | 3.23 [0.08 to 16.70] | 0.00 [0.00 to 24.71] | 7.69 [1.08 to 24.10] | 5.74 [1.26 to 15.53]
  Oropharyngeal pain,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Oropharyngeal pain,Week 44 | 2.78 [0.00 to 99.94] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 24.91] | 2.59 [0.40 to 8.31]
  Oropharyngeal pain,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Oropharyngeal pain,Week 45 | 2.70 [0.00 to 39.00] | 11.11 [1.38 to 34.71] | 5.16 [1.79 to 11.30] | 4.86 [2.54 to 8.33]
  Oropharyngeal pain,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Oropharyngeal pain,Week 46 | 3.85 [0.10 to 19.64] | 3.85 [0.10 to 19.64] | 7.46 [0.18 to 35.54] | 5.88 [1.23 to 16.24]
  Oropharyngeal pain,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Oropharyngeal pain,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.71] | 2.33 [0.00 to 25.06]
  Oropharyngeal pain,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Oropharyngeal pain,Week 48 |  |  | 18.75 [0.00 to 99.99] | 18.75 [0.00 to 99.99]
  Rhinorrhoea,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rhinorrhoea,Week 40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Rhinorrhoea,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Rhinorrhoea,Week 41 |  | 6.59 [0.46 to 25.51] |  | 6.59 [0.46 to 25.51]
  Rhinorrhoea,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Rhinorrhoea,Week 42 | 3.55 [0.00 to 90.30] | 6.98 [0.00 to 87.92] | 7.69 [0.19 to 36.17] | 5.08 [1.26 to 13.14]
  Rhinorrhoea,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Rhinorrhoea,Week 43 | 16.13 [5.45 to 33.73] | 0.00 [0.00 to 24.71] | 10.26 [1.39 to 31.54] | 10.66 [4.95 to 19.36]
  Rhinorrhoea,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Rhinorrhoea,Week 44 | 16.67 [6.37 to 32.81] | 0.00 [0.00 to 21.80] | 10.77 [4.44 to 20.94] | 11.21 [6.10 to 18.40]
  Rhinorrhoea,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Rhinorrhoea,Week 45 | 16.22 [8.67 to 26.61] | 11.11 [1.38 to 34.71] | 10.32 [2.41 to 26.28] | 12.15 [7.21 to 18.78]
  Rhinorrhoea,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Rhinorrhoea,Week 46 | 7.69 [0.95 to 25.13] | 3.85 [0.10 to 19.64] | 8.96 [0.58 to 34.08] | 7.56 [3.52 to 13.87]
  Rhinorrhoea,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Rhinorrhoea,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 15.00 [0.00 to 100] | 6.98 [0.00 to 60.43]
  Rhinorrhoea,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Rhinorrhoea,Week 48 |  |  | 18.75 [0.30 to 72.31] | 18.75 [0.30 to 72.31]
  Wheezing,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Wheezing,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Wheezing,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Wheezing,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Wheezing,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Wheezing,Week 42 | 0.71 [0.01 to 4.40] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.85 [0.10 to 3.03]
  Wheezing,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Wheezing,Week 43 | 0.00 [0.00 to 11.22] | 15.38 [1.92 to 45.45] | 0.00 [0.00 to 4.62] | 1.64 [0.00 to 25.52]
  Wheezing,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Wheezing,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 24.91] | 1.72 [0.18 to 6.35]
  Wheezing,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Wheezing,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Wheezing,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Wheezing,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Wheezing,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Wheezing,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Wheezing,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Wheezing,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Dry throat,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dry throat,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Dry throat,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Dry throat,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Dry throat,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Dry throat,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Dry throat,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Dry throat,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Dry throat,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Dry throat,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.86 [0.00 to 7.14]
  Dry throat,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Dry throat,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Dry throat,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Dry throat,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Dry throat,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Dry throat,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Dry throat,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Dry throat,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Dyspnoea,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dyspnoea,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Dyspnoea,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Dyspnoea,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Dyspnoea,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Dyspnoea,Week 42 | 0.00 [0.00 to 2.58] | 4.65 [0.00 to 74.17] | 0.00 [0.00 to 6.85] | 0.85 [0.00 to 8.26]
  Dyspnoea,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Dyspnoea,Week 43 | 0.00 [0.00 to 11.22] | 7.69 [0.19 to 36.03] | 0.00 [0.00 to 4.62] | 0.82 [0.00 to 13.55]
  Dyspnoea,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Dyspnoea,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Dyspnoea,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Dyspnoea,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Dyspnoea,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Dyspnoea,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Dyspnoea,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Dyspnoea,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Dyspnoea,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Dyspnoea,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Increased upper airway secretion,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Increased upper airway secretion,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Increased upper airway secretion,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Increased upper airway secretion,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Increased upper airway secretion,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Increased upper airway secretion,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Increased upper airway secretion,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Increased upper airway secretion,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 1.28 [0.03 to 6.94] | 0.82 [0.02 to 4.48]
  Increased upper airway secretion,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Increased upper airway secretion,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Increased upper airway secretion,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Increased upper airway secretion,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Increased upper airway secretion,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Increased upper airway secretion,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Increased upper airway secretion,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Increased upper airway secretion,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Increased upper airway secretion,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Increased upper airway secretion,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Sneezing,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Sneezing,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Sneezing,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Sneezing,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Sneezing,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Sneezing,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Sneezing,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Sneezing,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 1.28 [0.03 to 6.94] | 0.82 [0.02 to 4.48]
  Sneezing,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Sneezing,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 1.54 [0.04 to 8.28] | 1.72 [0.21 to 6.09]
  Sneezing,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Sneezing,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Sneezing,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Sneezing,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Sneezing,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Sneezing,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Sneezing,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Sneezing,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Throat clearing,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Throat clearing,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Throat clearing,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Throat clearing,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Throat clearing,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Throat clearing,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Throat clearing,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Throat clearing,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Throat clearing,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Throat clearing,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Throat clearing,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Throat clearing,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Throat clearing,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Throat clearing,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Throat clearing,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Throat clearing,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 5.00 [0.00 to 99.98] | 2.33 [0.00 to 27.06]
  Throat clearing,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Throat clearing,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

20. Secondary Outcome: Weekly Percentage of Subjects Reporting Respiratory, Thoracic and Mediastinal Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were cough, dysphonia, epistaxis, nasal congestion, oropharyngeal pain, rhinorrhoea, and wheezing.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 15.79 [0.00 to 100]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 36.00 [17.97 to 57.48]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 8.82 [0.01 to 58.08]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 4.76 [0.58 to 16.16]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 16.67 [0.00 to 100]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Cough,Week 46: number analyzed (Participants) | 3
  Cough,Week 46 | 0.00 [0.00 to 70.76]
  Cough,Week 47: number analyzed (Participants) | 19
  Cough,Week 47 | 15.79 [0.00 to 100]
  Cough,Week 48: number analyzed (Participants) | 25
  Cough,Week 48 | 20.00 [6.83 to 40.70]
  Cough,Week 49: number analyzed (Participants) | 34
  Cough,Week 49 | 8.82 [0.01 to 58.08]
  Cough,Week 50: number analyzed (Participants) | 42
  Cough,Week 50 | 4.76 [0.58 to 16.16]
  Cough,Week 51: number analyzed (Participants) | 12
  Cough,Week 51 | 0.00 [0.00 to 26.46]
  Cough,Week 52: number analyzed (Participants) | 4
  Cough,Week 52 | 0.00 [0.00 to 60.24]
  Dysphonia,Week 46: number analyzed (Participants) | 3
  Dysphonia,Week 46 | 0.00 [0.00 to 70.76]
  Dysphonia,Week 47: number analyzed (Participants) | 19
  Dysphonia,Week 47 | 5.26 [0.00 to 100]
  Dysphonia,Week 48: number analyzed (Participants) | 25
  Dysphonia,Week 48 | 8.00 [0.98 to 26.03]
  Dysphonia,Week 49: number analyzed (Participants) | 34
  Dysphonia,Week 49 | 0.00 [0.00 to 10.28]
  Dysphonia,Week 50: number analyzed (Participants) | 42
  Dysphonia,Week 50 | 0.00 [0.00 to 8.41]
  Dysphonia,Week 51: number analyzed (Participants) | 12
  Dysphonia,Week 51 | 0.00 [0.00 to 26.46]
  Dysphonia,Week 52: number analyzed (Participants) | 4
  Dysphonia,Week 52 | 0.00 [0.00 to 60.24]
  Epistaxis,Week 46: number analyzed (Participants) | 3
  Epistaxis,Week 46 | 0.00 [0.00 to 70.76]
  Epistaxis,Week 47: number analyzed (Participants) | 19
  Epistaxis,Week 47 | 5.26 [0.00 to 95.26]
  Epistaxis,Week 48: number analyzed (Participants) | 25
  Epistaxis,Week 48 | 0.00 [0.00 to 13.72]
  Epistaxis,Week 49: number analyzed (Participants) | 34
  Epistaxis,Week 49 | 0.00 [0.00 to 10.28]
  Epistaxis,Week 50: number analyzed (Participants) | 42
  Epistaxis,Week 50 | 0.00 [0.00 to 8.41]
  Epistaxis,Week 51: number analyzed (Participants) | 12
  Epistaxis,Week 51 | 0.00 [0.00 to 26.46]
  Epistaxis,Week 52: number analyzed (Participants) | 4
  Epistaxis,Week 52 | 0.00 [0.00 to 60.24]
  Nasal congestion,Week 46: number analyzed (Participants) | 3
  Nasal congestion,Week 46 | 0.00 [0.00 to 70.76]
  Nasal congestion,Week 47: number analyzed (Participants) | 19
  Nasal congestion,Week 47 | 0.00 [0.00 to 17.65]
  Nasal congestion,Week 48: number analyzed (Participants) | 25
  Nasal congestion,Week 48 | 12.00 [2.55 to 31.22]
  Nasal congestion,Week 49: number analyzed (Participants) | 34
  Nasal congestion,Week 49 | 2.94 [0.00 to 67.58]
  Nasal congestion,Week 50: number analyzed (Participants) | 42
  Nasal congestion,Week 50 | 0.00 [0.00 to 8.41]
  Nasal congestion,Week 51: number analyzed (Participants) | 12
  Nasal congestion,Week 51 | 0.00 [0.00 to 26.46]
  Nasal congestion,Week 52: number analyzed (Participants) | 4
  Nasal congestion,Week 52 | 0.00 [0.00 to 60.24]
  Oropharyngeal pain,Week 46: number analyzed (Participants) | 3
  Oropharyngeal pain,Week 46 | 0.00 [0.00 to 70.76]
  Oropharyngeal pain,Week 47: number analyzed (Participants) | 19
  Oropharyngeal pain,Week 47 | 0.00 [0.00 to 17.65]
  Oropharyngeal pain,Week 48: number analyzed (Participants) | 25
  Oropharyngeal pain,Week 48 | 0.00 [0.00 to 13.72]
  Oropharyngeal pain,Week 49: number analyzed (Participants) | 34
  Oropharyngeal pain,Week 49 | 0.00 [0.00 to 10.28]
  Oropharyngeal pain,Week 50: number analyzed (Participants) | 42
  Oropharyngeal pain,Week 50 | 0.00 [0.00 to 8.41]
  Oropharyngeal pain,Week 51: number analyzed (Participants) | 12
  Oropharyngeal pain,Week 51 | 0.00 [0.00 to 26.46]
  Oropharyngeal pain,Week 52: number analyzed (Participants) | 4
  Oropharyngeal pain,Week 52 | 0.00 [0.00 to 60.24]
  Rhinorrhoea,Week 46: number analyzed (Participants) | 3
  Rhinorrhoea,Week 46 | 0.00 [0.00 to 70.76]
  Rhinorrhoea,Week 47: number analyzed (Participants) | 19
  Rhinorrhoea,Week 47 | 5.26 [0.00 to 100]
  Rhinorrhoea,Week 48: number analyzed (Participants) | 25
  Rhinorrhoea,Week 48 | 20.00 [6.83 to 40.70]
  Rhinorrhoea,Week 49: number analyzed (Participants) | 34
  Rhinorrhoea,Week 49 | 5.88 [0.00 to 77.51]
  Rhinorrhoea,Week 50: number analyzed (Participants) | 42
  Rhinorrhoea,Week 50 | 2.38 [0.06 to 12.57]
  Rhinorrhoea,Week 51: number analyzed (Participants) | 12
  Rhinorrhoea,Week 51 | 8.33 [0.00 to 100]
  Rhinorrhoea,Week 52: number analyzed (Participants) | 4
  Rhinorrhoea,Week 52 | 0.00 [0.00 to 60.24]
  Wheezing,Week 46: number analyzed (Participants) | 3
  Wheezing,Week 46 | 0.00 [0.00 to 70.76]
  Wheezing,Week 47: number analyzed (Participants) | 19
  Wheezing,Week 47 | 5.26 [0.00 to 100]
  Wheezing,Week 48: number analyzed (Participants) | 25
  Wheezing,Week 48 | 4.00 [0.10 to 20.35]
  Wheezing,Week 49: number analyzed (Participants) | 34
  Wheezing,Week 49 | 0.00 [0.00 to 10.28]
  Wheezing,Week 50: number analyzed (Participants) | 42
  Wheezing,Week 50 | 0.00 [0.00 to 8.41]
  Wheezing,Week 51: number analyzed (Participants) | 12
  Wheezing,Week 51 | 0.00 [0.00 to 26.46]
  Wheezing,Week 52: number analyzed (Participants) | 4
  Wheezing,Week 52 | 0.00 [0.00 to 60.24]
  Sneezing,Week 46: number analyzed (Participants) | 3
  Sneezing,Week 46 | 0.00 [0.00 to 70.76]
  Sneezing,Week 47: number analyzed (Participants) | 19
  Sneezing,Week 47 | 0.00 [0.00 to 17.65]
  Sneezing,Week 48: number analyzed (Participants) | 25
  Sneezing,Week 48 | 0.00 [0.00 to 13.72]
  Sneezing,Week 49: number analyzed (Participants) | 34
  Sneezing,Week 49 | 0.00 [0.00 to 10.28]
  Sneezing,Week 50: number analyzed (Participants) | 42
  Sneezing,Week 50 | 0.00 [0.00 to 8.41]
  Sneezing,Week 51: number analyzed (Participants) | 12
  Sneezing,Week 51 | 8.33 [0.21 to 38.48]
  Sneezing,Week 52: number analyzed (Participants) | 4
  Sneezing,Week 52 | 0.00 [0.00 to 60.24]

21. Secondary Outcome: Weekly Percentage of Subjects Reporting Skin and Subcutaneous Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were rash and rash generalised.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 1.10 [0.00 to 21.06] |  | 1.10 [0.00 to 21.06]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 3.85 [0.11 to 19.24] | 1.27 [0.02 to 7.52]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 3.23 [0.08 to 16.70] | 7.69 [0.19 to 36.03] | 0.00 [0.00 to 4.62] | 1.64 [0.00 to 14.48]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 28.63] | 1.72 [0.15 to 6.81]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 6.76 [1.90 to 16.31] | 0.00 [0.00 to 18.53] | 1.29 [0.00 to 35.42] | 2.83 [0.20 to 11.67]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Rash,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rash,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Rash,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Rash,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Rash,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Rash,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 1.92 [0.05 to 10.26] | 0.42 [0.00 to 3.83]
  Rash,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Rash,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Rash,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Rash,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 3.08 [0.00 to 28.63] | 1.72 [0.15 to 6.81]
  Rash,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Rash,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 19.47] | 0.81 [0.03 to 3.98]
  Rash,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Rash,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Rash,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Rash,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Rash,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Rash,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Rash generalised,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rash generalised,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Rash generalised,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Rash generalised,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Rash generalised,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Rash generalised,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Rash generalised,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Rash generalised,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Rash generalised,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Rash generalised,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Rash generalised,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Rash generalised,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Rash generalised,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Rash generalised,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Rash generalised,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Rash generalised,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Rash generalised,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Rash generalised,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Erythema,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Erythema,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Erythema,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Erythema,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Erythema,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Erythema,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 1.92 [0.05 to 10.26] | 0.42 [0.00 to 3.83]
  Erythema,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Erythema,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Erythema,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Erythema,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Erythema,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Erythema,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.65 [0.00 to 19.47] | 0.40 [0.00 to 4.07]
  Erythema,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Erythema,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Erythema,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Erythema,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Erythema,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Erythema,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Hyperhidrosis,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hyperhidrosis,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Hyperhidrosis,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Hyperhidrosis,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Hyperhidrosis,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Hyperhidrosis,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Hyperhidrosis,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Hyperhidrosis,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Hyperhidrosis,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Hyperhidrosis,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Hyperhidrosis,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Hyperhidrosis,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Hyperhidrosis,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Hyperhidrosis,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Hyperhidrosis,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Hyperhidrosis,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Hyperhidrosis,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Hyperhidrosis,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Pruritus,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pruritus,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Pruritus,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Pruritus,Week 41 |  | 1.10 [0.00 to 21.06] |  | 1.10 [0.00 to 21.06]
  Pruritus,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Pruritus,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Pruritus,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Pruritus,Week 43 | 3.23 [0.08 to 16.70] | 7.69 [0.19 to 36.03] | 0.00 [0.00 to 4.62] | 1.64 [0.00 to 14.48]
  Pruritus,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Pruritus,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Pruritus,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Pruritus,Week 45 | 2.70 [0.00 to 85.98] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.81 [0.03 to 4.10]
  Pruritus,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Pruritus,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Pruritus,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Pruritus,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Pruritus,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Pruritus,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Pruritus generalised,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pruritus generalised,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Pruritus generalised,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Pruritus generalised,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Pruritus generalised,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Pruritus generalised,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Pruritus generalised,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Pruritus generalised,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Pruritus generalised,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Pruritus generalised,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Pruritus generalised,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Pruritus generalised,Week 45 | 2.70 [0.00 to 39.00] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.81 [0.00 to 5.90]
  Pruritus generalised,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Pruritus generalised,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Pruritus generalised,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Pruritus generalised,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Pruritus generalised,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Pruritus generalised,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

22. Secondary Outcome: Weekly Percentage of Subjects Reporting Skin and Subcutaneous Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were rash and rash generalised.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 0.00 [0.00 to 17.65]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 4.00 [0.10 to 20.35]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 0.00 [0.00 to 10.28]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 0.00 [0.00 to 8.41]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 0.00 [0.00 to 26.46]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Rash,Week 46: number analyzed (Participants) | 3
  Rash,Week 46 | 0.00 [0.00 to 70.76]
  Rash,Week 47: number analyzed (Participants) | 19
  Rash,Week 47 | 0.00 [0.00 to 17.65]
  Rash,Week 48: number analyzed (Participants) | 25
  Rash,Week 48 | 4.00 [0.10 to 20.35]
  Rash,Week 49: number analyzed (Participants) | 34
  Rash,Week 49 | 0.00 [0.00 to 10.28]
  Rash,Week 50: number analyzed (Participants) | 42
  Rash,Week 50 | 0.00 [0.00 to 8.41]
  Rash,Week 51: number analyzed (Participants) | 12
  Rash,Week 51 | 0.00 [0.00 to 26.46]
  Rash,Week 52: number analyzed (Participants) | 4
  Rash,Week 52 | 0.00 [0.00 to 60.24]
  Rash generalised,Week 46: number analyzed (Participants) | 3
  Rash generalised,Week 46 | 0.00 [0.00 to 70.76]
  Rash generalised,Week 47: number analyzed (Participants) | 19
  Rash generalised,Week 47 | 0.00 [0.00 to 17.65]
  Rash generalised,Week 48: number analyzed (Participants) | 25
  Rash generalised,Week 48 | 0.00 [0.00 to 13.72]
  Rash generalised,Week 49: number analyzed (Participants) | 34
  Rash generalised,Week 49 | 0.00 [0.00 to 10.28]
  Rash generalised,Week 50: number analyzed (Participants) | 42
  Rash generalised,Week 50 | 0.00 [0.00 to 8.41]
  Rash generalised,Week 51: number analyzed (Participants) | 12
  Rash generalised,Week 51 | 0.00 [0.00 to 26.46]
  Rash generalised,Week 52: number analyzed (Participants) | 4
  Rash generalised,Week 52 | 0.00 [0.00 to 60.24]

23. Secondary Outcome: Weekly Percentage of Subjects Reporting Cardiac Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for cardiac disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Tachycardia,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tachycardia,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Tachycardia,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Tachycardia,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Tachycardia,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Tachycardia,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Tachycardia,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Tachycardia,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Tachycardia,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Tachycardia,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Tachycardia,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Tachycardia,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Tachycardia,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Tachycardia,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Tachycardia,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Tachycardia,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Tachycardia,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Tachycardia,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

24. Secondary Outcome: Weekly Percentage of Subjects Reporting Cardiac Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for cardiac disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

25. Secondary Outcome: Weekly Percentage of Subjects Reporting Ear and Labyrinth Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for ear and labyrinth disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 2.20 [0.01 to 16.50] |  | 2.20 [0.01 to 16.50]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 1.54 [0.04 to 8.28] | 1.72 [0.21 to 6.09]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 0.00 [0.00 to 4.86] | 11.11 [1.38 to 34.71] | 0.00 [0.00 to 2.35] | 0.81 [0.00 to 7.97]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Ear haemorrhage,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear haemorrhage,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear haemorrhage,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Ear haemorrhage,Week 41 |  | 1.10 [0.00 to 20.56] |  | 1.10 [0.00 to 20.56]
  Ear haemorrhage,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Ear haemorrhage,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Ear haemorrhage,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Ear haemorrhage,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Ear haemorrhage,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Ear haemorrhage,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Ear haemorrhage,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Ear haemorrhage,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Ear haemorrhage,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Ear haemorrhage,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Ear haemorrhage,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Ear haemorrhage,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Ear haemorrhage,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Ear haemorrhage,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Ear pain,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear pain,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear pain,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Ear pain,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Ear pain,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Ear pain,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Ear pain,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Ear pain,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Ear pain,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Ear pain,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 1.54 [0.04 to 8.28] | 0.86 [0.02 to 4.71]
  Ear pain,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Ear pain,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Ear pain,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Ear pain,Week 46 | 0.00 [0.00 to 13.23] | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 5.36] | 0.84 [0.00 to 7.70]
  Ear pain,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Ear pain,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Ear pain,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Ear pain,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Ear pruritus,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear pruritus,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear pruritus,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Ear pruritus,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Ear pruritus,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Ear pruritus,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Ear pruritus,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Ear pruritus,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Ear pruritus,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Ear pruritus,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.86 [0.00 to 7.14]
  Ear pruritus,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Ear pruritus,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Ear pruritus,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Ear pruritus,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Ear pruritus,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Ear pruritus,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Ear pruritus,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Ear pruritus,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Tinnitus,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tinnitus,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Tinnitus,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Tinnitus,Week 41 |  | 1.10 [0.00 to 21.06] |  | 1.10 [0.00 to 21.06]
  Tinnitus,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Tinnitus,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Tinnitus,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Tinnitus,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Tinnitus,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Tinnitus,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Tinnitus,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Tinnitus,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Tinnitus,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Tinnitus,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Tinnitus,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Tinnitus,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Tinnitus,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Tinnitus,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Vertigo,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Vertigo,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Vertigo,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Vertigo,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Vertigo,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Vertigo,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Vertigo,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Vertigo,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Vertigo,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Vertigo,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Vertigo,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Vertigo,Week 45 | 0.00 [0.00 to 4.86] | 11.11 [1.38 to 34.71] | 0.00 [0.00 to 2.35] | 0.81 [0.00 to 7.97]
  Vertigo,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Vertigo,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Vertigo,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Vertigo,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Vertigo,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Vertigo,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

26. Secondary Outcome: Weekly Percentage of Subjects Reporting Ear and Labyrinth Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for ear and labyrinth disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

27. Secondary Outcome: Weekly Percentage of Subjects Reporting Eye Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for eye disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 4.65 [0.00 to 74.17] | 0.00 [0.00 to 6.85] | 0.85 [0.00 to 8.26]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.86 [0.00 to 7.14]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Eye discharge,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Eye discharge,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Eye discharge,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Eye discharge,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Eye discharge,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Eye discharge,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Eye discharge,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Eye discharge,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Eye discharge,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Eye discharge,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Eye discharge,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Eye discharge,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Eye discharge,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Eye discharge,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Eye discharge,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Eye discharge,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Eye discharge,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Eye discharge,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Eye pruritus,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Eye pruritus,Week 40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Eye pruritus,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Eye pruritus,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Eye pruritus,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Eye pruritus,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Eye pruritus,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Eye pruritus,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Eye pruritus,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Eye pruritus,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Eye pruritus,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Eye pruritus,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Eye pruritus,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Eye pruritus,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Eye pruritus,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Eye pruritus,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Eye pruritus,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Eye pruritus,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Lacrimation increased,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Lacrimation increased,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Lacrimation increased,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Lacrimation increased,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Lacrimation increased,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Lacrimation increased,Week 42 | 0.00 [0.00 to 2.58] | 2.33 [0.00 to 47.90] | 0.00 [0.00 to 6.85] | 0.42 [0.00 to 4.20]
  Lacrimation increased,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Lacrimation increased,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Lacrimation increased,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Lacrimation increased,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Lacrimation increased,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Lacrimation increased,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Lacrimation increased,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Lacrimation increased,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Lacrimation increased,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Lacrimation increased,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Lacrimation increased,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Lacrimation increased,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Swelling of eyelid,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Swelling of eyelid,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Swelling of eyelid,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Swelling of eyelid,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Swelling of eyelid,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Swelling of eyelid,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Swelling of eyelid,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Swelling of eyelid,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Swelling of eyelid,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Swelling of eyelid,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.86 [0.00 to 7.14]
  Swelling of eyelid,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Swelling of eyelid,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Swelling of eyelid,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Swelling of eyelid,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Swelling of eyelid,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Swelling of eyelid,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Swelling of eyelid,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Swelling of eyelid,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

28. Secondary Outcome: Weekly Percentage of Subjects Reporting Eye Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for eye disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Week 46: number analyzed (Participants) | 3
  Any,Week 46 | 0.00 [0.00 to 70.76]
  Any,Week 47: number analyzed (Participants) | 19
  Any,Week 47 | 10.53 [0.00 to 99.89]
  Any,Week 48: number analyzed (Participants) | 25
  Any,Week 48 | 0.00 [0.00 to 13.72]
  Any,Week 49: number analyzed (Participants) | 34
  Any,Week 49 | 0.00 [0.00 to 10.28]
  Any,Week 50: number analyzed (Participants) | 42
  Any,Week 50 | 0.00 [0.00 to 8.41]
  Any,Week 51: number analyzed (Participants) | 12
  Any,Week 51 | 0.00 [0.00 to 26.46]
  Any,Week 52: number analyzed (Participants) | 4
  Any,Week 52 | 0.00 [0.00 to 60.24]
  Eye pruritus,Week 46: number analyzed (Participants) | 3
  Eye pruritus,Week 46 | 0.00 [0.00 to 70.76]
  Eye pruritus,Week 47: number analyzed (Participants) | 19
  Eye pruritus,Week 47 | 10.53 [0.00 to 99.89]
  Eye pruritus,Week 48: number analyzed (Participants) | 25
  Eye pruritus,Week 48 | 0.00 [0.00 to 13.72]
  Eye pruritus,Week 49: number analyzed (Participants) | 34
  Eye pruritus,Week 49 | 0.00 [0.00 to 10.28]
  Eye pruritus,Week 50: number analyzed (Participants) | 42
  Eye pruritus,Week 50 | 0.00 [0.00 to 8.41]
  Eye pruritus,Week 51: number analyzed (Participants) | 12
  Eye pruritus,Week 51 | 0.00 [0.00 to 26.46]
  Eye pruritus,Week 52: number analyzed (Participants) | 4
  Eye pruritus,Week 52 | 0.00 [0.00 to 60.24]

29. Secondary Outcome: Weekly Percentage of Subjects Reporting Injury, Poisoning and Procedural Complications by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for injury, poisoning and procedural complications.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 0.00 [0.00 to 4.86] | 5.56 [0.14 to 27.29] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 4.05]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Muscle strain,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Muscle strain,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Muscle strain,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Muscle strain,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Muscle strain,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Muscle strain,Week 42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 1.55]
  Muscle strain,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Muscle strain,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Muscle strain,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Muscle strain,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Muscle strain,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Muscle strain,Week 45 | 0.00 [0.00 to 4.86] | 5.56 [0.14 to 27.29] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 4.05]
  Muscle strain,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Muscle strain,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Muscle strain,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Muscle strain,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Muscle strain,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Muscle strain,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

30. Secondary Outcome: Weekly Percentage of Subjects Reporting Injury, Poisoning and Procedural Complications by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for injury, poisoning and procedural complications.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

31. Secondary Outcome: Weekly Percentage of Subjects Reporting Investigations by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for investigations.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.00 [0.00 to 2.58] | 4.65 [0.00 to 74.17] | 0.00 [0.00 to 6.85] | 0.85 [0.00 to 8.26]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 7.69 [0.19 to 36.03] | 0.00 [0.00 to 4.62] | 0.82 [0.00 to 13.55]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Heart rate increased,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Heart rate increased,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Heart rate increased,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Heart rate increased,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Heart rate increased,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Heart rate increased,Week 42 | 0.00 [0.00 to 2.58] | 4.65 [0.00 to 74.17] | 0.00 [0.00 to 6.85] | 0.85 [0.00 to 8.26]
  Heart rate increased,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Heart rate increased,Week 43 | 0.00 [0.00 to 11.22] | 7.69 [0.19 to 36.03] | 0.00 [0.00 to 4.62] | 0.82 [0.00 to 13.55]
  Heart rate increased,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Heart rate increased,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Heart rate increased,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Heart rate increased,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.40 [0.00 to 2.98]
  Heart rate increased,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Heart rate increased,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Heart rate increased,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Heart rate increased,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Heart rate increased,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Heart rate increased,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

32. Secondary Outcome: Weekly Percentage of Subjects Reporting Investigations by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for investigations.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

33. Secondary Outcome: Weekly Percentage of Subjects Reporting Vascular Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for vascular disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Any,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Any,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Any,Week 42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.42 [0.01 to 2.34]
  Any,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Any,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Any,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Any,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Any,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Any,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Any,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Any,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Any,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Any,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Any,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Any,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  Hot flush,Week 40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hot flush,Week 40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Hot flush,Week 41: number analyzed (Participants) | 0 | 91 | 0 | 91
  Hot flush,Week 41 |  | 0.00 [0.00 to 3.97] |  | 0.00 [0.00 to 3.97]
  Hot flush,Week 42: number analyzed (Participants) | 141 | 43 | 52 | 236
  Hot flush,Week 42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 8.22] | 0.00 [0.00 to 6.85] | 0.42 [0.01 to 2.34]
  Hot flush,Week 43: number analyzed (Participants) | 31 | 13 | 78 | 122
  Hot flush,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 2.98]
  Hot flush,Week 44: number analyzed (Participants) | 36 | 15 | 65 | 116
  Hot flush,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 21.80] | 0.00 [0.00 to 5.52] | 0.00 [0.00 to 3.13]
  Hot flush,Week 45: number analyzed (Participants) | 74 | 18 | 155 | 247
  Hot flush,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 2.35] | 0.00 [0.00 to 1.48]
  Hot flush,Week 46: number analyzed (Participants) | 26 | 26 | 67 | 119
  Hot flush,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 5.36] | 0.00 [0.00 to 3.05]
  Hot flush,Week 47: number analyzed (Participants) | 21 | 2 | 20 | 43
  Hot flush,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 16.84] | 0.00 [0.00 to 8.22]
  Hot flush,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  Hot flush,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]

34. Secondary Outcome: Weekly Percentage of Subjects Reporting Vascular Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for vascular disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

35. Primary Outcome: Cumulative Percentage of Subjects Reporting Any Adverse Events of Interest (AEIs) and/or Adverse Events (AEs) Using Adverse Drug Reaction (ADR) Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between Intenational Organization for Standardization (ISO) weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Week 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Week 40-40 |  | 32.86 [12.23 to 59.90] |  | 32.86 [12.23 to 59.90]
  Week 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Week 40-41 |  | 34.78 [7.27 to 73.22] |  | 34.78 [7.27 to 73.22]
  Week 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Week 40-42 | 45.39 [36.99 to 53.98] | 34.31 [11.18 to 64.77] | 44.23 [0.11 to 99.54] | 39.55 [30.15 to 49.55]
  Week 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Week 40-43 | 45.35 [37.76 to 53.10] | 34.56 [12.27 to 63.37] | 46.15 [14.72 to 80.10] | 41.04 [33.11 to 49.33]
  Week 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Week 40-44 | 47.12 [35.40 to 59.06] | 33.62 [13.15 to 59.93] | 42.56 [35.53 to 49.83] | 40.79 [34.98 to 46.79]
  Week 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Week 40-45 | 43.97 [26.40 to 62.73] | 36.00 [14.36 to 62.87] | 46.29 [24.41 to 69.27] | 42.63 [37.13 to 48.27]
  Week 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Week 40-46 | 42.53 [22.10 to 65.02] | 36.59 [15.78 to 61.90] | 45.08 [28.25 to 62.79] | 41.96 [36.86 to 47.19]
  Week 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Week 40-47 | 42.25 [22.24 to 64.31] | 36.69 [15.84 to 62.00] | 46.22 [25.61 to 67.83] | 42.43 [36.88 to 48.13]
  Week 40-48 | 42.25 [22.24 to 64.31] | 36.69 [15.84 to 62.00] | 47.46 [23.20 to 72.64] | 43.02 [36.81 to 49.39]
  Week 40-49 | 42.25 [22.24 to 64.31] | 36.69 [15.84 to 62.00] | 47.46 [23.20 to 72.64] | 43.02 [36.81 to 49.39]
  Week 40-50 | 42.25 [22.24 to 64.31] | 36.69 [15.84 to 62.00] | 47.46 [23.20 to 72.64] | 43.02 [36.81 to 49.39]
  Week 40-51 | 42.25 [22.24 to 64.31] | 36.69 [15.84 to 62.00] | 47.46 [23.20 to 72.64] | 43.02 [36.81 to 49.39]
  Week 40-52 | 42.25 [22.24 to 64.31] | 36.69 [15.84 to 62.00] | 47.46 [23.20 to 72.64] | 43.02 [36.81 to 49.39]

36. Primary Outcome: Cumulative Percentage of Subjects Reporting Any AEIs and/or AEs Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any, Weeks 40-46: number analyzed (Participants) | 3
  Any, Weeks 40-46 | 33.33 [0.84 to 90.57]
  Any, Weeks 40-47: number analyzed (Participants) | 22
  Any, Weeks 40-47 | 45.45 [0.84 to 76.22]
  Any, Weeks 40-48: number analyzed (Participants) | 47
  Any, Weeks 40-48 | 44.68 [0.84 to 62.55]
  Any, Weeks 40-49: number analyzed (Participants) | 81
  Any, Weeks 40-49 | 30.86 [0.84 to 42.11]
  Any, Weeks 40-50: number analyzed (Participants) | 123
  Any, Weeks 40-50 | 23.58 [0.84 to 32.07]
  Any, Weeks 40-51: number analyzed (Participants) | 135
  Any, Weeks 40-51 | 23.70 [0.84 to 33.21]
  Any, Weeks 40-52 | 23.74 [0.84 to 32.89]

37. Primary Outcome: Cumulative Percentage of Subjects Reporting Gastrointestinal Disorders by MedDRA Preferred Term [PT], Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were diarrhoea, nausea, and vomiting.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 2.48 [0.14 to 10.81] |  | 2.48 [0.14 to 10.81]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 2.13 [0.00 to 57.89] | 4.41 [0.02 to 29.40] | 7.69 [0.19 to 36.17] | 4.03 [1.17 to 9.74]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 3.49 [0.00 to 98.14] | 4.61 [0.02 to 29.48] | 8.46 [3.32 to 17.07] | 5.20 [2.02 to 10.70]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 5.29 [0.00 to 42.00] | 4.74 [0.04 to 28.55] | 7.18 [3.98 to 11.75] | 5.67 [2.98 to 9.67]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 6.38 [0.05 to 37.11] | 5.20 [0.05 to 30.53] | 5.71 [1.68 to 13.59] | 5.78 [3.36 to 9.18]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 6.49 [0.09 to 34.29] | 5.07 [0.11 to 26.00] | 6.47 [4.01 to 9.81] | 6.09 [3.99 to 8.84]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 6.69 [0.14 to 33.10] | 5.04 [0.12 to 25.46] | 6.64 [3.91 to 10.42] | 6.23 [4.13 to 8.96]
  Any,Weeks 40-48 | 6.69 [0.14 to 33.10] | 5.04 [0.12 to 25.46] | 6.84 [4.06 to 10.69] | 6.32 [4.24 to 9.01]
  Any,Weeks 40-49 | 6.69 [0.14 to 33.10] | 5.04 [0.12 to 25.46] | 6.84 [4.06 to 10.69] | 6.32 [4.24 to 9.01]
  Any,Weeks 40-50 | 6.69 [0.14 to 33.10] | 5.04 [0.12 to 25.46] | 6.84 [4.06 to 10.69] | 6.32 [4.24 to 9.01]
  Any,Weeks 40-51 | 6.69 [0.14 to 33.10] | 5.04 [0.12 to 25.46] | 6.84 [4.06 to 10.69] | 6.32 [4.24 to 9.01]
  Any,Weeks 40-52 | 6.69 [0.14 to 33.10] | 5.04 [0.12 to 25.46] | 6.84 [4.06 to 10.69] | 6.32 [4.24 to 9.01]
  Diarrhoea,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Diarrhoea,Weeks 40-40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Diarrhoea,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Diarrhoea,Weeks 40-41 |  | 2.48 [0.14 to 10.81] |  | 2.48 [0.14 to 10.81]
  Diarrhoea,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Diarrhoea,Weeks 40-42 | 0.00 [0.00 to 2.58] | 3.43 [0.09 to 17.62] | 3.85 [0.11 to 19.24] | 2.27 [0.36 to 7.25]
  Diarrhoea,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Diarrhoea,Weeks 40-43 | 1.16 [0.00 to 98.31] | 3.23 [0.16 to 14.35] | 4.62 [0.01 to 34.55] | 2.89 [0.98 to 6.48]
  Diarrhoea,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Diarrhoea,Weeks 40-44 | 1.44 [0.00 to 22.84] | 3.45 [0.18 to 15.24] | 4.10 [1.03 to 10.63] | 2.99 [1.40 to 5.56]
  Diarrhoea,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Diarrhoea,Weeks 40-45 | 1.77 [0.00 to 17.14] | 3.60 [0.21 to 15.27] | 3.71 [0.67 to 11.07] | 3.06 [1.61 to 5.24]
  Diarrhoea,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Diarrhoea,Weeks 40-46 | 1.95 [0.00 to 16.30] | 3.26 [0.40 to 11.22] | 4.08 [1.93 to 7.46] | 3.20 [2.02 to 4.79]
  Diarrhoea,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Diarrhoea,Weeks 40-47 | 1.82 [0.00 to 14.00] | 3.24 [0.42 to 10.98] | 3.89 [2.28 to 6.16] | 3.07 [1.95 to 4.57]
  Diarrhoea,Weeks 40-48 | 1.82 [0.00 to 14.00] | 3.24 [0.42 to 10.98] | 3.97 [2.37 to 6.21] | 3.11 [1.99 to 4.61]
  Diarrhoea,Weeks 40-49 | 1.82 [0.00 to 14.00] | 3.24 [0.42 to 10.98] | 3.97 [2.37 to 6.21] | 3.11 [1.99 to 4.61]
  Diarrhoea,Weeks 40-50 | 1.82 [0.00 to 14.00] | 3.24 [0.42 to 10.98] | 3.97 [2.37 to 6.21] | 3.11 [1.99 to 4.61]
  Diarrhoea,Weeks 40-51 | 1.82 [0.00 to 14.00] | 3.24 [0.42 to 10.98] | 3.97 [2.37 to 6.21] | 3.11 [1.99 to 4.61]
  Diarrhoea,Weeks 40-52 | 1.82 [0.00 to 14.00] | 3.24 [0.42 to 10.98] | 3.97 [2.37 to 6.21] | 3.11 [1.99 to 4.61]
  Nausea,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Nausea,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Nausea,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Nausea,Weeks 40-41 |  | 0.62 [0.00 to 17.42] |  | 0.62 [0.00 to 17.42]
  Nausea,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Nausea,Weeks 40-42 | 2.13 [0.00 to 57.89] | 1.47 [0.00 to 28.09] | 3.85 [0.11 to 19.24] | 2.02 [0.50 to 5.32]
  Nausea,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Nausea,Weeks 40-43 | 2.33 [0.00 to 61.91] | 1.84 [0.00 to 31.06] | 3.08 [0.24 to 12.22] | 2.31 [0.79 to 5.18]
  Nausea,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Nausea,Weeks 40-44 | 3.37 [0.04 to 19.87] | 1.72 [0.00 to 26.54] | 3.08 [1.05 to 6.89] | 2.68 [1.31 to 4.83]
  Nausea,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Nausea,Weeks 40-45 | 3.90 [0.12 to 19.29] | 1.60 [0.00 to 22.17] | 2.29 [0.99 to 4.45] | 2.61 [1.33 to 4.57]
  Nausea,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Nausea,Weeks 40-46 | 3.90 [0.19 to 17.32] | 1.81 [0.00 to 21.35] | 2.88 [0.36 to 9.96] | 2.90 [1.57 to 4.87]
  Nausea,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Nausea,Weeks 40-47 | 4.26 [0.19 to 19.12] | 1.80 [0.00 to 20.98] | 2.97 [0.26 to 11.52] | 3.07 [1.57 to 5.34]
  Nausea,Weeks 40-48 | 4.26 [0.19 to 19.12] | 1.80 [0.00 to 20.98] | 2.87 [0.34 to 10.12] | 3.02 [1.57 to 5.21]
  Nausea,Weeks 40-49 | 4.26 [0.19 to 19.12] | 1.80 [0.00 to 20.98] | 2.87 [0.34 to 10.12] | 3.02 [1.57 to 5.21]
  Nausea,Weeks 40-50 | 4.26 [0.19 to 19.12] | 1.80 [0.00 to 20.98] | 2.87 [0.34 to 10.12] | 3.02 [1.57 to 5.21]
  Nausea,Weeks 40-51 | 4.26 [0.19 to 19.12] | 1.80 [0.00 to 20.98] | 2.87 [0.34 to 10.12] | 3.02 [1.57 to 5.21]
  Nausea,Weeks 40-52 | 4.26 [0.19 to 19.12] | 1.80 [0.00 to 20.98] | 2.87 [0.34 to 10.12] | 3.02 [1.57 to 5.21]
  Vomiting,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Vomiting,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Vomiting,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Vomiting,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Vomiting,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Vomiting,Weeks 40-42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 1.79] | 5.77 [0.15 to 27.99] | 1.01 [0.03 to 5.13]
  Vomiting,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Vomiting,Weeks 40-43 | 1.16 [0.00 to 37.75] | 0.00 [0.00 to 1.69] | 4.62 [0.35 to 18.05] | 1.54 [0.12 to 6.23]
  Vomiting,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Vomiting,Weeks 40-44 | 1.44 [0.04 to 7.62] | 0.00 [0.00 to 1.58] | 4.10 [1.79 to 7.92] | 1.73 [0.39 to 4.82]
  Vomiting,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Vomiting,Weeks 40-45 | 1.77 [0.09 to 8.03] | 0.00 [0.00 to 1.46] | 3.14 [0.82 to 8.06] | 1.81 [0.68 to 3.87]
  Vomiting,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Vomiting,Weeks 40-46 | 1.62 [0.18 to 5.94] | 0.00 [0.00 to 1.33] | 2.88 [0.23 to 11.45] | 1.70 [0.61 to 3.71]
  Vomiting,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Vomiting,Weeks 40-47 | 1.52 [0.25 to 4.80] | 0.00 [0.00 to 1.32] | 2.97 [0.16 to 13.12] | 1.72 [0.61 to 3.80]
  Vomiting,Weeks 40-48 | 1.52 [0.25 to 4.80] | 0.00 [0.00 to 1.32] | 3.09 [0.36 to 10.85] | 1.79 [0.71 to 3.70]
  Vomiting,Weeks 40-49 | 1.52 [0.25 to 4.80] | 0.00 [0.00 to 1.32] | 3.09 [0.36 to 10.85] | 1.79 [0.71 to 3.70]
  Vomiting,Weeks 40-50 | 1.52 [0.25 to 4.80] | 0.00 [0.00 to 1.32] | 3.09 [0.36 to 10.85] | 1.79 [0.71 to 3.70]
  Vomiting,Weeks 40-51 | 1.52 [0.25 to 4.80] | 0.00 [0.00 to 1.32] | 3.09 [0.36 to 10.85] | 1.79 [0.71 to 3.70]
  Vomiting,Weeks 40-52 | 1.52 [0.25 to 4.80] | 0.00 [0.00 to 1.32] | 3.09 [0.36 to 10.85] | 1.79 [0.71 to 3.70]
  Abdominal discomfort,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Abdominal discomfort,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Abdominal discomfort,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Abdominal discomfort,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Abdominal discomfort,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Abdominal discomfort,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Abdominal discomfort,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Abdominal discomfort,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Abdominal discomfort,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Abdominal discomfort,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Abdominal discomfort,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Abdominal discomfort,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.42]
  Abdominal discomfort,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Abdominal discomfort,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.10 [0.00 to 0.70]
  Abdominal discomfort,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Abdominal discomfort,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.10 [0.00 to 0.66]
  Abdominal discomfort,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Abdominal discomfort,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Abdominal discomfort,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Abdominal discomfort,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Abdominal discomfort,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Abdominal pain,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Abdominal pain,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Abdominal pain,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Abdominal pain,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Abdominal pain,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Abdominal pain,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Abdominal pain,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Abdominal pain,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 2.31 [0.18 to 9.24] | 0.58 [0.01 to 3.82]
  Abdominal pain,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Abdominal pain,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 1.54 [0.32 to 4.43] | 0.47 [0.01 to 2.54]
  Abdominal pain,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Abdominal pain,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.86 [0.01 to 5.38] | 0.34 [0.01 to 1.83]
  Abdominal pain,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Abdominal pain,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.72 [0.00 to 6.36] | 0.30 [0.01 to 1.67]
  Abdominal pain,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Abdominal pain,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.69 [0.00 to 6.61] | 0.29 [0.01 to 1.63]
  Abdominal pain,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.66 [0.00 to 6.86] | 0.28 [0.01 to 1.62]
  Abdominal pain,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.66 [0.00 to 6.86] | 0.28 [0.01 to 1.62]
  Abdominal pain,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.66 [0.00 to 6.86] | 0.28 [0.01 to 1.62]
  Abdominal pain,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.66 [0.00 to 6.86] | 0.28 [0.01 to 1.62]
  Abdominal pain,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.66 [0.00 to 6.86] | 0.28 [0.01 to 1.62]
  Gingival bleeding,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Gingival bleeding,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Gingival bleeding,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Gingival bleeding,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Gingival bleeding,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Gingival bleeding,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Gingival bleeding,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Gingival bleeding,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Gingival bleeding,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Gingival bleeding,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Gingival bleeding,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Gingival bleeding,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Gingival bleeding,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Gingival bleeding,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Gingival bleeding,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Gingival bleeding,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Gingival bleeding,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Gingival bleeding,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Gingival bleeding,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Gingival bleeding,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Gingival bleeding,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lip swelling,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Lip swelling,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Lip swelling,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Lip swelling,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Lip swelling,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Lip swelling,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Lip swelling,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Lip swelling,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Lip swelling,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Lip swelling,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Lip swelling,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Lip swelling,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Lip swelling,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Lip swelling,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Lip swelling,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Lip swelling,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Lip swelling,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lip swelling,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lip swelling,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lip swelling,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lip swelling,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Stomatitis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Stomatitis,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Stomatitis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Stomatitis,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Stomatitis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Stomatitis,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Stomatitis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Stomatitis,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Stomatitis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Stomatitis,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Stomatitis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Stomatitis,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Stomatitis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Stomatitis,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Stomatitis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Stomatitis,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Stomatitis,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Stomatitis,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Stomatitis,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Stomatitis,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Stomatitis,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tongue discomfort,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tongue discomfort,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Tongue discomfort,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Tongue discomfort,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Tongue discomfort,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Tongue discomfort,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Tongue discomfort,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Tongue discomfort,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Tongue discomfort,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Tongue discomfort,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Tongue discomfort,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Tongue discomfort,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Tongue discomfort,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Tongue discomfort,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Tongue discomfort,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Tongue discomfort,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Tongue discomfort,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tongue discomfort,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tongue discomfort,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tongue discomfort,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tongue discomfort,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]

38. Primary Outcome: Cumulative Percentage of Subjects Reporting Gastrointestinal Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were diarrhoea, nausea, and vomiting.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 33.33 [0.84 to 90.57]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 13.64 [1.21 to 44.80]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 6.38 [0.00 to 84.50]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 3.70 [0.49 to 12.42]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 3.25 [0.01 to 23.49]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 2.96 [0.01 to 22.21]
  Any,Weeks 40-52 | 2.88 [0.01 to 22.02]
  Diarrhoea,Weeks 40-46: number analyzed (Participants) | 3
  Diarrhoea,Weeks 40-46 | 33.33 [0.84 to 90.57]
  Diarrhoea,Weeks 40-47: number analyzed (Participants) | 22
  Diarrhoea,Weeks 40-47 | 4.55 [0.00 to 86.65]
  Diarrhoea,Weeks 40-48: number analyzed (Participants) | 47
  Diarrhoea,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Diarrhoea,Weeks 40-49: number analyzed (Participants) | 81
  Diarrhoea,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Diarrhoea,Weeks 40-50: number analyzed (Participants) | 123
  Diarrhoea,Weeks 40-50 | 1.63 [0.01 to 12.28]
  Diarrhoea,Weeks 40-51: number analyzed (Participants) | 135
  Diarrhoea,Weeks 40-51 | 1.48 [0.00 to 11.58]
  Diarrhoea,Weeks 40-52 | 1.44 [0.00 to 11.48]
  Nausea,Weeks 40-46: number analyzed (Participants) | 3
  Nausea,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Nausea,Weeks 40-47: number analyzed (Participants) | 22
  Nausea,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Nausea,Weeks 40-48: number analyzed (Participants) | 47
  Nausea,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Nausea,Weeks 40-49: number analyzed (Participants) | 81
  Nausea,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Nausea,Weeks 40-50: number analyzed (Participants) | 123
  Nausea,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Nausea,Weeks 40-51: number analyzed (Participants) | 135
  Nausea,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Nausea,Weeks 40-52 | 0.00 [0.00 to 2.62]
  Vomiting,Weeks 40-46: number analyzed (Participants) | 3
  Vomiting,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Vomiting,Weeks 40-47: number analyzed (Participants) | 22
  Vomiting,Weeks 40-47 | 4.55 [0.00 to 100]
  Vomiting,Weeks 40-48: number analyzed (Participants) | 47
  Vomiting,Weeks 40-48 | 2.13 [0.00 to 99.99]
  Vomiting,Weeks 40-49: number analyzed (Participants) | 81
  Vomiting,Weeks 40-49 | 1.23 [0.00 to 38.50]
  Vomiting,Weeks 40-50: number analyzed (Participants) | 123
  Vomiting,Weeks 40-50 | 0.81 [0.00 to 27.14]
  Vomiting,Weeks 40-51: number analyzed (Participants) | 135
  Vomiting,Weeks 40-51 | 0.74 [0.00 to 25.43]
  Vomiting,Weeks 40-52 | 0.72 [0.00 to 25.02]
  Abdominal pain,Weeks 40-46: number analyzed (Participants) | 3
  Abdominal pain,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Abdominal pain,Weeks 40-47: number analyzed (Participants) | 22
  Abdominal pain,Weeks 40-47 | 4.55 [0.00 to 86.65]
  Abdominal pain,Weeks 40-48: number analyzed (Participants) | 47
  Abdominal pain,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Abdominal pain,Weeks 40-49: number analyzed (Participants) | 81
  Abdominal pain,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Abdominal pain,Weeks 40-50: number analyzed (Participants) | 123
  Abdominal pain,Weeks 40-50 | 0.81 [0.02 to 4.45]
  Abdominal pain,Weeks 40-51: number analyzed (Participants) | 135
  Abdominal pain,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Abdominal pain,Weeks 40-52 | 0.72 [0.02 to 3.94]

39. Primary Outcome: Cumulative Percentage of Subjects Reporting General Disorders and Administration Site Conditions by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were chills, face oedema, fatigue, injection site erythema, injection site pain, injection site swelling, and pyrexia.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 25.71 [16.01 to 37.56] |  | 25.71 [16.01 to 37.56]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 27.95 [6.70 to 60.73] |  | 27.95 [6.70 to 60.73]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 31.21 [18.49 to 46.39] | 27.45 [10.68 to 50.73] | 26.92 [0.28 to 88.26] | 28.72 [23.30 to 34.62]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 29.07 [0.46 to 88.60] | 26.73 [10.78 to 48.84] | 26.92 [8.05 to 55.09] | 27.55 [22.75 to 32.77]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 31.25 [15.06 to 51.66] | 26.29 [11.02 to 47.35] | 24.10 [18.28 to 30.73] | 27.24 [22.33 to 32.60]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 27.66 [6.51 to 60.56] | 28.00 [13.58 to 46.73] | 28.00 [7.70 to 58.39] | 27.89 [21.77 to 34.69]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 26.62 [5.17 to 61.91] | 27.90 [14.72 to 44.61] | 28.06 [8.81 to 56.01] | 27.57 [21.54 to 34.28]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 26.75 [6.31 to 59.00] | 27.70 [14.69 to 44.20] | 29.06 [8.31 to 59.38] | 27.97 [21.82 to 34.80]
  Any,Weeks 40-48 | 26.75 [6.31 to 59.00] | 27.70 [14.69 to 44.20] | 30.24 [7.34 to 64.15] | 28.49 [21.83 to 35.92]
  Any,Weeks 40-49 | 26.75 [6.31 to 59.00] | 27.70 [14.69 to 44.20] | 30.24 [7.34 to 64.15] | 28.49 [21.83 to 35.92]
  Any,Weeks 40-50 | 26.75 [6.31 to 59.00] | 27.70 [14.69 to 44.20] | 30.24 [7.34 to 64.15] | 28.49 [21.83 to 35.92]
  Any,Weeks 40-51 | 26.75 [6.31 to 59.00] | 27.70 [14.69 to 44.20] | 30.24 [7.34 to 64.15] | 28.49 [21.83 to 35.92]
  Any,Weeks 40-52 | 26.75 [6.31 to 59.00] | 27.70 [14.69 to 44.20] | 30.24 [7.34 to 64.15] | 28.49 [21.83 to 35.92]
  Chills,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Chills,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Chills,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Chills,Weeks 40-41 |  | 1.86 [0.00 to 44.30] |  | 1.86 [0.00 to 44.30]
  Chills,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Chills,Weeks 40-42 | 0.71 [0.01 to 4.40] | 2.45 [0.00 to 42.75] | 1.92 [0.05 to 10.26] | 1.76 [0.09 to 7.99]
  Chills,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Chills,Weeks 40-43 | 0.58 [0.00 to 20.94] | 2.30 [0.00 to 37.38] | 3.08 [0.24 to 12.22] | 1.93 [0.31 to 6.16]
  Chills,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Chills,Weeks 40-44 | 1.44 [0.00 to 18.59] | 2.16 [0.00 to 32.16] | 2.56 [0.72 to 6.37] | 2.05 [0.66 to 4.75]
  Chills,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Chills,Weeks 40-45 | 1.42 [0.01 to 10.19] | 2.40 [0.00 to 31.64] | 2.29 [0.99 to 4.45] | 2.04 [0.88 to 3.99]
  Chills,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Chills,Weeks 40-46 | 1.30 [0.00 to 9.76] | 2.54 [0.00 to 28.80] | 2.88 [0.36 to 9.96] | 2.30 [1.00 to 4.47]
  Chills,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Chills,Weeks 40-47 | 1.52 [0.04 to 7.92] | 2.52 [0.00 to 28.33] | 2.97 [0.26 to 11.52] | 2.39 [1.10 to 4.51]
  Chills,Weeks 40-48 | 1.52 [0.04 to 7.92] | 2.52 [0.00 to 28.33] | 2.87 [0.34 to 10.12] | 2.36 [1.10 to 4.38]
  Chills,Weeks 40-49 | 1.52 [0.04 to 7.92] | 2.52 [0.00 to 28.33] | 2.87 [0.34 to 10.12] | 2.36 [1.10 to 4.38]
  Chills,Weeks 40-50 | 1.52 [0.04 to 7.92] | 2.52 [0.00 to 28.33] | 2.87 [0.34 to 10.12] | 2.36 [1.10 to 4.38]
  Chills,Weeks 40-51 | 1.52 [0.04 to 7.92] | 2.52 [0.00 to 28.33] | 2.87 [0.34 to 10.12] | 2.36 [1.10 to 4.38]
  Chills,Weeks 40-52 | 1.52 [0.04 to 7.92] | 2.52 [0.00 to 28.33] | 2.87 [0.34 to 10.12] | 2.36 [1.10 to 4.38]
  Face oedema,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Face oedema,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Face oedema,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Face oedema,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Face oedema,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Face oedema,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Face oedema,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Face oedema,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.77 [0.02 to 4.21] | 0.19 [0.00 to 1.28]
  Face oedema,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Face oedema,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.00 [0.00 to 1.58] | 0.51 [0.01 to 2.82] | 0.31 [0.03 to 1.21]
  Face oedema,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Face oedema,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 1.82] | 0.23 [0.02 to 0.85]
  Face oedema,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Face oedema,Weeks 40-46 | 0.32 [0.00 to 10.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 2.15] | 0.20 [0.02 to 0.77]
  Face oedema,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Face oedema,Weeks 40-47 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 2.24] | 0.19 [0.02 to 0.75]
  Face oedema,Weeks 40-48 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.74]
  Face oedema,Weeks 40-49 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.74]
  Face oedema,Weeks 40-50 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.74]
  Face oedema,Weeks 40-51 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.74]
  Face oedema,Weeks 40-52 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.74]
  Fatigue,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Fatigue,Weeks 40-40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Fatigue,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Fatigue,Weeks 40-41 |  | 6.21 [0.58 to 22.47] |  | 6.21 [0.58 to 22.47]
  Fatigue,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Fatigue,Weeks 40-42 | 2.84 [0.04 to 16.88] | 6.86 [1.33 to 19.37] | 3.85 [0.11 to 19.24] | 5.04 [2.31 to 9.40]
  Fatigue,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Fatigue,Weeks 40-43 | 2.91 [0.45 to 9.29] | 7.37 [1.58 to 19.91] | 6.92 [1.05 to 21.30] | 5.78 [3.21 to 9.49]
  Fatigue,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Fatigue,Weeks 40-44 | 4.33 [0.06 to 24.57] | 7.76 [1.72 to 20.58] | 7.18 [2.35 to 16.05] | 6.46 [3.93 to 9.90]
  Fatigue,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Fatigue,Weeks 40-45 | 4.26 [0.55 to 14.24] | 8.40 [1.72 to 22.87] | 6.86 [0.60 to 25.02] | 6.46 [3.85 to 10.07]
  Fatigue,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Fatigue,Weeks 40-46 | 3.90 [0.43 to 13.80] | 7.97 [2.29 to 18.89] | 7.43 [0.75 to 25.84] | 6.49 [3.88 to 10.10]
  Fatigue,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Fatigue,Weeks 40-47 | 3.95 [0.58 to 12.73] | 7.91 [2.33 to 18.52] | 7.78 [0.88 to 26.02] | 6.61 [3.99 to 10.19]
  Fatigue,Weeks 40-48 | 3.95 [0.58 to 12.73] | 7.91 [2.33 to 18.52] | 7.51 [1.16 to 22.81] | 6.51 [4.03 to 9.85]
  Fatigue,Weeks 40-49 | 3.95 [0.58 to 12.73] | 7.91 [2.33 to 18.52] | 7.51 [1.16 to 22.81] | 6.51 [4.03 to 9.85]
  Fatigue,Weeks 40-50 | 3.95 [0.58 to 12.73] | 7.91 [2.33 to 18.52] | 7.51 [1.16 to 22.81] | 6.51 [4.03 to 9.85]
  Fatigue,Weeks 40-51 | 3.95 [0.58 to 12.73] | 7.91 [2.33 to 18.52] | 7.51 [1.16 to 22.81] | 6.51 [4.03 to 9.85]
  Fatigue,Weeks 40-52 | 3.95 [0.58 to 12.73] | 7.91 [2.33 to 18.52] | 7.51 [1.16 to 22.81] | 6.51 [4.03 to 9.85]
  Injection site erythema,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site erythema,Weeks 40-40 |  | 8.57 [0.03 to 50.40] |  | 8.57 [0.03 to 50.40]
  Injection site erythema,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Injection site erythema,Weeks 40-41 |  | 8.07 [4.37 to 13.41] |  | 8.07 [4.37 to 13.41]
  Injection site erythema,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Injection site erythema,Weeks 40-42 | 0.71 [0.01 to 4.40] | 8.82 [2.52 to 20.82] | 5.77 [0.15 to 27.99] | 5.54 [1.60 to 13.30]
  Injection site erythema,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Injection site erythema,Weeks 40-43 | 1.16 [0.00 to 37.75] | 8.29 [1.84 to 21.89] | 6.15 [0.45 to 23.69] | 5.39 [2.13 to 10.99]
  Injection site erythema,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Injection site erythema,Weeks 40-44 | 1.44 [0.00 to 12.02] | 8.19 [1.91 to 21.22] | 6.15 [3.22 to 10.50] | 5.35 [2.72 to 9.34]
  Injection site erythema,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Injection site erythema,Weeks 40-45 | 1.77 [0.09 to 8.03] | 7.60 [1.17 to 23.10] | 5.71 [2.36 to 11.32] | 4.99 [2.90 to 7.92]
  Injection site erythema,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Injection site erythema,Weeks 40-46 | 2.27 [0.05 to 12.17] | 7.61 [1.51 to 21.09] | 5.76 [2.62 to 10.76] | 5.19 [3.30 to 7.73]
  Injection site erythema,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Injection site erythema,Weeks 40-47 | 3.04 [0.03 to 18.73] | 7.55 [1.45 to 21.25] | 5.49 [2.61 to 10.00] | 5.27 [3.52 to 7.54]
  Injection site erythema,Weeks 40-48 | 3.04 [0.03 to 18.73] | 7.55 [1.45 to 21.25] | 5.52 [2.42 to 10.58] | 5.28 [3.52 to 7.57]
  Injection site erythema,Weeks 40-49 | 3.04 [0.03 to 18.73] | 7.55 [1.45 to 21.25] | 5.52 [2.42 to 10.58] | 5.28 [3.52 to 7.57]
  Injection site erythema,Weeks 40-50 | 3.04 [0.03 to 18.73] | 7.55 [1.45 to 21.25] | 5.52 [2.42 to 10.58] | 5.28 [3.52 to 7.57]
  Injection site erythema,Weeks 40-51 | 3.04 [0.03 to 18.73] | 7.55 [1.45 to 21.25] | 5.52 [2.42 to 10.58] | 5.28 [3.52 to 7.57]
  Injection site erythema,Weeks 40-52 | 3.04 [0.03 to 18.73] | 7.55 [1.45 to 21.25] | 5.52 [2.42 to 10.58] | 5.28 [3.52 to 7.57]
  Injection site pain,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site pain,Weeks 40-40 |  | 17.14 [9.18 to 28.03] |  | 17.14 [9.18 to 28.03]
  Injection site pain,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Injection site pain,Weeks 40-41 |  | 18.01 [4.65 to 41.50] |  | 18.01 [4.65 to 41.50]
  Injection site pain,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Injection site pain,Weeks 40-42 | 28.37 [7.46 to 59.80] | 16.67 [3.53 to 41.60] | 15.38 [0.28 to 63.30] | 20.65 [12.25 to 31.42]
  Injection site pain,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Injection site pain,Weeks 40-43 | 26.16 [0.02 to 94.78] | 16.13 [2.91 to 42.60] | 10.00 [0.68 to 36.93] | 17.92 [9.29 to 29.82]
  Injection site pain,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Injection site pain,Weeks 40-44 | 25.48 [9.68 to 48.07] | 15.95 [3.05 to 41.46] | 8.72 [4.24 to 15.49] | 16.85 [9.12 to 27.40]
  Injection site pain,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Injection site pain,Weeks 40-45 | 21.63 [2.65 to 59.28] | 17.20 [6.38 to 34.25] | 13.71 [1.03 to 46.65] | 17.23 [10.65 to 25.69]
  Injection site pain,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Injection site pain,Weeks 40-46 | 20.13 [1.26 to 63.88] | 16.67 [5.95 to 33.88] | 14.39 [1.71 to 43.62] | 16.78 [10.78 to 24.38]
  Injection site pain,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Injection site pain,Weeks 40-47 | 19.76 [1.27 to 62.83] | 16.55 [5.74 to 34.13] | 15.10 [1.45 to 47.74] | 16.95 [10.93 to 24.55]
  Injection site pain,Weeks 40-48 | 19.76 [1.27 to 62.83] | 16.55 [5.74 to 34.13] | 16.78 [1.01 to 56.72] | 17.64 [11.18 to 25.83]
  Injection site pain,Weeks 40-49 | 19.76 [1.27 to 62.83] | 16.55 [5.74 to 34.13] | 16.78 [1.01 to 56.72] | 17.64 [11.18 to 25.83]
  Injection site pain,Weeks 40-50 | 19.76 [1.27 to 62.83] | 16.55 [5.74 to 34.13] | 16.78 [1.01 to 56.72] | 17.64 [11.18 to 25.83]
  Injection site pain,Weeks 40-51 | 19.76 [1.27 to 62.83] | 16.55 [5.74 to 34.13] | 16.78 [1.01 to 56.72] | 17.64 [11.18 to 25.83]
  Injection site pain,Weeks 40-52 | 19.76 [1.27 to 62.83] | 16.55 [5.74 to 34.13] | 16.78 [1.01 to 56.72] | 17.64 [11.18 to 25.83]
  Injection site swelling,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site swelling,Weeks 40-40 |  | 11.43 [1.34 to 36.13] |  | 11.43 [1.34 to 36.13]
  Injection site swelling,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Injection site swelling,Weeks 40-41 |  | 10.56 [6.27 to 16.37] |  | 10.56 [6.27 to 16.37]
  Injection site swelling,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Injection site swelling,Weeks 40-42 | 4.96 [0.48 to 18.09] | 10.29 [5.11 to 17.97] | 5.77 [0.15 to 27.99] | 7.81 [4.57 to 12.30]
  Injection site swelling,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Injection site swelling,Weeks 40-43 | 6.40 [0.00 to 85.72] | 9.68 [3.63 to 19.89] | 6.15 [0.45 to 23.69] | 7.71 [4.99 to 11.28]
  Injection site swelling,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Injection site swelling,Weeks 40-44 | 5.29 [0.85 to 16.23] | 9.91 [4.60 to 18.06] | 5.13 [2.49 to 9.23] | 6.93 [4.73 to 9.73]
  Injection site swelling,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Injection site swelling,Weeks 40-45 | 4.61 [2.48 to 7.75] | 10.40 [6.19 to 16.11] | 5.71 [3.53 to 8.69] | 6.69 [4.81 to 9.02]
  Injection site swelling,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Injection site swelling,Weeks 40-46 | 4.55 [2.51 to 7.51] | 10.87 [7.40 to 15.24] | 6.24 [2.36 to 12.98] | 6.99 [4.86 to 9.69]
  Injection site swelling,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Injection site swelling,Weeks 40-47 | 5.17 [3.04 to 8.14] | 10.79 [7.31 to 15.19] | 6.86 [2.09 to 15.94] | 7.38 [5.32 to 9.92]
  Injection site swelling,Weeks 40-48 | 5.17 [3.04 to 8.14] | 10.79 [7.31 to 15.19] | 7.28 [1.72 to 18.91] | 7.55 [5.38 to 10.23]
  Injection site swelling,Weeks 40-49 | 5.17 [3.04 to 8.14] | 10.79 [7.31 to 15.19] | 7.28 [1.72 to 18.91] | 7.55 [5.38 to 10.23]
  Injection site swelling,Weeks 40-50 | 5.17 [3.04 to 8.14] | 10.79 [7.31 to 15.19] | 7.28 [1.72 to 18.91] | 7.55 [5.38 to 10.23]
  Injection site swelling,Weeks 40-51 | 5.17 [3.04 to 8.14] | 10.79 [7.31 to 15.19] | 7.28 [1.72 to 18.91] | 7.55 [5.38 to 10.23]
  Injection site swelling,Weeks 40-52 | 5.17 [3.04 to 8.14] | 10.79 [7.31 to 15.19] | 7.28 [1.72 to 18.91] | 7.55 [5.38 to 10.23]
  Pyrexia,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pyrexia,Weeks 40-40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Pyrexia,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Pyrexia,Weeks 40-41 |  | 1.24 [0.00 to 10.80] |  | 1.24 [0.00 to 10.80]
  Pyrexia,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Pyrexia,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.98 [0.00 to 12.72] | 5.77 [0.15 to 27.99] | 1.26 [0.07 to 5.60]
  Pyrexia,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Pyrexia,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.92 [0.00 to 13.10] | 10.00 [0.68 to 36.93] | 2.89 [0.09 to 14.40]
  Pyrexia,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Pyrexia,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.86 [0.00 to 13.44] | 7.69 [4.37 to 12.37] | 2.83 [0.32 to 10.09]
  Pyrexia,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Pyrexia,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.80 [0.00 to 13.75] | 6.29 [1.62 to 15.81] | 2.83 [0.51 to 8.52]
  Pyrexia,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Pyrexia,Weeks 40-46 | 0.65 [0.00 to 6.66] | 0.72 [0.00 to 14.00] | 6.47 [3.06 to 11.80] | 3.10 [0.87 to 7.65]
  Pyrexia,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Pyrexia,Weeks 40-47 | 0.61 [0.00 to 5.98] | 0.72 [0.00 to 14.01] | 6.41 [2.64 to 12.69] | 3.07 [0.86 to 7.56]
  Pyrexia,Weeks 40-48 | 0.61 [0.00 to 5.98] | 0.72 [0.00 to 14.01] | 6.40 [2.99 to 11.76] | 3.11 [0.92 to 7.51]
  Pyrexia,Weeks 40-49 | 0.61 [0.00 to 5.98] | 0.72 [0.00 to 14.01] | 6.40 [2.99 to 11.76] | 3.11 [0.92 to 7.51]
  Pyrexia,Weeks 40-50 | 0.61 [0.00 to 5.98] | 0.72 [0.00 to 14.01] | 6.40 [2.99 to 11.76] | 3.11 [0.92 to 7.51]
  Pyrexia,Weeks 40-51 | 0.61 [0.00 to 5.98] | 0.72 [0.00 to 14.01] | 6.40 [2.99 to 11.76] | 3.11 [0.92 to 7.51]
  Pyrexia,Weeks 40-52 | 0.61 [0.00 to 5.98] | 0.72 [0.00 to 14.01] | 6.40 [2.99 to 11.76] | 3.11 [0.92 to 7.51]
  Discomfort,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Discomfort,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Discomfort,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Discomfort,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Discomfort,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Discomfort,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Discomfort,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Discomfort,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Discomfort,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Discomfort,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Discomfort,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Discomfort,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 8.11] | 0.11 [0.00 to 0.84]
  Discomfort,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Discomfort,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.10 [0.00 to 0.70]
  Discomfort,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Discomfort,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.10 [0.00 to 0.66]
  Discomfort,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Discomfort,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Discomfort,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Discomfort,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Discomfort,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Feeling cold,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Feeling cold,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Feeling cold,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Feeling cold,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Feeling cold,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Feeling cold,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Feeling cold,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Feeling cold,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Feeling cold,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Feeling cold,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Feeling cold,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Feeling cold,Weeks 40-45 | 0.35 [0.00 to 5.88] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.79]
  Feeling cold,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Feeling cold,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.68]
  Feeling cold,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Feeling cold,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.64]
  Feeling cold,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling cold,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling cold,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling cold,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling cold,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling hot,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Feeling hot,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Feeling hot,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Feeling hot,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Feeling hot,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Feeling hot,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Feeling hot,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Feeling hot,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Feeling hot,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Feeling hot,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Feeling hot,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Feeling hot,Weeks 40-45 | 0.35 [0.00 to 5.88] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.79]
  Feeling hot,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Feeling hot,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.68]
  Feeling hot,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Feeling hot,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.64]
  Feeling hot,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling hot,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling hot,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling hot,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Feeling hot,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Influenza like illness,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Influenza like illness,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Influenza like illness,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Influenza like illness,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Influenza like illness,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Influenza like illness,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Influenza like illness,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Influenza like illness,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Influenza like illness,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Influenza like illness,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Influenza like illness,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Influenza like illness,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.42]
  Influenza like illness,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Influenza like illness,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.20 [0.02 to 0.78]
  Influenza like illness,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Influenza like illness,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.19 [0.02 to 0.73]
  Influenza like illness,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.19 [0.02 to 0.71]
  Influenza like illness,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.19 [0.02 to 0.71]
  Influenza like illness,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.19 [0.02 to 0.71]
  Influenza like illness,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.19 [0.02 to 0.71]
  Influenza like illness,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.19 [0.02 to 0.71]
  Injection site haematoma,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site haematoma,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Injection site haematoma,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Injection site haematoma,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Injection site haematoma,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Injection site haematoma,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Injection site haematoma,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Injection site haematoma,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Injection site haematoma,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Injection site haematoma,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Injection site haematoma,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Injection site haematoma,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Injection site haematoma,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Injection site haematoma,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Injection site haematoma,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Injection site haematoma,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Injection site haematoma,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Injection site haematoma,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Injection site haematoma,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Injection site haematoma,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Injection site haematoma,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Injection site pruritus,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site pruritus,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Injection site pruritus,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Injection site pruritus,Weeks 40-41 |  | 0.62 [0.00 to 17.42] |  | 0.62 [0.00 to 17.42]
  Injection site pruritus,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Injection site pruritus,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Injection site pruritus,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Injection site pruritus,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Injection site pruritus,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Injection site pruritus,Weeks 40-44 | 0.48 [0.00 to 12.12] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.31 [0.02 to 1.38]
  Injection site pruritus,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Injection site pruritus,Weeks 40-45 | 0.35 [0.00 to 5.88] | 1.20 [0.00 to 17.05] | 0.29 [0.00 to 8.11] | 0.57 [0.06 to 2.15]
  Injection site pruritus,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Injection site pruritus,Weeks 40-46 | 0.32 [0.00 to 4.64] | 1.09 [0.00 to 13.30] | 0.24 [0.00 to 5.63] | 0.50 [0.06 to 1.79]
  Injection site pruritus,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Injection site pruritus,Weeks 40-47 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.23 [0.00 to 5.17] | 0.48 [0.06 to 1.70]
  Injection site pruritus,Weeks 40-48 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.22 [0.00 to 4.76] | 0.47 [0.06 to 1.67]
  Injection site pruritus,Weeks 40-49 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.22 [0.00 to 4.76] | 0.47 [0.06 to 1.67]
  Injection site pruritus,Weeks 40-50 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.22 [0.00 to 4.76] | 0.47 [0.06 to 1.67]
  Injection site pruritus,Weeks 40-51 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.22 [0.00 to 4.76] | 0.47 [0.06 to 1.67]
  Injection site pruritus,Weeks 40-52 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.22 [0.00 to 4.76] | 0.47 [0.06 to 1.67]
  Injection site warmth,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Injection site warmth,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Injection site warmth,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Injection site warmth,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Injection site warmth,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Injection site warmth,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Injection site warmth,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Injection site warmth,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Injection site warmth,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Injection site warmth,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Injection site warmth,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Injection site warmth,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.91]
  Injection site warmth,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Injection site warmth,Weeks 40-46 | 0.32 [0.00 to 10.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.81]
  Injection site warmth,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Injection site warmth,Weeks 40-47 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.78]
  Injection site warmth,Weeks 40-48 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Injection site warmth,Weeks 40-49 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Injection site warmth,Weeks 40-50 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Injection site warmth,Weeks 40-51 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Injection site warmth,Weeks 40-52 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Malaise,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Malaise,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Malaise,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Malaise,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Malaise,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Malaise,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Malaise,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Malaise,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Malaise,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Malaise,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Malaise,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Malaise,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Malaise,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Malaise,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Malaise,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Malaise,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Malaise,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Malaise,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Malaise,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Malaise,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Malaise,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Mucous membrane disorder,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Mucous membrane disorder,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Mucous membrane disorder,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Mucous membrane disorder,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Mucous membrane disorder,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Mucous membrane disorder,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Mucous membrane disorder,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Mucous membrane disorder,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Mucous membrane disorder,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Mucous membrane disorder,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.00 to 22.01] | 0.16 [0.00 to 1.34]
  Mucous membrane disorder,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Mucous membrane disorder,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.57 [0.03 to 2.60] | 0.23 [0.03 to 0.82]
  Mucous membrane disorder,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Mucous membrane disorder,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.48 [0.06 to 1.72] | 0.20 [0.02 to 0.72]
  Mucous membrane disorder,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Mucous membrane disorder,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.46 [0.06 to 1.64] | 0.19 [0.02 to 0.69]
  Mucous membrane disorder,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.05 to 1.59] | 0.19 [0.02 to 0.68]
  Mucous membrane disorder,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.05 to 1.59] | 0.19 [0.02 to 0.68]
  Mucous membrane disorder,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.05 to 1.59] | 0.19 [0.02 to 0.68]
  Mucous membrane disorder,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.05 to 1.59] | 0.19 [0.02 to 0.68]
  Mucous membrane disorder,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.05 to 1.59] | 0.19 [0.02 to 0.68]
  Peripheral swelling,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Peripheral swelling,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Peripheral swelling,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Peripheral swelling,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Peripheral swelling,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Peripheral swelling,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Peripheral swelling,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Peripheral swelling,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Peripheral swelling,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Peripheral swelling,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.29]
  Peripheral swelling,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Peripheral swelling,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.91]
  Peripheral swelling,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Peripheral swelling,Weeks 40-46 | 0.32 [0.00 to 10.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 8.39] | 0.20 [0.01 to 1.03]
  Peripheral swelling,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Peripheral swelling,Weeks 40-47 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 7.65] | 0.19 [0.01 to 0.98]
  Peripheral swelling,Weeks 40-48 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.19 [0.01 to 0.96]
  Peripheral swelling,Weeks 40-49 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.19 [0.01 to 0.96]
  Peripheral swelling,Weeks 40-50 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.19 [0.01 to 0.96]
  Peripheral swelling,Weeks 40-51 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.19 [0.01 to 0.96]
  Peripheral swelling,Weeks 40-52 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.19 [0.01 to 0.96]

40. Primary Outcome: Cumulative Percentage of Subjects Reporting General Disorders and Administration Site Conditions by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were chills, face oedema, fatigue, injection site erythema, injection site pain, injection site swelling, and pyrexia.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 31.82 [0.00 to 99.83]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 17.02 [7.65 to 30.81]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 11.11 [5.21 to 20.05]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 8.94 [4.54 to 15.47]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 8.89 [4.52 to 15.35]
  Any,Weeks 40-52 | 9.35 [4.67 to 16.31]
  Chills,Weeks 40-46: number analyzed (Participants) | 3
  Chills,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Chills,Weeks 40-47: number analyzed (Participants) | 22
  Chills,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Chills,Weeks 40-48: number analyzed (Participants) | 47
  Chills,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Chills,Weeks 40-49: number analyzed (Participants) | 81
  Chills,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Chills,Weeks 40-50: number analyzed (Participants) | 123
  Chills,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Chills,Weeks 40-51: number analyzed (Participants) | 135
  Chills,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Chills,Weeks 40-52 | 0.00 [0.00 to 2.62]
  Face oedema,Weeks 40-46: number analyzed (Participants) | 3
  Face oedema,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Face oedema,Weeks 40-47: number analyzed (Participants) | 22
  Face oedema,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Face oedema,Weeks 40-48: number analyzed (Participants) | 47
  Face oedema,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Face oedema,Weeks 40-49: number analyzed (Participants) | 81
  Face oedema,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Face oedema,Weeks 40-50: number analyzed (Participants) | 123
  Face oedema,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Face oedema,Weeks 40-51: number analyzed (Participants) | 135
  Face oedema,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Face oedema,Weeks 40-52 | 0.00 [0.00 to 2.62]
  Fatigue,Weeks 40-46: number analyzed (Participants) | 3
  Fatigue,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Fatigue,Weeks 40-47: number analyzed (Participants) | 22
  Fatigue,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Fatigue,Weeks 40-48: number analyzed (Participants) | 47
  Fatigue,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Fatigue,Weeks 40-49: number analyzed (Participants) | 81
  Fatigue,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Fatigue,Weeks 40-50: number analyzed (Participants) | 123
  Fatigue,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Fatigue,Weeks 40-51: number analyzed (Participants) | 135
  Fatigue,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Fatigue,Weeks 40-52 | 0.72 [0.02 to 3.94]
  Injection site erythema,Weeks 40-46: number analyzed (Participants) | 3
  Injection site erythema,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Injection site erythema,Weeks 40-47: number analyzed (Participants) | 22
  Injection site erythema,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Injection site erythema,Weeks 40-48: number analyzed (Participants) | 47
  Injection site erythema,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Injection site erythema,Weeks 40-49: number analyzed (Participants) | 81
  Injection site erythema,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Injection site erythema,Weeks 40-50: number analyzed (Participants) | 123
  Injection site erythema,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Injection site erythema,Weeks 40-51: number analyzed (Participants) | 135
  Injection site erythema,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Injection site erythema,Weeks 40-52 | 0.00 [0.00 to 2.62]
  Injection site pain,Weeks 40-46: number analyzed (Participants) | 3
  Injection site pain,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Injection site pain,Weeks 40-47: number analyzed (Participants) | 22
  Injection site pain,Weeks 40-47 | 27.27 [0.01 to 96.64]
  Injection site pain,Weeks 40-48: number analyzed (Participants) | 47
  Injection site pain,Weeks 40-48 | 14.89 [6.20 to 28.31]
  Injection site pain,Weeks 40-49: number analyzed (Participants) | 81
  Injection site pain,Weeks 40-49 | 8.64 [3.55 to 17.00]
  Injection site pain,Weeks 40-50: number analyzed (Participants) | 123
  Injection site pain,Weeks 40-50 | 5.69 [2.32 to 11.37]
  Injection site pain,Weeks 40-51: number analyzed (Participants) | 135
  Injection site pain,Weeks 40-51 | 5.19 [2.11 to 10.39]
  Injection site pain,Weeks 40-52 | 5.04 [2.05 to 10.10]
  Injection site swelling,Weeks 40-46: number analyzed (Participants) | 3
  Injection site swelling,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Injection site swelling,Weeks 40-47: number analyzed (Participants) | 22
  Injection site swelling,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Injection site swelling,Weeks 40-48: number analyzed (Participants) | 47
  Injection site swelling,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Injection site swelling,Weeks 40-49: number analyzed (Participants) | 81
  Injection site swelling,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Injection site swelling,Weeks 40-50: number analyzed (Participants) | 123
  Injection site swelling,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Injection site swelling,Weeks 40-51: number analyzed (Participants) | 135
  Injection site swelling,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Injection site swelling,Weeks 40-52 | 0.00 [0.00 to 2.62]
  Pyrexia,Weeks 40-46: number analyzed (Participants) | 3
  Pyrexia,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Pyrexia,Weeks 40-47: number analyzed (Participants) | 22
  Pyrexia,Weeks 40-47 | 9.09 [0.00 to 98.76]
  Pyrexia,Weeks 40-48: number analyzed (Participants) | 47
  Pyrexia,Weeks 40-48 | 6.38 [0.00 to 54.84]
  Pyrexia,Weeks 40-49: number analyzed (Participants) | 81
  Pyrexia,Weeks 40-49 | 4.94 [0.94 to 14.29]
  Pyrexia,Weeks 40-50: number analyzed (Participants) | 123
  Pyrexia,Weeks 40-50 | 4.88 [0.81 to 14.85]
  Pyrexia,Weeks 40-51: number analyzed (Participants) | 135
  Pyrexia,Weeks 40-51 | 4.44 [0.83 to 13.00]
  Pyrexia,Weeks 40-52 | 5.04 [1.00 to 14.30]

41. Primary Outcome: Cumulative Percentage of Subjects Reporting Immune System Disorders by MedDRA PT, Using ADR Card, Post Dose 1, by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were anaphylactic reaction and hypersensitivity.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 0.00]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 0.00]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.00]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.00]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.00]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.35 [0.00 to 5.88] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.11 to 0.00]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.10 to 0.00]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.10 to 0.00]
  Any,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Any,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Any,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Any,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Any,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Anaphylactic reaction,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Anaphylactic reaction,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Anaphylactic reaction,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Anaphylactic reaction,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Anaphylactic reaction,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Anaphylactic reaction,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Anaphylactic reaction,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Anaphylactic reaction,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Anaphylactic reaction,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.00]
  Anaphylactic reaction,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.00]
  Hypersensitivity,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hypersensitivity,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 0.00]
  Hypersensitivity,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Hypersensitivity,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 0.00]
  Hypersensitivity,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Hypersensitivity,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.00]
  Hypersensitivity,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Hypersensitivity,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.00]
  Hypersensitivity,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Hypersensitivity,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.00]
  Hypersensitivity,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Hypersensitivity,Weeks 40-45 | 0.35 [0.00 to 5.88] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.11 to 0.00]
  Hypersensitivity,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Hypersensitivity,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.10 to 0.00]
  Hypersensitivity,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Hypersensitivity,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.10 to 0.00]
  Hypersensitivity,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Hypersensitivity,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Hypersensitivity,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Hypersensitivity,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]
  Hypersensitivity,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.09 to 0.00]

42. Primary Outcome: Cumulative Percentage of Subjects Reporting Immune System Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were anaphylactic reaction and hypersensitivity.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

43. Primary Outcome: Cumulative Percentage of Subjects Reporting Infections and Infestations by MedDRA PT, Using ADR Card, Post Dose 1, by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were conjunctivitis and rhinitis.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 8.57 [0.31 to 37.07] |  | 8.57 [0.31 to 37.07]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 8.70 [1.37 to 25.91] |  | 8.70 [1.37 to 25.91]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.71 [0.01 to 4.40] | 7.84 [1.03 to 25.06] | 1.92 [0.05 to 10.26] | 4.53 [0.81 to 13.48]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 1.74 [0.00 to 85.49] | 7.83 [1.22 to 23.66] | 3.85 [0.30 to 15.16] | 4.82 [1.57 to 10.92]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 2.88 [0.00 to 26.08] | 7.76 [1.39 to 22.35] | 4.62 [1.57 to 10.25] | 5.20 [2.41 to 9.61]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 4.61 [0.02 to 31.32] | 8.00 [1.85 to 20.84] | 5.14 [0.31 to 21.15] | 5.78 [3.11 to 9.69]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 4.55 [0.04 to 27.57] | 7.97 [2.19 to 19.25] | 5.76 [0.18 to 27.12] | 5.99 [3.31 to 9.87]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 4.56 [0.06 to 25.49] | 7.91 [2.17 to 19.14] | 6.18 [0.20 to 28.60] | 6.13 [3.45 to 9.95]
  Any,Weeks 40-48 | 4.56 [0.06 to 25.49] | 7.91 [2.17 to 19.14] | 6.40 [0.22 to 29.12] | 6.23 [3.52 to 10.08]
  Any,Weeks 40-49 | 4.56 [0.06 to 25.49] | 7.91 [2.17 to 19.14] | 6.40 [0.22 to 29.12] | 6.23 [3.52 to 10.08]
  Any,Weeks 40-50 | 4.56 [0.06 to 25.49] | 7.91 [2.17 to 19.14] | 6.40 [0.22 to 29.12] | 6.23 [3.52 to 10.08]
  Any,Weeks 40-51 | 4.56 [0.06 to 25.49] | 7.91 [2.17 to 19.14] | 6.40 [0.22 to 29.12] | 6.23 [3.52 to 10.08]
  Any,Weeks 40-52 | 4.56 [0.06 to 25.49] | 7.91 [2.17 to 19.14] | 6.40 [0.22 to 29.12] | 6.23 [3.52 to 10.08]
  Conjunctivitis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Conjunctivitis,Weeks 40-40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Conjunctivitis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Conjunctivitis,Weeks 40-41 |  | 3.73 [0.22 to 15.88] |  | 3.73 [0.22 to 15.88]
  Conjunctivitis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Conjunctivitis,Weeks 40-42 | 0.71 [0.01 to 4.40] | 3.92 [0.21 to 16.93] | 0.00 [0.00 to 6.85] | 2.27 [0.40 to 6.90]
  Conjunctivitis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Conjunctivitis,Weeks 40-43 | 1.16 [0.00 to 37.75] | 4.15 [0.24 to 17.56] | 0.77 [0.02 to 4.21] | 2.31 [0.55 to 6.23]
  Conjunctivitis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Conjunctivitis,Weeks 40-44 | 1.92 [0.01 to 13.68] | 3.88 [0.37 to 14.38] | 1.03 [0.00 to 11.31] | 2.36 [0.77 to 5.44]
  Conjunctivitis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Conjunctivitis,Weeks 40-45 | 3.55 [0.02 to 22.81] | 3.60 [0.51 to 11.82] | 2.00 [0.00 to 16.82] | 2.95 [1.29 to 5.71]
  Conjunctivitis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Conjunctivitis,Weeks 40-46 | 3.57 [0.05 to 20.55] | 3.99 [0.61 to 12.61] | 2.64 [0.00 to 22.96] | 3.30 [1.51 to 6.19]
  Conjunctivitis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Conjunctivitis,Weeks 40-47 | 3.65 [0.08 to 19.45] | 3.96 [0.63 to 12.36] | 2.75 [0.00 to 21.86] | 3.35 [1.60 to 6.12]
  Conjunctivitis,Weeks 40-48 | 3.65 [0.08 to 19.45] | 3.96 [0.63 to 12.36] | 2.87 [0.00 to 22.55] | 3.40 [1.63 to 6.18]
  Conjunctivitis,Weeks 40-49 | 3.65 [0.08 to 19.45] | 3.96 [0.63 to 12.36] | 2.87 [0.00 to 22.55] | 3.40 [1.63 to 6.18]
  Conjunctivitis,Weeks 40-50 | 3.65 [0.08 to 19.45] | 3.96 [0.63 to 12.36] | 2.87 [0.00 to 22.55] | 3.40 [1.63 to 6.18]
  Conjunctivitis,Weeks 40-51 | 3.65 [0.08 to 19.45] | 3.96 [0.63 to 12.36] | 2.87 [0.00 to 22.55] | 3.40 [1.63 to 6.18]
  Conjunctivitis,Weeks 40-52 | 3.65 [0.08 to 19.45] | 3.96 [0.63 to 12.36] | 2.87 [0.00 to 22.55] | 3.40 [1.63 to 6.18]
  Rhinitis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rhinitis,Weeks 40-40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Rhinitis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Rhinitis,Weeks 40-41 |  | 5.59 [0.73 to 18.36] |  | 5.59 [0.73 to 18.36]
  Rhinitis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Rhinitis,Weeks 40-42 | 0.71 [0.01 to 4.40] | 4.90 [0.34 to 19.50] | 1.92 [0.05 to 10.26] | 3.02 [0.61 to 8.70]
  Rhinitis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Rhinitis,Weeks 40-43 | 1.16 [0.00 to 37.75] | 4.61 [0.20 to 20.63] | 2.31 [0.18 to 9.24] | 2.89 [0.88 to 6.87]
  Rhinitis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Rhinitis,Weeks 40-44 | 1.92 [0.00 to 17.01] | 4.74 [0.39 to 18.08] | 2.56 [0.59 to 7.01] | 3.15 [1.36 to 6.13]
  Rhinitis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Rhinitis,Weeks 40-45 | 2.13 [0.06 to 11.14] | 5.20 [1.07 to 14.51] | 2.57 [0.04 to 14.91] | 3.17 [1.54 to 5.75]
  Rhinitis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Rhinitis,Weeks 40-46 | 1.95 [0.09 to 9.11] | 4.71 [0.66 to 15.28] | 2.88 [0.06 to 15.48] | 3.10 [1.58 to 5.41]
  Rhinitis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Rhinitis,Weeks 40-47 | 1.82 [0.11 to 8.03] | 4.68 [0.63 to 15.35] | 2.97 [0.05 to 17.00] | 3.07 [1.53 to 5.44]
  Rhinitis,Weeks 40-48 | 1.82 [0.11 to 8.03] | 4.68 [0.63 to 15.35] | 2.87 [0.07 to 15.15] | 3.02 [1.54 to 5.28]
  Rhinitis,Weeks 40-49 | 1.82 [0.11 to 8.03] | 4.68 [0.63 to 15.35] | 2.87 [0.07 to 15.15] | 3.02 [1.54 to 5.28]
  Rhinitis,Weeks 40-50 | 1.82 [0.11 to 8.03] | 4.68 [0.63 to 15.35] | 2.87 [0.07 to 15.15] | 3.02 [1.54 to 5.28]
  Rhinitis,Weeks 40-51 | 1.82 [0.11 to 8.03] | 4.68 [0.63 to 15.35] | 2.87 [0.07 to 15.15] | 3.02 [1.54 to 5.28]
  Rhinitis,Weeks 40-52 | 1.82 [0.11 to 8.03] | 4.68 [0.63 to 15.35] | 2.87 [0.07 to 15.15] | 3.02 [1.54 to 5.28]
  Bronchitis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Bronchitis,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Bronchitis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Bronchitis,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Bronchitis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Bronchitis,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Bronchitis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Bronchitis,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Bronchitis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Bronchitis,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.01 to 2.82] | 0.16 [0.00 to 0.87]
  Bronchitis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Bronchitis,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 1.82] | 0.11 [0.00 to 0.63]
  Bronchitis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Bronchitis,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 2.15] | 0.10 [0.00 to 0.56]
  Bronchitis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Bronchitis,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 2.24] | 0.10 [0.00 to 0.55]
  Bronchitis,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Bronchitis,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Bronchitis,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Bronchitis,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Bronchitis,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Ear infection,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear infection,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear infection,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Ear infection,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Ear infection,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Ear infection,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Ear infection,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Ear infection,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Ear infection,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Ear infection,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.01 to 2.82] | 0.16 [0.00 to 0.87]
  Ear infection,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Ear infection,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 1.82] | 0.11 [0.00 to 0.63]
  Ear infection,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Ear infection,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 2.15] | 0.10 [0.00 to 0.56]
  Ear infection,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Ear infection,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 2.24] | 0.10 [0.00 to 0.55]
  Ear infection,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Ear infection,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Ear infection,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Ear infection,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Ear infection,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Herpes simplex,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Herpes simplex,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Herpes simplex,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Herpes simplex,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Herpes simplex,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Herpes simplex,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Herpes simplex,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Herpes simplex,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Herpes simplex,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Herpes simplex,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Herpes simplex,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Herpes simplex,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Herpes simplex,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Herpes simplex,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Herpes simplex,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Herpes simplex,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Herpes simplex,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Herpes simplex,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Herpes simplex,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Herpes simplex,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Herpes simplex,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Hordeolum,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hordeolum,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Hordeolum,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Hordeolum,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Hordeolum,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Hordeolum,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Hordeolum,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Hordeolum,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Hordeolum,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Hordeolum,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Hordeolum,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Hordeolum,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.42]
  Hordeolum,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Hordeolum,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.00 [0.00 to 0.37]
  Hordeolum,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Hordeolum,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 7.65] | 0.10 [0.00 to 0.76]
  Hordeolum,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Hordeolum,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Hordeolum,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Hordeolum,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Hordeolum,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Laryngitis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Laryngitis,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Laryngitis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Laryngitis,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Laryngitis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Laryngitis,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Laryngitis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Laryngitis,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Laryngitis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Laryngitis,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Laryngitis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Laryngitis,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 10.35] | 0.11 [0.00 to 0.92]
  Laryngitis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Laryngitis,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 8.39] | 0.10 [0.00 to 0.81]
  Laryngitis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Laryngitis,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 7.65] | 0.10 [0.00 to 0.76]
  Laryngitis,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Laryngitis,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Laryngitis,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Laryngitis,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Laryngitis,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Nasopharyngitis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Nasopharyngitis,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Nasopharyngitis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Nasopharyngitis,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Nasopharyngitis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Nasopharyngitis,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Nasopharyngitis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Nasopharyngitis,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Nasopharyngitis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Nasopharyngitis,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Nasopharyngitis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Nasopharyngitis,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.42]
  Nasopharyngitis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Nasopharyngitis,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.00 [0.00 to 0.37]
  Nasopharyngitis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Nasopharyngitis,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.00 [0.00 to 0.35]
  Nasopharyngitis,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Nasopharyngitis,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Nasopharyngitis,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Nasopharyngitis,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Nasopharyngitis,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 7.27] | 0.09 [0.00 to 0.75]
  Oral herpes,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Oral herpes,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Oral herpes,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Oral herpes,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Oral herpes,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Oral herpes,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Oral herpes,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Oral herpes,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Oral herpes,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Oral herpes,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Oral herpes,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Oral herpes,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Oral herpes,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Oral herpes,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Oral herpes,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Oral herpes,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Oral herpes,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Oral herpes,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Oral herpes,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Oral herpes,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Oral herpes,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Upper respiratory tract infection,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Upper respiratory tract infection,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Upper respiratory tract infection,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Upper respiratory tract infection,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Upper respiratory tract infection,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Upper respiratory tract infection,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Upper respiratory tract infection,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Upper respiratory tract infection,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.77 [0.02 to 4.21] | 0.19 [0.00 to 1.28]
  Upper respiratory tract infection,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Upper respiratory tract infection,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.01 to 2.82] | 0.16 [0.00 to 0.87]
  Upper respiratory tract infection,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Upper respiratory tract infection,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 1.82] | 0.11 [0.00 to 0.63]
  Upper respiratory tract infection,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Upper respiratory tract infection,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 2.15] | 0.10 [0.00 to 0.56]
  Upper respiratory tract infection,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Upper respiratory tract infection,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 2.24] | 0.10 [0.00 to 0.55]
  Upper respiratory tract infection,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Upper respiratory tract infection,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Upper respiratory tract infection,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Upper respiratory tract infection,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Upper respiratory tract infection,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]

44. Primary Outcome: Cumulative Percentage of Subjects Reporting Infections and Infestations by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were conjunctivitis and rhinitis.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 6.38 [0.00 to 54.84]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 3.70 [0.71 to 10.79]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 3.25 [0.55 to 9.99]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 2.96 [0.56 to 8.74]
  Any,Weeks 40-52 | 2.88 [0.58 to 8.26]
  Conjunctivitis,Weeks 40-46: number analyzed (Participants) | 3
  Conjunctivitis,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Conjunctivitis,Weeks 40-47: number analyzed (Participants) | 22
  Conjunctivitis,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Conjunctivitis,Weeks 40-48: number analyzed (Participants) | 47
  Conjunctivitis,Weeks 40-48 | 4.26 [0.00 to 40.16]
  Conjunctivitis,Weeks 40-49: number analyzed (Participants) | 81
  Conjunctivitis,Weeks 40-49 | 2.47 [0.30 to 8.64]
  Conjunctivitis,Weeks 40-50: number analyzed (Participants) | 123
  Conjunctivitis,Weeks 40-50 | 2.44 [0.42 to 7.53]
  Conjunctivitis,Weeks 40-51: number analyzed (Participants) | 135
  Conjunctivitis,Weeks 40-51 | 2.22 [0.42 to 6.58]
  Conjunctivitis,Weeks 40-52 | 2.16 [0.44 to 6.22]
  Rhinitis,Weeks 40-46: number analyzed (Participants) | 3
  Rhinitis,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Rhinitis,Weeks 40-47: number analyzed (Participants) | 22
  Rhinitis,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Rhinitis,Weeks 40-48: number analyzed (Participants) | 47
  Rhinitis,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Rhinitis,Weeks 40-49: number analyzed (Participants) | 81
  Rhinitis,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Rhinitis,Weeks 40-50: number analyzed (Participants) | 123
  Rhinitis,Weeks 40-50 | 0.81 [0.02 to 4.45]
  Rhinitis,Weeks 40-51: number analyzed (Participants) | 135
  Rhinitis,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Rhinitis,Weeks 40-52 | 0.72 [0.02 to 3.94]

45. Primary Outcome: Cumulative Percentage of Subjects Reporting Metabolism and Nutrition Disorders by MedDRA PT, Using ADR Card, Post Dose 1, by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEI listed on the ADR card was decreased appetite.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.71 [0.01 to 4.40] | 0.49 [0.00 to 6.53] | 3.85 [0.11 to 19.24] | 1.01 [0.20 to 2.97]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.58 [0.00 to 20.94] | 0.46 [0.00 to 6.74] | 8.46 [0.60 to 31.78] | 2.50 [0.11 to 11.76]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.96 [0.00 to 7.53] | 0.43 [0.00 to 6.92] | 8.21 [4.76 to 12.98] | 2.99 [0.34 to 10.65]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 1.77 [0.09 to 8.03] | 0.40 [0.00 to 7.09] | 6.29 [0.63 to 22.23] | 3.17 [0.66 to 9.02]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 1.95 [0.10 to 8.87] | 0.36 [0.00 to 7.23] | 5.28 [0.10 to 27.37] | 2.90 [0.60 to 8.21]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.03 [0.06 to 28.27] | 2.87 [0.64 to 7.94]
  Any,Weeks 40-48 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Any,Weeks 40-49 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Any,Weeks 40-50 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Any,Weeks 40-51 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Any,Weeks 40-52 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Decreased appetite,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Decreased appetite,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Decreased appetite,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Decreased appetite,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Decreased appetite,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Decreased appetite,Weeks 40-42 | 0.71 [0.01 to 4.40] | 0.49 [0.00 to 6.53] | 3.85 [0.11 to 19.24] | 1.01 [0.20 to 2.97]
  Decreased appetite,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Decreased appetite,Weeks 40-43 | 0.58 [0.00 to 20.94] | 0.46 [0.00 to 6.74] | 8.46 [0.60 to 31.78] | 2.50 [0.11 to 11.76]
  Decreased appetite,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Decreased appetite,Weeks 40-44 | 0.96 [0.00 to 7.53] | 0.43 [0.00 to 6.92] | 8.21 [4.76 to 12.98] | 2.99 [0.34 to 10.65]
  Decreased appetite,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Decreased appetite,Weeks 40-45 | 1.77 [0.09 to 8.03] | 0.40 [0.00 to 7.09] | 6.29 [0.63 to 22.23] | 3.17 [0.66 to 9.02]
  Decreased appetite,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Decreased appetite,Weeks 40-46 | 1.95 [0.10 to 8.87] | 0.36 [0.00 to 7.23] | 5.28 [0.10 to 27.37] | 2.90 [0.60 to 8.21]
  Decreased appetite,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Decreased appetite,Weeks 40-47 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.03 [0.06 to 28.27] | 2.87 [0.64 to 7.94]
  Decreased appetite,Weeks 40-48 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Decreased appetite,Weeks 40-49 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Decreased appetite,Weeks 40-50 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Decreased appetite,Weeks 40-51 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]
  Decreased appetite,Weeks 40-52 | 2.13 [0.10 to 9.83] | 0.36 [0.00 to 7.23] | 5.30 [0.27 to 22.74] | 3.02 [0.81 to 7.64]

46. Primary Outcome: Cumulative Percentage of Subjects Reporting Metabolism and Nutrition Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEI listed on the ADR card was decreased appetite.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 4.55 [0.00 to 86.65]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 4.26 [0.00 to 40.16]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 2.47 [0.30 to 8.64]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 2.44 [0.42 to 7.53]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 2.22 [0.42 to 6.58]
  Any,Weeks 40-52 | 2.16 [0.44 to 6.22]
  Decreased appetite,Weeks 40-46: number analyzed (Participants) | 3
  Decreased appetite,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Decreased appetite,Weeks 40-47: number analyzed (Participants) | 22
  Decreased appetite,Weeks 40-47 | 4.55 [0.00 to 86.65]
  Decreased appetite,Weeks 40-48: number analyzed (Participants) | 47
  Decreased appetite,Weeks 40-48 | 4.26 [0.00 to 40.16]
  Decreased appetite,Weeks 40-49: number analyzed (Participants) | 81
  Decreased appetite,Weeks 40-49 | 2.47 [0.30 to 8.64]
  Decreased appetite,Weeks 40-50: number analyzed (Participants) | 123
  Decreased appetite,Weeks 40-50 | 2.44 [0.42 to 7.53]
  Decreased appetite,Weeks 40-51: number analyzed (Participants) | 135
  Decreased appetite,Weeks 40-51 | 2.22 [0.42 to 6.58]
  Decreased appetite,Weeks 40-52 | 2.16 [0.44 to 6.22]

47. Primary Outcome: Cumulative Percentage of Subjects Reporting Musculoskeletal and Connective Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were arthropathy and myalgia.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 6.83 [0.05 to 39.06] |  | 6.83 [0.05 to 39.06]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 11.35 [0.10 to 56.46] | 5.88 [0.02 to 38.78] | 7.69 [0.19 to 36.17] | 8.06 [3.59 to 15.14]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 9.30 [0.00 to 98.75] | 6.91 [0.29 to 29.90] | 7.69 [0.55 to 29.13] | 7.90 [4.20 to 13.29]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 11.06 [3.48 to 24.62] | 6.90 [0.40 to 27.87] | 6.15 [2.06 to 13.66] | 8.03 [4.88 to 12.30]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 10.99 [3.84 to 23.27] | 7.60 [0.91 to 25.06] | 7.14 [0.51 to 27.33] | 8.50 [5.54 to 12.37]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 11.04 [4.44 to 21.74] | 8.33 [1.48 to 23.91] | 7.43 [0.50 to 28.64] | 8.79 [5.87 to 12.53]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 10.64 [3.62 to 22.86] | 8.27 [1.50 to 23.61] | 7.32 [0.74 to 25.51] | 8.62 [5.90 to 12.07]
  Any,Weeks 40-48 | 10.64 [3.62 to 22.86] | 8.27 [1.50 to 23.61] | 8.39 [0.26 to 37.24] | 9.06 [5.82 to 13.29]
  Any,Weeks 40-49 | 10.64 [3.62 to 22.86] | 8.27 [1.50 to 23.61] | 8.39 [0.26 to 37.24] | 9.06 [5.82 to 13.29]
  Any,Weeks 40-50 | 10.64 [3.62 to 22.86] | 8.27 [1.50 to 23.61] | 8.39 [0.26 to 37.24] | 9.06 [5.82 to 13.29]
  Any,Weeks 40-51 | 10.64 [3.62 to 22.86] | 8.27 [1.50 to 23.61] | 8.39 [0.26 to 37.24] | 9.06 [5.82 to 13.29]
  Any,Weeks 40-52 | 10.64 [3.62 to 22.86] | 8.27 [1.50 to 23.61] | 8.39 [0.26 to 37.24] | 9.06 [5.82 to 13.29]
  Arthropathy,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Arthropathy,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Arthropathy,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Arthropathy,Weeks 40-41 |  | 1.86 [0.00 to 15.87] |  | 1.86 [0.00 to 15.87]
  Arthropathy,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Arthropathy,Weeks 40-42 | 1.42 [0.02 to 8.68] | 1.96 [0.04 to 10.99] | 0.00 [0.00 to 6.85] | 1.51 [0.52 to 3.40]
  Arthropathy,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Arthropathy,Weeks 40-43 | 1.16 [0.00 to 37.75] | 2.76 [0.24 to 10.75] | 0.00 [0.00 to 2.80] | 1.54 [0.36 to 4.23]
  Arthropathy,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Arthropathy,Weeks 40-44 | 3.37 [0.01 to 23.06] | 2.59 [0.30 to 9.13] | 0.51 [0.00 to 22.01] | 2.20 [0.68 to 5.22]
  Arthropathy,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Arthropathy,Weeks 40-45 | 3.19 [0.04 to 18.56] | 3.20 [0.30 to 12.02] | 1.71 [0.00 to 27.48] | 2.61 [0.99 to 5.51]
  Arthropathy,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Arthropathy,Weeks 40-46 | 3.25 [0.09 to 16.56] | 3.62 [0.32 to 13.84] | 1.68 [0.00 to 23.32] | 2.70 [1.09 to 5.47]
  Arthropathy,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Arthropathy,Weeks 40-47 | 3.34 [0.15 to 15.29] | 3.60 [0.33 to 13.54] | 1.83 [0.00 to 20.37] | 2.78 [1.22 to 5.36]
  Arthropathy,Weeks 40-48 | 3.34 [0.15 to 15.29] | 3.60 [0.33 to 13.54] | 2.43 [0.00 to 29.22] | 3.02 [1.27 to 5.98]
  Arthropathy,Weeks 40-49 | 3.34 [0.15 to 15.29] | 3.60 [0.33 to 13.54] | 2.43 [0.00 to 29.22] | 3.02 [1.27 to 5.98]
  Arthropathy,Weeks 40-50 | 3.34 [0.15 to 15.29] | 3.60 [0.33 to 13.54] | 2.43 [0.00 to 29.22] | 3.02 [1.27 to 5.98]
  Arthropathy,Weeks 40-51 | 3.34 [0.15 to 15.29] | 3.60 [0.33 to 13.54] | 2.43 [0.00 to 29.22] | 3.02 [1.27 to 5.98]
  Arthropathy,Weeks 40-52 | 3.34 [0.15 to 15.29] | 3.60 [0.33 to 13.54] | 2.43 [0.00 to 29.22] | 3.02 [1.27 to 5.98]
  Myalgia,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Myalgia,Weeks 40-40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Myalgia,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Myalgia,Weeks 40-41 |  | 5.59 [0.07 to 31.12] |  | 5.59 [0.07 to 31.12]
  Myalgia,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Myalgia,Weeks 40-42 | 9.93 [0.09 to 50.96] | 4.41 [0.00 to 35.58] | 7.69 [0.19 to 36.17] | 6.80 [2.81 to 13.43]
  Myalgia,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Myalgia,Weeks 40-43 | 8.14 [0.00 to 97.65] | 4.61 [0.02 to 30.64] | 6.92 [0.50 to 26.44] | 6.36 [2.91 to 11.83]
  Myalgia,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Myalgia,Weeks 40-44 | 8.17 [0.63 to 30.15] | 4.74 [0.06 to 26.99] | 5.13 [2.49 to 9.23] | 5.98 [3.20 to 10.06]
  Myalgia,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Myalgia,Weeks 40-45 | 8.51 [1.71 to 23.33] | 5.20 [0.28 to 21.98] | 5.71 [0.71 to 19.10] | 6.46 [4.09 to 9.63]
  Myalgia,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Myalgia,Weeks 40-46 | 8.77 [2.71 to 19.96] | 5.43 [0.59 to 19.03] | 6.00 [0.68 to 20.51] | 6.69 [4.44 to 9.62]
  Myalgia,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Myalgia,Weeks 40-47 | 8.21 [1.64 to 22.59] | 5.40 [0.57 to 18.99] | 5.95 [0.95 to 18.16] | 6.51 [4.39 to 9.25]
  Myalgia,Weeks 40-48 | 8.21 [1.64 to 22.59] | 5.40 [0.57 to 18.99] | 6.84 [0.36 to 28.26] | 6.89 [4.33 to 10.30]
  Myalgia,Weeks 40-49 | 8.21 [1.64 to 22.59] | 5.40 [0.57 to 18.99] | 6.84 [0.36 to 28.26] | 6.89 [4.33 to 10.30]
  Myalgia,Weeks 40-50 | 8.21 [1.64 to 22.59] | 5.40 [0.57 to 18.99] | 6.84 [0.36 to 28.26] | 6.89 [4.33 to 10.30]
  Myalgia,Weeks 40-51 | 8.21 [1.64 to 22.59] | 5.40 [0.57 to 18.99] | 6.84 [0.36 to 28.26] | 6.89 [4.33 to 10.30]
  Myalgia,Weeks 40-52 | 8.21 [1.64 to 22.59] | 5.40 [0.57 to 18.99] | 6.84 [0.36 to 28.26] | 6.89 [4.33 to 10.30]
  Limb discomfort,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Limb discomfort,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Limb discomfort,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Limb discomfort,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Limb discomfort,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Limb discomfort,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Limb discomfort,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Limb discomfort,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Limb discomfort,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Limb discomfort,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Limb discomfort,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Limb discomfort,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Limb discomfort,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Limb discomfort,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Limb discomfort,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Limb discomfort,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Limb discomfort,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Limb discomfort,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Limb discomfort,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Limb discomfort,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Limb discomfort,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Musculoskeletal pain,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Musculoskeletal pain,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Musculoskeletal pain,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Musculoskeletal pain,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Musculoskeletal pain,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Musculoskeletal pain,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Musculoskeletal pain,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Musculoskeletal pain,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Musculoskeletal pain,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Musculoskeletal pain,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Musculoskeletal pain,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Musculoskeletal pain,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Musculoskeletal pain,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Musculoskeletal pain,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Musculoskeletal pain,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Musculoskeletal pain,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Musculoskeletal pain,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Musculoskeletal pain,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Musculoskeletal pain,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Musculoskeletal pain,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Musculoskeletal pain,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Pain in extremity,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pain in extremity,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Pain in extremity,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Pain in extremity,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Pain in extremity,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Pain in extremity,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Pain in extremity,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Pain in extremity,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.77 [0.02 to 4.21] | 0.39 [0.05 to 1.39]
  Pain in extremity,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Pain in extremity,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.51 [0.01 to 2.82] | 0.31 [0.04 to 1.13]
  Pain in extremity,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Pain in extremity,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.80 [0.10 to 2.86] | 0.29 [0.00 to 1.82] | 0.34 [0.07 to 0.99]
  Pain in extremity,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Pain in extremity,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.72 [0.09 to 2.59] | 0.24 [0.00 to 2.15] | 0.30 [0.06 to 0.87]
  Pain in extremity,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Pain in extremity,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.72 [0.09 to 2.57] | 0.23 [0.00 to 2.24] | 0.29 [0.06 to 0.84]
  Pain in extremity,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.72 [0.09 to 2.57] | 0.22 [0.00 to 2.33] | 0.28 [0.06 to 0.82]
  Pain in extremity,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.72 [0.09 to 2.57] | 0.22 [0.00 to 2.33] | 0.28 [0.06 to 0.82]
  Pain in extremity,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.72 [0.09 to 2.57] | 0.22 [0.00 to 2.33] | 0.28 [0.06 to 0.82]
  Pain in extremity,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.72 [0.09 to 2.57] | 0.22 [0.00 to 2.33] | 0.28 [0.06 to 0.82]
  Pain in extremity,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.72 [0.09 to 2.57] | 0.22 [0.00 to 2.33] | 0.28 [0.06 to 0.82]
  Rheumatic disorder,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rheumatic disorder,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Rheumatic disorder,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Rheumatic disorder,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Rheumatic disorder,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Rheumatic disorder,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Rheumatic disorder,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Rheumatic disorder,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Rheumatic disorder,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Rheumatic disorder,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Rheumatic disorder,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Rheumatic disorder,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Rheumatic disorder,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Rheumatic disorder,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.72 [0.00 to 9.03] | 0.00 [0.00 to 0.88] | 0.20 [0.00 to 1.39]
  Rheumatic disorder,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Rheumatic disorder,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.84] | 0.19 [0.00 to 1.34]
  Rheumatic disorder,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Rheumatic disorder,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Rheumatic disorder,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Rheumatic disorder,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Rheumatic disorder,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Synovial cyst,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Synovial cyst,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Synovial cyst,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Synovial cyst,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Synovial cyst,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Synovial cyst,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Synovial cyst,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Synovial cyst,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Synovial cyst,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Synovial cyst,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.00 to 22.01] | 0.16 [0.00 to 1.34]
  Synovial cyst,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Synovial cyst,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 8.11] | 0.11 [0.00 to 0.84]
  Synovial cyst,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Synovial cyst,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.10 [0.00 to 0.70]
  Synovial cyst,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Synovial cyst,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.10 [0.00 to 0.66]
  Synovial cyst,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Synovial cyst,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Synovial cyst,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Synovial cyst,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Synovial cyst,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]

48. Primary Outcome: Cumulative Percentage of Subjects Reporting Musculoskeletal and Connective Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were arthropathy and myalgia.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 4.55 [0.00 to 86.65]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 0.81 [0.02 to 4.45]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Any,Weeks 40-52 | 0.72 [0.02 to 3.94]
  Arthropathy,Weeks 40-46: number analyzed (Participants) | 3
  Arthropathy,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Arthropathy,Weeks 40-47: number analyzed (Participants) | 22
  Arthropathy,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Arthropathy,Weeks 40-48: number analyzed (Participants) | 47
  Arthropathy,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Arthropathy,Weeks 40-49: number analyzed (Participants) | 81
  Arthropathy,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Arthropathy,Weeks 40-50: number analyzed (Participants) | 123
  Arthropathy,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Arthropathy,Weeks 40-51: number analyzed (Participants) | 135
  Arthropathy,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Arthropathy,Weeks 40-52 | 0.00 [0.00 to 2.62]
  Myalgia,Weeks 40-46: number analyzed (Participants) | 3
  Myalgia,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Myalgia,Weeks 40-47: number analyzed (Participants) | 22
  Myalgia,Weeks 40-47 | 4.55 [0.00 to 86.65]
  Myalgia,Weeks 40-48: number analyzed (Participants) | 47
  Myalgia,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Myalgia,Weeks 40-49: number analyzed (Participants) | 81
  Myalgia,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Myalgia,Weeks 40-50: number analyzed (Participants) | 123
  Myalgia,Weeks 40-50 | 0.81 [0.02 to 4.45]
  Myalgia,Weeks 40-51: number analyzed (Participants) | 135
  Myalgia,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Myalgia,Weeks 40-52 | 0.72 [0.02 to 3.94]

49. Primary Outcome: Cumulative Percentage of Subjects Reporting Nervous System Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were febrile convulsion and headache.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 6.83 [1.53 to 18.20] |  | 6.83 [1.53 to 18.20]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 5.67 [0.00 to 68.10] | 6.37 [1.38 to 17.25] | 1.92 [0.05 to 10.26] | 5.54 [3.25 to 8.74]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 6.40 [0.00 to 85.72] | 6.45 [1.56 to 16.67] | 5.38 [0.40 to 20.90] | 6.17 [4.19 to 8.70]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 8.17 [0.32 to 34.96] | 6.47 [1.76 to 15.84] | 4.10 [1.79 to 7.92] | 6.30 [4.05 to 9.28]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 9.57 [0.70 to 34.96] | 6.80 [1.93 to 16.33] | 6.57 [1.02 to 20.19] | 7.60 [4.91 to 11.12]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 8.77 [1.25 to 27.02] | 7.61 [1.89 to 19.29] | 6.95 [0.84 to 23.06] | 7.69 [5.20 to 10.88]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 8.21 [1.64 to 22.61] | 7.91 [1.75 to 21.01] | 6.86 [1.15 to 20.43] | 7.57 [5.29 to 10.42]
  Any,Weeks 40-48 | 8.21 [1.64 to 22.61] | 7.91 [1.75 to 21.01] | 7.95 [0.59 to 29.68] | 8.02 [5.33 to 11.49]
  Any,Weeks 40-49 | 8.21 [1.64 to 22.61] | 7.91 [1.75 to 21.01] | 7.95 [0.59 to 29.68] | 8.02 [5.33 to 11.49]
  Any,Weeks 40-50 | 8.21 [1.64 to 22.61] | 7.91 [1.75 to 21.01] | 7.95 [0.59 to 29.68] | 8.02 [5.33 to 11.49]
  Any,Weeks 40-51 | 8.21 [1.64 to 22.61] | 7.91 [1.75 to 21.01] | 7.95 [0.59 to 29.68] | 8.02 [5.33 to 11.49]
  Any,Weeks 40-52 | 8.21 [1.64 to 22.61] | 7.91 [1.75 to 21.01] | 7.95 [0.59 to 29.68] | 8.02 [5.33 to 11.49]
  Febrile convulsion,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Febrile convulsion,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Febrile convulsion,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Febrile convulsion,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Febrile convulsion,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Febrile convulsion,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Febrile convulsion,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Febrile convulsion,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Febrile convulsion,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Febrile convulsion,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Febrile convulsion,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Febrile convulsion,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.42]
  Febrile convulsion,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Febrile convulsion,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.00 [0.00 to 0.37]
  Febrile convulsion,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Febrile convulsion,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.00 [0.00 to 0.35]
  Febrile convulsion,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.35]
  Febrile convulsion,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.35]
  Febrile convulsion,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.35]
  Febrile convulsion,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.35]
  Febrile convulsion,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.00 [0.00 to 0.35]
  Headache,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Headache,Weeks 40-40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Headache,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Headache,Weeks 40-41 |  | 6.21 [1.37 to 16.71] |  | 6.21 [1.37 to 16.71]
  Headache,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Headache,Weeks 40-42 | 4.96 [0.48 to 18.09] | 5.88 [1.30 to 15.88] | 1.92 [0.05 to 10.26] | 5.04 [3.10 to 7.67]
  Headache,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Headache,Weeks 40-43 | 5.81 [0.00 to 63.02] | 5.99 [1.42 to 15.70] | 5.38 [0.40 to 20.90] | 5.78 [3.93 to 8.15]
  Headache,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Headache,Weeks 40-44 | 7.69 [0.39 to 31.51] | 6.03 [1.58 to 15.11] | 4.10 [1.79 to 7.92] | 5.98 [3.97 to 8.61]
  Headache,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Headache,Weeks 40-45 | 8.51 [1.02 to 27.75] | 6.40 [1.59 to 16.37] | 5.71 [2.34 to 11.38] | 6.80 [4.81 to 9.30]
  Headache,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Headache,Weeks 40-46 | 7.79 [1.46 to 22.06] | 7.25 [1.39 to 20.44] | 6.24 [1.71 to 15.26] | 6.99 [5.02 to 9.44]
  Headache,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Headache,Weeks 40-47 | 7.29 [1.66 to 19.22] | 7.55 [1.25 to 22.42] | 6.18 [2.16 to 13.41] | 6.90 [5.02 to 9.21]
  Headache,Weeks 40-48 | 7.29 [1.66 to 19.22] | 7.55 [1.25 to 22.42] | 7.28 [1.08 to 22.49] | 7.36 [5.12 to 10.18]
  Headache,Weeks 40-49 | 7.29 [1.66 to 19.22] | 7.55 [1.25 to 22.42] | 7.28 [1.08 to 22.49] | 7.36 [5.12 to 10.18]
  Headache,Weeks 40-50 | 7.29 [1.66 to 19.22] | 7.55 [1.25 to 22.42] | 7.28 [1.08 to 22.49] | 7.36 [5.12 to 10.18]
  Headache,Weeks 40-51 | 7.29 [1.66 to 19.22] | 7.55 [1.25 to 22.42] | 7.28 [1.08 to 22.49] | 7.36 [5.12 to 10.18]
  Headache,Weeks 40-52 | 7.29 [1.66 to 19.22] | 7.55 [1.25 to 22.42] | 7.28 [1.08 to 22.49] | 7.36 [5.12 to 10.18]
  Aphonia,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Aphonia,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Aphonia,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Aphonia,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Aphonia,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Aphonia,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Aphonia,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Aphonia,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Aphonia,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Aphonia,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Aphonia,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Aphonia,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 8.11] | 0.11 [0.00 to 0.84]
  Aphonia,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Aphonia,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.10 [0.00 to 0.70]
  Aphonia,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Aphonia,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.10 [0.00 to 0.66]
  Aphonia,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Aphonia,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Aphonia,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Aphonia,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Aphonia,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Dizziness,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dizziness,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Dizziness,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Dizziness,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Dizziness,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Dizziness,Weeks 40-42 | 0.71 [0.00 to 97.40] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.41]
  Dizziness,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Dizziness,Weeks 40-43 | 0.58 [0.00 to 86.72] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.68]
  Dizziness,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Dizziness,Weeks 40-44 | 0.48 [0.00 to 12.12] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.20]
  Dizziness,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Dizziness,Weeks 40-45 | 1.06 [0.00 to 16.76] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 8.11] | 0.45 [0.02 to 2.20]
  Dizziness,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Dizziness,Weeks 40-46 | 0.97 [0.00 to 13.40] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.40 [0.02 to 1.85]
  Dizziness,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Dizziness,Weeks 40-47 | 0.91 [0.00 to 11.33] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.38 [0.02 to 1.72]
  Dizziness,Weeks 40-48 | 0.91 [0.00 to 11.33] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.38 [0.02 to 1.69]
  Dizziness,Weeks 40-49 | 0.91 [0.00 to 11.33] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.38 [0.02 to 1.69]
  Dizziness,Weeks 40-50 | 0.91 [0.00 to 11.33] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.38 [0.02 to 1.69]
  Dizziness,Weeks 40-51 | 0.91 [0.00 to 11.33] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.38 [0.02 to 1.69]
  Dizziness,Weeks 40-52 | 0.91 [0.00 to 11.33] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.38 [0.02 to 1.69]
  Poor quality sleep,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Poor quality sleep,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Poor quality sleep,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Poor quality sleep,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Poor quality sleep,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Poor quality sleep,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Poor quality sleep,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Poor quality sleep,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Poor quality sleep,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Poor quality sleep,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Poor quality sleep,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Poor quality sleep,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Poor quality sleep,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Poor quality sleep,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Poor quality sleep,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Poor quality sleep,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Poor quality sleep,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Poor quality sleep,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Poor quality sleep,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Poor quality sleep,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Poor quality sleep,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Somnolence,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Somnolence,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Somnolence,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Somnolence,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Somnolence,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Somnolence,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Somnolence,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Somnolence,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Somnolence,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Somnolence,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Somnolence,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Somnolence,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 8.11] | 0.11 [0.00 to 0.84]
  Somnolence,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Somnolence,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.10 [0.00 to 0.70]
  Somnolence,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Somnolence,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.10 [0.00 to 0.66]
  Somnolence,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Somnolence,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Somnolence,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Somnolence,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Somnolence,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Tremor,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tremor,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Tremor,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Tremor,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Tremor,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Tremor,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Tremor,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Tremor,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Tremor,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Tremor,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Tremor,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Tremor,Weeks 40-45 | 0.35 [0.00 to 5.88] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.79]
  Tremor,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Tremor,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.68]
  Tremor,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Tremor,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.64]
  Tremor,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Tremor,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Tremor,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Tremor,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Tremor,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]

50. Primary Outcome: Cumulative Percentage of Subjects Reporting Nervous System Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were febrile convulsion and headache.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

51. Primary Outcome: Cumulative Percentage of Subjects Reporting Psychiatric Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEI listed on the ADR card was irritability.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 1.96 [0.00 to 35.78] | 1.92 [0.05 to 10.26] | 1.26 [0.02 to 7.26]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.00 [0.00 to 2.12] | 2.30 [0.00 to 37.38] | 3.85 [0.30 to 15.16] | 1.93 [0.19 to 7.28]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.48 [0.00 to 15.39] | 2.16 [0.00 to 32.16] | 3.59 [1.46 to 7.26] | 2.05 [0.51 to 5.40]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.71 [0.00 to 7.80] | 2.00 [0.00 to 27.03] | 2.29 [0.34 to 7.45] | 1.70 [0.55 to 3.92]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.97 [0.00 to 8.41] | 1.81 [0.00 to 21.35] | 2.40 [0.19 to 9.65] | 1.80 [0.71 to 3.72]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.91 [0.00 to 7.18] | 1.80 [0.00 to 20.98] | 2.52 [0.54 to 7.09] | 1.82 [0.78 to 3.57]
  Any,Weeks 40-48 | 0.91 [0.00 to 7.18] | 1.80 [0.00 to 20.98] | 2.43 [0.40 to 7.64] | 1.79 [0.76 to 3.54]
  Any,Weeks 40-49 | 0.91 [0.00 to 7.18] | 1.80 [0.00 to 20.98] | 2.43 [0.40 to 7.64] | 1.79 [0.76 to 3.54]
  Any,Weeks 40-50 | 0.91 [0.00 to 7.18] | 1.80 [0.00 to 20.98] | 2.43 [0.40 to 7.64] | 1.79 [0.76 to 3.54]
  Any,Weeks 40-51 | 0.91 [0.00 to 7.18] | 1.80 [0.00 to 20.98] | 2.43 [0.40 to 7.64] | 1.79 [0.76 to 3.54]
  Any,Weeks 40-52 | 0.91 [0.00 to 7.18] | 1.80 [0.00 to 20.98] | 2.43 [0.40 to 7.64] | 1.79 [0.76 to 3.54]
  Irritability,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Irritability,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Irritability,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Irritability,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Irritability,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Irritability,Weeks 40-42 | 0.00 [0.00 to 2.58] | 1.47 [0.00 to 28.09] | 1.92 [0.05 to 10.26] | 1.01 [0.03 to 5.49]
  Irritability,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Irritability,Weeks 40-43 | 0.00 [0.00 to 2.12] | 1.84 [0.00 to 31.06] | 3.85 [0.30 to 15.16] | 1.73 [0.18 to 6.51]
  Irritability,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Irritability,Weeks 40-44 | 0.48 [0.00 to 15.39] | 1.72 [0.00 to 26.54] | 3.59 [1.46 to 7.26] | 1.89 [0.49 to 4.92]
  Irritability,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Irritability,Weeks 40-45 | 0.71 [0.00 to 7.80] | 1.60 [0.00 to 22.17] | 2.29 [0.34 to 7.45] | 1.59 [0.53 to 3.62]
  Irritability,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Irritability,Weeks 40-46 | 0.97 [0.00 to 8.41] | 1.45 [0.00 to 17.40] | 2.40 [0.19 to 9.65] | 1.70 [0.67 to 3.51]
  Irritability,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Irritability,Weeks 40-47 | 0.91 [0.00 to 7.18] | 1.44 [0.00 to 17.09] | 2.52 [0.54 to 7.09] | 1.72 [0.75 to 3.37]
  Irritability,Weeks 40-48 | 0.91 [0.00 to 7.18] | 1.44 [0.00 to 17.09] | 2.43 [0.40 to 7.64] | 1.70 [0.73 to 3.34]
  Irritability,Weeks 40-49 | 0.91 [0.00 to 7.18] | 1.44 [0.00 to 17.09] | 2.43 [0.40 to 7.64] | 1.70 [0.73 to 3.34]
  Irritability,Weeks 40-50 | 0.91 [0.00 to 7.18] | 1.44 [0.00 to 17.09] | 2.43 [0.40 to 7.64] | 1.70 [0.73 to 3.34]
  Irritability,Weeks 40-51 | 0.91 [0.00 to 7.18] | 1.44 [0.00 to 17.09] | 2.43 [0.40 to 7.64] | 1.70 [0.73 to 3.34]
  Irritability,Weeks 40-52 | 0.91 [0.00 to 7.18] | 1.44 [0.00 to 17.09] | 2.43 [0.40 to 7.64] | 1.70 [0.73 to 3.34]
  Insomnia,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Insomnia,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Insomnia,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Insomnia,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Insomnia,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Insomnia,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Insomnia,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Insomnia,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Insomnia,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Insomnia,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Insomnia,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Insomnia,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Insomnia,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Insomnia,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Insomnia,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Insomnia,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Insomnia,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Insomnia,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Insomnia,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Insomnia,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Insomnia,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Mood swings,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Mood swings,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Mood swings,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Mood swings,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Mood swings,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Mood swings,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Mood swings,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Mood swings,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Mood swings,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Mood swings,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.00 to 22.01] | 0.16 [0.00 to 1.34]
  Mood swings,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Mood swings,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 8.11] | 0.11 [0.00 to 0.84]
  Mood swings,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Mood swings,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 5.63] | 0.10 [0.00 to 0.70]
  Mood swings,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Mood swings,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.10 [0.00 to 0.66]
  Mood swings,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Mood swings,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Mood swings,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Mood swings,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Mood swings,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Sleep disorder,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Sleep disorder,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Sleep disorder,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Sleep disorder,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Sleep disorder,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Sleep disorder,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Sleep disorder,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Sleep disorder,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Sleep disorder,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Sleep disorder,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Sleep disorder,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Sleep disorder,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Sleep disorder,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Sleep disorder,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Sleep disorder,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Sleep disorder,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Sleep disorder,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Sleep disorder,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Sleep disorder,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Sleep disorder,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Sleep disorder,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]

52. Primary Outcome: Cumulative Percentage of Subjects Reporting Psychiatric Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEI listed on the ADR card was irritability.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 4.26 [0.00 to 40.16]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 4.94 [0.59 to 16.86]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 3.25 [0.35 to 11.68]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 2.96 [0.32 to 10.76]
  Any,Weeks 40-52 | 2.88 [0.31 to 10.46]
  Irritability,Weeks 40-46: number analyzed (Participants) | 3
  Irritability,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Irritability,Weeks 40-47: number analyzed (Participants) | 22
  Irritability,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Irritability,Weeks 40-48: number analyzed (Participants) | 47
  Irritability,Weeks 40-48 | 4.26 [0.00 to 40.16]
  Irritability,Weeks 40-49: number analyzed (Participants) | 81
  Irritability,Weeks 40-49 | 4.94 [0.59 to 16.86]
  Irritability,Weeks 40-50: number analyzed (Participants) | 123
  Irritability,Weeks 40-50 | 3.25 [0.35 to 11.68]
  Irritability,Weeks 40-51: number analyzed (Participants) | 135
  Irritability,Weeks 40-51 | 2.96 [0.32 to 10.76]
  Irritability,Weeks 40-52 | 2.88 [0.31 to 10.46]

53. Primary Outcome: Cumulative Percentage of Subjects Reporting Respiratory, Thoracic and Mediastinal Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were cough, dysphonia, epistaxis, nasal congestion, oropharyngeal pain, rhinorrhoea, and wheezing.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 8.57 [0.31 to 37.07] |  | 8.57 [0.31 to 37.07]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 11.18 [1.36 to 35.08] |  | 11.18 [1.36 to 35.08]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 9.93 [0.87 to 34.53] | 10.78 [1.35 to 33.71] | 26.92 [0.28 to 88.26] | 12.59 [6.42 to 21.49]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 11.63 [0.00 to 88.89] | 11.52 [1.74 to 33.76] | 26.15 [8.21 to 52.91] | 15.22 [7.32 to 26.68]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 13.94 [1.58 to 43.03] | 11.21 [2.04 to 30.99] | 23.59 [17.82 to 30.18] | 15.91 [9.50 to 24.32]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 15.60 [2.23 to 44.35] | 12.00 [2.45 to 31.67] | 22.57 [15.58 to 30.91] | 17.35 [12.31 to 23.41]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 14.94 [3.31 to 37.29] | 11.59 [3.01 to 27.99] | 22.30 [15.71 to 30.10] | 17.08 [12.48 to 22.55]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 14.59 [4.03 to 33.60] | 11.51 [3.04 to 27.60] | 22.65 [13.27 to 34.59] | 17.15 [12.50 to 22.67]
  Any,Weeks 40-48 | 14.59 [4.03 to 33.60] | 11.51 [3.04 to 27.60] | 22.96 [12.87 to 35.99] | 17.36 [12.64 to 22.96]
  Any,Weeks 40-49 | 14.59 [4.03 to 33.60] | 11.51 [3.04 to 27.60] | 22.96 [12.87 to 35.99] | 17.36 [12.64 to 22.96]
  Any,Weeks 40-50 | 14.59 [4.03 to 33.60] | 11.51 [3.04 to 27.60] | 22.96 [12.87 to 35.99] | 17.36 [12.64 to 22.96]
  Any,Weeks 40-51 | 14.59 [4.03 to 33.60] | 11.51 [3.04 to 27.60] | 22.96 [12.87 to 35.99] | 17.36 [12.64 to 22.96]
  Any,Weeks 40-52 | 14.59 [4.03 to 33.60] | 11.51 [3.04 to 27.60] | 22.96 [12.87 to 35.99] | 17.36 [12.64 to 22.96]
  Cough,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Cough,Weeks 40-40 |  | 7.14 [0.27 to 31.53] |  | 7.14 [0.27 to 31.53]
  Cough,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Cough,Weeks 40-41 |  | 4.35 [0.09 to 22.77] |  | 4.35 [0.09 to 22.77]
  Cough,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Cough,Weeks 40-42 | 2.84 [0.04 to 16.88] | 4.41 [0.22 to 19.28] | 15.38 [0.28 to 63.30] | 5.29 [1.74 to 11.93]
  Cough,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Cough,Weeks 40-43 | 3.49 [0.05 to 20.00] | 4.15 [0.19 to 18.61] | 15.38 [9.66 to 22.76] | 6.74 [1.90 to 16.23]
  Cough,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Cough,Weeks 40-44 | 3.37 [1.36 to 6.81] | 3.88 [0.14 to 18.39] | 14.36 [9.76 to 20.08] | 6.93 [2.42 to 14.99]
  Cough,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Cough,Weeks 40-45 | 3.90 [1.27 to 8.90] | 4.40 [0.49 to 15.44] | 10.86 [4.37 to 21.39] | 6.80 [3.44 to 11.85]
  Cough,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Cough,Weeks 40-46 | 3.57 [1.80 to 6.30] | 3.99 [0.39 to 14.69] | 10.55 [4.21 to 20.90] | 6.59 [3.39 to 11.38]
  Cough,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Cough,Weeks 40-47 | 3.65 [1.89 to 6.30] | 3.96 [0.38 to 14.67] | 10.53 [3.58 to 22.65] | 6.61 [3.43 to 11.32]
  Cough,Weeks 40-48 | 3.65 [1.89 to 6.30] | 3.96 [0.38 to 14.67] | 10.60 [3.48 to 23.18] | 6.70 [3.53 to 11.37]
  Cough,Weeks 40-49 | 3.65 [1.89 to 6.30] | 3.96 [0.38 to 14.67] | 10.60 [3.48 to 23.18] | 6.70 [3.53 to 11.37]
  Cough,Weeks 40-50 | 3.65 [1.89 to 6.30] | 3.96 [0.38 to 14.67] | 10.60 [3.48 to 23.18] | 6.70 [3.53 to 11.37]
  Cough,Weeks 40-51 | 3.65 [1.89 to 6.30] | 3.96 [0.38 to 14.67] | 10.60 [3.48 to 23.18] | 6.70 [3.53 to 11.37]
  Cough,Weeks 40-52 | 3.65 [1.89 to 6.30] | 3.96 [0.38 to 14.67] | 10.60 [3.48 to 23.18] | 6.70 [3.53 to 11.37]
  Dysphonia,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dysphonia,Weeks 40-40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Dysphonia,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Dysphonia,Weeks 40-41 |  | 2.48 [0.14 to 10.81] |  | 2.48 [0.14 to 10.81]
  Dysphonia,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Dysphonia,Weeks 40-42 | 1.42 [0.02 to 8.68] | 3.43 [0.09 to 17.62] | 3.85 [0.11 to 19.24] | 2.77 [1.05 to 5.86]
  Dysphonia,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Dysphonia,Weeks 40-43 | 1.74 [0.03 to 10.34] | 3.23 [0.16 to 14.35] | 3.08 [0.24 to 12.22] | 2.70 [1.40 to 4.67]
  Dysphonia,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Dysphonia,Weeks 40-44 | 1.44 [0.30 to 4.16] | 3.02 [0.26 to 11.63] | 2.56 [0.59 to 7.01] | 2.36 [1.33 to 3.87]
  Dysphonia,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Dysphonia,Weeks 40-45 | 1.06 [0.14 to 3.71] | 3.60 [0.21 to 15.27] | 2.57 [1.18 to 4.83] | 2.38 [1.29 to 4.00]
  Dysphonia,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Dysphonia,Weeks 40-46 | 0.97 [0.07 to 4.10] | 3.26 [0.40 to 11.22] | 2.40 [1.16 to 4.37] | 2.20 [1.29 to 3.49]
  Dysphonia,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Dysphonia,Weeks 40-47 | 1.22 [0.33 to 3.08] | 3.24 [0.42 to 10.98] | 2.29 [1.10 to 4.17] | 2.20 [1.38 to 3.33]
  Dysphonia,Weeks 40-48 | 1.22 [0.33 to 3.08] | 3.24 [0.42 to 10.98] | 2.21 [1.06 to 4.02] | 2.17 [1.35 to 3.29]
  Dysphonia,Weeks 40-49 | 1.22 [0.33 to 3.08] | 3.24 [0.42 to 10.98] | 2.21 [1.06 to 4.02] | 2.17 [1.35 to 3.29]
  Dysphonia,Weeks 40-50 | 1.22 [0.33 to 3.08] | 3.24 [0.42 to 10.98] | 2.21 [1.06 to 4.02] | 2.17 [1.35 to 3.29]
  Dysphonia,Weeks 40-51 | 1.22 [0.33 to 3.08] | 3.24 [0.42 to 10.98] | 2.21 [1.06 to 4.02] | 2.17 [1.35 to 3.29]
  Dysphonia,Weeks 40-52 | 1.22 [0.33 to 3.08] | 3.24 [0.42 to 10.98] | 2.21 [1.06 to 4.02] | 2.17 [1.35 to 3.29]
  Epistaxis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Epistaxis,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Epistaxis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Epistaxis,Weeks 40-41 |  | 1.24 [0.01 to 8.05] |  | 1.24 [0.01 to 8.05]
  Epistaxis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Epistaxis,Weeks 40-42 | 0.00 [0.00 to 2.58] | 1.47 [0.01 to 10.56] | 0.00 [0.00 to 6.85] | 0.76 [0.04 to 3.42]
  Epistaxis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Epistaxis,Weeks 40-43 | 0.58 [0.00 to 86.72] | 1.84 [0.00 to 14.96] | 0.00 [0.00 to 2.80] | 0.96 [0.08 to 3.95]
  Epistaxis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Epistaxis,Weeks 40-44 | 0.48 [0.00 to 12.12] | 1.72 [0.01 to 12.04] | 0.00 [0.00 to 1.87] | 0.79 [0.08 to 2.98]
  Epistaxis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Epistaxis,Weeks 40-45 | 0.35 [0.00 to 5.88] | 1.60 [0.03 to 9.43] | 1.14 [0.00 to 12.47] | 1.02 [0.32 to 2.40]
  Epistaxis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Epistaxis,Weeks 40-46 | 0.32 [0.00 to 4.64] | 1.45 [0.07 to 6.84] | 0.96 [0.00 to 9.17] | 0.90 [0.31 to 2.01]
  Epistaxis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Epistaxis,Weeks 40-47 | 0.30 [0.00 to 3.90] | 1.44 [0.07 to 6.68] | 0.92 [0.00 to 7.97] | 0.86 [0.31 to 1.90]
  Epistaxis,Weeks 40-48 | 0.30 [0.00 to 3.90] | 1.44 [0.07 to 6.68] | 0.88 [0.00 to 7.39] | 0.85 [0.31 to 1.86]
  Epistaxis,Weeks 40-49 | 0.30 [0.00 to 3.90] | 1.44 [0.07 to 6.68] | 0.88 [0.00 to 7.39] | 0.85 [0.31 to 1.86]
  Epistaxis,Weeks 40-50 | 0.30 [0.00 to 3.90] | 1.44 [0.07 to 6.68] | 0.88 [0.00 to 7.39] | 0.85 [0.31 to 1.86]
  Epistaxis,Weeks 40-51 | 0.30 [0.00 to 3.90] | 1.44 [0.07 to 6.68] | 0.88 [0.00 to 7.39] | 0.85 [0.31 to 1.86]
  Epistaxis,Weeks 40-52 | 0.30 [0.00 to 3.90] | 1.44 [0.07 to 6.68] | 0.88 [0.00 to 7.39] | 0.85 [0.31 to 1.86]
  Nasal congestion,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Nasal congestion,Weeks 40-40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Nasal congestion,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Nasal congestion,Weeks 40-41 |  | 3.73 [0.00 to 29.85] |  | 3.73 [0.00 to 29.85]
  Nasal congestion,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Nasal congestion,Weeks 40-42 | 2.84 [0.04 to 16.88] | 3.92 [0.07 to 21.23] | 15.38 [0.28 to 63.30] | 5.04 [1.52 to 11.85]
  Nasal congestion,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Nasal congestion,Weeks 40-43 | 2.91 [0.45 to 9.29] | 4.15 [0.19 to 18.61] | 10.77 [0.72 to 39.43] | 5.39 [1.89 to 11.74]
  Nasal congestion,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Nasal congestion,Weeks 40-44 | 3.85 [0.21 to 16.51] | 4.31 [0.34 to 16.84] | 10.26 [6.38 to 15.40] | 5.98 [2.91 to 10.73]
  Nasal congestion,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Nasal congestion,Weeks 40-45 | 3.55 [0.72 to 10.14] | 4.00 [0.27 to 16.33] | 8.00 [5.38 to 11.35] | 5.44 [3.17 to 8.64]
  Nasal congestion,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Nasal congestion,Weeks 40-46 | 3.25 [0.46 to 10.64] | 3.62 [0.17 to 16.30] | 8.15 [5.71 to 11.21] | 5.39 [3.02 to 8.80]
  Nasal congestion,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Nasal congestion,Weeks 40-47 | 3.04 [0.31 to 11.21] | 3.60 [0.16 to 16.32] | 8.01 [5.64 to 10.96] | 5.27 [2.90 to 8.70]
  Nasal congestion,Weeks 40-48 | 3.04 [0.31 to 11.21] | 3.60 [0.16 to 16.32] | 8.17 [5.82 to 11.08] | 5.38 [3.01 to 8.77]
  Nasal congestion,Weeks 40-49 | 3.04 [0.31 to 11.21] | 3.60 [0.16 to 16.32] | 8.17 [5.82 to 11.08] | 5.38 [3.01 to 8.77]
  Nasal congestion,Weeks 40-50 | 3.04 [0.31 to 11.21] | 3.60 [0.16 to 16.32] | 8.17 [5.82 to 11.08] | 5.38 [3.01 to 8.77]
  Nasal congestion,Weeks 40-51 | 3.04 [0.31 to 11.21] | 3.60 [0.16 to 16.32] | 8.17 [5.82 to 11.08] | 5.38 [3.01 to 8.77]
  Nasal congestion,Weeks 40-52 | 3.04 [0.31 to 11.21] | 3.60 [0.16 to 16.32] | 8.17 [5.82 to 11.08] | 5.38 [3.01 to 8.77]
  Oropharyngeal pain,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Oropharyngeal pain,Weeks 40-40 |  | 5.71 [0.22 to 25.74] |  | 5.71 [0.22 to 25.74]
  Oropharyngeal pain,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Oropharyngeal pain,Weeks 40-41 |  | 5.59 [0.11 to 28.89] |  | 5.59 [0.11 to 28.89]
  Oropharyngeal pain,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Oropharyngeal pain,Weeks 40-42 | 3.55 [0.04 to 20.80] | 5.88 [0.61 to 20.68] | 1.92 [0.05 to 10.26] | 4.53 [2.13 to 8.35]
  Oropharyngeal pain,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Oropharyngeal pain,Weeks 40-43 | 3.49 [0.05 to 20.00] | 5.53 [0.42 to 21.36] | 5.38 [0.40 to 20.90] | 4.82 [2.86 to 7.54]
  Oropharyngeal pain,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Oropharyngeal pain,Weeks 40-44 | 3.37 [1.25 to 7.18] | 5.17 [0.25 to 22.45] | 4.62 [2.13 to 8.58] | 4.41 [2.85 to 6.48]
  Oropharyngeal pain,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Oropharyngeal pain,Weeks 40-45 | 3.19 [1.05 to 7.26] | 5.60 [0.77 to 18.10] | 4.86 [2.65 to 8.09] | 4.54 [3.24 to 6.16]
  Oropharyngeal pain,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Oropharyngeal pain,Weeks 40-46 | 3.25 [1.24 to 6.82] | 5.43 [0.80 to 17.17] | 5.28 [1.62 to 12.31] | 4.70 [3.28 to 6.48]
  Oropharyngeal pain,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Oropharyngeal pain,Weeks 40-47 | 3.04 [1.09 to 6.60] | 5.40 [0.77 to 17.24] | 5.26 [2.14 to 10.55] | 4.60 [3.24 to 6.31]
  Oropharyngeal pain,Weeks 40-48 | 3.04 [1.09 to 6.60] | 5.40 [0.77 to 17.24] | 5.74 [1.33 to 15.20] | 4.81 [3.17 to 6.97]
  Oropharyngeal pain,Weeks 40-49 | 3.04 [1.09 to 6.60] | 5.40 [0.77 to 17.24] | 5.74 [1.33 to 15.20] | 4.81 [3.17 to 6.97]
  Oropharyngeal pain,Weeks 40-50 | 3.04 [1.09 to 6.60] | 5.40 [0.77 to 17.24] | 5.74 [1.33 to 15.20] | 4.81 [3.17 to 6.97]
  Oropharyngeal pain,Weeks 40-51 | 3.04 [1.09 to 6.60] | 5.40 [0.77 to 17.24] | 5.74 [1.33 to 15.20] | 4.81 [3.17 to 6.97]
  Oropharyngeal pain,Weeks 40-52 | 3.04 [1.09 to 6.60] | 5.40 [0.77 to 17.24] | 5.74 [1.33 to 15.20] | 4.81 [3.17 to 6.97]
  Rhinorrhoea,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rhinorrhoea,Weeks 40-40 |  | 4.29 [0.17 to 19.69] |  | 4.29 [0.17 to 19.69]
  Rhinorrhoea,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Rhinorrhoea,Weeks 40-41 |  | 5.59 [1.62 to 13.39] |  | 5.59 [1.62 to 13.39]
  Rhinorrhoea,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Rhinorrhoea,Weeks 40-42 | 3.55 [0.00 to 90.30] | 5.88 [1.30 to 15.88] | 7.69 [0.19 to 36.17] | 5.29 [2.45 to 9.80]
  Rhinorrhoea,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Rhinorrhoea,Weeks 40-43 | 5.81 [0.00 to 99.97] | 5.53 [1.56 to 13.44] | 9.23 [0.64 to 34.38] | 6.55 [2.99 to 12.19]
  Rhinorrhoea,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Rhinorrhoea,Weeks 40-44 | 7.69 [0.00 to 56.43] | 5.17 [1.62 to 11.95] | 9.74 [5.97 to 14.80] | 7.40 [3.92 to 12.50]
  Rhinorrhoea,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Rhinorrhoea,Weeks 40-45 | 9.93 [0.04 to 55.87] | 5.60 [1.92 to 12.31] | 10.00 [7.01 to 13.72] | 8.73 [5.35 to 13.27]
  Rhinorrhoea,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Rhinorrhoea,Weeks 40-46 | 9.74 [0.09 to 49.87] | 5.43 [2.16 to 11.03] | 9.83 [6.20 to 14.62] | 8.59 [5.53 to 12.59]
  Rhinorrhoea,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Rhinorrhoea,Weeks 40-47 | 9.12 [0.19 to 42.57] | 5.40 [2.17 to 10.88] | 10.07 [4.58 to 18.56] | 8.52 [5.66 to 12.21]
  Rhinorrhoea,Weeks 40-48 | 9.12 [0.19 to 42.57] | 5.40 [2.17 to 10.88] | 10.38 [4.53 to 19.56] | 8.68 [5.80 to 12.38]
  Rhinorrhoea,Weeks 40-49 | 9.12 [0.19 to 42.57] | 5.40 [2.17 to 10.88] | 10.38 [4.53 to 19.56] | 8.68 [5.80 to 12.38]
  Rhinorrhoea,Weeks 40-50 | 9.12 [0.19 to 42.57] | 5.40 [2.17 to 10.88] | 10.38 [4.53 to 19.56] | 8.68 [5.80 to 12.38]
  Rhinorrhoea,Weeks 40-51 | 9.12 [0.19 to 42.57] | 5.40 [2.17 to 10.88] | 10.38 [4.53 to 19.56] | 8.68 [5.80 to 12.38]
  Rhinorrhoea,Weeks 40-52 | 9.12 [0.19 to 42.57] | 5.40 [2.17 to 10.88] | 10.38 [4.53 to 19.56] | 8.68 [5.80 to 12.38]
  Wheezing,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Wheezing,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Wheezing,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Wheezing,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Wheezing,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Wheezing,Weeks 40-42 | 0.71 [0.01 to 4.40] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.50 [0.06 to 1.81]
  Wheezing,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Wheezing,Weeks 40-43 | 0.58 [0.00 to 20.94] | 1.38 [0.00 to 24.20] | 0.00 [0.00 to 2.80] | 0.77 [0.03 to 3.82]
  Wheezing,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Wheezing,Weeks 40-44 | 0.48 [0.00 to 3.76] | 1.29 [0.00 to 20.54] | 1.03 [0.00 to 11.81] | 0.94 [0.20 to 2.68]
  Wheezing,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Wheezing,Weeks 40-45 | 0.35 [0.00 to 5.12] | 1.20 [0.00 to 17.05] | 0.57 [0.03 to 2.60] | 0.68 [0.16 to 1.89]
  Wheezing,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Wheezing,Weeks 40-46 | 0.32 [0.00 to 5.39] | 1.09 [0.00 to 13.30] | 0.48 [0.06 to 1.72] | 0.60 [0.15 to 1.60]
  Wheezing,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Wheezing,Weeks 40-47 | 0.30 [0.00 to 5.54] | 1.08 [0.00 to 13.06] | 0.46 [0.06 to 1.64] | 0.57 [0.14 to 1.56]
  Wheezing,Weeks 40-48 | 0.30 [0.00 to 5.54] | 1.08 [0.00 to 13.06] | 0.44 [0.05 to 1.59] | 0.57 [0.14 to 1.53]
  Wheezing,Weeks 40-49 | 0.30 [0.00 to 5.54] | 1.08 [0.00 to 13.06] | 0.44 [0.05 to 1.59] | 0.57 [0.14 to 1.53]
  Wheezing,Weeks 40-50 | 0.30 [0.00 to 5.54] | 1.08 [0.00 to 13.06] | 0.44 [0.05 to 1.59] | 0.57 [0.14 to 1.53]
  Wheezing,Weeks 40-51 | 0.30 [0.00 to 5.54] | 1.08 [0.00 to 13.06] | 0.44 [0.05 to 1.59] | 0.57 [0.14 to 1.53]
  Wheezing,Weeks 40-52 | 0.30 [0.00 to 5.54] | 1.08 [0.00 to 13.06] | 0.44 [0.05 to 1.59] | 0.57 [0.14 to 1.53]
  Dry throat,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dry throat,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Dry throat,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Dry throat,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Dry throat,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Dry throat,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Dry throat,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Dry throat,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Dry throat,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Dry throat,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.29]
  Dry throat,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Dry throat,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.91]
  Dry throat,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Dry throat,Weeks 40-46 | 0.32 [0.00 to 10.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.81]
  Dry throat,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Dry throat,Weeks 40-47 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.78]
  Dry throat,Weeks 40-48 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Dry throat,Weeks 40-49 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Dry throat,Weeks 40-50 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Dry throat,Weeks 40-51 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Dry throat,Weeks 40-52 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Dyspnoea,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Dyspnoea,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Dyspnoea,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Dyspnoea,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Dyspnoea,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Dyspnoea,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.98 [0.00 to 19.61] | 0.00 [0.00 to 6.85] | 0.50 [0.00 to 3.97]
  Dyspnoea,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Dyspnoea,Weeks 40-43 | 0.00 [0.00 to 2.12] | 1.38 [0.00 to 24.20] | 0.00 [0.00 to 2.80] | 0.58 [0.00 to 4.52]
  Dyspnoea,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Dyspnoea,Weeks 40-44 | 0.00 [0.00 to 1.76] | 1.29 [0.00 to 20.54] | 0.00 [0.00 to 1.87] | 0.47 [0.00 to 3.29]
  Dyspnoea,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Dyspnoea,Weeks 40-45 | 0.00 [0.00 to 1.30] | 1.20 [0.00 to 17.05] | 0.00 [0.00 to 1.05] | 0.34 [0.00 to 2.41]
  Dyspnoea,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Dyspnoea,Weeks 40-46 | 0.00 [0.00 to 1.19] | 1.09 [0.00 to 13.30] | 0.00 [0.00 to 0.88] | 0.30 [0.00 to 2.08]
  Dyspnoea,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Dyspnoea,Weeks 40-47 | 0.00 [0.00 to 1.11] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.84] | 0.29 [0.00 to 2.00]
  Dyspnoea,Weeks 40-48 | 0.00 [0.00 to 1.11] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.28 [0.00 to 1.98]
  Dyspnoea,Weeks 40-49 | 0.00 [0.00 to 1.11] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.28 [0.00 to 1.98]
  Dyspnoea,Weeks 40-50 | 0.00 [0.00 to 1.11] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.28 [0.00 to 1.98]
  Dyspnoea,Weeks 40-51 | 0.00 [0.00 to 1.11] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.28 [0.00 to 1.98]
  Dyspnoea,Weeks 40-52 | 0.00 [0.00 to 1.11] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.28 [0.00 to 1.98]
  Increased upper airway secretion,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Increased upper airway secretion,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Increased upper airway secretion,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Increased upper airway secretion,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Increased upper airway secretion,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Increased upper airway secretion,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Increased upper airway secretion,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Increased upper airway secretion,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.77 [0.02 to 4.21] | 0.19 [0.00 to 1.28]
  Increased upper airway secretion,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Increased upper airway secretion,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.01 to 2.82] | 0.16 [0.00 to 0.87]
  Increased upper airway secretion,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Increased upper airway secretion,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 1.82] | 0.11 [0.00 to 0.63]
  Increased upper airway secretion,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Increased upper airway secretion,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.24 [0.00 to 2.15] | 0.10 [0.00 to 0.56]
  Increased upper airway secretion,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Increased upper airway secretion,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 2.24] | 0.10 [0.00 to 0.55]
  Increased upper airway secretion,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Increased upper airway secretion,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Increased upper airway secretion,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Increased upper airway secretion,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Increased upper airway secretion,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 2.33] | 0.09 [0.00 to 0.54]
  Sneezing,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Sneezing,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Sneezing,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Sneezing,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Sneezing,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Sneezing,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Sneezing,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Sneezing,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.77 [0.02 to 4.21] | 0.19 [0.00 to 1.28]
  Sneezing,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Sneezing,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.00 [0.00 to 1.58] | 1.03 [0.12 to 3.66] | 0.47 [0.05 to 1.73]
  Sneezing,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Sneezing,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.00 [0.00 to 1.46] | 0.57 [0.01 to 3.61] | 0.34 [0.04 to 1.23]
  Sneezing,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Sneezing,Weeks 40-46 | 0.32 [0.00 to 10.19] | 0.00 [0.00 to 1.33] | 0.48 [0.00 to 4.27] | 0.30 [0.03 to 1.13]
  Sneezing,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Sneezing,Weeks 40-47 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.46 [0.00 to 4.44] | 0.29 [0.03 to 1.10]
  Sneezing,Weeks 40-48 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 4.62] | 0.28 [0.03 to 1.09]
  Sneezing,Weeks 40-49 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 4.62] | 0.28 [0.03 to 1.09]
  Sneezing,Weeks 40-50 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 4.62] | 0.28 [0.03 to 1.09]
  Sneezing,Weeks 40-51 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 4.62] | 0.28 [0.03 to 1.09]
  Sneezing,Weeks 40-52 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 4.62] | 0.28 [0.03 to 1.09]
  Throat clearing,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Throat clearing,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Throat clearing,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Throat clearing,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Throat clearing,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Throat clearing,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Throat clearing,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Throat clearing,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Throat clearing,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Throat clearing,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Throat clearing,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Throat clearing,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.42]
  Throat clearing,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Throat clearing,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.00 [0.00 to 0.37]
  Throat clearing,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Throat clearing,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.23 [0.00 to 5.17] | 0.10 [0.00 to 0.66]
  Throat clearing,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Throat clearing,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Throat clearing,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Throat clearing,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]
  Throat clearing,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.22 [0.00 to 4.76] | 0.09 [0.00 to 0.64]

54. Primary Outcome: Cumulative Percentage of Subjects Reporting Respiratory, Thoracic and Mediastinal Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were cough, dysphonia, epistaxis, nasal congestion, oropharyngeal pain, rhinorrhoea, and wheezing.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 13.64 [0.00 to 100]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 25.53 [5.89 to 57.29]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 18.52 [8.61 to 32.71]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 13.82 [8.26 to 21.20]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 14.07 [6.54 to 25.27]
  Any,Weeks 40-52 | 13.67 [6.04 to 25.29]
  Cough,Weeks 40-46: number analyzed (Participants) | 3
  Cough,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Cough,Weeks 40-47: number analyzed (Participants) | 22
  Cough,Weeks 40-47 | 13.64 [0.00 to 100]
  Cough,Weeks 40-48: number analyzed (Participants) | 47
  Cough,Weeks 40-48 | 17.02 [0.00 to 90.61]
  Cough,Weeks 40-49: number analyzed (Participants) | 81
  Cough,Weeks 40-49 | 13.58 [1.89 to 39.84]
  Cough,Weeks 40-50: number analyzed (Participants) | 123
  Cough,Weeks 40-50 | 10.57 [3.50 to 23.04]
  Cough,Weeks 40-51: number analyzed (Participants) | 135
  Cough,Weeks 40-51 | 9.63 [2.90 to 22.07]
  Cough,Weeks 40-52 | 9.35 [2.66 to 22.05]
  Dysphonia,Weeks 40-46: number analyzed (Participants) | 3
  Dysphonia,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Dysphonia,Weeks 40-47: number analyzed (Participants) | 22
  Dysphonia,Weeks 40-47 | 4.55 [0.00 to 100]
  Dysphonia,Weeks 40-48: number analyzed (Participants) | 47
  Dysphonia,Weeks 40-48 | 6.38 [0.00 to 84.50]
  Dysphonia,Weeks 40-49: number analyzed (Participants) | 81
  Dysphonia,Weeks 40-49 | 3.70 [0.49 to 12.42]
  Dysphonia,Weeks 40-50: number analyzed (Participants) | 123
  Dysphonia,Weeks 40-50 | 2.44 [0.37 to 7.90]
  Dysphonia,Weeks 40-51: number analyzed (Participants) | 135
  Dysphonia,Weeks 40-51 | 2.22 [0.30 to 7.50]
  Dysphonia,Weeks 40-52 | 2.16 [0.27 to 7.48]
  Epistaxis,Weeks 40-46: number analyzed (Participants) | 3
  Epistaxis,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Epistaxis,Weeks 40-47: number analyzed (Participants) | 22
  Epistaxis,Weeks 40-47 | 4.55 [0.00 to 86.65]
  Epistaxis,Weeks 40-48: number analyzed (Participants) | 47
  Epistaxis,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Epistaxis,Weeks 40-49: number analyzed (Participants) | 81
  Epistaxis,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Epistaxis,Weeks 40-50: number analyzed (Participants) | 123
  Epistaxis,Weeks 40-50 | 0.81 [0.02 to 4.45]
  Epistaxis,Weeks 40-51: number analyzed (Participants) | 135
  Epistaxis,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Epistaxis,Weeks 40-52 | 0.72 [0.02 to 3.94]
  Nasal congestion,Weeks 40-46: number analyzed (Participants) | 3
  Nasal congestion,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Nasal congestion,Weeks 40-47: number analyzed (Participants) | 22
  Nasal congestion,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Nasal congestion,Weeks 40-48: number analyzed (Participants) | 47
  Nasal congestion,Weeks 40-48 | 6.38 [0.00 to 54.84]
  Nasal congestion,Weeks 40-49: number analyzed (Participants) | 81
  Nasal congestion,Weeks 40-49 | 4.94 [0.59 to 16.86]
  Nasal congestion,Weeks 40-50: number analyzed (Participants) | 123
  Nasal congestion,Weeks 40-50 | 3.25 [0.35 to 11.68]
  Nasal congestion,Weeks 40-51: number analyzed (Participants) | 135
  Nasal congestion,Weeks 40-51 | 2.96 [0.32 to 10.76]
  Nasal congestion,Weeks 40-52 | 2.88 [0.31 to 10.46]
  Oropharyngeal pain,Weeks 40-46: number analyzed (Participants) | 3
  Oropharyngeal pain,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Oropharyngeal pain,Weeks 40-47: number analyzed (Participants) | 22
  Oropharyngeal pain,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Oropharyngeal pain,Weeks 40-48: number analyzed (Participants) | 47
  Oropharyngeal pain,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Oropharyngeal pain,Weeks 40-49: number analyzed (Participants) | 81
  Oropharyngeal pain,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Oropharyngeal pain,Weeks 40-50: number analyzed (Participants) | 123
  Oropharyngeal pain,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Oropharyngeal pain,Weeks 40-51: number analyzed (Participants) | 135
  Oropharyngeal pain,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Oropharyngeal pain,Weeks 40-52 | 0.00 [0.00 to 2.62]
  Rhinorrhoea,Weeks 40-46: number analyzed (Participants) | 3
  Rhinorrhoea,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Rhinorrhoea,Weeks 40-47: number analyzed (Participants) | 22
  Rhinorrhoea,Weeks 40-47 | 4.55 [0.00 to 100]
  Rhinorrhoea,Weeks 40-48: number analyzed (Participants) | 47
  Rhinorrhoea,Weeks 40-48 | 12.77 [3.33 to 30.49]
  Rhinorrhoea,Weeks 40-49: number analyzed (Participants) | 81
  Rhinorrhoea,Weeks 40-49 | 9.88 [1.33 to 30.59]
  Rhinorrhoea,Weeks 40-50: number analyzed (Participants) | 123
  Rhinorrhoea,Weeks 40-50 | 7.32 [1.89 to 18.28]
  Rhinorrhoea,Weeks 40-51: number analyzed (Participants) | 135
  Rhinorrhoea,Weeks 40-51 | 7.41 [0.60 to 27.31]
  Rhinorrhoea,Weeks 40-52 | 7.19 [0.54 to 27.20]
  Wheezing,Weeks 40-46: number analyzed (Participants) | 3
  Wheezing,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Wheezing,Weeks 40-47: number analyzed (Participants) | 22
  Wheezing,Weeks 40-47 | 4.55 [0.00 to 100]
  Wheezing,Weeks 40-48: number analyzed (Participants) | 47
  Wheezing,Weeks 40-48 | 4.26 [0.00 to 97.64]
  Wheezing,Weeks 40-49: number analyzed (Participants) | 81
  Wheezing,Weeks 40-49 | 2.47 [0.01 to 18.68]
  Wheezing,Weeks 40-50: number analyzed (Participants) | 123
  Wheezing,Weeks 40-50 | 1.63 [0.01 to 12.28]
  Wheezing,Weeks 40-51: number analyzed (Participants) | 135
  Wheezing,Weeks 40-51 | 1.48 [0.00 to 11.58]
  Wheezing,Weeks 40-52 | 1.44 [0.00 to 11.48]
  Sneezing,Weeks 40-46: number analyzed (Participants) | 3
  Sneezing,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Sneezing,Weeks 40-47: number analyzed (Participants) | 22
  Sneezing,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Sneezing,Weeks 40-48: number analyzed (Participants) | 47
  Sneezing,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Sneezing,Weeks 40-49: number analyzed (Participants) | 81
  Sneezing,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Sneezing,Weeks 40-50: number analyzed (Participants) | 123
  Sneezing,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Sneezing,Weeks 40-51: number analyzed (Participants) | 135
  Sneezing,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Sneezing,Weeks 40-52 | 0.72 [0.02 to 3.94]

55. Primary Outcome: Cumulative Percentage of Subjects Reporting Skin and Subcutaneous Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. The pre-defined AEIs listed on the ADR card were rash and rash generalised.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 2.86 [0.12 to 13.38] |  | 2.86 [0.12 to 13.38]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 1.86 [0.11 to 8.11] |  | 1.86 [0.11 to 8.11]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 1.96 [0.11 to 8.66] | 3.85 [0.11 to 19.24] | 1.51 [0.27 to 4.66]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.58 [0.00 to 86.72] | 2.30 [0.08 to 11.24] | 1.54 [0.12 to 6.20] | 1.54 [0.43 to 3.85]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.48 [0.00 to 12.12] | 2.16 [0.15 to 9.00] | 2.05 [0.28 to 6.91] | 1.57 [0.66 to 3.15]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 2.13 [0.00 to 23.40] | 2.00 [0.23 to 7.13] | 1.71 [0.00 to 14.61] | 1.93 [0.77 to 3.97]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 1.95 [0.00 to 18.56] | 2.17 [0.27 to 7.54] | 1.44 [0.00 to 12.96] | 1.80 [0.74 to 3.63]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 1.82 [0.00 to 15.58] | 2.16 [0.28 to 7.38] | 1.37 [0.00 to 11.80] | 1.72 [0.74 to 3.38]
  Any,Weeks 40-48 | 1.82 [0.00 to 15.58] | 2.16 [0.28 to 7.38] | 1.32 [0.00 to 11.51] | 1.70 [0.72 to 3.36]
  Any,Weeks 40-49 | 1.82 [0.00 to 15.58] | 2.16 [0.28 to 7.38] | 1.32 [0.00 to 11.51] | 1.70 [0.72 to 3.36]
  Any,Weeks 40-50 | 1.82 [0.00 to 15.58] | 2.16 [0.28 to 7.38] | 1.32 [0.00 to 11.51] | 1.70 [0.72 to 3.36]
  Any,Weeks 40-51 | 1.82 [0.00 to 15.58] | 2.16 [0.28 to 7.38] | 1.32 [0.00 to 11.51] | 1.70 [0.72 to 3.36]
  Any,Weeks 40-52 | 1.82 [0.00 to 15.58] | 2.16 [0.28 to 7.38] | 1.32 [0.00 to 11.51] | 1.70 [0.72 to 3.36]
  Rash,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rash,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Rash,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Rash,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Rash,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Rash,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 1.92 [0.05 to 10.26] | 0.50 [0.04 to 2.11]
  Rash,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Rash,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.77 [0.02 to 4.21] | 0.39 [0.05 to 1.39]
  Rash,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Rash,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 1.54 [0.04 to 8.18] | 0.63 [0.15 to 1.73]
  Rash,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Rash,Weeks 40-45 | 0.35 [0.00 to 5.88] | 0.40 [0.00 to 7.09] | 1.14 [0.00 to 9.92] | 0.68 [0.20 to 1.69]
  Rash,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Rash,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.36 [0.00 to 7.23] | 0.96 [0.00 to 8.78] | 0.60 [0.17 to 1.52]
  Rash,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Rash,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.36 [0.00 to 7.23] | 0.92 [0.00 to 7.98] | 0.57 [0.16 to 1.43]
  Rash,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.36 [0.00 to 7.23] | 0.88 [0.00 to 7.79] | 0.57 [0.16 to 1.42]
  Rash,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.36 [0.00 to 7.23] | 0.88 [0.00 to 7.79] | 0.57 [0.16 to 1.42]
  Rash,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.36 [0.00 to 7.23] | 0.88 [0.00 to 7.79] | 0.57 [0.16 to 1.42]
  Rash,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.36 [0.00 to 7.23] | 0.88 [0.00 to 7.79] | 0.57 [0.16 to 1.42]
  Rash,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.36 [0.00 to 7.23] | 0.88 [0.00 to 7.79] | 0.57 [0.16 to 1.42]
  Rash generalised,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Rash generalised,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Rash generalised,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Rash generalised,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Rash generalised,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Rash generalised,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Rash generalised,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Rash generalised,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Rash generalised,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Rash generalised,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Rash generalised,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Rash generalised,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.00 [0.00 to 0.42]
  Rash generalised,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Rash generalised,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Rash generalised,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Rash generalised,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Rash generalised,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Rash generalised,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Rash generalised,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Rash generalised,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Rash generalised,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Erythema,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Erythema,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Erythema,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Erythema,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Erythema,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Erythema,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 1.92 [0.05 to 10.26] | 0.25 [0.00 to 2.11]
  Erythema,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Erythema,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.77 [0.02 to 4.21] | 0.19 [0.00 to 1.28]
  Erythema,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Erythema,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.01 to 2.82] | 0.16 [0.00 to 0.87]
  Erythema,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Erythema,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.57 [0.00 to 5.05] | 0.23 [0.02 to 0.86]
  Erythema,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Erythema,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.00 [0.00 to 1.33] | 0.48 [0.00 to 4.46] | 0.20 [0.02 to 0.77]
  Erythema,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Erythema,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.46 [0.00 to 4.05] | 0.19 [0.02 to 0.74]
  Erythema,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 3.95] | 0.19 [0.02 to 0.73]
  Erythema,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 3.95] | 0.19 [0.02 to 0.73]
  Erythema,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 3.95] | 0.19 [0.02 to 0.73]
  Erythema,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 3.95] | 0.19 [0.02 to 0.73]
  Erythema,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.00 [0.00 to 1.32] | 0.44 [0.00 to 3.95] | 0.19 [0.02 to 0.73]
  Hyperhidrosis,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hyperhidrosis,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Hyperhidrosis,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Hyperhidrosis,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Hyperhidrosis,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Hyperhidrosis,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Hyperhidrosis,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Hyperhidrosis,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Hyperhidrosis,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Hyperhidrosis,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Hyperhidrosis,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Hyperhidrosis,Weeks 40-45 | 0.35 [0.00 to 5.88] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.79]
  Hyperhidrosis,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Hyperhidrosis,Weeks 40-46 | 0.32 [0.00 to 4.64] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.68]
  Hyperhidrosis,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Hyperhidrosis,Weeks 40-47 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.64]
  Hyperhidrosis,Weeks 40-48 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Hyperhidrosis,Weeks 40-49 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Hyperhidrosis,Weeks 40-50 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Hyperhidrosis,Weeks 40-51 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Hyperhidrosis,Weeks 40-52 | 0.30 [0.00 to 3.90] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.63]
  Pruritus,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pruritus,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Pruritus,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Pruritus,Weeks 40-41 |  | 1.24 [0.01 to 8.05] |  | 1.24 [0.01 to 8.05]
  Pruritus,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Pruritus,Weeks 40-42 | 0.00 [0.00 to 2.58] | 1.47 [0.01 to 10.56] | 0.00 [0.00 to 6.85] | 0.76 [0.04 to 3.42]
  Pruritus,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Pruritus,Weeks 40-43 | 0.58 [0.00 to 86.72] | 1.84 [0.00 to 14.96] | 0.00 [0.00 to 2.80] | 0.96 [0.08 to 3.95]
  Pruritus,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Pruritus,Weeks 40-44 | 0.48 [0.00 to 12.12] | 1.72 [0.01 to 12.04] | 0.00 [0.00 to 1.87] | 0.79 [0.08 to 2.98]
  Pruritus,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Pruritus,Weeks 40-45 | 1.06 [0.00 to 10.50] | 1.60 [0.03 to 9.43] | 0.00 [0.00 to 1.05] | 0.79 [0.15 to 2.42]
  Pruritus,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Pruritus,Weeks 40-46 | 0.97 [0.00 to 8.41] | 1.81 [0.03 to 10.38] | 0.00 [0.00 to 0.88] | 0.80 [0.13 to 2.54]
  Pruritus,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Pruritus,Weeks 40-47 | 0.91 [0.00 to 7.18] | 1.80 [0.03 to 10.15] | 0.00 [0.00 to 0.84] | 0.77 [0.13 to 2.41]
  Pruritus,Weeks 40-48 | 0.91 [0.00 to 7.18] | 1.80 [0.03 to 10.15] | 0.00 [0.00 to 0.81] | 0.75 [0.13 to 2.39]
  Pruritus,Weeks 40-49 | 0.91 [0.00 to 7.18] | 1.80 [0.03 to 10.15] | 0.00 [0.00 to 0.81] | 0.75 [0.13 to 2.39]
  Pruritus,Weeks 40-50 | 0.91 [0.00 to 7.18] | 1.80 [0.03 to 10.15] | 0.00 [0.00 to 0.81] | 0.75 [0.13 to 2.39]
  Pruritus,Weeks 40-51 | 0.91 [0.00 to 7.18] | 1.80 [0.03 to 10.15] | 0.00 [0.00 to 0.81] | 0.75 [0.13 to 2.39]
  Pruritus,Weeks 40-52 | 0.91 [0.00 to 7.18] | 1.80 [0.03 to 10.15] | 0.00 [0.00 to 0.81] | 0.75 [0.13 to 2.39]
  Pruritus generalised,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Pruritus generalised,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Pruritus generalised,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Pruritus generalised,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Pruritus generalised,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Pruritus generalised,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Pruritus generalised,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Pruritus generalised,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Pruritus generalised,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Pruritus generalised,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Pruritus generalised,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Pruritus generalised,Weeks 40-45 | 0.71 [0.00 to 11.46] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.23 [0.00 to 1.58]
  Pruritus generalised,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Pruritus generalised,Weeks 40-46 | 0.65 [0.00 to 9.11] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.20 [0.00 to 1.36]
  Pruritus generalised,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Pruritus generalised,Weeks 40-47 | 0.61 [0.00 to 7.67] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.19 [0.00 to 1.27]
  Pruritus generalised,Weeks 40-48 | 0.61 [0.00 to 7.67] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.26]
  Pruritus generalised,Weeks 40-49 | 0.61 [0.00 to 7.67] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.26]
  Pruritus generalised,Weeks 40-50 | 0.61 [0.00 to 7.67] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.26]
  Pruritus generalised,Weeks 40-51 | 0.61 [0.00 to 7.67] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.26]
  Pruritus generalised,Weeks 40-52 | 0.61 [0.00 to 7.67] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.26]

56. Primary Outcome: Cumulative Percentage of Subjects Reporting Skin and Subcutaneous Tissue Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were rash and rash generalised.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 0.81 [0.02 to 4.45]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Any,Weeks 40-52 | 0.72 [0.02 to 3.94]
  Rash,Weeks 40-46: number analyzed (Participants) | 3
  Rash,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Rash,Weeks 40-47: number analyzed (Participants) | 22
  Rash,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Rash,Weeks 40-48: number analyzed (Participants) | 47
  Rash,Weeks 40-48 | 2.13 [0.00 to 22.05]
  Rash,Weeks 40-49: number analyzed (Participants) | 81
  Rash,Weeks 40-49 | 1.23 [0.03 to 6.69]
  Rash,Weeks 40-50: number analyzed (Participants) | 123
  Rash,Weeks 40-50 | 0.81 [0.02 to 4.45]
  Rash,Weeks 40-51: number analyzed (Participants) | 135
  Rash,Weeks 40-51 | 0.74 [0.02 to 4.06]
  Rash,Weeks 40-52 | 0.72 [0.02 to 3.94]
  Rash generalised,Weeks 40-46: number analyzed (Participants) | 3
  Rash generalised,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Rash generalised,Weeks 40-47: number analyzed (Participants) | 22
  Rash generalised,Weeks 40-47 | 0.00 [0.00 to 15.44]
  Rash generalised,Weeks 40-48: number analyzed (Participants) | 47
  Rash generalised,Weeks 40-48 | 0.00 [0.00 to 7.55]
  Rash generalised,Weeks 40-49: number analyzed (Participants) | 81
  Rash generalised,Weeks 40-49 | 0.00 [0.00 to 4.45]
  Rash generalised,Weeks 40-50: number analyzed (Participants) | 123
  Rash generalised,Weeks 40-50 | 0.00 [0.00 to 2.95]
  Rash generalised,Weeks 40-51: number analyzed (Participants) | 135
  Rash generalised,Weeks 40-51 | 0.00 [0.00 to 2.70]
  Rash generalised,Weeks 40-52 | 0.00 [0.00 to 2.62]

57. Primary Outcome: Cumulative Percentage of Subjects Reporting Cardiac Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for cardiac disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Any,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Any,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Any,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Any,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Any,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Tachycardia,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tachycardia,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Tachycardia,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Tachycardia,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Tachycardia,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Tachycardia,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Tachycardia,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Tachycardia,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Tachycardia,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Tachycardia,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Tachycardia,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Tachycardia,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Tachycardia,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Tachycardia,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Tachycardia,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Tachycardia,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Tachycardia,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Tachycardia,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Tachycardia,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Tachycardia,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Tachycardia,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]

58. Primary Outcome: Cumulative Percentage of Subjects Reporting Cardiac Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for cardiac disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

59. Primary Outcome: Cumulative Percentage of Subjects Reporting Ear and Labyrinth Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for ear and labyrinth disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 1.24 [0.01 to 8.05] |  | 1.24 [0.01 to 8.05]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.98 [0.06 to 4.38] | 0.00 [0.00 to 6.85] | 0.50 [0.05 to 1.99]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.92 [0.08 to 3.65] | 0.00 [0.00 to 2.80] | 0.39 [0.03 to 1.63]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.86 [0.10 to 3.08] | 0.51 [0.01 to 2.82] | 0.63 [0.17 to 1.60]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.35 [0.00 to 10.83] | 1.60 [0.03 to 9.43] | 0.29 [0.00 to 1.82] | 0.68 [0.13 to 2.03]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.32 [0.00 to 10.19] | 1.81 [0.03 to 10.38] | 0.24 [0.00 to 2.15] | 0.70 [0.11 to 2.31]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.30 [0.00 to 9.75] | 1.80 [0.03 to 10.15] | 0.23 [0.00 to 2.24] | 0.67 [0.10 to 2.24]
  Any,Weeks 40-48 | 0.30 [0.00 to 9.75] | 1.80 [0.03 to 10.15] | 0.22 [0.00 to 2.33] | 0.66 [0.10 to 2.22]
  Any,Weeks 40-49 | 0.30 [0.00 to 9.75] | 1.80 [0.03 to 10.15] | 0.22 [0.00 to 2.33] | 0.66 [0.10 to 2.22]
  Any,Weeks 40-50 | 0.30 [0.00 to 9.75] | 1.80 [0.03 to 10.15] | 0.22 [0.00 to 2.33] | 0.66 [0.10 to 2.22]
  Any,Weeks 40-51 | 0.30 [0.00 to 9.75] | 1.80 [0.03 to 10.15] | 0.22 [0.00 to 2.33] | 0.66 [0.10 to 2.22]
  Any,Weeks 40-52 | 0.30 [0.00 to 9.75] | 1.80 [0.03 to 10.15] | 0.22 [0.00 to 2.33] | 0.66 [0.10 to 2.22]
  Ear haemorrhage,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear haemorrhage,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear haemorrhage,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Ear haemorrhage,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Ear haemorrhage,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Ear haemorrhage,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Ear haemorrhage,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Ear haemorrhage,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Ear haemorrhage,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Ear haemorrhage,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Ear haemorrhage,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Ear haemorrhage,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Ear haemorrhage,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Ear haemorrhage,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Ear haemorrhage,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Ear haemorrhage,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Ear haemorrhage,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Ear haemorrhage,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Ear haemorrhage,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Ear haemorrhage,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Ear haemorrhage,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Ear pain,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear pain,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear pain,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Ear pain,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Ear pain,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Ear pain,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Ear pain,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Ear pain,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Ear pain,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Ear pain,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.51 [0.01 to 2.82] | 0.16 [0.00 to 0.87]
  Ear pain,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Ear pain,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.00 [0.00 to 1.46] | 0.29 [0.00 to 1.82] | 0.11 [0.00 to 0.63]
  Ear pain,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Ear pain,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.24 [0.00 to 2.15] | 0.20 [0.02 to 0.72]
  Ear pain,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Ear pain,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.23 [0.00 to 2.24] | 0.19 [0.02 to 0.69]
  Ear pain,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.68]
  Ear pain,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.68]
  Ear pain,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.68]
  Ear pain,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.68]
  Ear pain,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.22 [0.00 to 2.33] | 0.19 [0.02 to 0.68]
  Ear pruritus,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Ear pruritus,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Ear pruritus,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Ear pruritus,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Ear pruritus,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Ear pruritus,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Ear pruritus,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Ear pruritus,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Ear pruritus,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Ear pruritus,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.29]
  Ear pruritus,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Ear pruritus,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.91]
  Ear pruritus,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Ear pruritus,Weeks 40-46 | 0.32 [0.00 to 10.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.81]
  Ear pruritus,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Ear pruritus,Weeks 40-47 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.78]
  Ear pruritus,Weeks 40-48 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Ear pruritus,Weeks 40-49 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Ear pruritus,Weeks 40-50 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Ear pruritus,Weeks 40-51 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Ear pruritus,Weeks 40-52 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Tinnitus,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Tinnitus,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Tinnitus,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Tinnitus,Weeks 40-41 |  | 0.62 [0.00 to 17.42] |  | 0.62 [0.00 to 17.42]
  Tinnitus,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Tinnitus,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Tinnitus,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Tinnitus,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Tinnitus,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Tinnitus,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Tinnitus,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Tinnitus,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Tinnitus,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Tinnitus,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Tinnitus,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Tinnitus,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Tinnitus,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tinnitus,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tinnitus,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tinnitus,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Tinnitus,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Vertigo,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Vertigo,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Vertigo,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Vertigo,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Vertigo,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Vertigo,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Vertigo,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Vertigo,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Vertigo,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Vertigo,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Vertigo,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Vertigo,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.80 [0.00 to 11.66] | 0.00 [0.00 to 1.05] | 0.23 [0.00 to 1.61]
  Vertigo,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Vertigo,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.72 [0.00 to 9.03] | 0.00 [0.00 to 0.88] | 0.20 [0.00 to 1.39]
  Vertigo,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Vertigo,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.84] | 0.19 [0.00 to 1.34]
  Vertigo,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Vertigo,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Vertigo,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Vertigo,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]
  Vertigo,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.72 [0.00 to 8.86] | 0.00 [0.00 to 0.81] | 0.19 [0.00 to 1.32]

60. Primary Outcome: Cumulative Percentage of Subjects Reporting Ear and Labyrinth Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for ear and labyrinth disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

61. Primary Outcome: Cumulative Percentage of Subjects Reporting Eye Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for eye disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 1.47 [0.01 to 10.56] | 0.00 [0.00 to 6.85] | 0.76 [0.04 to 3.42]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.00 [0.00 to 2.12] | 1.38 [0.02 to 8.51] | 0.00 [0.00 to 2.80] | 0.58 [0.03 to 2.71]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.48 [0.00 to 15.39] | 1.29 [0.04 to 6.74] | 0.00 [0.00 to 1.87] | 0.63 [0.08 to 2.25]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.35 [0.00 to 10.83] | 1.20 [0.08 to 5.23] | 0.00 [0.00 to 1.05] | 0.45 [0.05 to 1.66]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.32 [0.00 to 10.19] | 1.09 [0.14 to 3.80] | 0.00 [0.00 to 0.88] | 0.40 [0.05 to 1.45]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.30 [0.00 to 9.75] | 1.08 [0.14 to 3.72] | 0.00 [0.00 to 0.84] | 0.38 [0.04 to 1.40]
  Any,Weeks 40-48 | 0.30 [0.00 to 9.75] | 1.08 [0.14 to 3.72] | 0.00 [0.00 to 0.81] | 0.38 [0.04 to 1.38]
  Any,Weeks 40-49 | 0.30 [0.00 to 9.75] | 1.08 [0.14 to 3.72] | 0.00 [0.00 to 0.81] | 0.38 [0.04 to 1.38]
  Any,Weeks 40-50 | 0.30 [0.00 to 9.75] | 1.08 [0.14 to 3.72] | 0.00 [0.00 to 0.81] | 0.38 [0.04 to 1.38]
  Any,Weeks 40-51 | 0.30 [0.00 to 9.75] | 1.08 [0.14 to 3.72] | 0.00 [0.00 to 0.81] | 0.38 [0.04 to 1.38]
  Any,Weeks 40-52 | 0.30 [0.00 to 9.75] | 1.08 [0.14 to 3.72] | 0.00 [0.00 to 0.81] | 0.38 [0.04 to 1.38]
  Eye discharge,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Eye discharge,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Eye discharge,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Eye discharge,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Eye discharge,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Eye discharge,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Eye discharge,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Eye discharge,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Eye discharge,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Eye discharge,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Eye discharge,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Eye discharge,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Eye discharge,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Eye discharge,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Eye discharge,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Eye discharge,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Eye discharge,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Eye discharge,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Eye discharge,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Eye discharge,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Eye discharge,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Eye pruritus,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Eye pruritus,Weeks 40-40 |  | 1.43 [0.04 to 7.70] |  | 1.43 [0.04 to 7.70]
  Eye pruritus,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Eye pruritus,Weeks 40-41 |  | 0.62 [0.00 to 5.51] |  | 0.62 [0.00 to 5.51]
  Eye pruritus,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Eye pruritus,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 6.53] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 1.73]
  Eye pruritus,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Eye pruritus,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 6.74] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.43]
  Eye pruritus,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Eye pruritus,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 6.92] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.09]
  Eye pruritus,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Eye pruritus,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 7.09] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.83]
  Eye pruritus,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Eye pruritus,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.74]
  Eye pruritus,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Eye pruritus,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.71]
  Eye pruritus,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Eye pruritus,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Eye pruritus,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Eye pruritus,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Eye pruritus,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 7.23] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.70]
  Lacrimation increased,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Lacrimation increased,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Lacrimation increased,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Lacrimation increased,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Lacrimation increased,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Lacrimation increased,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.49 [0.00 to 10.27] | 0.00 [0.00 to 6.85] | 0.25 [0.00 to 2.00]
  Lacrimation increased,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Lacrimation increased,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.46 [0.00 to 8.71] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.52]
  Lacrimation increased,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Lacrimation increased,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.43 [0.00 to 7.29] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.11]
  Lacrimation increased,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Lacrimation increased,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Lacrimation increased,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Lacrimation increased,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Lacrimation increased,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Lacrimation increased,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Lacrimation increased,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lacrimation increased,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lacrimation increased,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lacrimation increased,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Lacrimation increased,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Swelling of eyelid,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Swelling of eyelid,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Swelling of eyelid,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Swelling of eyelid,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Swelling of eyelid,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Swelling of eyelid,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Swelling of eyelid,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Swelling of eyelid,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Swelling of eyelid,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Swelling of eyelid,Weeks 40-44 | 0.48 [0.00 to 15.39] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 1.29]
  Swelling of eyelid,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Swelling of eyelid,Weeks 40-45 | 0.35 [0.00 to 10.83] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.91]
  Swelling of eyelid,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Swelling of eyelid,Weeks 40-46 | 0.32 [0.00 to 10.19] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.81]
  Swelling of eyelid,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Swelling of eyelid,Weeks 40-47 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.78]
  Swelling of eyelid,Weeks 40-48 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Swelling of eyelid,Weeks 40-49 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Swelling of eyelid,Weeks 40-50 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Swelling of eyelid,Weeks 40-51 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]
  Swelling of eyelid,Weeks 40-52 | 0.30 [0.00 to 9.75] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.76]

62. Primary Outcome: Cumulative Percentage of Subjects Reporting Eye Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for eye disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  Any,Weeks 40-46: number analyzed (Participants) | 3
  Any,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Any,Weeks 40-47: number analyzed (Participants) | 22
  Any,Weeks 40-47 | 9.09 [0.00 to 98.76]
  Any,Weeks 40-48: number analyzed (Participants) | 47
  Any,Weeks 40-48 | 4.26 [0.00 to 40.16]
  Any,Weeks 40-49: number analyzed (Participants) | 81
  Any,Weeks 40-49 | 2.47 [0.30 to 8.64]
  Any,Weeks 40-50: number analyzed (Participants) | 123
  Any,Weeks 40-50 | 1.63 [0.20 to 5.75]
  Any,Weeks 40-51: number analyzed (Participants) | 135
  Any,Weeks 40-51 | 1.48 [0.18 to 5.25]
  Any,Weeks 40-52 | 1.44 [0.17 to 5.10]
  Eye pruritus,Weeks 40-46: number analyzed (Participants) | 3
  Eye pruritus,Weeks 40-46 | 0.00 [0.00 to 70.76]
  Eye pruritus,Weeks 40-47: number analyzed (Participants) | 22
  Eye pruritus,Weeks 40-47 | 9.09 [0.00 to 98.76]
  Eye pruritus,Weeks 40-50: number analyzed (Participants) | 123
  Eye pruritus,Weeks 40-50 | 1.63 [0.20 to 5.75]
  Eye pruritus,Weeks 40-51: number analyzed (Participants) | 135
  Eye pruritus,Weeks 40-51 | 1.48 [0.18 to 5.25]
  Eye pruritus,Weeks 40-52 | 1.44 [0.17 to 5.10]

63. Primary Outcome: Cumulative Percentage of Subjects Reporting Injury, Poisoning and Procedural Complications by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for injury, poisoning and procedural complications.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Any,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Any,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Any,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Any,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Any,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Muscle strain,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Muscle strain,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Muscle strain,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Muscle strain,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Muscle strain,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Muscle strain,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 0.92]
  Muscle strain,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Muscle strain,Weeks 40-43 | 0.00 [0.00 to 2.12] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 0.71]
  Muscle strain,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Muscle strain,Weeks 40-44 | 0.00 [0.00 to 1.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.00 [0.00 to 0.58]
  Muscle strain,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Muscle strain,Weeks 40-45 | 0.00 [0.00 to 1.30] | 0.40 [0.00 to 5.98] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.81]
  Muscle strain,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Muscle strain,Weeks 40-46 | 0.00 [0.00 to 1.19] | 0.36 [0.00 to 4.60] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Muscle strain,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Muscle strain,Weeks 40-47 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.67]
  Muscle strain,Weeks 40-48 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Muscle strain,Weeks 40-49 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Muscle strain,Weeks 40-50 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Muscle strain,Weeks 40-51 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]
  Muscle strain,Weeks 40-52 | 0.00 [0.00 to 1.11] | 0.36 [0.00 to 4.51] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.66]

64. Primary Outcome: Cumulative Percentage of Subjects Reporting Injury, Poisoning and Procedural Complications by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for injury, poisoning and procedural complications.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

65. Primary Outcome: Cumulative Percentage of Subjects Reporting Investigations by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for investigations.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.98 [0.00 to 19.61] | 0.00 [0.00 to 6.85] | 0.50 [0.00 to 3.97]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.00 [0.00 to 2.12] | 1.38 [0.00 to 24.20] | 0.00 [0.00 to 2.80] | 0.58 [0.00 to 4.52]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.00 [0.00 to 1.76] | 1.29 [0.00 to 20.54] | 0.00 [0.00 to 1.87] | 0.47 [0.00 to 3.29]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.35 [0.00 to 5.88] | 1.20 [0.00 to 17.05] | 0.00 [0.00 to 1.05] | 0.45 [0.02 to 2.20]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.32 [0.00 to 4.64] | 1.09 [0.00 to 13.30] | 0.00 [0.00 to 0.88] | 0.40 [0.02 to 1.88]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.84] | 0.38 [0.02 to 1.79]
  Any,Weeks 40-48 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Any,Weeks 40-49 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Any,Weeks 40-50 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Any,Weeks 40-51 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Any,Weeks 40-52 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Heart rate increased,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Heart rate increased,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Heart rate increased,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Heart rate increased,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Heart rate increased,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Heart rate increased,Weeks 40-42 | 0.00 [0.00 to 2.58] | 0.98 [0.00 to 19.61] | 0.00 [0.00 to 6.85] | 0.50 [0.00 to 3.97]
  Heart rate increased,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Heart rate increased,Weeks 40-43 | 0.00 [0.00 to 2.12] | 1.38 [0.00 to 24.20] | 0.00 [0.00 to 2.80] | 0.58 [0.00 to 4.52]
  Heart rate increased,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Heart rate increased,Weeks 40-44 | 0.00 [0.00 to 1.76] | 1.29 [0.00 to 20.54] | 0.00 [0.00 to 1.87] | 0.47 [0.00 to 3.29]
  Heart rate increased,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Heart rate increased,Weeks 40-45 | 0.35 [0.00 to 5.88] | 1.20 [0.00 to 17.05] | 0.00 [0.00 to 1.05] | 0.45 [0.02 to 2.20]
  Heart rate increased,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Heart rate increased,Weeks 40-46 | 0.32 [0.00 to 4.64] | 1.09 [0.00 to 13.30] | 0.00 [0.00 to 0.88] | 0.40 [0.02 to 1.88]
  Heart rate increased,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Heart rate increased,Weeks 40-47 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.84] | 0.38 [0.02 to 1.79]
  Heart rate increased,Weeks 40-48 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Heart rate increased,Weeks 40-49 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Heart rate increased,Weeks 40-50 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Heart rate increased,Weeks 40-51 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]
  Heart rate increased,Weeks 40-52 | 0.30 [0.00 to 3.90] | 1.08 [0.00 to 13.06] | 0.00 [0.00 to 0.81] | 0.38 [0.02 to 1.77]

66. Primary Outcome: Cumulative Percentage of Subjects Reporting Investigations by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52.There were no predefined AEIs listed on the ADR card for investigations.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

67. Primary Outcome: Cumulative Percentage of Subjects Reporting Vascular Disorders by MedDRA PT, Using ADR Card, Post Dose 1 by Vaccine Group and Overall
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. There were no predefined AEIs listed on the ADR card for vascular disorders.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  Any,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Any,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Any,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Any,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Any,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Any,Weeks 40-42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.25 [0.01 to 1.42]
  Any,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Any,Weeks 40-43 | 0.58 [0.00 to 20.94] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.25]
  Any,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Any,Weeks 40-44 | 0.48 [0.00 to 3.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 0.99]
  Any,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Any,Weeks 40-45 | 0.35 [0.00 to 5.12] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.77]
  Any,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Any,Weeks 40-46 | 0.32 [0.00 to 5.39] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Any,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Any,Weeks 40-47 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.68]
  Any,Weeks 40-48 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Any,Weeks 40-49 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Any,Weeks 40-50 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Any,Weeks 40-51 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Any,Weeks 40-52 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Hot flush,Weeks 40-40: number analyzed (Participants) | 0 | 70 | 0 | 70
  Hot flush,Weeks 40-40 |  | 0.00 [0.00 to 5.13] |  | 0.00 [0.00 to 5.13]
  Hot flush,Weeks 40-41: number analyzed (Participants) | 0 | 161 | 0 | 161
  Hot flush,Weeks 40-41 |  | 0.00 [0.00 to 2.27] |  | 0.00 [0.00 to 2.27]
  Hot flush,Weeks 40-42: number analyzed (Participants) | 141 | 204 | 52 | 397
  Hot flush,Weeks 40-42 | 0.71 [0.01 to 4.40] | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 6.85] | 0.25 [0.01 to 1.42]
  Hot flush,Weeks 40-43: number analyzed (Participants) | 172 | 217 | 130 | 519
  Hot flush,Weeks 40-43 | 0.58 [0.00 to 20.94] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 2.80] | 0.19 [0.00 to 1.25]
  Hot flush,Weeks 40-44: number analyzed (Participants) | 208 | 232 | 195 | 635
  Hot flush,Weeks 40-44 | 0.48 [0.00 to 3.76] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 1.87] | 0.16 [0.00 to 0.99]
  Hot flush,Weeks 40-45: number analyzed (Participants) | 282 | 250 | 350 | 882
  Hot flush,Weeks 40-45 | 0.35 [0.00 to 5.12] | 0.00 [0.00 to 1.46] | 0.00 [0.00 to 1.05] | 0.11 [0.00 to 0.77]
  Hot flush,Weeks 40-46: number analyzed (Participants) | 308 | 276 | 417 | 1001
  Hot flush,Weeks 40-46 | 0.32 [0.00 to 5.39] | 0.00 [0.00 to 1.33] | 0.00 [0.00 to 0.88] | 0.10 [0.00 to 0.70]
  Hot flush,Weeks 40-47: number analyzed (Participants) | 329 | 278 | 437 | 1044
  Hot flush,Weeks 40-47 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.84] | 0.10 [0.00 to 0.68]
  Hot flush,Weeks 40-48 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Hot flush,Weeks 40-49 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Hot flush,Weeks 40-50 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Hot flush,Weeks 40-51 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]
  Hot flush,Weeks 40-52 | 0.30 [0.00 to 5.54] | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 0.81] | 0.09 [0.00 to 0.67]

68. Primary Outcome: Cumulative Percentage of Subjects Reporting Vascular Disorders by MedDRA PT, Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. There were no predefined AEIs listed on the ADR card for vascular disorders.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects | 0 [0 to 2.62]

69. Secondary Outcome: Weekly Percentage of Subjects Reporting Any AEs, Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°36 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: Analysis was performed the enrolled subjects who were vaccinated with the first dose of GSK's quadrivalent seasonal influenza vaccine and who returned the ADR card.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 44.23 [0.11 to 99.54] | 44.23 [0.11 to 99.54]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 47.44 [36.01 to 59.07] | 47.44 [36.01 to 59.07]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 33.33 [10.12 to 64.74] | 33.33 [10.12 to 64.74]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 47.13 [10.74 to 86.08] | 47.13 [10.74 to 86.08]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 31.03 [13.11 to 54.42] | 31.03 [13.11 to 54.42]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 70.59 [0.00 to 100] | 70.59 [0.00 to 100]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 81.25 [0.01 to 100] | 81.25 [0.01 to 100]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 46.15 [0.35 to 99.22] |  | 46.15 [0.35 to 99.22]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 41.46 [0.08 to 99.36] |  | 41.46 [0.08 to 99.36]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 47.58 [38.54 to 56.74] | 50.00 [0.43 to 99.57] |  | 47.83 [39.26 to 56.49]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 33.33 [0.84 to 90.57] | 33.33 [0.84 to 90.57] |  | 33.33 [4.33 to 77.72]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 50.00 [6.76 to 93.24] | 60.00 [14.66 to 94.73] | 50.00 [18.71 to 81.29]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 87.50 [47.35 to 99.68] | 55.88 [43.32 to 67.92] | 56.96 [35.12 to 76.98]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 50.00 [23.04 to 76.96] | 44.74 [28.62 to 61.70] | 46.15 [20.68 to 73.21]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 100 [15.81 to 100] | 100 [2.50 to 100] | 66.67 [9.43 to 99.16] | 83.33 [22.88 to 99.95]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 25.00 [12.33 to 41.82] |  | 25.00 [12.33 to 41.82]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 32.00 [0.06 to 96.94] |  | 32.00 [0.06 to 96.94]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 29.41 [0.00 to 100] | 24.14 [0.76 to 77.59] |  | 26.09 [10.20 to 48.46]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 46.43 [27.51 to 66.13] | 40.00 [12.16 to 73.76] |  | 44.74 [15.59 to 76.89]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 57.14 [0.28 to 99.96] | 9.09 [0.23 to 41.28] |  | 45.65 [1.56 to 96.94]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 36.62 [1.04 to 92.67] | 50.00 [18.71 to 81.29] |  | 38.27 [18.79 to 60.98]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 26.92 [11.57 to 47.79] | 33.33 [9.92 to 65.11] |  | 28.95 [3.80 to 71.27]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 31.58 [12.58 to 56.55] | 0.00 [0.00 to 97.50] |  | 30.00 [3.86 to 73.12]

70. Secondary Outcome: Weekly Percentage of Subjects Reporting Gastrointestinal Disorders (MedDRA Primary System Organ Class [SOC]), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°38 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 69
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 7.69 [0.19 to 36.17] | 7.69 [0.19 to 36.17]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 8.97 [0.05 to 50.25] | 8.97 [0.05 to 50.25]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 3.33 [0.41 to 11.53] | 3.33 [0.41 to 11.53]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 5.75 [0.79 to 18.58] | 5.75 [0.79 to 18.58]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 6.90 [0.00 to 49.97] | 6.90 [0.00 to 49.97]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 11.76 [0.00 to 83.56] | 11.76 [0.00 to 83.56]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 3.85 [0.00 to 45.20] |  | 3.85 [0.00 to 45.20]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 1.61 [0.20 to 5.70] | 14.29 [0.00 to 100] |  | 2.90 [0.00 to 29.19]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 33.33 [0.84 to 90.57] |  | 16.67 [0.00 to 100]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 25.00 [0.63 to 80.59] | 20.00 [0.51 to 71.64] | 20.00 [2.52 to 55.61]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 25.00 [3.19 to 65.09] | 1.47 [0.04 to 7.92] | 3.80 [0.00 to 50.11]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 7.14 [0.18 to 33.87] | 13.16 [4.41 to 28.09] | 11.54 [0.02 to 66.50]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 2.27 [0.06 to 12.02] |  | 2.27 [0.06 to 12.02]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 4.00 [0.00 to 34.94] |  | 4.00 [0.00 to 34.94]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 5.88 [0.00 to 94.68] | 10.34 [0.51 to 40.58] |  | 8.70 [2.42 to 20.79]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 10.71 [2.27 to 28.23] | 0.00 [0.00 to 30.85] |  | 7.89 [0.00 to 97.58]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 14.29 [0.00 to 80.69] | 0.00 [0.00 to 28.49] |  | 10.87 [0.26 to 47.98]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 9.86 [4.06 to 19.26] | 0.00 [0.00 to 30.85] |  | 8.64 [2.48 to 20.40]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 7.69 [0.95 to 25.13] | 0.00 [0.00 to 26.46] |  | 5.26 [0.00 to 96.53]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 10.53 [1.30 to 33.14] | 0.00 [0.00 to 97.50] |  | 10.00 [1.23 to 31.70]

71. Secondary Outcome: Weekly Percentage of Subjects Reporting General Disorders and Administration Site Conditions (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°40 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 69
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 26.92 [0.28 to 88.26] | 26.92 [0.28 to 88.26]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 26.92 [17.50 to 38.16] | 26.92 [17.50 to 38.16]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 16.67 [6.34 to 32.90] | 16.67 [6.34 to 32.90]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 24.14 [15.60 to 34.50] | 24.14 [15.60 to 34.50]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 24.14 [2.85 to 64.50] | 24.14 [2.85 to 64.50]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 47.06 [22.98 to 72.19] | 47.06 [22.98 to 72.19]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 62.50 [2.31 to 99.81] | 62.50 [2.31 to 99.81]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 42.31 [1.05 to 96.43] |  | 42.31 [1.05 to 96.43]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 36.59 [0.25 to 96.81] |  | 36.59 [0.25 to 96.81]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 33.06 [24.88 to 42.08] | 42.86 [17.66 to 71.14] |  | 34.06 [26.21 to 42.61]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 33.33 [0.84 to 90.57] |  | 16.67 [0.00 to 100]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 50.00 [6.76 to 93.24] | 40.00 [5.27 to 85.34] | 40.00 [12.16 to 73.76]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 62.50 [24.49 to 91.48] | 44.12 [32.08 to 56.68] | 44.30 [31.16 to 58.06]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 35.71 [12.76 to 64.86] | 31.58 [17.50 to 48.65] | 32.69 [14.19 to 56.24]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 100 [15.81 to 100] | 0.00 [0.00 to 97.50] | 66.67 [9.43 to 99.16] | 66.67 [7.08 to 99.52]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 15.91 [6.64 to 30.07] |  | 15.91 [6.64 to 30.07]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 24.00 [0.07 to 89.80] |  | 24.00 [0.07 to 89.80]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 17.65 [0.00 to 100] | 17.24 [0.70 to 61.56] |  | 17.39 [7.82 to 31.42]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 21.43 [8.30 to 40.95] | 10.00 [0.25 to 44.50] |  | 18.42 [0.00 to 91.91]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 42.86 [0.00 to 100] | 9.09 [0.23 to 41.28] |  | 34.78 [1.29 to 89.85]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 18.31 [0.00 to 96.43] | 40.00 [12.16 to 73.76] |  | 20.99 [2.46 to 58.55]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 15.38 [4.36 to 34.87] | 16.67 [2.09 to 48.41] |  | 15.79 [6.02 to 31.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 21.05 [6.05 to 45.57] | 0.00 [0.00 to 97.50] |  | 20.00 [3.08 to 52.97]

72. Secondary Outcome: Weekly Percentage of Subjects Reporting Immune System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°42 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 5.96]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 4.15]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 23.16] |  | 0.00 [0.00 to 2.64]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.94] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 28.49] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 1.41 [0.00 to 23.79] | 0.00 [0.00 to 30.85] |  | 1.23 [0.03 to 6.69]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

73. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Infections and Infestations (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°44 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 1.92 [0.05 to 10.26] | 1.92 [0.05 to 10.26]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 5.13 [0.75 to 16.35] | 5.13 [0.75 to 16.35]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 6.67 [0.01 to 46.29] | 6.67 [0.01 to 46.29]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 3.45 [0.02 to 21.98] | 3.45 [0.02 to 21.98]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 6.90 [0.00 to 49.97] | 6.90 [0.00 to 49.97]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 17.65 [3.80 to 43.43] | 17.65 [3.80 to 43.43]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 11.54 [0.00 to 87.11] |  | 11.54 [0.00 to 87.11]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 12.20 [0.05 to 62.92] |  | 12.20 [0.05 to 62.92]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.81 [0.02 to 4.41] | 0.00 [0.00 to 23.16] |  | 0.72 [0.02 to 3.97]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 33.33 [0.84 to 90.57] |  | 16.67 [0.00 to 100]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 25.00 [0.63 to 80.59] | 0.00 [0.00 to 52.18] | 10.00 [0.00 to 78.43]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 12.50 [0.32 to 52.65] | 8.82 [3.31 to 18.22] | 8.86 [3.64 to 17.41]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 7.14 [0.18 to 33.87] | 10.53 [2.94 to 24.80] | 9.62 [0.41 to 39.32]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 6.82 [1.43 to 18.66] |  | 6.82 [1.43 to 18.66]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 6.00 [0.45 to 23.11] |  | 6.00 [0.45 to 23.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 6.90 [0.37 to 28.25] |  | 4.35 [0.17 to 20.04]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 7.14 [0.88 to 23.50] | 0.00 [0.00 to 30.85] |  | 5.26 [0.00 to 90.58]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 8.57 [1.80 to 23.06] | 0.00 [0.00 to 28.49] |  | 6.52 [0.54 to 24.21]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 9.86 [0.00 to 68.01] | 10.00 [0.25 to 44.50] |  | 9.88 [3.78 to 20.08]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 3.85 [0.10 to 19.64] | 8.33 [0.21 to 38.48] |  | 5.26 [0.00 to 70.17]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 5.26 [0.13 to 26.03] | 0.00 [0.00 to 97.50] |  | 5.00 [0.13 to 24.87]

74. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Metabolism and Nutrition Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°46 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 3.85 [0.11 to 19.24] | 3.85 [0.11 to 19.24]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 11.54 [1.53 to 35.14] | 11.54 [1.53 to 35.14]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 6.67 [1.85 to 16.20] | 6.67 [1.85 to 16.20]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 6.90 [1.95 to 16.58] | 6.90 [1.95 to 16.58]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 12.50 [0.00 to 99.41] | 12.50 [0.00 to 99.41]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 2.44 [0.00 to 24.59] |  | 2.44 [0.00 to 24.59]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.81 [0.02 to 4.41] | 0.00 [0.00 to 23.16] |  | 0.72 [0.02 to 3.97]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 20.00 [0.51 to 71.64] | 10.00 [0.00 to 66.77]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.94] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 2.86 [0.00 to 82.04] | 0.00 [0.00 to 28.49] |  | 2.17 [0.00 to 20.88]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 4.23 [0.00 to 57.27] | 0.00 [0.00 to 30.85] |  | 3.70 [0.18 to 16.55]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 26.46] |  | 2.63 [0.00 to 79.87]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 5.26 [0.13 to 26.03] | 0.00 [0.00 to 97.50] |  | 5.00 [0.13 to 24.87]

75. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Musculoskeletal and Connective Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°48 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 7.69 [0.19 to 36.17] | 7.69 [0.19 to 36.17]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 7.69 [1.08 to 24.10] | 7.69 [1.08 to 24.10]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 1.67 [0.00 to 55.06] | 1.67 [0.00 to 55.06]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 3.45 [0.07 to 18.45] | 3.45 [0.07 to 18.45]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 3.45 [0.00 to 56.00] | 3.45 [0.00 to 56.00]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 5.88 [0.00 to 98.47] | 5.88 [0.00 to 98.47]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 37.50 [0.00 to 100] | 37.50 [0.00 to 100]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 3.85 [0.00 to 45.20] |  | 3.85 [0.00 to 45.20]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 12.20 [0.00 to 80.65] |  | 12.20 [0.00 to 80.65]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 12.90 [7.56 to 20.11] | 0.00 [0.00 to 23.16] |  | 11.59 [5.18 to 21.48]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 25.00 [0.63 to 80.59] | 20.00 [0.51 to 71.64] | 20.00 [2.52 to 55.61]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 12.50 [0.32 to 52.65] | 14.71 [7.28 to 25.39] | 13.92 [7.16 to 23.55]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 21.43 [4.66 to 50.80] | 13.16 [4.41 to 28.09] | 15.38 [0.01 to 80.48]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 6.82 [1.43 to 18.66] |  | 6.82 [1.43 to 18.66]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 4.00 [0.00 to 34.94] |  | 4.00 [0.00 to 34.94]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 3.45 [0.09 to 17.76] |  | 2.17 [0.06 to 11.53]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 30.00 [6.67 to 65.25] |  | 7.89 [0.00 to 100]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 20.00 [0.00 to 92.27] | 0.00 [0.00 to 28.49] |  | 15.22 [0.84 to 53.59]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 11.27 [0.16 to 52.91] | 20.00 [2.52 to 55.61] |  | 12.35 [4.17 to 26.40]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 11.54 [2.45 to 30.15] | 8.33 [0.21 to 38.48] |  | 10.53 [0.61 to 39.92]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 5.26 [0.13 to 26.03] | 0.00 [0.00 to 97.50] |  | 5.00 [0.13 to 24.87]

76. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Nervous System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°50 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 1.92 [0.05 to 10.26] | 1.92 [0.05 to 10.26]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 7.69 [1.08 to 24.10] | 7.69 [1.08 to 24.10]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 1.67 [0.04 to 8.94] | 1.67 [0.04 to 8.94]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 5.75 [0.11 to 29.55] | 5.75 [0.11 to 29.55]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 3.45 [0.00 to 56.00] | 3.45 [0.00 to 56.00]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 5.88 [0.00 to 98.47] | 5.88 [0.00 to 98.47]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 37.50 [0.19 to 97.69] | 37.50 [0.19 to 97.69]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 7.69 [0.00 to 72.14] |  | 7.69 [0.00 to 72.14]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 12.20 [3.66 to 27.56] |  | 12.20 [3.66 to 27.56]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 4.84 [1.80 to 10.23] | 0.00 [0.00 to 23.16] |  | 4.35 [1.61 to 9.22]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 33.33 [0.84 to 90.57] |  | 16.67 [0.00 to 100]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 25.00 [0.63 to 80.59] | 0.00 [0.00 to 52.18] | 10.00 [0.00 to 78.43]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 12.50 [0.32 to 52.65] | 14.71 [7.28 to 25.39] | 13.92 [7.16 to 23.55]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 28.57 [8.39 to 58.10] | 13.16 [4.41 to 28.09] | 17.31 [0.00 to 99.06]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 100 [2.50 to 100] | 0.00 [0.00 to 70.76] | 16.67 [0.00 to 96.87]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 4.55 [0.56 to 15.47] |  | 4.55 [0.56 to 15.47]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 4.00 [0.00 to 48.56] |  | 4.00 [0.00 to 48.56]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 11.76 [0.00 to 99.87] | 6.90 [0.37 to 28.25] |  | 8.70 [2.19 to 21.73]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 10.71 [2.27 to 28.23] | 0.00 [0.00 to 30.85] |  | 7.89 [0.00 to 97.58]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 17.14 [0.00 to 96.14] | 0.00 [0.00 to 28.49] |  | 13.04 [0.16 to 59.60]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 14.08 [0.51 to 54.36] | 10.00 [0.25 to 44.50] |  | 13.58 [6.73 to 23.52]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

77. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Psychiatric Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°52 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 1.92 [0.05 to 10.26] | 1.92 [0.05 to 10.26]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 5.13 [0.75 to 16.35] | 5.13 [0.75 to 16.35]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 3.33 [0.00 to 34.01] | 3.33 [0.00 to 34.01]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 1.15 [0.03 to 6.40] | 1.15 [0.03 to 6.40]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 6.90 [0.11 to 35.38] | 6.90 [0.11 to 35.38]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 5.88 [0.00 to 100] | 5.88 [0.00 to 100]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 7.14 [0.00 to 99.99] |  | 0.72 [0.00 to 28.91]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 10.34 [0.51 to 40.58] |  | 6.52 [0.24 to 29.16]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 10.00 [0.25 to 44.50] |  | 2.63 [0.00 to 99.98]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 2.86 [0.00 to 82.04] | 0.00 [0.00 to 28.49] |  | 2.17 [0.00 to 20.88]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 1.41 [0.00 to 23.79] | 0.00 [0.00 to 30.85] |  | 1.23 [0.03 to 6.69]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 26.46] |  | 2.63 [0.00 to 79.87]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

78. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Respiratory, Thoracic and Mediastinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°54 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 26.92 [0.28 to 88.26] | 26.92 [0.28 to 88.26]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 25.64 [16.42 to 36.79] | 25.64 [16.42 to 36.79]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 18.33 [8.34 to 32.80] | 18.33 [8.34 to 32.80]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 22.99 [2.17 to 65.07] | 22.99 [2.17 to 65.07]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 17.24 [4.06 to 41.32] | 17.24 [4.06 to 41.32]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 35.29 [0.00 to 100] | 35.29 [0.00 to 100]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 31.25 [0.00 to 99.95] | 31.25 [0.00 to 99.95]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 15.38 [0.00 to 94.70] |  | 15.38 [0.00 to 94.70]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 17.07 [0.02 to 81.68] |  | 17.07 [0.02 to 81.68]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 9.68 [5.10 to 16.29] | 14.29 [0.00 to 100] |  | 10.14 [4.97 to 17.88]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 33.33 [0.84 to 90.57] | 33.33 [0.84 to 90.57] |  | 33.33 [4.33 to 77.72]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 25.00 [0.63 to 80.59] | 20.00 [0.51 to 71.64] | 20.00 [2.52 to 55.61]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 25.00 [3.19 to 65.09] | 19.12 [10.59 to 30.47] | 18.99 [11.03 to 29.38]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 14.29 [1.78 to 42.81] | 23.68 [11.44 to 40.24] | 21.15 [0.09 to 84.06]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 4.55 [0.56 to 15.47] |  | 4.55 [0.56 to 15.47]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 10.00 [0.65 to 37.24] |  | 10.00 [0.65 to 37.24]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 11.76 [0.00 to 99.87] | 6.90 [0.37 to 28.25] |  | 8.70 [2.19 to 21.73]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 17.86 [6.06 to 36.89] | 20.00 [2.52 to 55.61] |  | 18.42 [7.74 to 34.33]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 25.71 [12.49 to 43.26] | 0.00 [0.00 to 28.49] |  | 19.57 [1.20 to 62.87]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 21.13 [5.90 to 46.18] | 20.00 [2.52 to 55.61] |  | 20.99 [12.73 to 31.46]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 7.69 [0.95 to 25.13] | 0.00 [0.00 to 26.46] |  | 5.26 [0.00 to 96.53]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 10.53 [1.30 to 33.14] | 0.00 [0.00 to 97.50] |  | 10.00 [1.23 to 31.70]

79. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Skin and Subcutaneous Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°56 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 3.85 [0.11 to 19.24] | 3.85 [0.11 to 19.24]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 3.33 [0.00 to 33.03] | 3.33 [0.00 to 33.03]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 2.30 [0.00 to 52.37] | 2.30 [0.00 to 52.37]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 23.16] |  | 0.00 [0.00 to 2.64]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 7.14 [0.18 to 33.87] | 0.00 [0.00 to 9.25] | 1.92 [0.00 to 99.80]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 4.55 [0.56 to 15.47] |  | 4.55 [0.56 to 15.47]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 2.00 [0.00 to 27.58] |  | 2.00 [0.00 to 27.58]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 3.45 [0.09 to 17.76] |  | 2.17 [0.06 to 11.53]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 3.57 [0.09 to 18.35] | 10.00 [0.25 to 44.50] |  | 5.26 [0.00 to 85.52]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 28.49] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 7.04 [2.33 to 15.67] | 0.00 [0.00 to 30.85] |  | 6.17 [2.03 to 13.82]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

80. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Cardiac Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°58 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 5.96]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 4.15]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 3.85 [0.00 to 45.20] |  | 3.85 [0.00 to 45.20]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 23.16] |  | 0.00 [0.00 to 2.64]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.94] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 28.49] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 0.00 [0.00 to 5.06] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 4.45]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

81. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Ear and Labyrinth Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°60 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 1.67 [0.04 to 8.94] | 1.67 [0.04 to 8.94]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 4.15]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 2.44 [0.00 to 24.59] |  | 2.44 [0.00 to 24.59]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 23.16] |  | 0.00 [0.00 to 2.64]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 25.00 [3.19 to 65.09] | 0.00 [0.00 to 5.28] | 2.53 [0.00 to 66.57]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 7.14 [0.18 to 33.87] | 0.00 [0.00 to 9.25] | 1.92 [0.00 to 99.80]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 2.00 [0.00 to 27.58] |  | 2.00 [0.00 to 27.58]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.94] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 2.86 [0.00 to 82.04] | 0.00 [0.00 to 28.49] |  | 2.17 [0.00 to 20.88]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 0.00 [0.00 to 5.06] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 4.45]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

82. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Eye Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°62 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 5.96]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 4.15]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 23.16] |  | 0.00 [0.00 to 2.64]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 2.27 [0.06 to 12.02] |  | 2.27 [0.06 to 12.02]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 6.90 [0.37 to 28.25] |  | 4.35 [0.17 to 20.04]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 2.86 [0.00 to 82.04] | 0.00 [0.00 to 28.49] |  | 2.17 [0.00 to 20.88]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 0.00 [0.00 to 5.06] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 4.45]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

83. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Injury, Poisoning and Procedural Complications (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°64 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 5.96]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 4.15]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 23.16] |  | 0.00 [0.00 to 2.64]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 12.50 [0.32 to 52.65] | 0.00 [0.00 to 5.28] | 1.27 [0.00 to 41.55]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.94] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 28.49] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 0.00 [0.00 to 5.06] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 4.45]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

84. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Investigations (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°66 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 5.96]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 4.15]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.00 [0.00 to 2.93] | 7.14 [0.00 to 99.99] |  | 0.72 [0.00 to 28.91]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 33.33 [0.84 to 90.57] |  | 16.67 [0.00 to 100]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 3.45 [0.09 to 17.76] |  | 2.17 [0.06 to 11.53]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 28.49] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 1.41 [0.00 to 23.79] | 0.00 [0.00 to 30.85] |  | 1.23 [0.03 to 6.69]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

85. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Vascular Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1, by Vaccine Group and Overall, and by Age Category
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°68 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Week 42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Week 42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Week 43: number analyzed (Participants) | 0 | 0 | 78 | 78
  6 months to 17 years,Week 43 |  |  | 0.00 [0.00 to 4.62] | 0.00 [0.00 to 4.62]
  6 months to 17 years,Week 44: number analyzed (Participants) | 0 | 0 | 60 | 60
  6 months to 17 years,Week 44 |  |  | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 5.96]
  6 months to 17 years,Week 45: number analyzed (Participants) | 0 | 0 | 87 | 87
  6 months to 17 years,Week 45 |  |  | 0.00 [0.00 to 4.15] | 0.00 [0.00 to 4.15]
  6 months to 17 years,Week 46: number analyzed (Participants) | 0 | 0 | 29 | 29
  6 months to 17 years,Week 46 |  |  | 0.00 [0.00 to 11.94] | 0.00 [0.00 to 11.94]
  6 months to 17 years,Week 47: number analyzed (Participants) | 0 | 0 | 17 | 17
  6 months to 17 years,Week 47 |  |  | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 19.51]
  6 months to 17 years,Week 48: number analyzed (Participants) | 0 | 0 | 16 | 16
  6 months to 17 years,Week 48 |  |  | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 20.59]
  18-65 years,Week 40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Week 40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Week 41: number analyzed (Participants) | 0 | 41 | 0 | 41
  18-65 years,Week 41 |  | 0.00 [0.00 to 8.60] |  | 0.00 [0.00 to 8.60]
  18-65 years,Week 42: number analyzed (Participants) | 124 | 14 | 0 | 138
  18-65 years,Week 42 | 0.81 [0.02 to 4.41] | 0.00 [0.00 to 23.16] |  | 0.72 [0.02 to 3.97]
  18-65 years,Week 43: number analyzed (Participants) | 3 | 3 | 0 | 6
  18-65 years,Week 43 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 45.93]
  18-65 years,Week 44: number analyzed (Participants) | 1 | 4 | 5 | 10
  18-65 years,Week 44 | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 60.24] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]
  18-65 years,Week 45: number analyzed (Participants) | 3 | 8 | 68 | 79
  18-65 years,Week 45 | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 5.28] | 0.00 [0.00 to 4.56]
  18-65 years,Week 46: number analyzed (Participants) | 0 | 14 | 38 | 52
  18-65 years,Week 46 |  | 0.00 [0.00 to 23.16] | 0.00 [0.00 to 9.25] | 0.00 [0.00 to 6.85]
  18-65 years,Week 47: number analyzed (Participants) | 2 | 1 | 3 | 6
  18-65 years,Week 47 | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 45.93]
  >65 years,Week 40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Week 40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Week 41: number analyzed (Participants) | 0 | 50 | 0 | 50
  >65 years,Week 41 |  | 0.00 [0.00 to 7.11] |  | 0.00 [0.00 to 7.11]
  >65 years,Week 42: number analyzed (Participants) | 17 | 29 | 0 | 46
  >65 years,Week 42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 11.94] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 43: number analyzed (Participants) | 28 | 10 | 0 | 38
  >65 years,Week 43 | 0.00 [0.00 to 12.34] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 44: number analyzed (Participants) | 35 | 11 | 0 | 46
  >65 years,Week 44 | 0.00 [0.00 to 10.00] | 0.00 [0.00 to 28.49] |  | 0.00 [0.00 to 7.71]
  >65 years,Week 45: number analyzed (Participants) | 71 | 10 | 0 | 81
  >65 years,Week 45 | 0.00 [0.00 to 5.06] | 0.00 [0.00 to 30.85] |  | 0.00 [0.00 to 4.45]
  >65 years,Week 46: number analyzed (Participants) | 26 | 12 | 0 | 38
  >65 years,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 26.46] |  | 0.00 [0.00 to 9.25]
  >65 years,Week 47: number analyzed (Participants) | 19 | 1 | 0 | 20
  >65 years,Week 47 | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 97.50] |  | 0.00 [0.00 to 16.84]

86. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any AEs Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°2 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 44.23 [0.11 to 99.54] | 44.23 [0.11 to 99.54]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 46.15 [14.72 to 80.10] | 46.15 [14.72 to 80.10]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 42.11 [34.99 to 49.47] | 42.11 [34.99 to 49.47]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 43.68 [28.34 to 59.96] | 43.68 [28.34 to 59.96]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 42.48 [29.17 to 56.65] | 42.48 [29.17 to 56.65]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 43.96 [23.26 to 66.33] | 43.96 [23.26 to 66.33]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 45.72 [20.08 to 73.17] | 45.72 [20.08 to 73.17]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 45.72 [20.08 to 73.17] | 45.72 [20.08 to 73.17]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 45.72 [20.08 to 73.17] | 45.72 [20.08 to 73.17]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 45.72 [20.08 to 73.17] | 45.72 [20.08 to 73.17]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 45.72 [20.08 to 73.17] | 45.72 [20.08 to 73.17]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 46.15 [0.35 to 99.22] |  | 46.15 [0.35 to 99.22]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 43.28 [1.27 to 96.39] |  | 43.28 [1.27 to 96.39]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 47.58 [38.54 to 56.74] | 44.44 [4.39 to 91.64] |  | 46.34 [32.14 to 60.99]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 47.24 [38.32 to 56.30] | 44.05 [4.66 to 90.87] |  | 45.97 [34.03 to 58.26]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 46.88 [29.25 to 65.09] | 44.32 [5.76 to 89.45] | 60.00 [14.66 to 94.73] | 46.15 [35.85 to 56.70]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 45.80 [8.30 to 87.53] | 47.92 [10.13 to 87.69] | 56.16 [44.05 to 67.76] | 49.00 [39.73 to 58.32]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 45.80 [8.30 to 87.53] | 48.18 [13.61 to 84.15] | 52.25 [42.56 to 61.82] | 48.58 [41.21 to 55.99]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 46.62 [23.72 to 70.61] | 48.65 [13.91 to 84.42] | 52.63 [43.06 to 62.06] | 49.16 [41.99 to 56.36]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 46.62 [23.72 to 70.61] | 48.65 [13.91 to 84.42] | 52.63 [43.06 to 62.06] | 49.16 [41.99 to 56.36]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 46.62 [23.72 to 70.61] | 48.65 [13.91 to 84.42] | 52.63 [43.06 to 62.06] | 49.16 [41.99 to 56.36]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 46.62 [23.72 to 70.61] | 48.65 [13.91 to 84.42] | 52.63 [43.06 to 62.06] | 49.16 [41.99 to 56.36]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 46.62 [23.72 to 70.61] | 48.65 [13.91 to 84.42] | 52.63 [43.06 to 62.06] | 49.16 [41.99 to 56.36]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 46.62 [23.72 to 70.61] | 48.65 [13.91 to 84.42] | 52.63 [43.06 to 62.06] | 49.16 [41.99 to 56.36]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 25.00 [12.33 to 41.82] |  | 25.00 [12.33 to 41.82]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 28.72 [1.77 to 79.09] |  | 28.72 [1.77 to 79.09]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 29.41 [0.00 to 100] | 27.64 [4.41 to 66.54] |  | 27.86 [12.90 to 47.58]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 40.00 [0.00 to 99.97] | 28.57 [4.53 to 68.14] |  | 31.46 [15.89 to 50.84]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 47.50 [18.69 to 77.61] | 27.08 [7.02 to 57.93] |  | 34.38 [20.23 to 50.89]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 42.38 [18.45 to 69.29] | 28.57 [6.49 to 62.62] |  | 35.41 [24.11 to 48.04]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 40.11 [16.85 to 67.22] | 28.92 [7.25 to 61.51] |  | 34.69 [24.92 to 45.51]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 39.29 [17.18 to 65.18] | 28.74 [7.49 to 60.56] |  | 34.44 [25.25 to 44.56]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 39.29 [17.18 to 65.18] | 28.74 [7.49 to 60.56] |  | 34.44 [25.25 to 44.56]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 39.29 [17.18 to 65.18] | 28.74 [7.49 to 60.56] |  | 34.44 [25.25 to 44.56]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 39.29 [17.18 to 65.18] | 28.74 [7.49 to 60.56] |  | 34.44 [25.25 to 44.56]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 39.29 [17.18 to 65.18] | 28.74 [7.49 to 60.56] |  | 34.44 [25.25 to 44.56]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 39.29 [17.18 to 65.18] | 28.74 [7.49 to 60.56] |  | 34.44 [25.25 to 44.56]

87. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Gastrointestinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°4 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 7.69 [0.19 to 36.17] | 7.69 [0.19 to 36.17]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 8.46 [3.32 to 17.07] | 8.46 [3.32 to 17.07]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 6.84 [3.69 to 11.42] | 6.84 [3.69 to 11.42]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 6.50 [3.90 to 10.08] | 6.50 [3.90 to 10.08]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 6.54 [3.28 to 11.46] | 6.54 [3.28 to 11.46]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 6.81 [3.04 to 12.85] | 6.81 [3.04 to 12.85]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 7.08 [2.85 to 14.16] | 7.08 [2.85 to 14.16]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 7.08 [2.85 to 14.16] | 7.08 [2.85 to 14.16]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 7.08 [2.85 to 14.16] | 7.08 [2.85 to 14.16]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 7.08 [2.85 to 14.16] | 7.08 [2.85 to 14.16]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 7.08 [2.85 to 14.16] | 7.08 [2.85 to 14.16]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 3.85 [0.00 to 45.20] |  | 3.85 [0.00 to 45.20]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 1.49 [0.01 to 10.39] |  | 1.49 [0.01 to 10.39]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 1.61 [0.20 to 5.70] | 3.70 [0.00 to 37.31] |  | 2.44 [0.21 to 9.46]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 1.57 [0.19 to 5.57] | 4.76 [0.00 to 51.14] |  | 2.84 [0.21 to 11.55]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 1.56 [0.19 to 5.53] | 5.68 [0.00 to 59.48] | 20.00 [0.51 to 71.64] | 3.62 [0.31 to 13.98]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 1.53 [0.19 to 5.41] | 7.29 [0.00 to 68.92] | 2.74 [0.33 to 9.55] | 3.67 [0.35 to 13.62]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 1.53 [0.19 to 5.41] | 7.27 [0.00 to 60.31] | 6.31 [2.57 to 12.56] | 4.83 [0.98 to 13.63]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 1.50 [0.08 to 6.80] | 7.21 [0.00 to 59.24] | 6.14 [2.50 to 12.24] | 4.75 [0.99 to 13.26]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 1.50 [0.08 to 6.80] | 7.21 [0.00 to 59.24] | 6.14 [2.50 to 12.24] | 4.75 [0.99 to 13.26]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 1.50 [0.08 to 6.80] | 7.21 [0.00 to 59.24] | 6.14 [2.50 to 12.24] | 4.75 [0.99 to 13.26]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 1.50 [0.08 to 6.80] | 7.21 [0.00 to 59.24] | 6.14 [2.50 to 12.24] | 4.75 [0.99 to 13.26]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 1.50 [0.08 to 6.80] | 7.21 [0.00 to 59.24] | 6.14 [2.50 to 12.24] | 4.75 [0.99 to 13.26]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 1.50 [0.08 to 6.80] | 7.21 [0.00 to 59.24] | 6.14 [2.50 to 12.24] | 4.75 [0.99 to 13.26]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 2.27 [0.06 to 12.02] |  | 2.27 [0.06 to 12.02]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 3.19 [0.24 to 12.75] |  | 3.19 [0.24 to 12.75]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 5.88 [0.00 to 94.68] | 4.88 [0.16 to 23.00] |  | 5.00 [1.42 to 12.14]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 8.89 [0.01 to 59.81] | 4.51 [0.33 to 17.92] |  | 5.62 [2.10 to 11.79]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 11.25 [3.20 to 26.18] | 4.17 [0.54 to 13.99] |  | 6.70 [2.88 to 12.90]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 10.60 [6.09 to 16.80] | 3.90 [0.72 to 11.49] |  | 7.21 [3.38 to 13.18]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 10.17 [5.80 to 16.22] | 3.61 [0.91 to 9.40] |  | 7.00 [3.24 to 12.89]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 10.20 [6.24 to 15.50] | 3.59 [0.92 to 9.26] |  | 7.16 [3.35 to 13.11]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 10.20 [6.24 to 15.50] | 3.59 [0.92 to 9.26] |  | 7.16 [3.35 to 13.11]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 10.20 [6.24 to 15.50] | 3.59 [0.92 to 9.26] |  | 7.16 [3.35 to 13.11]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 10.20 [6.24 to 15.50] | 3.59 [0.92 to 9.26] |  | 7.16 [3.35 to 13.11]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 10.20 [6.24 to 15.50] | 3.59 [0.92 to 9.26] |  | 7.16 [3.35 to 13.11]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 10.20 [6.24 to 15.50] | 3.59 [0.92 to 9.26] |  | 7.16 [3.35 to 13.11]

88. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any General Disorders and Administration Site Conditions (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°6 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 26.92 [0.28 to 88.26] | 26.92 [0.28 to 88.26]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 26.92 [8.05 to 55.09] | 26.92 [8.05 to 55.09]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 23.68 [17.83 to 30.38] | 23.68 [17.83 to 30.38]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 23.83 [18.93 to 29.29] | 23.83 [18.93 to 29.29]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 23.86 [19.19 to 29.04] | 23.86 [19.19 to 29.04]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 25.08 [16.20 to 35.81] | 25.08 [16.20 to 35.81]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 26.84 [11.26 to 48.19] | 26.84 [11.26 to 48.19]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 26.84 [11.26 to 48.19] | 26.84 [11.26 to 48.19]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 26.84 [11.26 to 48.19] | 26.84 [11.26 to 48.19]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 26.84 [11.26 to 48.19] | 26.84 [11.26 to 48.19]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 26.84 [11.26 to 48.19] | 26.84 [11.26 to 48.19]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 42.31 [1.05 to 96.43] |  | 42.31 [1.05 to 96.43]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 38.81 [2.16 to 90.96] |  | 38.81 [2.16 to 90.96]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 33.06 [24.88 to 42.08] | 39.51 [5.87 to 83.54] |  | 35.61 [21.75 to 51.49]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 32.28 [14.53 to 54.80] | 39.29 [6.21 to 82.59] |  | 35.07 [23.64 to 47.91]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 32.03 [10.00 to 62.27] | 39.77 [7.76 to 80.48] | 40.00 [5.27 to 85.34] | 35.29 [25.26 to 46.38]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 31.30 [2.25 to 81.21] | 41.67 [11.84 to 77.00] | 43.84 [32.24 to 55.95] | 37.67 [28.00 to 48.11]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 31.30 [2.25 to 81.21] | 40.91 [13.91 to 72.76] | 39.64 [30.48 to 49.37] | 36.93 [29.42 to 44.94]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 32.33 [16.16 to 52.33] | 40.54 [13.60 to 72.56] | 40.35 [31.27 to 49.95] | 37.43 [30.02 to 45.30]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 32.33 [16.16 to 52.33] | 40.54 [13.60 to 72.56] | 40.35 [31.27 to 49.95] | 37.43 [30.02 to 45.30]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 32.33 [16.16 to 52.33] | 40.54 [13.60 to 72.56] | 40.35 [31.27 to 49.95] | 37.43 [30.02 to 45.30]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 32.33 [16.16 to 52.33] | 40.54 [13.60 to 72.56] | 40.35 [31.27 to 49.95] | 37.43 [30.02 to 45.30]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 32.33 [16.16 to 52.33] | 40.54 [13.60 to 72.56] | 40.35 [31.27 to 49.95] | 37.43 [30.02 to 45.30]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 32.33 [16.16 to 52.33] | 40.54 [13.60 to 72.56] | 40.35 [31.27 to 49.95] | 37.43 [30.02 to 45.30]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 15.91 [6.64 to 30.07] |  | 15.91 [6.64 to 30.07]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 20.21 [0.90 to 67.30] |  | 20.21 [0.90 to 67.30]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 17.65 [0.00 to 100] | 19.51 [2.47 to 54.52] |  | 19.29 [8.10 to 35.82]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 20.00 [0.00 to 91.70] | 18.80 [3.70 to 47.08] |  | 19.10 [10.71 to 30.22]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 30.00 [2.61 to 77.58] | 18.06 [5.08 to 40.25] |  | 22.32 [12.73 to 34.68]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 24.50 [2.22 to 68.32] | 19.48 [4.44 to 46.28] |  | 21.97 [13.20 to 33.06]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 23.16 [2.41 to 64.26] | 19.28 [5.31 to 42.95] |  | 21.28 [13.22 to 31.39]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 22.96 [3.15 to 60.38] | 19.16 [5.45 to 42.20] |  | 21.21 [13.60 to 30.64]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 22.96 [3.15 to 60.38] | 19.16 [5.45 to 42.20] |  | 21.21 [13.60 to 30.64]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 22.96 [3.15 to 60.38] | 19.16 [5.45 to 42.20] |  | 21.21 [13.60 to 30.64]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 22.96 [3.15 to 60.38] | 19.16 [5.45 to 42.20] |  | 21.21 [13.60 to 30.64]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 22.96 [3.15 to 60.38] | 19.16 [5.45 to 42.20] |  | 21.21 [13.60 to 30.64]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 22.96 [3.15 to 60.38] | 19.16 [5.45 to 42.20] |  | 21.21 [13.60 to 30.64]

89. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Immune System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°8 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.80]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 0.00 [0.00 to 1.92] | 0.00 [0.00 to 1.92]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 1.32]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 0.00 [0.00 to 1.20] | 0.00 [0.00 to 1.20]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 0.00 [0.00 to 1.14] | 0.00 [0.00 to 1.14]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 4.45] |  | 0.00 [0.00 to 1.78]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 4.30] |  | 0.00 [0.00 to 1.73]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.66]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 0.00 [0.00 to 3.77] | 0.00 [0.00 to 4.93] | 0.00 [0.00 to 1.22]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 1.04]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 0.00 [0.00 to 3.85] |  | 0.00 [0.00 to 3.85]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 2.95] |  | 0.00 [0.00 to 2.60]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 2.05]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 2.53] |  | 0.00 [0.00 to 1.63]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 0.66 [0.02 to 3.63] | 0.00 [0.00 to 2.37] |  | 0.33 [0.01 to 1.90]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 0.56 [0.01 to 3.11] | 0.00 [0.00 to 2.20] |  | 0.29 [0.01 to 1.61]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 2.18] |  | 0.28 [0.01 to 1.53]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 2.18] |  | 0.28 [0.01 to 1.53]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 2.18] |  | 0.28 [0.01 to 1.53]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 2.18] |  | 0.28 [0.01 to 1.53]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 2.18] |  | 0.28 [0.01 to 1.53]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 0.51 [0.01 to 2.81] | 0.00 [0.00 to 2.18] |  | 0.28 [0.01 to 1.53]

90. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Infections and Infestations (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°10 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 1.92 [0.05 to 10.26] | 1.92 [0.05 to 10.26]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 3.85 [0.30 to 15.16] | 3.85 [0.30 to 15.16]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 4.74 [1.21 to 12.12] | 4.74 [1.21 to 12.12]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 4.33 [0.70 to 13.42] | 4.33 [0.70 to 13.42]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 4.58 [0.31 to 18.44] | 4.58 [0.31 to 18.44]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 5.26 [0.12 to 26.68] | 5.26 [0.12 to 26.68]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 5.60 [0.09 to 29.71] | 5.60 [0.09 to 29.71]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 5.60 [0.09 to 29.71] | 5.60 [0.09 to 29.71]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 5.60 [0.09 to 29.71] | 5.60 [0.09 to 29.71]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 5.60 [0.09 to 29.71] | 5.60 [0.09 to 29.71]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 5.60 [0.09 to 29.71] | 5.60 [0.09 to 29.71]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 11.54 [0.00 to 87.11] |  | 11.54 [0.00 to 87.11]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 11.94 [0.31 to 50.82] |  | 11.94 [0.31 to 50.82]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.81 [0.02 to 4.41] | 9.88 [0.03 to 56.84] |  | 4.39 [0.00 to 35.51]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.79 [0.02 to 4.31] | 10.71 [0.12 to 52.31] |  | 4.74 [0.04 to 28.25]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.78 [0.02 to 4.28] | 11.36 [0.27 to 49.65] | 0.00 [0.00 to 52.18] | 4.98 [0.13 to 24.63]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.76 [0.02 to 4.18] | 11.46 [0.46 to 45.77] | 8.22 [3.08 to 17.04] | 6.00 [0.79 to 19.61]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.76 [0.02 to 4.18] | 10.91 [0.70 to 40.17] | 9.01 [4.41 to 15.94] | 6.53 [1.32 to 18.21]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.75 [0.02 to 4.12] | 10.81 [0.69 to 39.88] | 8.77 [4.29 to 15.54] | 6.42 [1.33 to 17.73]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.75 [0.02 to 4.12] | 10.81 [0.69 to 39.88] | 8.77 [4.29 to 15.54] | 6.42 [1.33 to 17.73]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.75 [0.02 to 4.12] | 10.81 [0.69 to 39.88] | 8.77 [4.29 to 15.54] | 6.42 [1.33 to 17.73]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.75 [0.02 to 4.12] | 10.81 [0.69 to 39.88] | 8.77 [4.29 to 15.54] | 6.42 [1.33 to 17.73]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.75 [0.02 to 4.12] | 10.81 [0.69 to 39.88] | 8.77 [4.29 to 15.54] | 6.42 [1.33 to 17.73]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.75 [0.02 to 4.12] | 10.81 [0.69 to 39.88] | 8.77 [4.29 to 15.54] | 6.42 [1.33 to 17.73]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 6.82 [1.43 to 18.66] |  | 6.82 [1.43 to 18.66]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 6.38 [2.38 to 13.38] |  | 6.38 [2.38 to 13.38]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 6.50 [2.64 to 12.98] |  | 5.71 [2.50 to 10.95]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 4.44 [0.00 to 34.75] | 6.02 [2.63 to 11.51] |  | 5.62 [2.73 to 10.09]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 6.25 [2.06 to 13.99] | 5.56 [2.43 to 10.65] |  | 5.80 [3.13 to 9.72]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 7.95 [3.76 to 14.39] | 5.84 [2.71 to 10.80] |  | 6.89 [4.31 to 10.33]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 7.34 [3.12 to 14.25] | 6.02 [2.93 to 10.80] |  | 6.71 [4.30 to 9.89]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 7.14 [3.08 to 13.73] | 5.99 [2.91 to 10.74] |  | 6.61 [4.28 to 9.68]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 7.14 [3.08 to 13.73] | 5.99 [2.91 to 10.74] |  | 6.61 [4.28 to 9.68]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 7.14 [3.08 to 13.73] | 5.99 [2.91 to 10.74] |  | 6.61 [4.28 to 9.68]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 7.14 [3.08 to 13.73] | 5.99 [2.91 to 10.74] |  | 6.61 [4.28 to 9.68]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 7.14 [3.08 to 13.73] | 5.99 [2.91 to 10.74] |  | 6.61 [4.28 to 9.68]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 7.14 [3.08 to 13.73] | 5.99 [2.91 to 10.74] |  | 6.61 [4.28 to 9.68]

91. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Metabolism and Nutrition Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°12 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 3.85 [0.11 to 19.24] | 3.85 [0.11 to 19.24]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 8.46 [0.60 to 31.78] | 8.46 [0.60 to 31.78]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 7.89 [4.49 to 12.69] | 7.89 [4.49 to 12.69]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 7.58 [4.75 to 11.36] | 7.58 [4.75 to 11.36]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 6.86 [3.37 to 12.19] | 6.86 [3.37 to 12.19]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 6.50 [2.13 to 14.56] | 6.50 [2.13 to 14.56]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 6.78 [3.38 to 11.94] | 6.78 [3.38 to 11.94]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 6.78 [3.38 to 11.94] | 6.78 [3.38 to 11.94]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 6.78 [3.38 to 11.94] | 6.78 [3.38 to 11.94]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 6.78 [3.38 to 11.94] | 6.78 [3.38 to 11.94]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 6.78 [3.38 to 11.94] | 6.78 [3.38 to 11.94]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 1.49 [0.01 to 10.39] |  | 1.49 [0.01 to 10.39]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.81 [0.02 to 4.41] | 1.23 [0.00 to 12.57] |  | 0.98 [0.12 to 3.48]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.79 [0.02 to 4.31] | 1.19 [0.00 to 12.76] |  | 0.95 [0.11 to 3.38]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.78 [0.02 to 4.28] | 1.14 [0.00 to 13.03] | 20.00 [0.51 to 71.64] | 1.36 [0.23 to 4.22]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.76 [0.02 to 4.18] | 1.04 [0.00 to 13.56] | 1.37 [0.03 to 7.40] | 1.00 [0.21 to 2.89]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.76 [0.02 to 4.18] | 0.91 [0.00 to 14.27] | 0.90 [0.02 to 4.92] | 0.85 [0.18 to 2.47]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.75 [0.02 to 4.12] | 0.90 [0.00 to 14.30] | 0.88 [0.02 to 4.79] | 0.84 [0.17 to 2.43]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.75 [0.02 to 4.12] | 0.90 [0.00 to 14.30] | 0.88 [0.02 to 4.79] | 0.84 [0.17 to 2.43]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.75 [0.02 to 4.12] | 0.90 [0.00 to 14.30] | 0.88 [0.02 to 4.79] | 0.84 [0.17 to 2.43]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.75 [0.02 to 4.12] | 0.90 [0.00 to 14.30] | 0.88 [0.02 to 4.79] | 0.84 [0.17 to 2.43]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.75 [0.02 to 4.12] | 0.90 [0.00 to 14.30] | 0.88 [0.02 to 4.79] | 0.84 [0.17 to 2.43]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.75 [0.02 to 4.12] | 0.90 [0.00 to 14.30] | 0.88 [0.02 to 4.79] | 0.84 [0.17 to 2.43]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 0.00 [0.00 to 3.85] |  | 0.00 [0.00 to 3.85]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 2.95] |  | 0.00 [0.00 to 2.60]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 2.05]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 1.25 [0.00 to 27.29] | 0.00 [0.00 to 2.53] |  | 0.45 [0.00 to 4.19]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 2.65 [0.73 to 6.64] | 0.00 [0.00 to 2.37] |  | 1.31 [0.13 to 4.95]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 2.82 [0.92 to 6.47] | 0.00 [0.00 to 2.20] |  | 1.46 [0.15 to 5.49]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 3.06 [1.13 to 6.54] | 0.00 [0.00 to 2.18] |  | 1.65 [0.18 to 6.07]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 3.06 [1.13 to 6.54] | 0.00 [0.00 to 2.18] |  | 1.65 [0.18 to 6.07]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 3.06 [1.13 to 6.54] | 0.00 [0.00 to 2.18] |  | 1.65 [0.18 to 6.07]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 3.06 [1.13 to 6.54] | 0.00 [0.00 to 2.18] |  | 1.65 [0.18 to 6.07]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 3.06 [1.13 to 6.54] | 0.00 [0.00 to 2.18] |  | 1.65 [0.18 to 6.07]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 3.06 [1.13 to 6.54] | 0.00 [0.00 to 2.18] |  | 1.65 [0.18 to 6.07]

92. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Musculoskeletal and Connective Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°14 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 7.69 [0.19 to 36.17] | 7.69 [0.19 to 36.17]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 7.69 [0.55 to 29.13] | 7.69 [0.55 to 29.13]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 5.79 [2.93 to 10.12] | 5.79 [2.93 to 10.12]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 5.05 [2.23 to 9.66] | 5.05 [2.23 to 9.66]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 4.90 [2.77 to 7.96] | 4.90 [2.77 to 7.96]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 4.95 [2.86 to 7.92] | 4.95 [2.86 to 7.92]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 6.49 [0.78 to 21.64] | 6.49 [0.78 to 21.64]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 6.49 [0.78 to 21.64] | 6.49 [0.78 to 21.64]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 6.49 [0.78 to 21.64] | 6.49 [0.78 to 21.64]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 6.49 [0.78 to 21.64] | 6.49 [0.78 to 21.64]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 6.49 [0.78 to 21.64] | 6.49 [0.78 to 21.64]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 3.85 [0.00 to 45.20] |  | 3.85 [0.00 to 45.20]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 8.96 [0.04 to 51.75] |  | 8.96 [0.04 to 51.75]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 12.90 [7.56 to 20.11] | 7.41 [0.00 to 58.57] |  | 10.73 [4.36 to 21.03]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 12.60 [6.09 to 22.20] | 7.14 [0.00 to 59.06] |  | 10.43 [4.67 to 19.37]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 12.50 [4.46 to 26.00] | 7.95 [0.02 to 49.34] | 20.00 [0.51 to 71.64] | 10.86 [6.15 to 17.39]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 12.21 [1.37 to 38.68] | 8.33 [0.10 to 42.90] | 15.07 [7.77 to 25.36] | 11.67 [7.78 to 16.61]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 12.21 [1.37 to 38.68] | 10.00 [0.82 to 35.33] | 14.41 [8.47 to 22.35] | 12.22 [8.98 to 16.10]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 12.03 [0.49 to 47.47] | 9.91 [0.83 to 34.92] | 14.04 [8.24 to 21.79] | 12.01 [8.83 to 15.84]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 12.03 [0.49 to 47.47] | 9.91 [0.83 to 34.92] | 14.04 [8.24 to 21.79] | 12.01 [8.83 to 15.84]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 12.03 [0.49 to 47.47] | 9.91 [0.83 to 34.92] | 14.04 [8.24 to 21.79] | 12.01 [8.83 to 15.84]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 12.03 [0.49 to 47.47] | 9.91 [0.83 to 34.92] | 14.04 [8.24 to 21.79] | 12.01 [8.83 to 15.84]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 12.03 [0.49 to 47.47] | 9.91 [0.83 to 34.92] | 14.04 [8.24 to 21.79] | 12.01 [8.83 to 15.84]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 12.03 [0.49 to 47.47] | 9.91 [0.83 to 34.92] | 14.04 [8.24 to 21.79] | 12.01 [8.83 to 15.84]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 6.82 [1.43 to 18.66] |  | 6.82 [1.43 to 18.66]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 5.32 [0.15 to 25.86] |  | 5.32 [0.15 to 25.86]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 4.88 [0.21 to 21.80] |  | 4.29 [0.85 to 12.27]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 6.77 [1.11 to 20.35] |  | 5.06 [0.88 to 15.13]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 8.75 [0.29 to 38.30] | 6.25 [1.27 to 17.39] |  | 7.14 [3.84 to 11.95]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 9.93 [2.03 to 26.68] | 7.14 [1.52 to 19.35] |  | 8.52 [5.44 to 12.59]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 10.17 [3.14 to 22.97] | 7.23 [1.76 to 18.52] |  | 8.75 [5.98 to 12.25]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 9.69 [2.88 to 22.35] | 7.19 [1.79 to 18.25] |  | 8.54 [5.88 to 11.90]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 9.69 [2.88 to 22.35] | 7.19 [1.79 to 18.25] |  | 8.54 [5.88 to 11.90]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 9.69 [2.88 to 22.35] | 7.19 [1.79 to 18.25] |  | 8.54 [5.88 to 11.90]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 9.69 [2.88 to 22.35] | 7.19 [1.79 to 18.25] |  | 8.54 [5.88 to 11.90]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 9.69 [2.88 to 22.35] | 7.19 [1.79 to 18.25] |  | 8.54 [5.88 to 11.90]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 9.69 [2.88 to 22.35] | 7.19 [1.79 to 18.25] |  | 8.54 [5.88 to 11.90]

93. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Nervous System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°16 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 1.92 [0.05 to 10.26] | 1.92 [0.05 to 10.26]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 5.38 [0.40 to 20.90] | 5.38 [0.40 to 20.90]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 4.21 [1.84 to 8.13] | 4.21 [1.84 to 8.13]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 4.69 [1.31 to 11.52] | 4.69 [1.31 to 11.52]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 4.58 [1.86 to 9.19] | 4.58 [1.86 to 9.19]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 4.64 [2.09 to 8.78] | 4.64 [2.09 to 8.78]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 6.19 [1.88 to 14.44] | 6.19 [1.88 to 14.44]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 6.19 [1.88 to 14.44] | 6.19 [1.88 to 14.44]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 6.19 [1.88 to 14.44] | 6.19 [1.88 to 14.44]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 6.19 [1.88 to 14.44] | 6.19 [1.88 to 14.44]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 6.19 [1.88 to 14.44] | 6.19 [1.88 to 14.44]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 7.69 [0.00 to 72.14] |  | 7.69 [0.00 to 72.14]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 10.45 [3.70 to 22.05] |  | 10.45 [3.70 to 22.05]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 4.84 [1.80 to 10.23] | 8.64 [1.19 to 26.97] |  | 6.34 [2.11 to 14.10]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 4.72 [1.75 to 10.00] | 9.52 [1.88 to 26.03] |  | 6.64 [2.66 to 13.33]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 4.69 [1.73 to 9.94] | 10.23 [2.02 to 27.74] | 0.00 [0.00 to 52.18] | 6.79 [2.90 to 13.13]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 4.58 [0.58 to 15.42] | 10.42 [2.36 to 26.81] | 13.70 [6.77 to 23.75] | 8.67 [3.62 to 16.87]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 4.58 [0.58 to 15.42] | 12.73 [1.62 to 38.68] | 13.51 [7.77 to 21.31] | 9.94 [4.20 to 19.15]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 4.51 [0.22 to 19.67] | 13.51 [1.25 to 44.07] | 13.16 [7.56 to 20.77] | 10.06 [4.19 to 19.50]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 4.51 [0.22 to 19.67] | 13.51 [1.25 to 44.07] | 13.16 [7.56 to 20.77] | 10.06 [4.19 to 19.50]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 4.51 [0.22 to 19.67] | 13.51 [1.25 to 44.07] | 13.16 [7.56 to 20.77] | 10.06 [4.19 to 19.50]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 4.51 [0.22 to 19.67] | 13.51 [1.25 to 44.07] | 13.16 [7.56 to 20.77] | 10.06 [4.19 to 19.50]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 4.51 [0.22 to 19.67] | 13.51 [1.25 to 44.07] | 13.16 [7.56 to 20.77] | 10.06 [4.19 to 19.50]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 4.51 [0.22 to 19.67] | 13.51 [1.25 to 44.07] | 13.16 [7.56 to 20.77] | 10.06 [4.19 to 19.50]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 4.55 [0.56 to 15.47] |  | 4.55 [0.56 to 15.47]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 4.26 [0.11 to 21.52] |  | 4.26 [0.11 to 21.52]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 11.76 [0.00 to 99.87] | 4.88 [0.16 to 23.00] |  | 5.71 [1.58 to 13.99]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 11.11 [0.01 to 69.27] | 4.51 [0.33 to 17.92] |  | 6.18 [1.89 to 14.38]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 13.75 [3.37 to 33.39] | 4.17 [0.54 to 13.99] |  | 7.59 [2.74 to 16.09]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 13.91 [8.82 to 20.47] | 4.55 [0.54 to 15.58] |  | 9.18 [3.83 to 17.86]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 11.86 [6.25 to 19.87] | 4.22 [0.77 to 12.47] |  | 8.16 [3.80 to 14.93]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 10.71 [4.56 to 20.47] | 4.19 [0.79 to 12.26] |  | 7.71 [3.95 to 13.29]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 10.71 [4.56 to 20.47] | 4.19 [0.79 to 12.26] |  | 7.71 [3.95 to 13.29]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 10.71 [4.56 to 20.47] | 4.19 [0.79 to 12.26] |  | 7.71 [3.95 to 13.29]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 10.71 [4.56 to 20.47] | 4.19 [0.79 to 12.26] |  | 7.71 [3.95 to 13.29]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 10.71 [4.56 to 20.47] | 4.19 [0.79 to 12.26] |  | 7.71 [3.95 to 13.29]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 10.71 [4.56 to 20.47] | 4.19 [0.79 to 12.26] |  | 7.71 [3.95 to 13.29]

94. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Psychiatric Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°18 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 1.92 [0.05 to 10.26] | 1.92 [0.05 to 10.26]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 3.85 [0.30 to 15.16] | 3.85 [0.30 to 15.16]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 3.68 [1.23 to 8.30] | 3.68 [1.23 to 8.30]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 2.89 [1.25 to 5.64] | 2.89 [1.25 to 5.64]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 3.27 [1.58 to 5.93] | 3.27 [1.58 to 5.93]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 3.41 [1.59 to 6.30] | 3.41 [1.59 to 6.30]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 3.24 [1.63 to 5.73] | 3.24 [1.63 to 5.73]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 3.24 [1.63 to 5.73] | 3.24 [1.63 to 5.73]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 3.24 [1.63 to 5.73] | 3.24 [1.63 to 5.73]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 3.24 [1.63 to 5.73] | 3.24 [1.63 to 5.73]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 3.24 [1.63 to 5.73] | 3.24 [1.63 to 5.73]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 1.23 [0.00 to 31.16] |  | 0.49 [0.00 to 8.75]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 1.19 [0.00 to 28.59] |  | 0.47 [0.00 to 6.21]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 1.14 [0.00 to 25.56] | 0.00 [0.00 to 52.18] | 0.45 [0.00 to 4.86]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 1.04 [0.00 to 20.63] | 0.00 [0.00 to 4.93] | 0.33 [0.00 to 3.33]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 0.91 [0.00 to 14.64] | 0.00 [0.00 to 3.27] | 0.28 [0.00 to 2.72]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 0.00 [0.00 to 3.85] |  | 0.00 [0.00 to 3.85]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 2.44 [0.00 to 34.95] |  | 2.14 [0.01 to 14.95]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 3.01 [0.00 to 37.30] |  | 2.25 [0.01 to 15.77]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 1.25 [0.00 to 27.29] | 2.78 [0.00 to 31.28] |  | 2.23 [0.12 to 9.95]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 1.32 [0.05 to 6.55] | 2.60 [0.00 to 26.85] |  | 1.97 [0.24 to 6.92]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 1.69 [0.35 to 4.87] | 2.41 [0.00 to 22.57] |  | 2.04 [0.50 to 5.40]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 1.53 [0.32 to 4.41] | 2.40 [0.00 to 22.26] |  | 1.93 [0.44 to 5.32]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 1.53 [0.32 to 4.41] | 2.40 [0.00 to 22.26] |  | 1.93 [0.44 to 5.32]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 1.53 [0.32 to 4.41] | 2.40 [0.00 to 22.26] |  | 1.93 [0.44 to 5.32]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 1.53 [0.32 to 4.41] | 2.40 [0.00 to 22.26] |  | 1.93 [0.44 to 5.32]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 1.53 [0.32 to 4.41] | 2.40 [0.00 to 22.26] |  | 1.93 [0.44 to 5.32]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 1.53 [0.32 to 4.41] | 2.40 [0.00 to 22.26] |  | 1.93 [0.44 to 5.32]

95. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Respiratory, Thoracic and Mediastinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°20 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 26.92 [0.28 to 88.26] | 26.92 [0.28 to 88.26]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 26.15 [8.21 to 52.91] | 26.15 [8.21 to 52.91]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 23.68 [17.83 to 30.38] | 23.68 [17.83 to 30.38]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 23.47 [15.58 to 32.98] | 23.47 [15.58 to 32.98]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 22.88 [14.93 to 32.55] | 22.88 [14.93 to 32.55]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 23.53 [12.19 to 38.53] | 23.53 [12.19 to 38.53]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 23.89 [11.55 to 40.56] | 23.89 [11.55 to 40.56]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 23.89 [11.55 to 40.56] | 23.89 [11.55 to 40.56]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 23.89 [11.55 to 40.56] | 23.89 [11.55 to 40.56]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 23.89 [11.55 to 40.56] | 23.89 [11.55 to 40.56]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 23.89 [11.55 to 40.56] | 23.89 [11.55 to 40.56]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 15.38 [0.00 to 94.70] |  | 15.38 [0.00 to 94.70]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 16.42 [0.23 to 67.81] |  | 16.42 [0.23 to 67.81]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 9.68 [5.10 to 16.29] | 16.05 [0.15 to 69.39] |  | 12.20 [3.14 to 29.38]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 10.24 [1.20 to 32.87] | 16.67 [0.26 to 67.84] |  | 12.80 [4.40 to 27.04]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 10.16 [1.84 to 28.43] | 17.05 [0.38 to 65.95] | 20.00 [0.51 to 71.64] | 13.12 [5.29 to 25.56]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 9.92 [4.86 to 17.51] | 17.71 [0.69 to 62.94] | 19.18 [10.90 to 30.08] | 14.67 [7.13 to 25.61]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 9.92 [4.86 to 17.51] | 17.27 [1.28 to 55.73] | 20.72 [13.61 to 29.45] | 15.63 [7.93 to 26.51]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 9.77 [5.31 to 16.13] | 17.12 [1.31 to 55.05] | 20.18 [13.24 to 28.72] | 15.36 [7.98 to 25.72]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 9.77 [5.31 to 16.13] | 17.12 [1.31 to 55.05] | 20.18 [13.24 to 28.72] | 15.36 [7.98 to 25.72]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 9.77 [5.31 to 16.13] | 17.12 [1.31 to 55.05] | 20.18 [13.24 to 28.72] | 15.36 [7.98 to 25.72]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 9.77 [5.31 to 16.13] | 17.12 [1.31 to 55.05] | 20.18 [13.24 to 28.72] | 15.36 [7.98 to 25.72]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 9.77 [5.31 to 16.13] | 17.12 [1.31 to 55.05] | 20.18 [13.24 to 28.72] | 15.36 [7.98 to 25.72]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 9.77 [5.31 to 16.13] | 17.12 [1.31 to 55.05] | 20.18 [13.24 to 28.72] | 15.36 [7.98 to 25.72]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 4.55 [0.56 to 15.47] |  | 4.55 [0.56 to 15.47]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 7.45 [0.99 to 23.82] |  | 7.45 [0.99 to 23.82]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 11.76 [0.00 to 99.87] | 7.32 [1.65 to 19.37] |  | 7.86 [3.83 to 13.99]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 15.56 [0.01 to 83.16] | 8.27 [1.15 to 25.83] |  | 10.11 [4.17 to 19.71]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 20.00 [10.76 to 32.37] | 7.64 [1.89 to 19.37] |  | 12.05 [5.32 to 22.44]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 20.53 [14.40 to 27.86] | 8.44 [1.56 to 23.86] |  | 14.43 [6.84 to 25.58]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 18.64 [13.19 to 25.17] | 7.83 [2.26 to 18.54] |  | 13.41 [6.75 to 23.02]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 17.86 [12.76 to 23.95] | 7.78 [2.31 to 18.17] |  | 13.22 [7.02 to 21.97]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 17.86 [12.76 to 23.95] | 7.78 [2.31 to 18.17] |  | 13.22 [7.02 to 21.97]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 17.86 [12.76 to 23.95] | 7.78 [2.31 to 18.17] |  | 13.22 [7.02 to 21.97]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 17.86 [12.76 to 23.95] | 7.78 [2.31 to 18.17] |  | 13.22 [7.02 to 21.97]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 17.86 [12.76 to 23.95] | 7.78 [2.31 to 18.17] |  | 13.22 [7.02 to 21.97]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 17.86 [12.76 to 23.95] | 7.78 [2.31 to 18.17] |  | 13.22 [7.02 to 21.97]

96. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Skin and Subcutaneous Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°22 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 3.85 [0.11 to 19.24] | 3.85 [0.11 to 19.24]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 1.54 [0.12 to 6.20] | 1.54 [0.12 to 6.20]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 2.11 [0.25 to 7.46] | 2.11 [0.25 to 7.46]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 2.17 [0.00 to 19.17] | 2.17 [0.00 to 19.17]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 1.96 [0.00 to 15.98] | 1.96 [0.00 to 15.98]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 1.86 [0.01 to 13.26] | 1.86 [0.01 to 13.26]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 1.77 [0.01 to 11.97] | 1.77 [0.01 to 11.97]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 1.77 [0.01 to 11.97] | 1.77 [0.01 to 11.97]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 1.77 [0.01 to 11.97] | 1.77 [0.01 to 11.97]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 1.77 [0.01 to 11.97] | 1.77 [0.01 to 11.97]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 1.77 [0.01 to 11.97] | 1.77 [0.01 to 11.97]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 4.45] |  | 0.00 [0.00 to 1.78]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 4.30] |  | 0.00 [0.00 to 1.73]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.66]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 0.00 [0.00 to 3.77] | 0.00 [0.00 to 4.93] | 0.00 [0.00 to 1.22]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 0.91 [0.00 to 14.64] | 0.00 [0.00 to 3.27] | 0.28 [0.00 to 2.72]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 4.55 [0.56 to 15.47] |  | 4.55 [0.56 to 15.47]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 3.19 [0.24 to 12.75] |  | 3.19 [0.24 to 12.75]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 3.25 [0.46 to 10.67] |  | 2.86 [0.78 to 7.15]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 2.22 [0.00 to 18.70] | 3.76 [0.52 to 12.38] |  | 3.37 [1.25 to 7.19]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 1.25 [0.00 to 9.31] | 3.47 [0.69 to 10.00] |  | 2.68 [0.99 to 5.74]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 3.97 [1.47 to 8.45] | 3.25 [0.78 to 8.63] |  | 3.61 [1.81 to 6.36]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 3.39 [1.25 to 7.23] | 3.01 [0.81 to 7.61] |  | 3.21 [1.61 to 5.67]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 3.06 [1.13 to 6.54] | 2.99 [0.81 to 7.55] |  | 3.03 [1.52 to 5.36]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 3.06 [1.13 to 6.54] | 2.99 [0.81 to 7.55] |  | 3.03 [1.52 to 5.36]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 3.06 [1.13 to 6.54] | 2.99 [0.81 to 7.55] |  | 3.03 [1.52 to 5.36]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 3.06 [1.13 to 6.54] | 2.99 [0.81 to 7.55] |  | 3.03 [1.52 to 5.36]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 3.06 [1.13 to 6.54] | 2.99 [0.81 to 7.55] |  | 3.03 [1.52 to 5.36]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 3.06 [1.13 to 6.54] | 2.99 [0.81 to 7.55] |  | 3.03 [1.52 to 5.36]

97. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Any Cardiac Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°24 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.80]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 0.00 [0.00 to 1.92] | 0.00 [0.00 to 1.92]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 1.32]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 0.00 [0.00 to 1.20] | 0.00 [0.00 to 1.20]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 0.00 [0.00 to 1.14] | 0.00 [0.00 to 1.14]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 3.85 [0.00 to 45.20] |  | 3.85 [0.00 to 45.20]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 1.49 [0.01 to 10.39] |  | 1.49 [0.01 to 10.39]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 1.23 [0.00 to 12.57] |  | 0.49 [0.00 to 7.05]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 1.19 [0.00 to 12.76] |  | 0.47 [0.00 to 5.15]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 1.14 [0.00 to 13.03] | 0.00 [0.00 to 52.18] | 0.45 [0.00 to 4.17]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 1.04 [0.00 to 13.56] | 0.00 [0.00 to 4.93] | 0.33 [0.00 to 3.08]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 0.91 [0.00 to 14.27] | 0.00 [0.00 to 3.27] | 0.28 [0.00 to 2.71]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 0.00 [0.00 to 3.85] |  | 0.00 [0.00 to 3.85]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 2.95] |  | 0.00 [0.00 to 2.60]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 2.05]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 2.53] |  | 0.00 [0.00 to 1.63]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 0.00 [0.00 to 2.41] | 0.00 [0.00 to 2.37] |  | 0.00 [0.00 to 1.20]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 0.00 [0.00 to 2.06] | 0.00 [0.00 to 2.20] |  | 0.00 [0.00 to 1.07]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]

98. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Ear and Labyrinth Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°26 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.80]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 0.53 [0.01 to 2.90] | 0.53 [0.01 to 2.90]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 0.36 [0.01 to 1.99] | 0.36 [0.01 to 1.99]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 0.33 [0.01 to 1.81] | 0.33 [0.01 to 1.81]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 0.31 [0.01 to 1.71] | 0.31 [0.01 to 1.71]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 0.29 [0.01 to 1.63] | 0.29 [0.01 to 1.63]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 0.29 [0.01 to 1.63] | 0.29 [0.01 to 1.63]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 0.29 [0.01 to 1.63] | 0.29 [0.01 to 1.63]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 0.29 [0.01 to 1.63] | 0.29 [0.01 to 1.63]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 0.29 [0.01 to 1.63] | 0.29 [0.01 to 1.63]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 1.49 [0.01 to 10.39] |  | 1.49 [0.01 to 10.39]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 1.23 [0.00 to 12.57] |  | 0.49 [0.00 to 7.05]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 1.19 [0.00 to 12.76] |  | 0.47 [0.00 to 5.15]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 1.14 [0.00 to 13.03] | 0.00 [0.00 to 52.18] | 0.45 [0.00 to 4.17]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 3.13 [0.01 to 22.01] | 0.00 [0.00 to 4.93] | 1.00 [0.01 to 6.32]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 3.64 [0.02 to 24.24] | 0.00 [0.00 to 3.27] | 1.14 [0.01 to 7.51]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 3.60 [0.02 to 23.59] | 0.00 [0.00 to 3.18] | 1.12 [0.01 to 7.36]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 3.60 [0.02 to 23.59] | 0.00 [0.00 to 3.18] | 1.12 [0.01 to 7.36]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 3.60 [0.02 to 23.59] | 0.00 [0.00 to 3.18] | 1.12 [0.01 to 7.36]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 3.60 [0.02 to 23.59] | 0.00 [0.00 to 3.18] | 1.12 [0.01 to 7.36]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 3.60 [0.02 to 23.59] | 0.00 [0.00 to 3.18] | 1.12 [0.01 to 7.36]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 3.60 [0.02 to 23.59] | 0.00 [0.00 to 3.18] | 1.12 [0.01 to 7.36]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 1.06 [0.00 to 24.79] |  | 1.06 [0.00 to 24.79]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 0.81 [0.00 to 13.06] |  | 0.71 [0.00 to 5.16]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 0.75 [0.00 to 10.68] |  | 0.56 [0.00 to 4.11]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 1.25 [0.00 to 27.29] | 0.69 [0.00 to 8.71] |  | 0.89 [0.07 to 3.63]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 0.66 [0.00 to 18.74] | 0.65 [0.00 to 7.33] |  | 0.66 [0.04 to 3.00]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 0.56 [0.00 to 17.67] | 0.60 [0.00 to 6.05] |  | 0.58 [0.03 to 2.79]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 0.51 [0.00 to 16.86] | 0.60 [0.00 to 5.96] |  | 0.55 [0.02 to 2.78]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 0.51 [0.00 to 16.86] | 0.60 [0.00 to 5.96] |  | 0.55 [0.02 to 2.78]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 0.51 [0.00 to 16.86] | 0.60 [0.00 to 5.96] |  | 0.55 [0.02 to 2.78]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 0.51 [0.00 to 16.86] | 0.60 [0.00 to 5.96] |  | 0.55 [0.02 to 2.78]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 0.51 [0.00 to 16.86] | 0.60 [0.00 to 5.96] |  | 0.55 [0.02 to 2.78]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 0.51 [0.00 to 16.86] | 0.60 [0.00 to 5.96] |  | 0.55 [0.02 to 2.78]

99. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Eye Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°28 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.80]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 0.00 [0.00 to 1.92] | 0.00 [0.00 to 1.92]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 1.32]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 0.00 [0.00 to 1.20] | 0.00 [0.00 to 1.20]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 0.00 [0.00 to 1.14] | 0.00 [0.00 to 1.14]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 4.45] |  | 0.00 [0.00 to 1.78]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 4.30] |  | 0.00 [0.00 to 1.73]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.66]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 0.00 [0.00 to 3.77] | 0.00 [0.00 to 4.93] | 0.00 [0.00 to 1.22]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 1.04]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 1.03]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 2.27 [0.06 to 12.02] |  | 2.27 [0.06 to 12.02]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 1.06 [0.00 to 10.65] |  | 1.06 [0.00 to 10.65]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 2.44 [0.09 to 11.91] |  | 2.14 [0.40 to 6.41]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 2.26 [0.17 to 9.17] |  | 1.69 [0.22 to 5.80]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 1.25 [0.00 to 27.29] | 2.08 [0.28 to 7.10] |  | 1.79 [0.48 to 4.54]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 0.66 [0.00 to 18.74] | 1.95 [0.37 to 5.80] |  | 1.31 [0.18 to 4.43]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 0.56 [0.00 to 17.67] | 1.81 [0.37 to 5.19] |  | 1.17 [0.13 to 4.22]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 0.51 [0.00 to 16.86] | 1.80 [0.37 to 5.16] |  | 1.10 [0.10 to 4.29]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 0.51 [0.00 to 16.86] | 1.80 [0.37 to 5.16] |  | 1.10 [0.10 to 4.29]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 0.51 [0.00 to 16.86] | 1.80 [0.37 to 5.16] |  | 1.10 [0.10 to 4.29]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 0.51 [0.00 to 16.86] | 1.80 [0.37 to 5.16] |  | 1.10 [0.10 to 4.29]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 0.51 [0.00 to 16.86] | 1.80 [0.37 to 5.16] |  | 1.10 [0.10 to 4.29]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 0.51 [0.00 to 16.86] | 1.80 [0.37 to 5.16] |  | 1.10 [0.10 to 4.29]

100. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Injury, Poisoning and Procedural Complications (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°30 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.80]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 0.00 [0.00 to 1.92] | 0.00 [0.00 to 1.92]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 1.32]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 0.00 [0.00 to 1.20] | 0.00 [0.00 to 1.20]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 0.00 [0.00 to 1.14] | 0.00 [0.00 to 1.14]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 4.45] |  | 0.00 [0.00 to 1.78]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 4.30] |  | 0.00 [0.00 to 1.73]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 1.66]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 1.04 [0.00 to 20.63] | 0.00 [0.00 to 4.93] | 0.33 [0.00 to 3.33]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 0.91 [0.00 to 14.64] | 0.00 [0.00 to 3.27] | 0.28 [0.00 to 2.72]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 0.90 [0.00 to 14.30] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 2.66]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 0.00 [0.00 to 3.85] |  | 0.00 [0.00 to 3.85]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 2.95] |  | 0.00 [0.00 to 2.60]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 2.05]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 2.53] |  | 0.00 [0.00 to 1.63]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 0.00 [0.00 to 2.41] | 0.00 [0.00 to 2.37] |  | 0.00 [0.00 to 1.20]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 0.00 [0.00 to 2.06] | 0.00 [0.00 to 2.20] |  | 0.00 [0.00 to 1.07]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]

101. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Investigations (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°32 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.80]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 0.00 [0.00 to 1.92] | 0.00 [0.00 to 1.92]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 1.32]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 0.00 [0.00 to 1.20] | 0.00 [0.00 to 1.20]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 0.00 [0.00 to 1.14] | 0.00 [0.00 to 1.14]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.00 [0.00 to 2.93] | 1.23 [0.00 to 31.16] |  | 0.49 [0.00 to 8.75]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.00 [0.00 to 2.86] | 2.38 [0.00 to 49.63] |  | 0.95 [0.00 to 12.11]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.00 [0.00 to 2.84] | 2.27 [0.00 to 45.15] | 0.00 [0.00 to 52.18] | 0.90 [0.00 to 9.53]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.00 [0.00 to 2.78] | 2.08 [0.00 to 37.46] | 0.00 [0.00 to 4.93] | 0.67 [0.00 to 6.57]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.00 [0.00 to 2.78] | 1.82 [0.00 to 27.44] | 0.00 [0.00 to 3.27] | 0.57 [0.00 to 5.38]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.00 [0.00 to 2.74] | 1.80 [0.00 to 26.86] | 0.00 [0.00 to 3.18] | 0.56 [0.00 to 5.28]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.00 [0.00 to 2.74] | 1.80 [0.00 to 26.86] | 0.00 [0.00 to 3.18] | 0.56 [0.00 to 5.28]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.00 [0.00 to 2.74] | 1.80 [0.00 to 26.86] | 0.00 [0.00 to 3.18] | 0.56 [0.00 to 5.28]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.00 [0.00 to 2.74] | 1.80 [0.00 to 26.86] | 0.00 [0.00 to 3.18] | 0.56 [0.00 to 5.28]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.00 [0.00 to 2.74] | 1.80 [0.00 to 26.86] | 0.00 [0.00 to 3.18] | 0.56 [0.00 to 5.28]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.00 [0.00 to 2.74] | 1.80 [0.00 to 26.86] | 0.00 [0.00 to 3.18] | 0.56 [0.00 to 5.28]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 0.00 [0.00 to 3.85] |  | 0.00 [0.00 to 3.85]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 0.81 [0.00 to 13.06] |  | 0.71 [0.00 to 5.16]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 0.75 [0.00 to 10.68] |  | 0.56 [0.00 to 4.11]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 0.00 [0.00 to 4.51] | 0.69 [0.00 to 8.71] |  | 0.45 [0.01 to 2.85]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 0.66 [0.02 to 3.63] | 0.65 [0.00 to 7.33] |  | 0.66 [0.08 to 2.35]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 0.56 [0.01 to 3.11] | 0.60 [0.00 to 6.05] |  | 0.58 [0.07 to 2.09]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 0.51 [0.01 to 2.81] | 0.60 [0.00 to 5.96] |  | 0.55 [0.07 to 1.98]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 0.51 [0.01 to 2.81] | 0.60 [0.00 to 5.96] |  | 0.55 [0.07 to 1.98]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 0.51 [0.01 to 2.81] | 0.60 [0.00 to 5.96] |  | 0.55 [0.07 to 1.98]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 0.51 [0.01 to 2.81] | 0.60 [0.00 to 5.96] |  | 0.55 [0.07 to 1.98]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 0.51 [0.01 to 2.81] | 0.60 [0.00 to 5.96] |  | 0.55 [0.07 to 1.98]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 0.51 [0.01 to 2.81] | 0.60 [0.00 to 5.96] |  | 0.55 [0.07 to 1.98]

102. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Vascular Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Age Category
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Age strata were defined as "6 months to 17 years", "18 to 65 years" and ">65 years". All subjects who received the second dose of vaccine, were in the first age stratum: "6 months to 17 years". Please, refer to outcome n°34 for the overall (across age strata) post-dose 2 results.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  6 months to 17 years,Weeks 40-42: number analyzed (Participants) | 0 | 0 | 52 | 52
  6 months to 17 years,Weeks 40-42 |  |  | 0.00 [0.00 to 6.85] | 0.00 [0.00 to 6.85]
  6 months to 17 years,Weeks 40-43: number analyzed (Participants) | 0 | 0 | 130 | 130
  6 months to 17 years,Weeks 40-43 |  |  | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.80]
  6 months to 17 years,Weeks 40-44: number analyzed (Participants) | 0 | 0 | 190 | 190
  6 months to 17 years,Weeks 40-44 |  |  | 0.00 [0.00 to 1.92] | 0.00 [0.00 to 1.92]
  6 months to 17 years,Weeks 40-45: number analyzed (Participants) | 0 | 0 | 277 | 277
  6 months to 17 years,Weeks 40-45 |  |  | 0.00 [0.00 to 1.32] | 0.00 [0.00 to 1.32]
  6 months to 17 years,Weeks 40-46: number analyzed (Participants) | 0 | 0 | 306 | 306
  6 months to 17 years,Weeks 40-46 |  |  | 0.00 [0.00 to 1.20] | 0.00 [0.00 to 1.20]
  6 months to 17 years,Weeks 40-47: number analyzed (Participants) | 0 | 0 | 323 | 323
  6 months to 17 years,Weeks 40-47 |  |  | 0.00 [0.00 to 1.14] | 0.00 [0.00 to 1.14]
  6 months to 17 years,Weeks 40-48: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-48 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-49: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-49 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-50: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-50 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-51: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-51 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  6 months to 17 years,Weeks 40-52: number analyzed (Participants) | 0 | 0 | 339 | 339
  6 months to 17 years,Weeks 40-52 |  |  | 0.00 [0.00 to 1.08] | 0.00 [0.00 to 1.08]
  18-65 years,Weeks 40-40: number analyzed (Participants) | 0 | 26 | 0 | 26
  18-65 years,Weeks 40-40 |  | 0.00 [0.00 to 13.23] |  | 0.00 [0.00 to 13.23]
  18-65 years,Weeks 40-41: number analyzed (Participants) | 0 | 67 | 0 | 67
  18-65 years,Weeks 40-41 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  18-65 years,Weeks 40-42: number analyzed (Participants) | 124 | 81 | 0 | 205
  18-65 years,Weeks 40-42 | 0.81 [0.02 to 4.41] | 0.00 [0.00 to 4.45] |  | 0.49 [0.01 to 2.69]
  18-65 years,Weeks 40-43: number analyzed (Participants) | 127 | 84 | 0 | 211
  18-65 years,Weeks 40-43 | 0.79 [0.02 to 4.31] | 0.00 [0.00 to 4.30] |  | 0.47 [0.01 to 2.61]
  18-65 years,Weeks 40-44: number analyzed (Participants) | 128 | 88 | 5 | 221
  18-65 years,Weeks 40-44 | 0.78 [0.02 to 4.28] | 0.00 [0.00 to 4.11] | 0.00 [0.00 to 52.18] | 0.45 [0.01 to 2.50]
  18-65 years,Weeks 40-45: number analyzed (Participants) | 131 | 96 | 73 | 300
  18-65 years,Weeks 40-45 | 0.76 [0.02 to 4.18] | 0.00 [0.00 to 3.77] | 0.00 [0.00 to 4.93] | 0.33 [0.01 to 1.84]
  18-65 years,Weeks 40-46: number analyzed (Participants) | 131 | 110 | 111 | 352
  18-65 years,Weeks 40-46 | 0.76 [0.02 to 4.18] | 0.00 [0.00 to 3.30] | 0.00 [0.00 to 3.27] | 0.28 [0.00 to 1.72]
  18-65 years,Weeks 40-47: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-47 | 0.75 [0.02 to 4.12] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 1.71]
  18-65 years,Weeks 40-48: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-48 | 0.75 [0.02 to 4.12] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 1.71]
  18-65 years,Weeks 40-49: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-49 | 0.75 [0.02 to 4.12] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 1.71]
  18-65 years,Weeks 40-50: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-50 | 0.75 [0.02 to 4.12] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 1.71]
  18-65 years,Weeks 40-51: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-51 | 0.75 [0.02 to 4.12] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 1.71]
  18-65 years,Weeks 40-52: number analyzed (Participants) | 133 | 111 | 114 | 358
  18-65 years,Weeks 40-52 | 0.75 [0.02 to 4.12] | 0.00 [0.00 to 3.27] | 0.00 [0.00 to 3.18] | 0.28 [0.00 to 1.71]
  >65 years,Weeks 40-40: number analyzed (Participants) | 0 | 44 | 0 | 44
  >65 years,Weeks 40-40 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  >65 years,Weeks 40-41: number analyzed (Participants) | 0 | 94 | 0 | 94
  >65 years,Weeks 40-41 |  | 0.00 [0.00 to 3.85] |  | 0.00 [0.00 to 3.85]
  >65 years,Weeks 40-42: number analyzed (Participants) | 17 | 123 | 0 | 140
  >65 years,Weeks 40-42 | 0.00 [0.00 to 19.51] | 0.00 [0.00 to 2.95] |  | 0.00 [0.00 to 2.60]
  >65 years,Weeks 40-43: number analyzed (Participants) | 45 | 133 | 0 | 178
  >65 years,Weeks 40-43 | 0.00 [0.00 to 7.87] | 0.00 [0.00 to 2.74] |  | 0.00 [0.00 to 2.05]
  >65 years,Weeks 40-44: number analyzed (Participants) | 80 | 144 | 0 | 224
  >65 years,Weeks 40-44 | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 2.53] |  | 0.00 [0.00 to 1.63]
  >65 years,Weeks 40-45: number analyzed (Participants) | 151 | 154 | 0 | 305
  >65 years,Weeks 40-45 | 0.00 [0.00 to 2.41] | 0.00 [0.00 to 2.37] |  | 0.00 [0.00 to 1.20]
  >65 years,Weeks 40-46: number analyzed (Participants) | 177 | 166 | 0 | 343
  >65 years,Weeks 40-46 | 0.00 [0.00 to 2.06] | 0.00 [0.00 to 2.20] |  | 0.00 [0.00 to 1.07]
  >65 years,Weeks 40-47: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-47 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-48: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-48 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-49: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-49 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-50: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-50 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-51: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-51 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]
  >65 years,Weeks 40-52: number analyzed (Participants) | 196 | 167 | 0 | 363
  >65 years,Weeks 40-52 | 0.00 [0.00 to 1.86] | 0.00 [0.00 to 2.18] |  | 0.00 [0.00 to 1.01]

103. Secondary Outcome: Weekly Percentage of Subjects Reporting Any AEs, Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Risk status (At risk; Not at risk) was recorded for influenza-associated morbidity and mortality as per healthcare professional assessment.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 36.36 [0.00 to 100] |  | 36.36 [0.00 to 100]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 56.25 [0.00 to 100] | 30.30 [0.00 to 99.55] | 56.25 [0.73 to 99.82] | 43.08 [23.70 to 64.14]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 45.16 [27.32 to 63.97] | 40.00 [12.16 to 73.76] | 47.62 [6.49 to 91.59] | 45.16 [32.48 to 58.32]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 55.56 [0.01 to 100] | 25.00 [5.49 to 57.19] | 34.78 [4.15 to 80.55] | 43.66 [21.31 to 68.08]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 35.14 [0.51 to 94.16] | 58.33 [27.67 to 84.83] | 52.17 [17.17 to 85.61] | 45.51 [27.09 to 64.87]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 26.92 [11.57 to 47.79] | 38.89 [17.30 to 64.25] | 39.58 [20.92 to 60.77] | 35.87 [23.69 to 49.55]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 38.10 [18.11 to 61.56] | 0.00 [0.00 to 97.50] | 70.00 [0.00 to 100] | 46.88 [18.94 to 76.35]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 76.92 [23.37 to 99.35] | 76.92 [23.37 to 99.35]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 34.33 [22.95 to 47.19] |  | 34.33 [22.95 to 47.19]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 36.17 [0.29 to 96.34] |  | 36.17 [0.29 to 96.34]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 44.00 [35.14 to 53.16] | 40.00 [0.00 to 100] | 38.89 [0.08 to 98.92] | 42.69 [35.17 to 50.47]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 33.33 [0.84 to 90.57] | 47.37 [24.16 to 71.45] | 46.67 [33.67 to 60.00]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 35.71 [0.83 to 92.88] | 33.33 [6.20 to 72.97]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 83.33 [35.88 to 99.58] | 49.21 [32.01 to 66.54] | 52.17 [33.89 to 70.04]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 50.00 [15.70 to 84.30] | 36.84 [15.96 to 62.13] | 40.74 [22.39 to 61.20]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 100 [2.50 to 100] | 70.00 [0.76 to 100] | 72.73 [39.03 to 93.98]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 100 [29.24 to 100] | 100 [29.24 to 100]

104. Secondary Outcome: Weekly Percentage of Subjects Reporting Any AEs Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. Risk status (At risk; Not at risk) was recorded for influenza-associated morbidity and mortality as per healthcare professional assessment.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 66.67 [0.00 to 100]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 50.00 [11.81 to 88.19]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 15.38 [1.02 to 52.27]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 18.18 [0.46 to 67.75]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 25.00 [0.00 to 100]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 33.33 [0.84 to 90.57]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 50.00 [1.26 to 98.74]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 38.46 [0.00 to 100]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 42.11 [20.25 to 66.50]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 9.52 [0.00 to 65.04]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 6.45 [0.00 to 68.83]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 25.00 [0.63 to 80.59]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

105. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Gastrointestinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Risk status (At risk; Not at risk) was recorded for influenza-associated morbidity and mortality as per healthcare professional assessment.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 2.27 [0.00 to 99.42] |  | 2.27 [0.00 to 99.42]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 12.50 [0.00 to 99.41] | 15.15 [0.00 to 85.70] | 6.25 [0.16 to 30.23] | 12.31 [5.47 to 22.82]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 9.68 [2.04 to 25.75] | 10.00 [0.25 to 44.50] | 4.76 [0.00 to 100] | 8.06 [1.24 to 24.40]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 13.89 [0.00 to 87.39] | 8.33 [0.21 to 38.48] | 13.04 [0.00 to 91.75] | 12.68 [5.96 to 22.70]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 9.46 [3.89 to 18.52] | 8.33 [0.21 to 38.48] | 3.26 [0.02 to 21.52] | 6.18 [1.73 to 14.97]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 7.69 [0.95 to 25.13] | 0.00 [0.00 to 18.53] | 10.42 [2.04 to 28.30] | 7.61 [2.29 to 17.67]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 97.50] | 10.00 [0.00 to 99.13] | 9.38 [1.98 to 25.02]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 15.38 [0.58 to 57.61] | 15.38 [0.58 to 57.61]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 2.99 [0.36 to 10.37] |  | 2.99 [0.36 to 10.37]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 2.13 [0.01 to 16.09] |  | 2.13 [0.01 to 16.09]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 30.85] | 8.33 [0.13 to 41.57] | 2.34 [0.02 to 15.22]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 10.53 [3.96 to 21.52] | 10.00 [3.76 to 20.51]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 16.67 [0.42 to 64.12] | 4.76 [0.38 to 18.32] | 5.80 [1.37 to 15.21]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 12.50 [0.32 to 52.65] | 10.53 [0.00 to 68.41] | 11.11 [1.36 to 34.82]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 10.00 [0.00 to 88.98] | 9.09 [0.23 to 41.28]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

106. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Gastrointestinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: The weekly percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination at the same week. Vaccination period was defined between ISO weeks 46 and 52. The pre-defined AEIs listed on the ADR card were diarrhoea, nausea, and vomiting. Risk status (At risk; Not at risk) was recorded for influenza-associated morbidity and mortality as per healthcare professional assessment.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 16.67 [0.00 to 100]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 0.00 [0.00 to 45.93]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 0.00 [0.00 to 24.71]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 9.09 [0.00 to 92.61]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 50.00 [1.26 to 98.74]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 7.69 [0.00 to 90.25]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 0.00 [0.00 to 17.65]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 0.00 [0.00 to 16.11]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 0.00 [0.00 to 11.22]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

107. Secondary Outcome: Weekly Percentage of Subjects Reporting Any General Disorders and Administration Site Conditions (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 27.27 [0.00 to 100] |  | 27.27 [0.00 to 100]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 37.50 [0.00 to 100] | 24.24 [0.00 to 97.62] | 43.75 [1.42 to 96.32] | 32.31 [18.33 to 49.06]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 19.35 [7.45 to 37.47] | 20.00 [2.52 to 55.61] | 23.81 [2.15 to 67.11] | 20.97 [11.66 to 33.18]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 41.67 [0.00 to 100] | 25.00 [5.49 to 57.19] | 17.39 [0.43 to 66.04] | 30.99 [10.30 to 59.46]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 17.57 [0.00 to 96.81] | 50.00 [21.09 to 78.91] | 35.87 [2.46 to 86.88] | 29.21 [9.25 to 57.67]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 15.38 [4.36 to 34.87] | 27.78 [9.69 to 53.48] | 29.17 [3.75 to 71.88] | 25.00 [10.41 to 45.43]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 28.57 [11.28 to 52.18] | 0.00 [0.00 to 97.50] | 50.00 [0.01 to 99.99] | 34.38 [13.93 to 60.22]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 61.54 [3.60 to 99.52] | 61.54 [3.60 to 99.52]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 26.87 [11.49 to 47.81] |  | 26.87 [11.49 to 47.81]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 31.91 [0.49 to 91.50] |  | 31.91 [0.49 to 91.50]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 30.40 [22.49 to 39.26] | 30.00 [0.00 to 100] | 19.44 [0.18 to 77.39] | 28.07 [20.48 to 36.71]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 28.07 [16.56 to 42.15] | 26.67 [15.72 to 40.20]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 19.05 [1.16 to 61.85] | 17.78 [4.50 to 41.33]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 50.00 [11.81 to 88.19] | 28.57 [17.89 to 41.35] | 30.43 [19.92 to 42.69]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 25.00 [3.19 to 65.09] | 26.32 [0.24 to 88.00] | 25.93 [5.65 to 58.91]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 50.00 [18.71 to 81.29] | 45.45 [16.75 to 76.62]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 66.67 [9.43 to 99.16] | 66.67 [9.43 to 99.16]

108. Secondary Outcome: Weekly Percentage of Subjects Reporting Any General Disorders and Administration Site Conditions (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 33.33 [4.33 to 77.72]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 0.00 [0.00 to 45.93]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 7.69 [0.07 to 41.92]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 9.09 [0.23 to 41.28]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 33.33 [0.84 to 90.57]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 38.46 [0.00 to 100]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 5.26 [0.13 to 26.03]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 0.00 [0.00 to 16.11]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 3.23 [0.00 to 42.56]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 25.00 [0.63 to 80.59]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

109. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Immune System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 10.58] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 5.52]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 5.78]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 14.82] | 0.00 [0.00 to 5.06]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.93] | 0.56 [0.01 to 3.45]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 3.93]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 2.13]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 6.27] | 0.00 [0.00 to 5.96]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 5.21]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

110. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Immune System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: Analysis was to be performed on the enrolled subjects vaccinated with a second dose of GSK's quadrivalent seasonal influenza vaccine, and who returned the ADR card, i.e.: only Fluarix Tetra Group subjects who received the second dose. As no AEs were reported for the MedDRA Class considered, the "by risk status" analysis could not be performed.
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

111. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Infections and Infestations (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 9.09 [0.00 to 99.98] |  | 9.09 [0.00 to 99.98]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 6.06 [0.00 to 48.84] | 6.25 [0.16 to 30.23] | 4.62 [0.96 to 12.90]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 6.45 [0.79 to 21.42] | 10.00 [0.25 to 44.50] | 4.76 [0.00 to 47.50] | 6.45 [1.79 to 15.70]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 8.33 [1.75 to 22.47] | 8.33 [0.21 to 38.48] | 4.35 [0.00 to 56.70] | 7.04 [2.33 to 15.67]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 9.46 [0.00 to 69.82] | 8.33 [0.21 to 38.48] | 6.52 [1.82 to 15.81] | 7.87 [4.37 to 12.84]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 3.85 [0.10 to 19.64] | 11.11 [1.38 to 34.71] | 10.42 [0.85 to 36.63] | 8.70 [2.61 to 20.07]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 97.50] | 10.00 [0.00 to 99.13] | 6.25 [0.77 to 20.81]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 15.38 [0.00 to 100] | 15.38 [0.00 to 100]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 8.96 [3.36 to 18.48] |  | 8.96 [3.36 to 18.48]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 8.51 [0.02 to 53.58] |  | 8.51 [0.02 to 53.58]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.58 [0.01 to 3.22]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 5.26 [1.10 to 14.62] | 5.00 [1.04 to 13.92]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 7.14 [0.00 to 61.63] | 6.67 [0.07 to 36.62]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 16.67 [0.42 to 64.12] | 4.76 [0.00 to 55.81] | 5.80 [0.04 to 34.97]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 5.26 [0.00 to 73.64] | 3.70 [0.00 to 40.23]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 20.00 [0.00 to 99.56] | 18.18 [1.13 to 59.63]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

112. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Infections and Infestations (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 0.00 [0.00 to 45.93]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 50.00 [11.81 to 88.19]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 0.00 [0.00 to 24.71]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 0.00 [0.00 to 28.49]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 0.00 [0.00 to 24.71]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 0.00 [0.00 to 17.65]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 0.00 [0.00 to 16.11]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 3.23 [0.00 to 42.56]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

113. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Metabolism and Nutrition Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 6.25 [0.00 to 100] | 0.00 [0.00 to 10.58] | 6.25 [0.16 to 30.23] | 3.08 [0.07 to 16.12]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 30.85] | 4.76 [0.00 to 47.50] | 1.61 [0.00 to 17.38]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 26.46] | 17.39 [0.43 to 66.04] | 7.04 [0.78 to 23.94]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 4.05 [0.00 to 53.08] | 0.00 [0.00 to 26.46] | 4.35 [0.00 to 62.93] | 3.93 [0.46 to 13.64]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 1.09 [0.00 to 8.84]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 3.13 [0.08 to 16.22]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 15.38 [0.58 to 57.61] | 15.38 [0.58 to 57.61]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 2.13 [0.01 to 16.09] |  | 2.13 [0.01 to 16.09]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 2.78 [0.05 to 15.34] | 0.58 [0.00 to 7.25]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 14.04 [6.26 to 25.79] | 13.33 [5.94 to 24.59]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 2.38 [0.06 to 12.57] | 2.22 [0.06 to 11.77]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 3.17 [0.04 to 18.51] | 2.90 [0.26 to 11.06]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

114. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Metabolism and Nutrition Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 0.00 [0.00 to 45.93]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 0.00 [0.00 to 45.93]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 0.00 [0.00 to 24.71]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 9.09 [0.23 to 41.28]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 7.69 [0.00 to 90.25]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 5.26 [0.13 to 26.03]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 0.00 [0.00 to 16.11]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 0.00 [0.00 to 11.22]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

115. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Musculoskeletal and Connective Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 2.27 [0.00 to 99.42] |  | 2.27 [0.00 to 99.42]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 6.25 [0.00 to 100] | 3.03 [0.00 to 27.44] | 12.50 [1.15 to 41.43] | 6.15 [1.09 to 18.08]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 20.00 [2.52 to 55.61] | 4.76 [0.00 to 47.50] | 4.84 [0.01 to 34.50]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 19.44 [0.05 to 83.92] | 8.33 [0.21 to 38.48] | 4.35 [0.00 to 100] | 12.68 [2.83 to 32.16]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 10.81 [0.08 to 55.52] | 16.67 [2.09 to 48.41] | 8.70 [0.09 to 45.17] | 10.11 [5.74 to 16.19]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 11.54 [2.45 to 30.15] | 11.11 [1.38 to 34.71] | 8.33 [0.71 to 29.93] | 9.78 [4.57 to 17.76]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 4.76 [0.12 to 23.82] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 3.13 [0.08 to 16.22]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 46.15 [0.32 to 99.28] | 46.15 [0.32 to 99.28]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 5.97 [1.65 to 14.59] |  | 5.97 [1.65 to 14.59]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 12.77 [0.02 to 70.77] |  | 12.77 [0.02 to 70.77]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 12.00 [6.87 to 19.02] | 0.00 [0.00 to 30.85] | 5.56 [0.10 to 29.18] | 9.94 [5.24 to 16.73]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 33.33 [0.84 to 90.57] | 8.77 [2.91 to 19.30] | 10.00 [3.56 to 21.08]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 2.38 [0.00 to 63.98] | 2.22 [0.00 to 37.20]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 16.67 [0.42 to 64.12] | 7.94 [1.25 to 23.87] | 8.70 [3.21 to 18.10]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 25.00 [3.19 to 65.09] | 10.53 [0.25 to 46.86] | 14.81 [2.87 to 38.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 10.00 [0.00 to 88.98] | 9.09 [0.23 to 41.28]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

116. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Musculoskeletal and Connective Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 0.00 [0.00 to 45.93]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 0.00 [0.00 to 45.93]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 0.00 [0.00 to 24.71]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 0.00 [0.00 to 28.49]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 7.69 [0.00 to 90.25]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 0.00 [0.00 to 17.65]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 0.00 [0.00 to 16.11]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 0.00 [0.00 to 11.22]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

117. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Nervous System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 9.09 [0.00 to 99.98] |  | 9.09 [0.00 to 99.98]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 25.00 [0.00 to 100] | 6.06 [0.00 to 48.84] | 0.00 [0.00 to 20.59] | 9.23 [1.80 to 25.43]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 9.68 [2.04 to 25.75] | 10.00 [0.25 to 44.50] | 9.52 [0.00 to 75.08] | 9.68 [3.63 to 19.88]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 16.67 [0.00 to 98.03] | 8.33 [0.21 to 38.48] | 4.35 [0.00 to 56.70] | 11.27 [2.71 to 28.13]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 13.51 [0.84 to 47.92] | 8.33 [0.21 to 38.48] | 7.61 [0.09 to 40.43] | 10.11 [5.06 to 17.59]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 11.11 [1.38 to 34.71] | 8.33 [0.71 to 29.93] | 6.52 [0.91 to 20.73]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 38.46 [0.48 to 96.40] | 38.46 [0.48 to 96.40]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 5.97 [1.65 to 14.59] |  | 5.97 [1.65 to 14.59]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 6.38 [0.01 to 42.76] |  | 6.38 [0.01 to 42.76]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 3.20 [0.88 to 7.99] | 0.00 [0.00 to 30.85] | 2.78 [0.05 to 15.34] | 2.92 [0.96 to 6.69]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 7.02 [1.95 to 17.00] | 6.67 [1.85 to 16.20]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 16.67 [0.42 to 64.12] | 12.70 [2.19 to 35.21] | 13.04 [5.20 to 25.57]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 25.00 [3.19 to 65.09] | 10.53 [0.25 to 46.86] | 14.81 [2.87 to 38.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 100 [2.50 to 100] | 10.00 [0.00 to 88.98] | 18.18 [0.07 to 79.30]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 33.33 [0.84 to 90.57] | 33.33 [0.84 to 90.57]

118. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Nervous System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

119. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Psychiatric Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 12.12 [0.00 to 77.14] | 0.00 [0.00 to 20.59] | 6.15 [0.26 to 26.98]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 10.00 [0.25 to 44.50] | 0.00 [0.00 to 16.11] | 1.61 [0.00 to 21.62]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 26.46] | 4.35 [0.00 to 56.70] | 2.82 [0.34 to 9.81]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.93] | 0.56 [0.01 to 3.45]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 3.85 [0.10 to 19.64] | 0.00 [0.00 to 18.53] | 2.08 [0.00 to 51.95] | 2.17 [0.05 to 11.78]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 10.00 [0.00 to 99.13] | 3.13 [0.00 to 37.12]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 2.78 [0.05 to 15.34] | 0.58 [0.00 to 7.25]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 7.02 [1.95 to 17.00] | 6.67 [1.85 to 16.20]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 2.38 [0.00 to 63.98] | 2.22 [0.00 to 37.20]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 1.59 [0.00 to 12.80] | 1.45 [0.04 to 7.82]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 5.26 [0.00 to 73.64] | 3.70 [0.00 to 40.23]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

120. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Psychiatric Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 0.00 [0.00 to 45.93]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 0.00 [0.00 to 45.93]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 0.00 [0.00 to 24.71]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 0.00 [0.00 to 28.49]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 0.00 [0.00 to 24.71]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 10.53 [1.30 to 33.14]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 9.52 [0.00 to 65.04]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 0.00 [0.00 to 11.22]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

121. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Respiratory, Thoracic and Mediastinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 9.09 [0.00 to 99.98] |  | 9.09 [0.00 to 99.98]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 12.50 [0.00 to 99.41] | 9.09 [0.00 to 65.12] | 31.25 [1.75 to 83.28] | 15.38 [4.58 to 34.16]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 19.35 [7.45 to 37.47] | 30.00 [6.67 to 65.25] | 28.57 [0.00 to 99.80] | 24.19 [11.60 to 41.20]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 25.00 [12.12 to 42.20] | 8.33 [0.21 to 38.48] | 21.74 [0.00 to 99.72] | 21.13 [12.20 to 32.66]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 20.27 [7.81 to 39.06] | 25.00 [5.49 to 57.19] | 20.65 [4.48 to 49.35] | 20.79 [15.05 to 27.54]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 7.69 [0.95 to 25.13] | 11.11 [1.38 to 34.71] | 20.83 [10.47 to 34.99] | 15.22 [6.17 to 29.29]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 9.52 [1.17 to 30.38] | 0.00 [0.00 to 97.50] | 30.00 [0.00 to 100] | 15.63 [1.42 to 49.58]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 23.08 [0.65 to 76.63] | 23.08 [0.65 to 76.63]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 8.96 [3.36 to 18.48] |  | 8.96 [3.36 to 18.48]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 17.02 [0.45 to 64.71] |  | 17.02 [0.45 to 64.71]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 9.60 [5.06 to 16.17] | 10.00 [0.00 to 100] | 25.00 [0.16 to 87.94] | 12.87 [3.84 to 29.01]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 24.56 [2.20 to 68.56] | 23.33 [13.38 to 36.04]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 16.67 [0.35 to 65.58] | 15.56 [2.47 to 42.95]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 16.67 [0.42 to 64.12] | 22.22 [1.15 to 69.94] | 21.74 [4.99 to 50.53]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 21.05 [6.05 to 45.57] | 14.81 [2.31 to 41.47]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 30.00 [0.00 to 100] | 27.27 [1.29 to 79.30]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 66.67 [9.43 to 99.16] | 66.67 [9.43 to 99.16]

122. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Respiratory, Thoracic and Mediastinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 33.33 [0.00 to 100]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 33.33 [4.33 to 77.72]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 15.38 [1.02 to 52.27]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 9.09 [0.23 to 41.28]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 25.00 [0.00 to 100]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 7.69 [0.00 to 90.25]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 36.84 [16.29 to 61.64]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 4.76 [0.00 to 86.58]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 3.23 [0.00 to 42.56]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

123. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Skin and Subcutaneous Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 2.27 [0.00 to 99.42] |  | 2.27 [0.00 to 99.42]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 3.03 [0.00 to 27.44] | 12.50 [1.15 to 41.43] | 4.62 [0.56 to 15.72]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 3.23 [0.08 to 16.70] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 16.11] | 1.61 [0.02 to 9.93]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 26.46] | 4.35 [0.00 to 56.70] | 1.41 [0.00 to 11.12]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 6.76 [1.90 to 16.31] | 0.00 [0.00 to 26.46] | 2.17 [0.00 to 57.57] | 3.93 [0.40 to 14.32]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 3.93]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 2.99 [0.36 to 10.37] |  | 2.99 [0.36 to 10.37]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 2.13]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 33.33 [0.84 to 90.57] | 0.00 [0.00 to 6.27] | 1.67 [0.00 to 54.99]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 2.38 [0.00 to 63.98] | 2.22 [0.00 to 37.20]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 5.21]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 12.50 [0.32 to 52.65] | 0.00 [0.00 to 17.65] | 3.70 [0.00 to 31.71]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

124. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Skin and Subcutaneous Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 0.00 [0.00 to 45.93]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 0.00 [0.00 to 45.93]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 0.00 [0.00 to 24.71]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 0.00 [0.00 to 28.49]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 0.00 [0.00 to 24.71]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 5.26 [0.13 to 26.03]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 0.00 [0.00 to 16.11]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 0.00 [0.00 to 11.22]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

125. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Cardiac Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 10.58] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 5.52]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 5.78]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 14.82] | 0.00 [0.00 to 5.06]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.93] | 0.00 [0.00 to 2.05]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 3.93]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 1.49 [0.04 to 8.04] |  | 1.49 [0.04 to 8.04]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 2.13]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 6.27] | 0.00 [0.00 to 5.96]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 5.21]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

126. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Cardiac Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

127. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Ear and Labyrinth Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 2.27 [0.00 to 99.42] |  | 2.27 [0.00 to 99.42]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 10.58] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 5.52]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 5.78]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 26.46] | 4.35 [0.00 to 56.70] | 2.82 [0.34 to 9.81]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 0.00 [0.00 to 4.86] | 8.33 [0.21 to 38.48] | 0.00 [0.00 to 3.93] | 0.56 [0.00 to 5.76]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 5.56 [0.14 to 27.29] | 0.00 [0.00 to 7.40] | 1.09 [0.00 to 10.42]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 2.13 [0.01 to 16.09] |  | 2.13 [0.01 to 16.09]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 2.13]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 6.27] | 0.00 [0.00 to 5.96]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 16.67 [0.42 to 64.12] | 0.00 [0.00 to 5.69] | 1.45 [0.00 to 21.94]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

128. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Ear and Labyrinth Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 106
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

129. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Eye Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 6.06 [0.00 to 48.84] | 0.00 [0.00 to 20.59] | 3.08 [0.14 to 14.05]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 5.78]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 2.78 [0.00 to 84.65] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 14.82] | 1.41 [0.01 to 9.48]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.93] | 0.00 [0.00 to 2.05]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 3.93]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 1.49 [0.04 to 8.04] |  | 1.49 [0.04 to 8.04]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 2.13]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 6.27] | 0.00 [0.00 to 5.96]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 5.21]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

130. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Eye Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Week 46: number analyzed (Participants) | 1
  At risk,Week 46 | 0.00 [0.00 to 97.50]
  At risk,Week 47: number analyzed (Participants) | 6
  At risk,Week 47 | 16.67 [0.00 to 100]
  At risk,Week 48: number analyzed (Participants) | 6
  At risk,Week 48 | 0.00 [0.00 to 45.93]
  At risk,Week 49: number analyzed (Participants) | 13
  At risk,Week 49 | 0.00 [0.00 to 24.71]
  At risk,Week 50: number analyzed (Participants) | 11
  At risk,Week 50 | 0.00 [0.00 to 28.49]
  At risk,Week 51: number analyzed (Participants) | 8
  At risk,Week 51 | 0.00 [0.00 to 36.94]
  At risk,Week 52: number analyzed (Participants) | 3
  At risk,Week 52 | 0.00 [0.00 to 70.76]
  Not at risk,Week 46: number analyzed (Participants) | 2
  Not at risk,Week 46 | 0.00 [0.00 to 84.19]
  Not at risk,Week 47: number analyzed (Participants) | 13
  Not at risk,Week 47 | 7.69 [0.00 to 90.25]
  Not at risk,Week 48: number analyzed (Participants) | 19
  Not at risk,Week 48 | 0.00 [0.00 to 17.65]
  Not at risk,Week 49: number analyzed (Participants) | 21
  Not at risk,Week 49 | 0.00 [0.00 to 16.11]
  Not at risk,Week 50: number analyzed (Participants) | 31
  Not at risk,Week 50 | 0.00 [0.00 to 11.22]
  Not at risk,Week 51: number analyzed (Participants) | 4
  Not at risk,Week 51 | 0.00 [0.00 to 60.24]
  Not at risk,Week 52: number analyzed (Participants) | 1
  Not at risk,Week 52 | 0.00 [0.00 to 97.50]

131. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Injury, Poisoning and Procedural Complications (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 10.58] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 5.52]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 5.78]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 14.82] | 0.00 [0.00 to 5.06]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.93] | 0.00 [0.00 to 2.05]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 3.93]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 2.13]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 6.27] | 0.00 [0.00 to 5.96]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 16.67 [0.42 to 64.12] | 0.00 [0.00 to 5.69] | 1.45 [0.00 to 21.94]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

132. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Injury, Poisoning and Procedural Complications (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 106
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

133. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Investigations (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 6.06 [0.00 to 48.84] | 0.00 [0.00 to 20.59] | 3.08 [0.14 to 14.05]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 10.00 [0.25 to 44.50] | 0.00 [0.00 to 16.11] | 1.61 [0.00 to 21.62]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 14.82] | 0.00 [0.00 to 5.06]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 1.35 [0.00 to 21.52] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.93] | 0.56 [0.01 to 3.45]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 3.93]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 2.13]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 6.27] | 0.00 [0.00 to 5.96]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 5.21]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

134. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Investigations (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

135. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Vascular Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 105
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Week 40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Week 40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Week 41: number analyzed (Participants) | 0 | 44 | 0 | 44
  At risk,Week 41 |  | 0.00 [0.00 to 8.04] |  | 0.00 [0.00 to 8.04]
  At risk,Week 42: number analyzed (Participants) | 16 | 33 | 16 | 65
  At risk,Week 42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 10.58] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 5.52]
  At risk,Week 43: number analyzed (Participants) | 31 | 10 | 21 | 62
  At risk,Week 43 | 0.00 [0.00 to 11.22] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 5.78]
  At risk,Week 44: number analyzed (Participants) | 36 | 12 | 23 | 71
  At risk,Week 44 | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 14.82] | 0.00 [0.00 to 5.06]
  At risk,Week 45: number analyzed (Participants) | 74 | 12 | 92 | 178
  At risk,Week 45 | 0.00 [0.00 to 4.86] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 3.93] | 0.00 [0.00 to 2.05]
  At risk,Week 46: number analyzed (Participants) | 26 | 18 | 48 | 92
  At risk,Week 46 | 0.00 [0.00 to 13.23] | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 7.40] | 0.00 [0.00 to 3.93]
  At risk,Week 47: number analyzed (Participants) | 21 | 1 | 10 | 32
  At risk,Week 47 | 0.00 [0.00 to 16.11] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 10.89]
  At risk,Week 48: number analyzed (Participants) | 0 | 0 | 13 | 13
  At risk,Week 48 |  |  | 0.00 [0.00 to 24.71] | 0.00 [0.00 to 24.71]
  Not at risk,Week 40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Week 40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Week 41: number analyzed (Participants) | 0 | 47 | 0 | 47
  Not at risk,Week 41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  Not at risk,Week 42: number analyzed (Participants) | 125 | 10 | 36 | 171
  Not at risk,Week 42 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 9.74] | 0.58 [0.01 to 3.22]
  Not at risk,Week 43: number analyzed (Participants) | 0 | 3 | 57 | 60
  Not at risk,Week 43 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 6.27] | 0.00 [0.00 to 5.96]
  Not at risk,Week 44: number analyzed (Participants) | 0 | 3 | 42 | 45
  Not at risk,Week 44 |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 8.41] | 0.00 [0.00 to 7.87]
  Not at risk,Week 45: number analyzed (Participants) | 0 | 6 | 63 | 69
  Not at risk,Week 45 |  | 0.00 [0.00 to 45.93] | 0.00 [0.00 to 5.69] | 0.00 [0.00 to 5.21]
  Not at risk,Week 46: number analyzed (Participants) | 0 | 8 | 19 | 27
  Not at risk,Week 46 |  | 0.00 [0.00 to 36.94] | 0.00 [0.00 to 17.65] | 0.00 [0.00 to 12.77]
  Not at risk,Week 47: number analyzed (Participants) | 0 | 1 | 10 | 11
  Not at risk,Week 47 |  | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 30.85] | 0.00 [0.00 to 28.49]
  Not at risk,Week 48: number analyzed (Participants) | 0 | 0 | 3 | 3
  Not at risk,Week 48 |  |  | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 70.76]

136. Secondary Outcome: Weekly Percentage of Subjects Reporting Any Vascular Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 104
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

137. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any AEs Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e., week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Risk status (At risk; Not at risk) was recorded for influenza-associated morbidity and mortality as per healthcare professional assessment.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 34.04 [0.00 to 100] |  | 34.04 [0.00 to 100]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 56.25 [0.00 to 100] | 32.50 [0.00 to 100] | 56.25 [0.73 to 99.82] | 39.29 [16.38 to 66.30]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 48.94 [0.01 to 99.99] | 33.33 [0.00 to 100] | 51.35 [1.45 to 98.86] | 41.38 [24.45 to 59.95]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 51.81 [17.11 to 85.22] | 32.35 [0.00 to 100] | 45.00 [27.96 to 62.94] | 42.04 [30.32 to 54.46]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 43.95 [14.48 to 77.03] | 35.09 [0.00 to 100] | 49.34 [27.42 to 71.45] | 43.50 [34.29 to 53.05]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 41.53 [13.31 to 74.68] | 35.61 [0.00 to 100] | 47.00 [30.32 to 64.18] | 42.14 [33.74 to 50.88]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 41.18 [15.00 to 71.71] | 35.34 [0.00 to 100] | 48.10 [29.39 to 67.20] | 42.41 [33.83 to 51.34]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 41.18 [15.00 to 71.71] | 35.34 [0.00 to 100] | 49.78 [27.91 to 71.70] | 43.21 [33.66 to 53.15]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 41.18 [15.00 to 71.71] | 35.34 [0.00 to 100] | 49.78 [27.91 to 71.70] | 43.21 [33.66 to 53.15]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 41.18 [15.00 to 71.71] | 35.34 [0.00 to 100] | 49.78 [27.91 to 71.70] | 43.21 [33.66 to 53.15]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 41.18 [15.00 to 71.71] | 35.34 [0.00 to 100] | 49.78 [27.91 to 71.70] | 43.21 [33.66 to 53.15]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 41.18 [15.00 to 71.71] | 35.34 [0.00 to 100] | 49.78 [27.91 to 71.70] | 43.21 [33.66 to 53.15]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 34.33 [22.95 to 47.19] |  | 34.33 [22.95 to 47.19]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 35.09 [12.54 to 63.98] |  | 35.09 [12.54 to 63.98]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 44.00 [35.14 to 53.16] | 35.48 [16.02 to 59.26] | 38.89 [0.08 to 98.92] | 39.65 [32.94 to 46.66]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 44.00 [35.14 to 53.16] | 35.43 [16.17 to 58.94] | 44.09 [23.52 to 66.26] | 40.87 [35.21 to 46.71]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 44.00 [35.14 to 53.16] | 34.62 [12.67 to 62.80] | 41.48 [27.80 to 56.20] | 40.00 [34.92 to 45.24]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 44.00 [35.14 to 53.16] | 36.76 [23.53 to 51.64] | 43.94 [26.87 to 62.13] | 41.83 [37.27 to 46.49]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 44.00 [35.14 to 53.16] | 37.50 [26.97 to 48.98] | 43.32 [29.56 to 57.88] | 41.77 [37.34 to 46.30]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 44.00 [35.14 to 53.16] | 37.93 [28.18 to 48.46] | 44.49 [24.73 to 65.62] | 42.45 [38.02 to 46.98]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 44.00 [35.14 to 53.16] | 37.93 [28.18 to 48.46] | 45.22 [21.68 to 70.45] | 42.80 [37.59 to 48.14]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 44.00 [35.14 to 53.16] | 37.93 [28.18 to 48.46] | 45.22 [21.68 to 70.45] | 42.80 [37.59 to 48.14]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 44.00 [35.14 to 53.16] | 37.93 [28.18 to 48.46] | 45.22 [21.68 to 70.45] | 42.80 [37.59 to 48.14]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 44.00 [35.14 to 53.16] | 37.93 [28.18 to 48.46] | 45.22 [21.68 to 70.45] | 42.80 [37.59 to 48.14]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 44.00 [35.14 to 53.16] | 37.93 [28.18 to 48.46] | 45.22 [21.68 to 70.45] | 42.80 [37.59 to 48.14]

138. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any AEs Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a second dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 2 vaccination (i.e., week 46 for the second dose) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 46 and 52. Risk status (At risk; Not at risk) was recorded for influenza-associated morbidity and mortality as per healthcare professional assessment.
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 57.14 [0.00 to 100]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 53.85 [0.00 to 100]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 34.62 [2.53 to 85.04]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 29.73 [1.34 to 83.06]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 28.89 [0.63 to 86.72]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 29.17 [1.05 to 83.94]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 50.00 [1.26 to 98.74]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 40.00 [0.00 to 100]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 41.18 [0.03 to 99.64]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 29.09 [13.83 to 48.83]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 20.93 [7.66 to 41.13]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 21.11 [8.16 to 40.43]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 20.88 [8.20 to 39.75]

139. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Gastrointestinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 2.13 [0.00 to 99.46] |  | 2.13 [0.00 to 99.46]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 12.50 [0.00 to 99.41] | 7.50 [0.00 to 99.99] | 6.25 [0.16 to 30.23] | 8.04 [1.56 to 22.38]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 10.64 [0.00 to 69.52] | 7.78 [0.00 to 99.96] | 5.41 [0.00 to 99.49] | 8.05 [2.68 to 17.73]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 12.05 [2.62 to 31.07] | 7.84 [0.00 to 99.80] | 8.33 [0.41 to 34.04] | 9.39 [5.25 to 15.20]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 10.83 [4.92 to 19.92] | 7.89 [0.00 to 99.36] | 5.26 [0.60 to 18.20] | 8.04 [4.73 to 12.60]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 10.38 [4.74 to 19.08] | 6.82 [0.00 to 96.02] | 6.50 [1.41 to 17.58] | 7.96 [5.40 to 11.23]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 10.29 [5.05 to 18.12] | 6.77 [0.00 to 95.72] | 6.67 [1.89 to 16.02] | 8.04 [5.68 to 11.00]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 10.29 [5.05 to 18.12] | 6.77 [0.00 to 95.72] | 7.17 [2.28 to 16.25] | 8.21 [6.01 to 10.90]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 10.29 [5.05 to 18.12] | 6.77 [0.00 to 95.72] | 7.17 [2.28 to 16.25] | 8.21 [6.01 to 10.90]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 10.29 [5.05 to 18.12] | 6.77 [0.00 to 95.72] | 7.17 [2.28 to 16.25] | 8.21 [6.01 to 10.90]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 10.29 [5.05 to 18.12] | 6.77 [0.00 to 95.72] | 7.17 [2.28 to 16.25] | 8.21 [6.01 to 10.90]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 10.29 [5.05 to 18.12] | 6.77 [0.00 to 95.72] | 7.17 [2.28 to 16.25] | 8.21 [6.01 to 10.90]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 2.99 [0.36 to 10.37] |  | 2.99 [0.36 to 10.37]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 2.63 [0.49 to 7.85] |  | 2.63 [0.49 to 7.85]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.80 [0.02 to 4.38] | 2.42 [0.17 to 10.03] | 8.33 [0.13 to 41.57] | 2.46 [0.38 to 7.86]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.80 [0.02 to 4.38] | 2.36 [0.12 to 10.64] | 9.68 [2.05 to 25.70] | 3.77 [0.35 to 14.12]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.80 [0.02 to 4.38] | 2.31 [0.09 to 11.25] | 6.67 [3.09 to 12.28] | 3.33 [0.60 to 10.01]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.80 [0.02 to 4.38] | 2.94 [0.81 to 7.36] | 6.06 [2.54 to 11.91] | 3.70 [1.00 to 9.28]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.80 [0.02 to 4.38] | 3.47 [0.85 to 9.16] | 6.45 [3.57 to 10.59] | 4.12 [1.50 to 8.83]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.80 [0.02 to 4.38] | 3.45 [0.89 to 8.87] | 6.61 [3.75 to 10.66] | 4.23 [1.63 to 8.77]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.80 [0.02 to 4.38] | 3.45 [0.89 to 8.87] | 6.52 [3.70 to 10.53] | 4.20 [1.62 to 8.71]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.80 [0.02 to 4.38] | 3.45 [0.89 to 8.87] | 6.52 [3.70 to 10.53] | 4.20 [1.62 to 8.71]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.80 [0.02 to 4.38] | 3.45 [0.89 to 8.87] | 6.52 [3.70 to 10.53] | 4.20 [1.62 to 8.71]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.80 [0.02 to 4.38] | 3.45 [0.89 to 8.87] | 6.52 [3.70 to 10.53] | 4.20 [1.62 to 8.71]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.80 [0.02 to 4.38] | 3.45 [0.89 to 8.87] | 6.52 [3.70 to 10.53] | 4.20 [1.62 to 8.71]

140. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Gastrointestinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 14.29 [0.00 to 100]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 7.69 [0.00 to 100]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 3.85 [0.00 to 66.83]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 5.41 [0.00 to 81.93]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 4.44 [0.00 to 77.39]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 4.17 [0.00 to 76.38]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 50.00 [1.26 to 98.74]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 13.33 [0.00 to 97.21]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 5.88 [0.07 to 32.75]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 3.64 [0.44 to 12.53]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 2.33 [0.28 to 8.15]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 2.22 [0.27 to 7.80]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 2.20 [0.27 to 7.71]

141. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any General Disorders and Administration Site Conditions (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: The cumulative percentage of subjects was calculated as follows (per 100 subjects): the denominator was the number of subjects vaccinated with a first dose of the GSK's quadrivalent seasonal influenza vaccine at any point from dose 1 vaccination (i.e. week 40) up to the end of the week of interest; the numerator was the number of subjects among those vaccinated subjects, who reported the AE at least once on the ADR card within 7 days following vaccination. Vaccination period was defined between ISO weeks 40 and 52. No vaccination (Dose 1) was administered from ISO week 49 onwards. Risk status (At risk; Not at risk) was recorded for influenza-associated morbidity and mortality as per healthcare professional assessment.
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 25.53 [0.00 to 100] |  | 25.53 [0.00 to 100]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 37.50 [0.00 to 100] | 25.00 [0.00 to 100] | 43.75 [1.42 to 96.32] | 29.46 [13.05 to 51.01]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 25.53 [0.00 to 99.94] | 24.44 [0.00 to 100] | 32.43 [14.38 to 55.36] | 26.44 [15.77 to 39.59]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 32.53 [1.71 to 85.31] | 24.51 [0.00 to 99.96] | 26.67 [16.07 to 39.66] | 27.76 [19.07 to 37.87]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 25.48 [1.40 to 75.12] | 27.19 [0.00 to 99.99] | 32.24 [3.70 to 77.68] | 28.37 [17.36 to 41.65]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 24.04 [1.58 to 70.96] | 27.27 [0.00 to 99.90] | 31.50 [4.13 to 75.09] | 27.77 [16.90 to 40.95]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 24.51 [2.85 to 65.37] | 27.07 [0.00 to 99.87] | 32.38 [4.15 to 76.58] | 28.15 [17.34 to 41.19]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 24.51 [2.85 to 65.37] | 27.07 [0.00 to 99.87] | 34.08 [4.26 to 79.14] | 28.93 [17.28 to 43.04]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 24.51 [2.85 to 65.37] | 27.07 [0.00 to 99.87] | 34.08 [4.26 to 79.14] | 28.93 [17.28 to 43.04]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 24.51 [2.85 to 65.37] | 27.07 [0.00 to 99.87] | 34.08 [4.26 to 79.14] | 28.93 [17.28 to 43.04]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 24.51 [2.85 to 65.37] | 27.07 [0.00 to 99.87] | 34.08 [4.26 to 79.14] | 28.93 [17.28 to 43.04]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 24.51 [2.85 to 65.37] | 27.07 [0.00 to 99.87] | 34.08 [4.26 to 79.14] | 28.93 [17.28 to 43.04]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 26.87 [11.49 to 47.81] |  | 26.87 [11.49 to 47.81]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 28.95 [12.83 to 50.22] |  | 28.95 [12.83 to 50.22]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 30.40 [22.49 to 39.26] | 29.03 [14.04 to 48.34] | 19.44 [0.18 to 77.39] | 28.42 [23.06 to 34.27]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 30.40 [22.49 to 39.26] | 28.35 [10.83 to 52.51] | 24.73 [4.38 to 60.02] | 28.12 [23.18 to 33.47]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 30.40 [22.49 to 39.26] | 27.69 [8.22 to 56.49] | 22.96 [16.17 to 30.98] | 26.92 [20.63 to 33.98]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 30.40 [22.49 to 39.26] | 28.68 [13.37 to 48.65] | 24.75 [18.90 to 31.36] | 27.45 [22.67 to 32.65]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 30.40 [22.49 to 39.26] | 28.47 [13.11 to 48.63] | 24.88 [19.28 to 31.19] | 27.37 [23.07 to 31.99]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 30.40 [22.49 to 39.26] | 28.28 [12.28 to 49.64] | 25.99 [18.71 to 34.40] | 27.77 [23.41 to 32.46]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 30.40 [22.49 to 39.26] | 28.28 [12.28 to 49.64] | 26.52 [16.53 to 38.66] | 28.00 [23.48 to 32.87]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 30.40 [22.49 to 39.26] | 28.28 [12.28 to 49.64] | 26.52 [16.53 to 38.66] | 28.00 [23.48 to 32.87]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 30.40 [22.49 to 39.26] | 28.28 [12.28 to 49.64] | 26.52 [16.53 to 38.66] | 28.00 [23.48 to 32.87]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 30.40 [22.49 to 39.26] | 28.28 [12.28 to 49.64] | 26.52 [16.53 to 38.66] | 28.00 [23.48 to 32.87]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 30.40 [22.49 to 39.26] | 28.28 [12.28 to 49.64] | 26.52 [16.53 to 38.66] | 28.00 [23.48 to 32.87]

142. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any General Disorders and Administration Site Conditions (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 28.57 [2.18 to 76.83]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 15.38 [0.00 to 99.93]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 11.54 [2.45 to 30.15]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 10.81 [3.03 to 25.42]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 8.89 [2.48 to 21.22]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 10.42 [3.47 to 22.66]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 33.33 [0.00 to 100]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 17.65 [0.11 to 75.84]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 10.91 [4.11 to 22.25]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 8.14 [2.45 to 18.83]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 8.89 [2.85 to 19.86]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 8.79 [2.87 to 19.49]

143. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Immune System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 3.24]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 2.10]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 0.00 [0.00 to 4.35] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 1.49]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 0.64 [0.02 to 3.50] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 2.40] | 0.24 [0.01 to 1.35]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 0.55 [0.01 to 3.01] | 0.00 [0.00 to 2.76] | 0.00 [0.00 to 1.83] | 0.19 [0.00 to 1.11]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.74] | 0.18 [0.00 to 1.01]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.18 [0.00 to 1.00]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.18 [0.00 to 1.00]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.18 [0.00 to 1.00]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.18 [0.00 to 1.00]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 0.49 [0.01 to 2.70] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.18 [0.00 to 1.00]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.00 [0.00 to 3.18] |  | 0.00 [0.00 to 3.18]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 1.29]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 3.89] | 0.00 [0.00 to 1.06]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.70] | 0.00 [0.00 to 0.94]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.68] | 0.00 [0.00 to 1.85] | 0.00 [0.00 to 0.80]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.53] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 0.76]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.61] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]

144. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Immune System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

145. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Infections and Infestations (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 8.51 [0.00 to 99.99] |  | 8.51 [0.00 to 99.99]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 7.50 [0.00 to 97.14] | 6.25 [0.16 to 30.23] | 6.25 [1.56 to 15.94]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 4.26 [0.06 to 23.84] | 7.78 [0.00 to 95.50] | 5.41 [0.01 to 39.15] | 6.32 [2.58 to 12.60]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 6.02 [1.98 to 13.50] | 7.84 [0.00 to 91.81] | 5.00 [1.04 to 13.92] | 6.53 [3.78 to 10.39]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 7.64 [3.22 to 14.85] | 7.89 [0.00 to 87.38] | 5.92 [2.35 to 12.00] | 7.09 [4.84 to 9.97]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 7.10 [2.74 to 14.57] | 8.33 [0.00 to 83.24] | 7.00 [1.01 to 21.89] | 7.38 [5.11 to 10.24]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 6.86 [2.67 to 14.01] | 8.27 [0.00 to 82.34] | 7.14 [0.90 to 23.32] | 7.31 [4.99 to 10.26]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 6.86 [2.67 to 14.01] | 8.27 [0.00 to 82.34] | 7.62 [1.62 to 20.61] | 7.50 [5.26 to 10.31]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 6.86 [2.67 to 14.01] | 8.27 [0.00 to 82.34] | 7.62 [1.62 to 20.61] | 7.50 [5.26 to 10.31]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 6.86 [2.67 to 14.01] | 8.27 [0.00 to 82.34] | 7.62 [1.62 to 20.61] | 7.50 [5.26 to 10.31]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 6.86 [2.67 to 14.01] | 8.27 [0.00 to 82.34] | 7.62 [1.62 to 20.61] | 7.50 [5.26 to 10.31]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 6.86 [2.67 to 14.01] | 8.27 [0.00 to 82.34] | 7.62 [1.62 to 20.61] | 7.50 [5.26 to 10.31]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 8.96 [3.36 to 18.48] |  | 8.96 [3.36 to 18.48]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 8.77 [1.53 to 25.26] |  | 8.77 [1.53 to 25.26]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.80 [0.02 to 4.38] | 8.06 [0.50 to 31.40] | 0.00 [0.00 to 9.74] | 3.86 [0.09 to 19.92]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.80 [0.02 to 4.38] | 7.87 [0.35 to 33.05] | 3.23 [0.67 to 9.14] | 4.06 [0.34 to 15.55]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.80 [0.02 to 4.38] | 7.69 [0.24 to 34.68] | 4.44 [0.25 to 18.85] | 4.36 [0.76 to 13.14]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.80 [0.02 to 4.38] | 8.09 [0.76 to 28.36] | 4.55 [0.02 to 30.67] | 4.58 [1.01 to 12.49]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.80 [0.02 to 4.38] | 7.64 [0.36 to 31.76] | 4.61 [0.02 to 30.12] | 4.53 [1.07 to 12.02]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.80 [0.02 to 4.38] | 7.59 [0.33 to 32.18] | 5.29 [0.01 to 38.99] | 4.83 [1.16 to 12.69]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.80 [0.02 to 4.38] | 7.59 [0.33 to 32.18] | 5.22 [0.01 to 37.30] | 4.80 [1.17 to 12.53]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.80 [0.02 to 4.38] | 7.59 [0.33 to 32.18] | 5.22 [0.01 to 37.30] | 4.80 [1.17 to 12.53]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.80 [0.02 to 4.38] | 7.59 [0.33 to 32.18] | 5.22 [0.01 to 37.30] | 4.80 [1.17 to 12.53]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.80 [0.02 to 4.38] | 7.59 [0.33 to 32.18] | 5.22 [0.01 to 37.30] | 4.80 [1.17 to 12.53]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.80 [0.02 to 4.38] | 7.59 [0.33 to 32.18] | 5.22 [0.01 to 37.30] | 4.80 [1.17 to 12.53]

146. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Infections and Infestations (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 0.00 [0.00 to 40.96]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 23.08 [0.00 to 99.99]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 11.54 [0.21 to 51.85]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 8.11 [0.20 to 37.89]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 6.67 [0.29 to 28.75]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 6.25 [0.37 to 25.31]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 21.80]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 10.28]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 6.49]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 1.16 [0.03 to 6.31]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 1.11 [0.03 to 6.04]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 1.10 [0.03 to 5.97]

147. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Metabolism and Nutrition Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 6.25 [0.00 to 100] | 0.00 [0.00 to 4.51] | 6.25 [0.16 to 30.23] | 1.79 [0.02 to 11.20]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 2.13 [0.00 to 100] | 0.00 [0.00 to 4.02] | 5.41 [0.01 to 39.15] | 1.72 [0.03 to 9.75]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 2.41 [0.00 to 38.72] | 0.00 [0.00 to 3.55] | 10.00 [3.76 to 20.51] | 3.27 [0.31 to 12.24]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 3.18 [0.56 to 9.64] | 0.00 [0.00 to 3.18] | 6.58 [0.02 to 41.41] | 3.55 [0.76 to 9.87]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 3.28 [0.88 to 8.28] | 0.00 [0.00 to 2.76] | 5.00 [0.00 to 43.12] | 3.11 [0.70 to 8.49]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 3.43 [1.21 to 7.51] | 0.00 [0.00 to 2.74] | 4.76 [0.00 to 43.22] | 3.11 [0.78 to 8.12]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 3.43 [1.21 to 7.51] | 0.00 [0.00 to 2.74] | 5.38 [0.05 to 31.59] | 3.39 [1.11 to 7.74]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 3.43 [1.21 to 7.51] | 0.00 [0.00 to 2.74] | 5.38 [0.05 to 31.59] | 3.39 [1.11 to 7.74]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 3.43 [1.21 to 7.51] | 0.00 [0.00 to 2.74] | 5.38 [0.05 to 31.59] | 3.39 [1.11 to 7.74]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 3.43 [1.21 to 7.51] | 0.00 [0.00 to 2.74] | 5.38 [0.05 to 31.59] | 3.39 [1.11 to 7.74]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 3.43 [1.21 to 7.51] | 0.00 [0.00 to 2.74] | 5.38 [0.05 to 31.59] | 3.39 [1.11 to 7.74]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.88 [0.02 to 4.79] |  | 0.88 [0.02 to 4.79]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.81 [0.02 to 4.41] | 2.78 [0.05 to 15.34] | 0.70 [0.04 to 3.25]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.79 [0.02 to 4.31] | 9.68 [2.05 to 25.70] | 2.90 [0.04 to 17.14]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.77 [0.02 to 4.21] | 7.41 [3.61 to 13.20] | 2.82 [0.10 to 13.63]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 0.74 [0.01 to 4.27] | 6.06 [2.54 to 11.91] | 2.83 [0.23 to 11.23]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.82] | 5.53 [1.33 to 14.44] | 2.67 [0.21 to 10.65]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 5.29 [0.90 to 15.88] | 2.62 [0.20 to 10.48]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 5.22 [0.80 to 16.29] | 2.60 [0.20 to 10.44]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 5.22 [0.80 to 16.29] | 2.60 [0.20 to 10.44]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 5.22 [0.80 to 16.29] | 2.60 [0.20 to 10.44]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 5.22 [0.80 to 16.29] | 2.60 [0.20 to 10.44]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 5.22 [0.80 to 16.29] | 2.60 [0.20 to 10.44]

148. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Metabolism and Nutrition Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 0.00 [0.00 to 40.96]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 0.00 [0.00 to 24.71]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 0.00 [0.00 to 13.23]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 2.70 [0.07 to 14.16]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 2.22 [0.06 to 11.77]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 2.08 [0.05 to 11.07]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 6.67 [0.00 to 79.41]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 5.88 [0.07 to 32.75]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 3.64 [0.44 to 12.53]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 2.33 [0.28 to 8.15]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 2.22 [0.27 to 7.80]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 2.20 [0.27 to 7.71]

149. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Musculoskeletal and Connective Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 2.13 [0.00 to 99.46] |  | 2.13 [0.00 to 99.46]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 6.25 [0.00 to 100] | 2.50 [0.00 to 94.21] | 12.50 [1.15 to 41.43] | 4.46 [0.70 to 13.97]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 2.13 [0.00 to 100] | 4.44 [0.00 to 98.48] | 8.11 [0.01 to 53.94] | 4.60 [0.84 to 13.55]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 9.64 [0.23 to 43.70] | 4.90 [0.00 to 97.43] | 6.67 [1.21 to 19.31] | 6.94 [3.68 to 11.72]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 10.19 [1.52 to 30.44] | 6.14 [0.00 to 97.75] | 7.89 [0.10 to 41.07] | 8.27 [4.86 to 12.98]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 10.38 [2.47 to 26.20] | 6.82 [0.00 to 96.02] | 8.00 [0.15 to 39.06] | 8.54 [5.32 to 12.85]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 9.80 [2.20 to 25.43] | 6.77 [0.00 to 95.72] | 7.62 [0.19 to 35.69] | 8.23 [5.26 to 12.13]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 9.80 [2.20 to 25.43] | 6.77 [0.00 to 95.72] | 9.87 [0.11 to 49.43] | 9.11 [5.02 to 14.91]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 9.80 [2.20 to 25.43] | 6.77 [0.00 to 95.72] | 9.87 [0.11 to 49.43] | 9.11 [5.02 to 14.91]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 9.80 [2.20 to 25.43] | 6.77 [0.00 to 95.72] | 9.87 [0.11 to 49.43] | 9.11 [5.02 to 14.91]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 9.80 [2.20 to 25.43] | 6.77 [0.00 to 95.72] | 9.87 [0.11 to 49.43] | 9.11 [5.02 to 14.91]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 9.80 [2.20 to 25.43] | 6.77 [0.00 to 95.72] | 9.87 [0.11 to 49.43] | 9.11 [5.02 to 14.91]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 5.97 [1.65 to 14.59] |  | 5.97 [1.65 to 14.59]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 8.77 [1.53 to 25.26] |  | 8.77 [1.53 to 25.26]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 12.00 [6.87 to 19.02] | 8.06 [0.50 to 31.40] | 5.56 [0.10 to 29.18] | 9.47 [5.80 to 14.40]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 12.00 [6.87 to 19.02] | 8.66 [1.55 to 24.72] | 7.53 [1.63 to 20.21] | 9.57 [6.57 to 13.33]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 12.00 [6.87 to 19.02] | 8.46 [1.25 to 25.87] | 5.93 [2.59 to 11.34] | 8.72 [4.96 to 13.98]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 12.00 [6.87 to 19.02] | 8.82 [2.16 to 22.28] | 6.57 [1.95 to 15.45] | 8.71 [5.28 to 13.36]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 12.00 [6.87 to 19.02] | 9.72 [3.93 to 19.20] | 6.91 [2.02 to 16.36] | 9.05 [5.64 to 13.60]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 12.00 [6.87 to 19.02] | 9.66 [3.90 to 19.08] | 7.05 [2.32 to 15.70] | 9.05 [5.74 to 13.43]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 12.00 [6.87 to 19.02] | 9.66 [3.90 to 19.08] | 6.96 [2.38 to 15.22] | 9.00 [5.70 to 13.36]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 12.00 [6.87 to 19.02] | 9.66 [3.90 to 19.08] | 6.96 [2.38 to 15.22] | 9.00 [5.70 to 13.36]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 12.00 [6.87 to 19.02] | 9.66 [3.90 to 19.08] | 6.96 [2.38 to 15.22] | 9.00 [5.70 to 13.36]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 12.00 [6.87 to 19.02] | 9.66 [3.90 to 19.08] | 6.96 [2.38 to 15.22] | 9.00 [5.70 to 13.36]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 12.00 [6.87 to 19.02] | 9.66 [3.90 to 19.08] | 6.96 [2.38 to 15.22] | 9.00 [5.70 to 13.36]

150. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Musculoskeletal and Connective Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 0.00 [0.00 to 40.96]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 0.00 [0.00 to 24.71]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 0.00 [0.00 to 13.23]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 0.00 [0.00 to 9.49]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 0.00 [0.00 to 7.87]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 0.00 [0.00 to 7.40]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 6.67 [0.00 to 79.41]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 2.94 [0.04 to 17.37]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 1.82 [0.05 to 9.72]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 1.16 [0.03 to 6.31]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 1.11 [0.03 to 6.04]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 1.10 [0.03 to 5.97]

151. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Nervous System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 8.51 [0.00 to 99.99] |  | 8.51 [0.00 to 99.99]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 25.00 [0.00 to 100] | 7.50 [0.00 to 97.14] | 0.00 [0.00 to 20.59] | 8.93 [2.70 to 20.53]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 14.89 [0.00 to 99.25] | 7.78 [0.00 to 95.50] | 5.41 [0.01 to 39.15] | 9.20 [4.72 to 15.77]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 15.66 [1.96 to 46.07] | 7.84 [0.00 to 91.81] | 5.00 [1.04 to 13.92] | 9.80 [5.67 to 15.49]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 14.65 [6.92 to 26.01] | 7.89 [0.00 to 87.38] | 6.58 [0.29 to 28.35] | 9.93 [6.23 to 14.81]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 12.57 [4.16 to 27.09] | 8.33 [0.00 to 83.24] | 7.00 [0.26 to 31.01] | 9.32 [6.33 to 13.11]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 11.27 [2.87 to 27.49] | 8.27 [0.00 to 82.34] | 6.67 [0.32 to 28.17] | 8.78 [6.11 to 12.11]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 11.27 [2.87 to 27.49] | 8.27 [0.00 to 82.34] | 8.52 [0.18 to 40.41] | 9.46 [6.25 to 13.60]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 11.27 [2.87 to 27.49] | 8.27 [0.00 to 82.34] | 8.52 [0.18 to 40.41] | 9.46 [6.25 to 13.60]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 11.27 [2.87 to 27.49] | 8.27 [0.00 to 82.34] | 8.52 [0.18 to 40.41] | 9.46 [6.25 to 13.60]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 11.27 [2.87 to 27.49] | 8.27 [0.00 to 82.34] | 8.52 [0.18 to 40.41] | 9.46 [6.25 to 13.60]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 11.27 [2.87 to 27.49] | 8.27 [0.00 to 82.34] | 8.52 [0.18 to 40.41] | 9.46 [6.25 to 13.60]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 5.97 [1.65 to 14.59] |  | 5.97 [1.65 to 14.59]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 6.14 [1.10 to 17.96] |  | 6.14 [1.10 to 17.96]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 3.20 [0.88 to 7.99] | 5.65 [0.37 to 22.59] | 2.78 [0.05 to 15.34] | 4.21 [1.49 to 9.18]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 3.20 [0.88 to 7.99] | 5.51 [0.26 to 23.86] | 5.38 [1.19 to 14.58] | 4.64 [2.20 to 8.47]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 3.20 [0.88 to 7.99] | 5.38 [0.18 to 25.12] | 3.70 [1.21 to 8.43] | 4.10 [2.04 to 7.27]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 3.20 [0.88 to 7.99] | 5.88 [0.94 to 18.02] | 6.57 [1.95 to 15.45] | 5.45 [3.22 to 8.56]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 3.20 [0.88 to 7.99] | 6.94 [2.86 to 13.71] | 6.91 [2.02 to 16.36] | 5.97 [3.71 to 9.02]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 3.20 [0.88 to 7.99] | 7.59 [2.56 to 16.67] | 7.05 [2.32 to 15.70] | 6.24 [3.86 to 9.45]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 3.20 [0.88 to 7.99] | 7.59 [2.56 to 16.67] | 7.39 [2.13 to 17.55] | 6.40 [3.95 to 9.72]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 3.20 [0.88 to 7.99] | 7.59 [2.56 to 16.67] | 7.39 [2.13 to 17.55] | 6.40 [3.95 to 9.72]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 3.20 [0.88 to 7.99] | 7.59 [2.56 to 16.67] | 7.39 [2.13 to 17.55] | 6.40 [3.95 to 9.72]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 3.20 [0.88 to 7.99] | 7.59 [2.56 to 16.67] | 7.39 [2.13 to 17.55] | 6.40 [3.95 to 9.72]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 3.20 [0.88 to 7.99] | 7.59 [2.56 to 16.67] | 7.39 [2.13 to 17.55] | 6.40 [3.95 to 9.72]

152. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Nervous System Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

153. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Psychiatric Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 5.00 [0.00 to 99.75] | 0.00 [0.00 to 20.59] | 3.57 [0.10 to 18.07]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 5.56 [0.00 to 99.52] | 0.00 [0.00 to 9.49] | 2.87 [0.03 to 17.26]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 1.20 [0.00 to 27.53] | 4.90 [0.00 to 97.43] | 1.67 [0.04 to 8.94] | 2.86 [0.40 to 9.44]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 1.27 [0.04 to 6.71] | 4.39 [0.00 to 92.73] | 0.66 [0.00 to 8.80] | 1.89 [0.30 to 6.08]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 1.64 [0.34 to 4.72] | 3.79 [0.00 to 81.65] | 1.00 [0.00 to 16.86] | 1.94 [0.53 to 4.92]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 1.47 [0.30 to 4.24] | 3.76 [0.00 to 80.95] | 1.43 [0.06 to 6.92] | 2.01 [0.70 to 4.46]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 1.47 [0.30 to 4.24] | 3.76 [0.00 to 80.95] | 1.35 [0.03 to 7.32] | 1.96 [0.66 to 4.43]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 1.47 [0.30 to 4.24] | 3.76 [0.00 to 80.95] | 1.35 [0.03 to 7.32] | 1.96 [0.66 to 4.43]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 1.47 [0.30 to 4.24] | 3.76 [0.00 to 80.95] | 1.35 [0.03 to 7.32] | 1.96 [0.66 to 4.43]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 1.47 [0.30 to 4.24] | 3.76 [0.00 to 80.95] | 1.35 [0.03 to 7.32] | 1.96 [0.66 to 4.43]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 1.47 [0.30 to 4.24] | 3.76 [0.00 to 80.95] | 1.35 [0.03 to 7.32] | 1.96 [0.66 to 4.43]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.00 [0.00 to 3.18] |  | 0.00 [0.00 to 3.18]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.93] | 2.78 [0.05 to 15.34] | 0.35 [0.00 to 3.52]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.86] | 5.38 [1.19 to 14.58] | 1.45 [0.01 to 10.70]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.80] | 4.44 [1.28 to 10.75] | 1.54 [0.07 to 7.33]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.68] | 3.54 [1.43 to 7.15] | 1.53 [0.10 to 6.60]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.53] | 3.69 [1.60 to 7.13] | 1.65 [0.19 to 5.97]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 3.52 [1.53 to 6.83] | 1.61 [0.18 to 5.83]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 3.48 [1.51 to 6.74] | 1.60 [0.18 to 5.79]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 3.48 [1.51 to 6.74] | 1.60 [0.18 to 5.79]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 3.48 [1.51 to 6.74] | 1.60 [0.18 to 5.79]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 3.48 [1.51 to 6.74] | 1.60 [0.18 to 5.79]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 3.48 [1.51 to 6.74] | 1.60 [0.18 to 5.79]

154. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Psychiatric Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 0.00 [0.00 to 40.96]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 0.00 [0.00 to 24.71]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 0.00 [0.00 to 13.23]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 0.00 [0.00 to 9.49]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 0.00 [0.00 to 7.87]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 0.00 [0.00 to 7.40]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 21.80]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 5.88 [0.07 to 32.75]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 7.27 [0.65 to 26.14]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 4.65 [0.39 to 17.73]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 4.44 [0.37 to 17.05]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 4.40 [0.36 to 16.89]

155. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Respiratory, Thoracic and Mediastinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 8.51 [0.00 to 99.99] |  | 8.51 [0.00 to 99.99]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 12.50 [0.00 to 99.41] | 8.75 [0.00 to 99.35] | 31.25 [1.75 to 83.28] | 12.50 [3.59 to 28.74]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 17.02 [0.13 to 73.09] | 11.11 [0.00 to 99.86] | 29.73 [0.00 to 98.65] | 16.67 [6.65 to 32.12]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 20.48 [12.41 to 30.76] | 10.78 [0.00 to 99.23] | 26.67 [7.84 to 54.97] | 17.96 [9.63 to 29.30]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 20.38 [14.38 to 27.54] | 12.28 [0.00 to 99.36] | 23.03 [4.14 to 56.68] | 19.15 [13.30 to 26.21]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 18.58 [13.22 to 24.98] | 12.12 [0.00 to 97.62] | 22.50 [7.16 to 46.40] | 18.45 [13.70 to 24.01]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 17.65 [12.68 to 23.58] | 12.03 [0.00 to 97.36] | 22.86 [6.62 to 48.70] | 18.28 [13.54 to 23.84]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 17.65 [12.68 to 23.58] | 12.03 [0.00 to 97.36] | 22.87 [7.69 to 46.03] | 18.39 [13.80 to 23.75]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 17.65 [12.68 to 23.58] | 12.03 [0.00 to 97.36] | 22.87 [7.69 to 46.03] | 18.39 [13.80 to 23.75]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 17.65 [12.68 to 23.58] | 12.03 [0.00 to 97.36] | 22.87 [7.69 to 46.03] | 18.39 [13.80 to 23.75]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 17.65 [12.68 to 23.58] | 12.03 [0.00 to 97.36] | 22.87 [7.69 to 46.03] | 18.39 [13.80 to 23.75]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 17.65 [12.68 to 23.58] | 12.03 [0.00 to 97.36] | 22.87 [7.69 to 46.03] | 18.39 [13.80 to 23.75]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 8.96 [3.36 to 18.48] |  | 8.96 [3.36 to 18.48]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 12.28 [4.45 to 25.38] |  | 12.28 [4.45 to 25.38]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 9.60 [5.06 to 16.17] | 12.10 [3.48 to 27.87] | 25.00 [0.16 to 87.94] | 12.63 [6.85 to 20.72]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 9.60 [5.06 to 16.17] | 11.81 [3.08 to 28.40] | 24.73 [16.37 to 34.76] | 14.49 [6.58 to 26.33]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 9.60 [5.06 to 16.17] | 11.54 [2.65 to 29.25] | 22.22 [14.01 to 32.40] | 14.62 [8.24 to 23.28]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 9.60 [5.06 to 16.17] | 11.76 [3.37 to 27.20] | 22.22 [8.23 to 43.14] | 15.69 [9.73 to 23.39]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 9.60 [5.06 to 16.17] | 11.11 [2.28 to 29.50] | 22.12 [9.18 to 40.79] | 15.64 [9.72 to 23.28]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 9.60 [5.06 to 16.17] | 11.03 [2.15 to 29.85] | 22.47 [8.39 to 43.40] | 15.90 [9.76 to 23.85]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 9.60 [5.06 to 16.17] | 11.03 [2.15 to 29.85] | 23.04 [6.94 to 48.35] | 16.20 [9.72 to 24.69]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 9.60 [5.06 to 16.17] | 11.03 [2.15 to 29.85] | 23.04 [6.94 to 48.35] | 16.20 [9.72 to 24.69]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 9.60 [5.06 to 16.17] | 11.03 [2.15 to 29.85] | 23.04 [6.94 to 48.35] | 16.20 [9.72 to 24.69]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 9.60 [5.06 to 16.17] | 11.03 [2.15 to 29.85] | 23.04 [6.94 to 48.35] | 16.20 [9.72 to 24.69]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 9.60 [5.06 to 16.17] | 11.03 [2.15 to 29.85] | 23.04 [6.94 to 48.35] | 16.20 [9.72 to 24.69]

156. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Respiratory, Thoracic and Mediastinal Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 28.57 [0.00 to 100]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 30.77 [0.00 to 100]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 23.08 [0.70 to 76.09]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 18.92 [1.97 to 55.63]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 20.00 [0.96 to 66.16]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 18.75 [0.67 to 66.08]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 6.67 [0.00 to 79.41]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 23.53 [0.10 to 87.82]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 16.36 [7.00 to 30.49]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 11.63 [4.28 to 23.93]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 11.11 [4.26 to 22.44]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 10.99 [4.25 to 22.10]

157. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Skin and Subcutaneous Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 2.13 [0.00 to 99.46] |  | 2.13 [0.00 to 99.46]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 2.50 [0.00 to 94.21] | 12.50 [1.15 to 41.43] | 3.57 [0.42 to 12.48]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 2.13 [0.03 to 12.41] | 2.22 [0.00 to 86.59] | 5.41 [0.01 to 39.15] | 2.87 [0.94 to 6.58]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 1.20 [0.01 to 8.25] | 1.96 [0.00 to 75.07] | 5.00 [1.04 to 13.92] | 2.45 [0.80 to 5.62]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 3.82 [1.42 to 8.13] | 1.75 [0.00 to 63.29] | 3.29 [0.00 to 29.73] | 3.07 [1.42 to 5.73]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 3.28 [1.21 to 7.00] | 1.52 [0.00 to 47.97] | 2.50 [0.00 to 28.45] | 2.52 [1.05 to 5.03]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 2.94 [1.09 to 6.29] | 1.50 [0.00 to 47.23] | 2.38 [0.00 to 27.72] | 2.38 [1.02 to 4.65]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 2.94 [1.09 to 6.29] | 1.50 [0.00 to 47.23] | 2.24 [0.00 to 27.87] | 2.32 [0.95 to 4.70]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 2.94 [1.09 to 6.29] | 1.50 [0.00 to 47.23] | 2.24 [0.00 to 27.87] | 2.32 [0.95 to 4.70]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 2.94 [1.09 to 6.29] | 1.50 [0.00 to 47.23] | 2.24 [0.00 to 27.87] | 2.32 [0.95 to 4.70]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 2.94 [1.09 to 6.29] | 1.50 [0.00 to 47.23] | 2.24 [0.00 to 27.87] | 2.32 [0.95 to 4.70]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 2.94 [1.09 to 6.29] | 1.50 [0.00 to 47.23] | 2.24 [0.00 to 27.87] | 2.32 [0.95 to 4.70]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 2.99 [0.36 to 10.37] |  | 2.99 [0.36 to 10.37]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 1.75 [0.21 to 6.19] |  | 1.75 [0.21 to 6.19]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 1.61 [0.12 to 6.74] | 0.00 [0.00 to 9.74] | 0.70 [0.01 to 4.79]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 2.36 [0.38 to 7.46] | 0.00 [0.00 to 3.89] | 0.87 [0.03 to 4.43]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 2.31 [0.47 to 6.65] | 0.74 [0.00 to 30.06] | 1.03 [0.07 to 4.33]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 2.21 [0.46 to 6.31] | 0.51 [0.00 to 19.03] | 0.87 [0.06 to 3.70]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 2.78 [0.17 to 11.91] | 0.46 [0.00 to 16.65] | 1.03 [0.07 to 4.31]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 2.76 [0.18 to 11.54] | 0.44 [0.00 to 14.95] | 1.01 [0.08 to 4.15]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 2.76 [0.18 to 11.54] | 0.43 [0.00 to 14.44] | 1.00 [0.08 to 4.10]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 2.76 [0.18 to 11.54] | 0.43 [0.00 to 14.44] | 1.00 [0.08 to 4.10]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 2.76 [0.18 to 11.54] | 0.43 [0.00 to 14.44] | 1.00 [0.08 to 4.10]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 2.76 [0.18 to 11.54] | 0.43 [0.00 to 14.44] | 1.00 [0.08 to 4.10]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 2.76 [0.18 to 11.54] | 0.43 [0.00 to 14.44] | 1.00 [0.08 to 4.10]

158. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Skin and Subcutaneous Tissue Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 0.00 [0.00 to 40.96]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 0.00 [0.00 to 24.71]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 0.00 [0.00 to 13.23]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 0.00 [0.00 to 9.49]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 0.00 [0.00 to 7.87]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 0.00 [0.00 to 7.40]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 21.80]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 2.94 [0.04 to 17.37]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 1.82 [0.05 to 9.72]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 1.16 [0.03 to 6.31]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 1.11 [0.03 to 6.04]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 1.10 [0.03 to 5.97]

159. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Cardiac Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 3.24]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 2.10]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 0.00 [0.00 to 4.35] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 1.49]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 2.40] | 0.00 [0.00 to 0.87]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 2.76] | 0.00 [0.00 to 1.83] | 0.00 [0.00 to 0.71]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.74] | 0.00 [0.00 to 0.67]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 1.49 [0.04 to 8.04] |  | 1.49 [0.04 to 8.04]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.88 [0.02 to 4.79] |  | 0.88 [0.02 to 4.79]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.81 [0.02 to 4.41] | 0.00 [0.00 to 9.74] | 0.35 [0.00 to 2.41]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.79 [0.02 to 4.31] | 0.00 [0.00 to 3.89] | 0.29 [0.00 to 2.16]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.77 [0.02 to 4.21] | 0.00 [0.00 to 2.70] | 0.26 [0.00 to 1.83]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 0.74 [0.01 to 4.27] | 0.00 [0.00 to 1.85] | 0.22 [0.00 to 1.64]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.82] | 0.00 [0.00 to 1.69] | 0.21 [0.00 to 1.56]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.61] | 0.20 [0.00 to 1.52]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]

160. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Cardiac Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

161. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Ear and Labyrinth Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 2.13 [0.00 to 99.46] |  | 2.13 [0.00 to 99.46]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 1.25 [0.00 to 75.19] | 0.00 [0.00 to 20.59] | 0.89 [0.02 to 4.87]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 1.11 [0.00 to 62.70] | 0.00 [0.00 to 9.49] | 0.57 [0.01 to 3.61]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 1.20 [0.00 to 27.53] | 0.98 [0.00 to 49.52] | 1.67 [0.04 to 8.94] | 1.22 [0.25 to 3.54]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 0.64 [0.00 to 18.63] | 1.75 [0.00 to 63.29] | 0.66 [0.00 to 8.80] | 0.95 [0.16 to 2.98]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 0.55 [0.00 to 17.51] | 2.27 [0.00 to 62.91] | 0.50 [0.00 to 8.76] | 0.97 [0.11 to 3.52]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 0.49 [0.00 to 16.62] | 2.26 [0.00 to 62.10] | 0.48 [0.00 to 8.76] | 0.91 [0.09 to 3.45]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 0.49 [0.00 to 16.62] | 2.26 [0.00 to 62.10] | 0.45 [0.00 to 8.85] | 0.89 [0.09 to 3.42]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 0.49 [0.00 to 16.62] | 2.26 [0.00 to 62.10] | 0.45 [0.00 to 8.85] | 0.89 [0.09 to 3.42]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 0.49 [0.00 to 16.62] | 2.26 [0.00 to 62.10] | 0.45 [0.00 to 8.85] | 0.89 [0.09 to 3.42]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 0.49 [0.00 to 16.62] | 2.26 [0.00 to 62.10] | 0.45 [0.00 to 8.85] | 0.89 [0.09 to 3.42]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 0.49 [0.00 to 16.62] | 2.26 [0.00 to 62.10] | 0.45 [0.00 to 8.85] | 0.89 [0.09 to 3.42]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.88 [0.02 to 4.79] |  | 0.88 [0.02 to 4.79]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.81 [0.02 to 4.41] | 0.00 [0.00 to 9.74] | 0.35 [0.00 to 2.41]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.79 [0.02 to 4.31] | 0.00 [0.00 to 3.89] | 0.29 [0.00 to 2.16]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.77 [0.02 to 4.21] | 0.00 [0.00 to 2.70] | 0.26 [0.00 to 1.83]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 1.47 [0.04 to 7.88] | 0.00 [0.00 to 1.85] | 0.44 [0.02 to 2.21]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 1.39 [0.09 to 6.05] | 0.00 [0.00 to 1.69] | 0.41 [0.02 to 2.04]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 1.38 [0.09 to 5.86] | 0.00 [0.00 to 1.61] | 0.40 [0.02 to 1.98]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 1.38 [0.09 to 5.86] | 0.00 [0.00 to 1.59] | 0.40 [0.02 to 1.97]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 1.38 [0.09 to 5.86] | 0.00 [0.00 to 1.59] | 0.40 [0.02 to 1.97]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 1.38 [0.09 to 5.86] | 0.00 [0.00 to 1.59] | 0.40 [0.02 to 1.97]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 1.38 [0.09 to 5.86] | 0.00 [0.00 to 1.59] | 0.40 [0.02 to 1.97]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 1.38 [0.09 to 5.86] | 0.00 [0.00 to 1.59] | 0.40 [0.02 to 1.97]

162. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Ear and Labyrinth Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

163. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Eye Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 2.50 [0.00 to 94.21] | 0.00 [0.00 to 20.59] | 1.79 [0.05 to 9.29]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 2.22 [0.00 to 86.59] | 0.00 [0.00 to 9.49] | 1.15 [0.01 to 7.15]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 1.20 [0.00 to 27.53] | 1.96 [0.00 to 75.07] | 0.00 [0.00 to 5.96] | 1.22 [0.13 to 4.52]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 0.64 [0.00 to 18.63] | 1.75 [0.00 to 63.29] | 0.00 [0.00 to 2.40] | 0.71 [0.04 to 3.13]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 0.55 [0.00 to 17.51] | 1.52 [0.00 to 47.97] | 0.00 [0.00 to 1.83] | 0.58 [0.03 to 2.63]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 0.49 [0.00 to 16.62] | 1.50 [0.00 to 47.23] | 0.00 [0.00 to 1.74] | 0.55 [0.03 to 2.55]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 0.49 [0.00 to 16.62] | 1.50 [0.00 to 47.23] | 0.00 [0.00 to 1.64] | 0.54 [0.03 to 2.52]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 0.49 [0.00 to 16.62] | 1.50 [0.00 to 47.23] | 0.00 [0.00 to 1.64] | 0.54 [0.03 to 2.52]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 0.49 [0.00 to 16.62] | 1.50 [0.00 to 47.23] | 0.00 [0.00 to 1.64] | 0.54 [0.03 to 2.52]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 0.49 [0.00 to 16.62] | 1.50 [0.00 to 47.23] | 0.00 [0.00 to 1.64] | 0.54 [0.03 to 2.52]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 0.49 [0.00 to 16.62] | 1.50 [0.00 to 47.23] | 0.00 [0.00 to 1.64] | 0.54 [0.03 to 2.52]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 1.49 [0.04 to 8.04] |  | 1.49 [0.04 to 8.04]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.88 [0.02 to 4.79] |  | 0.88 [0.02 to 4.79]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.81 [0.02 to 4.41] | 0.00 [0.00 to 9.74] | 0.35 [0.00 to 2.41]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.79 [0.02 to 4.31] | 0.00 [0.00 to 3.89] | 0.29 [0.00 to 2.16]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.77 [0.02 to 4.21] | 0.00 [0.00 to 2.70] | 0.26 [0.00 to 1.83]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 0.74 [0.01 to 4.27] | 0.00 [0.00 to 1.85] | 0.22 [0.00 to 1.64]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.82] | 0.00 [0.00 to 1.69] | 0.21 [0.00 to 1.56]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.61] | 0.20 [0.00 to 1.52]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 4.89] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.51]

164. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Eye Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 139
Percentage of subjects
  At risk,Weeks 40-46: number analyzed (Participants) | 1
  At risk,Weeks 40-46 | 0.00 [0.00 to 97.50]
  At risk,Weeks 40-47: number analyzed (Participants) | 7
  At risk,Weeks 40-47 | 14.29 [0.00 to 100]
  At risk,Weeks 40-48: number analyzed (Participants) | 13
  At risk,Weeks 40-48 | 7.69 [0.00 to 90.25]
  At risk,Weeks 40-49: number analyzed (Participants) | 26
  At risk,Weeks 40-49 | 3.85 [0.10 to 19.72]
  At risk,Weeks 40-50: number analyzed (Participants) | 37
  At risk,Weeks 40-50 | 2.70 [0.07 to 14.16]
  At risk,Weeks 40-51: number analyzed (Participants) | 45
  At risk,Weeks 40-51 | 2.22 [0.06 to 11.77]
  At risk,Weeks 40-52: number analyzed (Participants) | 48
  At risk,Weeks 40-52 | 2.08 [0.05 to 11.07]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 2
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 84.19]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 15
  Not at risk,Weeks 40-47 | 6.67 [0.00 to 79.41]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 34
  Not at risk,Weeks 40-48 | 2.94 [0.04 to 17.37]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 55
  Not at risk,Weeks 40-49 | 1.82 [0.05 to 9.72]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 86
  Not at risk,Weeks 40-50 | 1.16 [0.03 to 6.31]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 90
  Not at risk,Weeks 40-51 | 1.11 [0.03 to 6.04]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 91
  Not at risk,Weeks 40-52 | 1.10 [0.03 to 5.97]

165. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Injury, Poisoning and Procedural Complications (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 3.24]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 2.10]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 0.00 [0.00 to 4.35] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 1.49]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 2.40] | 0.00 [0.00 to 0.87]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 2.76] | 0.00 [0.00 to 1.83] | 0.00 [0.00 to 0.71]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.74] | 0.00 [0.00 to 0.67]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.00 [0.00 to 3.18] |  | 0.00 [0.00 to 3.18]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 1.29]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 3.89] | 0.00 [0.00 to 1.06]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.70] | 0.00 [0.00 to 0.94]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 0.74 [0.00 to 20.74] | 0.00 [0.00 to 1.85] | 0.22 [0.00 to 2.05]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 17.92] | 0.00 [0.00 to 1.69] | 0.21 [0.00 to 1.88]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 17.61] | 0.00 [0.00 to 1.61] | 0.20 [0.00 to 1.83]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 17.61] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.82]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 17.61] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.82]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 17.61] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.82]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 17.61] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.82]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 0.69 [0.00 to 17.61] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.82]

166. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Injury, Poisoning and Procedural Complications (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

167. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Investigations (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 2.50 [0.00 to 94.21] | 0.00 [0.00 to 20.59] | 1.79 [0.05 to 9.29]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 3.33 [0.00 to 95.38] | 0.00 [0.00 to 9.49] | 1.72 [0.02 to 10.60]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 0.00 [0.00 to 4.35] | 2.94 [0.00 to 87.98] | 0.00 [0.00 to 5.96] | 1.22 [0.02 to 6.96]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 0.64 [0.02 to 3.50] | 2.63 [0.00 to 78.24] | 0.00 [0.00 to 2.40] | 0.95 [0.07 to 3.90]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 0.55 [0.01 to 3.01] | 2.27 [0.00 to 62.91] | 0.00 [0.00 to 1.83] | 0.78 [0.06 to 3.23]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 0.49 [0.01 to 2.70] | 2.26 [0.00 to 62.10] | 0.00 [0.00 to 1.74] | 0.73 [0.05 to 3.09]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 0.49 [0.01 to 2.70] | 2.26 [0.00 to 62.10] | 0.00 [0.00 to 1.64] | 0.71 [0.05 to 3.06]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 0.49 [0.01 to 2.70] | 2.26 [0.00 to 62.10] | 0.00 [0.00 to 1.64] | 0.71 [0.05 to 3.06]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 0.49 [0.01 to 2.70] | 2.26 [0.00 to 62.10] | 0.00 [0.00 to 1.64] | 0.71 [0.05 to 3.06]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 0.49 [0.01 to 2.70] | 2.26 [0.00 to 62.10] | 0.00 [0.00 to 1.64] | 0.71 [0.05 to 3.06]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 0.49 [0.01 to 2.70] | 2.26 [0.00 to 62.10] | 0.00 [0.00 to 1.64] | 0.71 [0.05 to 3.06]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.00 [0.00 to 3.18] |  | 0.00 [0.00 to 3.18]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 9.74] | 0.00 [0.00 to 1.29]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 3.89] | 0.00 [0.00 to 1.06]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.70] | 0.00 [0.00 to 0.94]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.68] | 0.00 [0.00 to 1.85] | 0.00 [0.00 to 0.80]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.53] | 0.00 [0.00 to 1.69] | 0.00 [0.00 to 0.76]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.61] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.00 [0.00 to 2.91] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.00 [0.00 to 0.74]

168. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Investigations (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

169. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Vascular Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 1 by Vaccine Group and Overall, by Risk Status
Description: as for outcome 137
Time Frame: Within 7 days post Dose 1 i.e. the day of vaccination and the following 6 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group | Total Group
Number analyzed (Participants) | 329 | 278 | 453 | 1060
Percentage of subjects
  At risk,Weeks 40-40: number analyzed (Participants) | 0 | 3 | 0 | 3
  At risk,Weeks 40-40 |  | 0.00 [0.00 to 70.76] |  | 0.00 [0.00 to 70.76]
  At risk,Weeks 40-41: number analyzed (Participants) | 0 | 47 | 0 | 47
  At risk,Weeks 40-41 |  | 0.00 [0.00 to 7.55] |  | 0.00 [0.00 to 7.55]
  At risk,Weeks 40-42: number analyzed (Participants) | 16 | 80 | 16 | 112
  At risk,Weeks 40-42 | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 4.51] | 0.00 [0.00 to 20.59] | 0.00 [0.00 to 3.24]
  At risk,Weeks 40-43: number analyzed (Participants) | 47 | 90 | 37 | 174
  At risk,Weeks 40-43 | 0.00 [0.00 to 7.55] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 9.49] | 0.00 [0.00 to 2.10]
  At risk,Weeks 40-44: number analyzed (Participants) | 83 | 102 | 60 | 245
  At risk,Weeks 40-44 | 0.00 [0.00 to 4.35] | 0.00 [0.00 to 3.55] | 0.00 [0.00 to 5.96] | 0.00 [0.00 to 1.49]
  At risk,Weeks 40-45: number analyzed (Participants) | 157 | 114 | 152 | 423
  At risk,Weeks 40-45 | 0.00 [0.00 to 2.32] | 0.00 [0.00 to 3.18] | 0.00 [0.00 to 2.40] | 0.00 [0.00 to 0.87]
  At risk,Weeks 40-46: number analyzed (Participants) | 183 | 132 | 200 | 515
  At risk,Weeks 40-46 | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 2.76] | 0.00 [0.00 to 1.83] | 0.00 [0.00 to 0.71]
  At risk,Weeks 40-47: number analyzed (Participants) | 204 | 133 | 210 | 547
  At risk,Weeks 40-47 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.74] | 0.00 [0.00 to 0.67]
  At risk,Weeks 40-48: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-48 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-49: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-49 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-50: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-50 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-51: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-51 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  At risk,Weeks 40-52: number analyzed (Participants) | 204 | 133 | 223 | 560
  At risk,Weeks 40-52 | 0.00 [0.00 to 1.79] | 0.00 [0.00 to 2.74] | 0.00 [0.00 to 1.64] | 0.00 [0.00 to 0.66]
  Not at risk,Weeks 40-40: number analyzed (Participants) | 0 | 67 | 0 | 67
  Not at risk,Weeks 40-40 |  | 0.00 [0.00 to 5.36] |  | 0.00 [0.00 to 5.36]
  Not at risk,Weeks 40-41: number analyzed (Participants) | 0 | 114 | 0 | 114
  Not at risk,Weeks 40-41 |  | 0.00 [0.00 to 3.18] |  | 0.00 [0.00 to 3.18]
  Not at risk,Weeks 40-42: number analyzed (Participants) | 125 | 124 | 36 | 285
  Not at risk,Weeks 40-42 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.93] | 0.00 [0.00 to 9.74] | 0.35 [0.01 to 1.94]
  Not at risk,Weeks 40-43: number analyzed (Participants) | 125 | 127 | 93 | 345
  Not at risk,Weeks 40-43 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.86] | 0.00 [0.00 to 3.89] | 0.29 [0.00 to 1.75]
  Not at risk,Weeks 40-44: number analyzed (Participants) | 125 | 130 | 135 | 390
  Not at risk,Weeks 40-44 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.80] | 0.00 [0.00 to 2.70] | 0.26 [0.00 to 1.55]
  Not at risk,Weeks 40-45: number analyzed (Participants) | 125 | 136 | 198 | 459
  Not at risk,Weeks 40-45 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.68] | 0.00 [0.00 to 1.85] | 0.22 [0.00 to 1.43]
  Not at risk,Weeks 40-46: number analyzed (Participants) | 125 | 144 | 217 | 486
  Not at risk,Weeks 40-46 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.53] | 0.00 [0.00 to 1.69] | 0.21 [0.00 to 1.37]
  Not at risk,Weeks 40-47: number analyzed (Participants) | 125 | 145 | 227 | 497
  Not at risk,Weeks 40-47 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.61] | 0.20 [0.00 to 1.35]
  Not at risk,Weeks 40-48: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-48 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.34]
  Not at risk,Weeks 40-49: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-49 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.34]
  Not at risk,Weeks 40-50: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-50 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.34]
  Not at risk,Weeks 40-51: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-51 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.34]
  Not at risk,Weeks 40-52: number analyzed (Participants) | 125 | 145 | 230 | 500
  Not at risk,Weeks 40-52 | 0.80 [0.02 to 4.38] | 0.00 [0.00 to 2.51] | 0.00 [0.00 to 1.59] | 0.20 [0.00 to 1.34]

170. Secondary Outcome: Cumulative Percentage of Subjects Reporting Any Vascular Disorders (MedDRA Primary SOC), Using ADR Card, Post Dose 2 in the Vaccinated_Fluarix Tetra Group, by Risk Status
Description: as for outcome 138
Time Frame: Within 7 days post Dose 2 i.e. the day of vaccination and the following 6 days
Population: as for outcome 110
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Unsolicited symptoms (i.e. AEIs and/or other AEs) were collected within 7 days post any vaccination. Serious adverse events related to the GSK's quadrivalent seasonal influenza vaccine, were collected over the whole study period (ISO weeks 40-52).
Arm/Group | Vaccinated_AlphaRix Tetra Group | Vaccinated_Influsplit Tetra Group | Vaccinated_Fluarix Tetra Group
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/278 | 0/453
Serious Adverse Events (participants affected / at risk) | 0/329 | 0/278 | 0/453
Other Adverse Events (participants affected / at risk) | 139/329 | 102/278 | 227/453
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccinated_AlphaRix Tetra Group (N=329) | Vaccinated_Influsplit Tetra Group (N=278) | Vaccinated_Fluarix Tetra Group (N=453)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (9) | 18 (20)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (14) | 5 (5) | 13 (13)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0) | 15 (15)
Chills (General disorders) | 5 (5) | 7 (7) | 13 (13)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 13 (13) | 22 (22) | 34 (36)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 10 (10) | 21 (21) | 25 (25)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 65 (65) | 46 (46) | 82 (83)
Injection site pruritus (General disorders) | 1 (1) | 3 (3) | 1 (1)
Injection site swelling (General disorders) | 17 (17) | 30 (30) | 33 (33)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucous membrane disorder (General disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 35 (36)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 12 (12) | 11 (11) | 16 (16)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 6 (6) | 13 (13) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 26 (27)
Arthropathy (Musculoskeletal and connective tissue disorders) | 11 (11) | 10 (10) | 11 (11)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (27) | 15 (15) | 32 (32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 24 (24) | 21 (21) | 33 (34)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 3 (3) | 4 (4) | 13 (15)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (11) | 57 (61)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 5 (5)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10) | 40 (41)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 15 (15) | 26 (26)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 30 (30) | 15 (15) | 52 (57)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (5)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT03688620/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03688620/SAP_001.pdf